CLINICAL TRIAL: NCT02951052
Title: A Phase III, Randomized, Multicenter, Parallel-group, Non-inferiority, Open-label Study Evaluating the Efficacy, Safety, and Tolerability of Switching to Long-acting Cabotegravir Plus Long-acting Rilpivirine From Current INI- NNRTI-, or PI-based Antiretroviral Regimen in HIV-1-infected Adults Who Are Virologically Suppressed
Brief Title: Study Evaluating the Efficacy, Safety, and Tolerability of Switching to Long-acting Cabotegravir Plus Long-acting Rilpivirine From Current Antiretroviral Regimen in Virologically Suppressed HIV-1-infected Adults
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201585; 2016-001647-39 (EudraCT Number)
Record Dates: First submitted 2016-09-15; First posted 2016-11-01 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: Long-acting cabotegravir; Virologic failure; long-acting rilpivirine; Antiretroviral
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — cabotegravir; Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- CAB LA + RPV LA every 4 weeks (Experimental): Eligible subjects receive Oral CAB 30 mg + RPV 25 mg once daily for four weeks, IM CAB LA 600 mg and RPV LA 900 mg for the first injection, and Week 4 onwards subjects will receive CAB LA (400 mg) + RPV LA (600 mg) injections every 4 weeks until withdrawal.
  Interventions: Drug: Cabotegravir (CAB) tablet; Drug: Rilpivirine (RPV) tablet; Drug: Cabotegravir - Injectable Suspension (CAB LA); Drug: Rilpivirine - Injectable Suspension (RPV LA)
- Current antiretroviral regimen (Active Comparator): Eligible subjects will continue their current anti-retroviral regimen (2 NRTIs plus an INI, NNRTI, or a PI) for 52 weeks. After 52 weeks subjects have the option to continue study participation by switching to CAB LA + RPV LA in the Extension Phase where they will follow the procedure of CAB LA + RPV LA arm.
  Interventions: Drug: 2 NRTIs plus an INI, NNRTI, or PI

INTERVENTIONS:
Drug: Cabotegravir (CAB) tablet — It is a white oval shaped film coated 30 mg tablets for oral administration. CAB Tablet is composed of cabotegravir sodium, lactose monohydrate, microcrystalline cellulose, hypromellose, sodium starch glycolate, magnesium stearate, and white film-coat
  Arms: CAB LA + RPV LA every 4 weeks
Drug: Rilpivirine (RPV) tablet — It is a 25 mg tablet with off-white, round, biconvex, film-coated and debossed on one side with "TMC" and the other side with "25". Each tablet contains RPV hydrochloride, and the inactive ingredients croscarmellose sodium, lactose monohydrate, magnesium stearate, polysorbate 20, povidone K30 and silicified microcrystalline cellulose
  Arms: CAB LA + RPV LA every 4 weeks
Drug: Cabotegravir - Injectable Suspension (CAB LA) — It is a sterile white to slightly pink suspension containing 200 mg/mL of CAB as free acid for administration by intramuscular (IM) injection. Each vial is for single-dose use containing a withdrawable volume of 2.0 mL, and does not require dilution prior to administration. CAB LA is composed of cabotegravir free acid, polysorbate 20, polyethylene glycol 3350, mannitol, and water for injection
  Arms: CAB LA + RPV LA every 4 weeks
Drug: Rilpivirine - Injectable Suspension (RPV LA) — It is a sterile white suspension containing 300 mg/mL of RPV as the free base. The route of administration is by intramuscular (IM) injection. Each vial contains a nominal fill of 2.0 mL, and does not require dilution prior to administration. RPV LA requires refrigeration and must be protected from light. RPV LA is composed of RPV free base, poloxamer 338, sodium dihydrogen phosphate monohydrate, citric acid monohydrate, glucose monohydrate, sodium hydroxide, water for injection.
  Arms: CAB LA + RPV LA every 4 weeks
Drug: 2 NRTIs plus an INI, NNRTI, or PI — Acceptable stable (initial or second) ARV regimens include 2 NRTIs plus:
  * INI with the exception of ABC/DTG/3TC (either the initial or second cART regimen)
  * NNRTI (either the initial or second cART regimen)
  * Boosted PI (or atazanavir [ATV] unboosted) (either the initial or second PI-based cART regimen)
  Arms: Current antiretroviral regimen

SUMMARY:
The Antiretroviral Therapy as Long Acting Suppression (ATLAS) study is being conducted to establish if human immunodeficiency virus type-1 (HIV-1) infected adult subjects with current viral suppression on a regimen with 2 nucleoside reverse transcriptase inhibitors (NRTIs) plus a third agent, remain suppressed upon switching to a two-drug intramuscular (IM) long-acting (LA) regimen of cabotegravir (CAB) and rilpivirine (RPV). This is a Phase 3, multi-phase, randomized, open label, active-controlled, multicenter, parallel-group, non-inferiority study in HIV-1, antiretroviral therapy (ART)-adult subjects who are stably suppressed on a current antiretroviral (ARV) regimen. This study is designed to demonstrate the non-inferior antiviral activity of switching to a two drug CAB LA 400 mg + RPV LA 600 mg regimen every 4 weeks (Q4W: monthly) compared with maintenance of current ARV regimen containing 2 NRTIs plus an INI, NNRTI, or a PI. Eligible subjects will be randomized (1:1) into the Maintenance Phase at Day 1 to either continue current ART or switch to initiate oral therapy with CAB 30 mg + RPV 25 mg once daily for 4 Weeks followed by Q4 weekly (monthly) CAB LA + RPV LA injections. Following the Maintenance phase at Week 52, subjects who were randomized to continue their current ART regimen will be given an option to switch to CAB LA + RPV LA injections. Those subjects would transition to LA dosing, beginning with 4 weeks oral CAB + RPV therapy at Week 52, and receive the first IM CAB LA + RPV LA injections at Week 56.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older (or ≥19 where required by local regulatory agencies), at the time of signing the informed consent.
* Must be on uninterrupted current regimen (either the initial or second ARV regimen) for at least 6 months prior to Screening. Any prior switch, defined as a change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability/safety, access to medications, or convenience/simplification, and must NOT have been done for treatment failure (HIV-1 RNA ≥400 c/mL).
* Acceptable stable (initial or second) ARV regimens prior to Screening include 2 NRTIs plus: INI with the exception of ABC/DTG/3TC (either the initial or second cART regimen);NNRTI (either the initial or second cART regimen);Boosted PI (or atazanavir [ATV] unboosted) (must be either the initial cART regimen or one historical within class switch is permitted due to safety/tolerability) The addition, removal, or switch of a drug(s) that has been used to treat HIV based on antiretroviral properties of the drug constitutes a change in ART with the following limited exceptions: Historical changes in formulations of ART drugs or booster drugs will not constitute a change in ART regimen if the data support similar exposures and efficacy, and the change must have been at least 3 months prior to Screening; Historical perinatal use of an NRTI when given in addition to an ongoing HAART will not be considered a change in ART regimen; A change in dosing scheme of the same drug from twice daily to once daily will not be considered a change in ART regimen if data support similar exposures and efficacy.
* Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: one within the 6 to 12 month window, and one within 6 months prior to Screening;
* Plasma HIV-1 RNA <50 c/mL at Screening;
* A female subjects is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at screen and a negative urine hCG test at Randomization), not lactating, and at least one of the following conditions applies:

  1. Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up; confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
  2. Reproductive potential and agrees to the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication, and until from 30 days prior to the first dose of study medication throughout the study, and for at least 30 days after discontinuation of all oral study medications and for at least 52 weeks after discontinuation of CAB LA and RPV LA. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form. Eligible subjects or their legal guardians (and next of kin when locally required), must sign a written Informed Consent Form before any protocol-specified assessments are conducted. Enrolment of subjects who are unable to provide direct informed consent is optional and will be based on local legal/regulatory requirements and site feasibility to conduct protocol procedures.
* Subjects enrolled in France must be affiliated to, or a beneficiary of, a social security category.
* All subjects participating in the study should be counselled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g., male condom) and on the risk of HIV transmission to an uninfected partner.

Exclusion Criteria:

* Within 6 months prior to Screening and after confirmed suppression to <50 c/mL on current ART regimen, any plasma HIV-1 RNA measurement ≥50 c/mL
* Within the 6 to 12 month window prior to Screening and after confirmed suppression to <50 c/mL, any plasma HIV-1 RNA measurement >200 c/mL, or 2 or more plasma HIV-1 RNA measurements ≥50 c/mL
* Any drug holiday during the window between initiating first HIV ART and 6 months prior to Screening, except for brief periods (less than 1 month) where all ART was stopped due to tolerability and/or safety concerns
* Any switch to a second line regimen, defined as change of a single drug or multiple drugs simultaneously, due to virologic failure to therapy (defined as a confirmed plasma HIV-1 RNA measurement ≥400 c/mL after initial suppression to <50 c/mL while on first line HIV therapy regimen)
* Abacavir/dolutegravir/lamivudine, (ABC/DTG/3TC) as current ART regimen
* A history of use of any regimen consisting of only single NNRTI therapy (even if only for peri-partum treatment), or only single or dual NRTI therapy prior to starting cART
* Subjects who are currently participating in or anticipate to be selected for any other interventional study
* Women who are pregnant, breastfeeding or plan to become pregnant or breastfeed during the study
* Any evidence of an active Center for Disease Control and Prevention (CDC) Stage 3 disease [CDC, 2014], except cutaneous Kaposi's sarcoma not requiring systemic therapy and historical or current CD4 cell counts less than 200 cells/mm^3
* Subjects with moderate to severe hepatic impairment
* Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the subjects ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the subject.
* Subjects determined by the Investigator to have a high risk of seizures, including subjects with an unstable or poorly controlled seizure disorder. A subject with a prior history of seizure may be considered for enrolment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrolment
* All subjects will be screened for syphilis (rapid plasma reagin [RPR]). Subjects with untreated syphilis infection, defined as a positive RPR without clear documentation of treatment, are excluded. Subjects with a serofast RPR result (persistence of a reactive nontreponemal syphilis test) despite history of adequate therapy and no evidence of re-exposure may enrol after consultation with the Medical Monitor. Subjects with a positive RPR test who have not been treated may be rescreened at least 30 days after completion of antibiotic treatment for syphilis
* Subjects who, in the investigator's judgment, pose a significant suicide risk. Subject's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk
* The subject has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV DNA as follows:•Subjects positive for HBsAg are excluded;
* Subjects negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded
* Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; subjects who are anticipated to require HCV treatment within 12 months must be excluded. (HCV treatment on study may be permitted post Week 48, following consultation with the medical monitor) Subjects with HCV co-infection will be allowed entry into phase 3 studies if: Liver enzymes meet entry criteria; HCV Disease has undergone appropriate work-up, and is not advanced, and will not require treatment prior to the Week 48 visit. Additional information (where available) on subjects with HCV co-infection at screening should include results from any liver biopsy, Fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment. In the event that recent biopsy or imaging data is not available or inconclusive, the Fib-4 score will be used to verify eligibility: Fib-4 score > 3.25 is exclusionary; Fib-4 scores 1.45 - 3.25 requires Medical Monitor consultation Fibrosis 4 Score Formula:( Age x AST ) / ( Platelets x ( sqr [ ALT ])
* Unstable liver disease (as defined by any of the following: presence of ascites,encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices,or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment)
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Ongoing or clinically relevant pancreatitis
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the subject prior to randomization
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the subject unable to receive study medication
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled
* Current or anticipated need for chronic anti-coagulation with the exception of the use of low dose acetylsalicylic acid (≤325mg).
* Any evidence of primary resistance based on the presence of any major known INI or NNRTI resistance-associated mutation, except for K103N, (International AIDS Society [IAS]-USA, 2015) by any historical resistance test result.
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening phase to verify a result
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the subject's participation in the study of an investigational compound
* Subject has estimated creatine clearance <50mL/min per 1.73m^2 via CKDEPI Method
* Alanine aminotransferase (ALT) ≥3 × ULN Exposure to an experimental drug or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study;
* Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; tuberculosis therapy with the exception of isoniazid (isonicotinylhydrazid,INH); anti-coagulation agents; Immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons. Note: Subjects using short term (e.g. ≤21 days) systemic corticosteroid treatment; topical, inhaled and intranasal corticosteroids are eligible for enrolment.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with any agent, except recognized ART as allowed above, with documented activity against HIV-1 within 28 days of study Day 1
* Use of medications which are associated with Torsade de Pointes.
* Current or prior history of etravirine (ETR)
* Current use of tipranavir/ritonavir or fosamprenavir/ritonavir
* Subjects receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2029-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (91):
- United States (31):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Rosario
- Australia (3):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Prahran, Victoria
- Canada (5):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
- France (5):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Denis
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tourcoing
- Germany (7):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, München
- Italy (2):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Milan
- GSK Investigational Site, Guadalajara, Mexico
- Russia (11):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Toliyatti
  - GSK Investigational Site, Yekaterinburg
- South Africa (7):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Middelburg
  - GSK Investigational Site, Pretorai
  - GSK Investigational Site, Winnie Mandela
- South Korea (4):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (10):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Elche Alicante
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo Pontevedra
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below).
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20382

REFERENCES:
- [Background] Swindells S, Lutz T, Van Zyl L, Porteiro N, Stoll M, Mitha E, Shon A, Benn P, Huang JO, Harrington CM, Hove K, Ford SL, Talarico CL, Chounta V, Crauwels H, Van Solingen-Ristea R, Vanveggel S, Margolis DA, Smith KY, Vandermeulen K, Spreen WR. Week 96 extension results of a Phase 3 study evaluating long-acting cabotegravir with rilpivirine for HIV-1 treatment. AIDS. 2022 Feb 1;36(2):185-194. doi: 10.1097/QAD.0000000000003025. PMID 34261093
- [Derived] Elliot ER, Polli JW, Patel P, Garside L, Grove R, Barnett V, Roberts J, Byrapuneni S, Crauwels H, Ford SL, Van Solingen-Ristea R, Birmingham E, D'Amico R, Baugh B, van Wyk J. Efficacy, Safety, and Pharmacokinetics by Body Mass Index Category in Phase 3/3b Long-Acting Cabotegravir Plus Rilpivirine Trials. J Infect Dis. 2024 Jul 25;230(1):e34-e42. doi: 10.1093/infdis/jiad580. PMID 39052748
- [Derived] Chounta V, Byrnes HF, Henry-Szatkowski M, Browning D, Donatti C, Lambert J. Psychometric Validation of the Perception of Injection (PIN) Questionnaire Using Data From Two Phase III, Open-Label, Active-Controlled, Non-Inferiority Studies in People Living With HIV. Adv Ther. 2023 Dec;40(12):5300-5314. doi: 10.1007/s12325-023-02656-1. Epub 2023 Sep 30. PMID 37776478
- [Derived] Moreno S, Rivero A, Ventayol P, Falco V, Torralba M, Schroeder M, Neches V, Vallejo-Aparicio LA, Mackenzie I, Turner M, Harrison C. Cabotegravir and Rilpivirine Long-Acting Antiretroviral Therapy Administered Every 2 Months is Cost-Effective for the Treatment of HIV-1 in Spain. Infect Dis Ther. 2023 Aug;12(8):2039-2055. doi: 10.1007/s40121-023-00840-y. Epub 2023 Jul 14. PMID 37452174
- [Derived] Chounta V, Snedecor SJ, Wu S, Van de Velde N. Indirect comparison of 48-week efficacy and safety of long-acting cabotegravir and rilpivirine maintenance every 8 weeks with daily oral standard of care antiretroviral therapy in participants with virologically suppressed HIV-1-infection. BMC Infect Dis. 2022 May 4;22(1):428. doi: 10.1186/s12879-022-07243-3. PMID 35508986
- [Derived] Rizzardini G, Overton ET, Orkin C, Swindells S, Arasteh K, Gorgolas Hernandez-Mora M, Pokrovsky V, Girard PM, Oka S, Andrade-Villanueva JF, Richmond GJ, Baumgarten A, Masia M, Latiff G, Griffith S, Harrington CM, Hudson KJ, St Clair M, Talarico CL, Patel P, Cutrell A, Van Eygen V, D'Amico R, Mrus JM, Wu S, Ford SL, Chow K, Roberts J, Wills A, Walters N, Vanveggel S, Van Solingen-Ristea R, Crauwels H, Smith KY, Spreen WR, Margolis DA. Long-Acting Injectable Cabotegravir + Rilpivirine for HIV Maintenance Therapy: Week 48 Pooled Analysis of Phase 3 ATLAS and FLAIR Trials. J Acquir Immune Defic Syndr. 2020 Dec 1;85(4):498-506. doi: 10.1097/QAI.0000000000002466. PMID 33136751
- [Derived] Swindells S, Andrade-Villanueva JF, Richmond GJ, Rizzardini G, Baumgarten A, Masia M, Latiff G, Pokrovsky V, Bredeek F, Smith G, Cahn P, Kim YS, Ford SL, Talarico CL, Patel P, Chounta V, Crauwels H, Parys W, Vanveggel S, Mrus J, Huang J, Harrington CM, Hudson KJ, Margolis DA, Smith KY, Williams PE, Spreen WR. Long-Acting Cabotegravir and Rilpivirine for Maintenance of HIV-1 Suppression. N Engl J Med. 2020 Mar 19;382(12):1112-1123. doi: 10.1056/NEJMoa1904398. Epub 2020 Mar 4. PMID 32130809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase III, randomized, open-label, active-controlled, multi-center, parallel-group, non-inferiority study to evaluate the antiviral activity and safety of two long-acting (LA) injectable drugs, cabotegravir (CAB) plus rilpivirine (RPV) when compared to current standard of care conducted in virologically suppressed human immunodeficiency.
Pre-assignment Details: A total of 618 participants were enrolled in the study. Two randomized participants did not receive study treatment. A total of 616 participants contributed to the Intent-to-treat exposed Population and Safety Population. The results presented are based on Week 48 primary analysis.
Groups:
- CAB LA+RPV LA (Q4W): During Maintenance phase (Day 1-Week 52), participants received oral CAB 30 milligram (mg)+RPV 25 mg once daily from Day 1 for 4 weeks. At Week 4B, the participants were given the last dose of oral CAB+RPV and the first dose of CAB LA 600 mg+RPV LA 900 mg injections within 2 hours of the final oral dose. Participants received intramuscular (IM) injections of CAB LA 400 mg and RPV LA 600 mg every four weeks (Q4W) through Week 52. After completion of Maintenance phase, participants who chose to enter Extension phase continued to receive both CAB LA and RPV LA. Participants withdrawn from study treatment who received at least one CAB LA+RPV LA injection were required to enter a 52-week long term follow-up period
- Current ART: During Maintenance phase (Day 1 - Week 52), participants continued to receive current antiretroviral therapy (ART) (protease inhibitor [PI] or integrase inhibitor [INI] or non-nucleoside reverse transcriptase inhibitor [NNRTI]) plus 2 NRTIs for 52 weeks. After completion of the Maintenance phase, participants who chose to enter the Extension phase switched to CAB LA+RPV LA
Period: Overall Study
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Started | 308 | 308
Completed | 281 | 290
Not Completed | 27 | 18
Not completed — Adverse Event | 13 | 5
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol-specified withdrawal criterion | 1 | 0
Not completed — Protocol Violation | 5 | 3
Not completed — Lack of Efficacy | 3 | 4
Not completed — Ongoing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART | Total
Number analyzed (Participants) | 308 | 308 | 616
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (9.99) | 43.2 (11.43) | 42.4 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 104 | 203
  Male | 209 | 204 | 413
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian (AI) or Alaska Native (AN) | 8 | 8 | 16
  Asian-Central South Asian Heritage | 1 | 0 | 1
  Asian-Japanese/East/South-East Asian Heritage | 21 | 13 | 34
  Black or African American | 62 | 77 | 139
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 214 | 207 | 421
  AI or AN & Black/African American | 0 | 1 | 1
  AI or AN & Black/African American & White | 1 | 1 | 2
  Black/African American or White | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virologic Failure (HIV-1 Ribonucleic Acid [RNA] >=50 Copies Per Millilter [mL]) Using Snapshot Algorithm at Week 48
Description: Number of participants with virologic failure endpoint (HIV-1 RNA>=50 c/mL) as per Food and Drug Administration (FDA) snapshot algorithm at Week 48 was assessed to demonstrate the non-inferior antiviral activity of switching to intramuscular (IM) CAB LA+RPV LA every 4 weeks compared to continuation of current ART regimen over 48 weeks in HIV-1 infected ART-experienced participants. The HIV-1 RNA >=50 copies/mL per snapshot algorithm was determined by the last available on-treatment HIV-1 RNA measurement within the analysis visit window of interest.
Time Frame: Week 48
Population: Intent-to treat exposed (ITT-E) participants included all randomized participants who received at least one dose of Investigational Product (IP) during the maintenance phase. Participants were analyzed according to the randomized treatment regardless of what treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants | 5 | 3
Statistical Analysis 1: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Non-Inferiority — Non-inferiority in the proportion of participants with virologic failure at Week 48 (per FDA's snapshot algorithm for assessing HIV-1 RNA >=50 copies/mL) can be concluded if the upper bound of a two-sided 95% confidence interval for the difference in failure rates between the two treatment arms (CAB - current ART) is not more than 6%; Adjusted difference in proportion = 0.6, 95% CI 2-sided [-1.2 to 2.5] — Adjusted difference in proportion was based on Cochran-Mantel Haenszel stratified analysis adjusting for the following baseline stratification factors: sex at birth (Male, Female) and Baseline third agent (PI, NNRTI, INI)

2. Secondary Outcome: Number of Participants With HIV-1 RNA <50 Copies/mL Using Snapshot Algorithm at Week 48
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Number of participants with plasma HIV-1 RNA <50 copies/mL at Week 48 using FDA snapshot algorithm was assessed to demonstrate antiviral and immunologic activity of switching to IM CAB LA+RPV LA every 4 weeks compared to continuation of current ART. The HIV-1 RNA <50 copies/mL per snapshot algorithm was determined by the last available on-treatment HIV-1 RNA measurement within the analysis visit window of interest.
Time Frame: Week 48
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants | 285 | 294
Statistical Analysis 1: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Non-Inferiority — Non-inferiority in the proportion of participants with HIV-1 RNA<50 c/mL at Week 48 (per FDA's snapshot algorithm) can be concluded if the lower bound of a two-sided 95% confidence interval for the difference in success rates between the two treatment arms (CAB - current ART) is more than -10%; Adjusted difference in proportion = -3.0, 95% CI 2-sided [-6.7 to 0.7] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With HIV-1 RNA <200 Copies/mL Using Snapshot Algorithm at Week 48
Description: Number of participants with plasma HIV-1 RNA <200 copies/mL at Week 48 using the snapshot algorithm was assessed based on the antiviral and immunologic activity of switching to IM CAB LA+RPV LA every 4 weeks compared to continuation of current ART.
Time Frame: Week 48
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants | 286 | 295

4. Secondary Outcome: Number of Participants With Confirmed Virologic Failure (CVF)
Description: The CVF is defined as rebound as indicated by two consecutive plasma HIV-1-RNA levels >=200 copies/mL after prior suppression to <200 copies/mL. The outcome displays only visits during which at least one new CVF occurs. Plasma samples were collected for quantitative analysis of HIV-1 RNA.
Time Frame: Weeks 8, 12, 20, 24, 32 and 40
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants
  Week 8 | 1 | 0
  Week 12 | 2 | 0
  Week 20 | 2 | 2
  Week 24 | 3 | 2
  Week 32 | 3 | 3
  Week 40 | 3 | 4

5. Secondary Outcome: Absolute Values for Plasma HIV-1 RNA at Week 48
Description: Logarithm to base 10 (log10) values for plasma HIV-1 RNA has been presented.
Time Frame: Week 48
Population: ITT-E population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 265 | 292
log10 copies/mL | 1.505 (0.0470) | 1.518 (0.1123)

6. Secondary Outcome: Change From Baseline Values for Plasma HIV-1 RNA
Description: Plasma for quantitative HIV-1 RNA were collected at indicated time points. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline was defined as: HIV-1 RNA(log 10) at Week 48 - HIV-1 RNA(log 10) at Baseline.
Time Frame: Baseline and Week 48
Population: ITT-E population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 265 | 292
log10 copies/mL | -0.013 (0.1940) | 0.012 (0.1201)

7. Secondary Outcome: Absolute Values for CD4+ Lymphocyte Count at Week 48
Description: Blood samples were collected and CD4+ cell count assessment by flow cyclometry was carried out to evaluate the immunologic activity of switching to IM CAB LA+RPV LA every 4 weeks compared to current ART.
Time Frame: Week 48
Population: ITT-E population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 263 | 290
Cells per cubic millimeter | 685.3 (262.97) | 716.7 (292.85)

8. Secondary Outcome: Change From Baseline Values for CD4+ Lymphocyte Count at Week 48
Description: Blood samples were collected and CD4+ cell count assessment by flow cyclometry was carried out to evaluate the immunologic activity of switching to IM CAB LA+RPV LA every 4 weeks compared to current ART.Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline was defined as post-dose visit value at Week 48 minus Baseline value.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-E population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 263 | 290
Cells per cubic millimeter | 9.9 (187.24) | 19.4 (168.80)

9. Secondary Outcome: Number of Participants With Disease Progression
Description: Disease progression was defined as HIV-associated conditions, acquired immunodeficiency syndrome (AIDS), and death through 48 Weeks. Data of participants who experienced disease progression to Centers for Disease Control and Prevention (CDC) Stage III or death has been presented.
Time Frame: Up to Week 48
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants | 8 | 8

10. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement. Safety Population comprised of all randomized participants who received at least one dose of IP during the maintenance phase of the study (on or after Day 1 visit). Participants will be assessed according to actual treatment received.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants
  Any non-SAE | 263 | 117
  Any SAE | 13 | 14

11. Secondary Outcome: Number of Participants With Severity of Adverse Events
Description: Severity of adverse events (AEs) were defined as per The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table) Version 2.0, November 2014. Severity grades for AEs were as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (Potentially life-threatening) and Grade 5 were all deaths related to an AE.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants
  Grade 1 | 101 | 115
  Grade 2 | 158 | 81
  Grade 3 | 27 | 19
  Grade 4 | 8 | 4
  Grade 5 | 0 | 1

12. Secondary Outcome: Absolute Values for Hematology Parameters Over Time Including Week 48: Basophil, Eosinophils, Leukocytes, Lymphocytes, Neutrophils, Monocytes, and Platelets
Description: Blood samples were collected for the analysis of hematology parameters including basophil, eosinophils, leukocytes, lymphocytes, neutrophils, monocytes, and platelets at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: Safety population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
10^9 cells per liter
  Basophils, Baseline, n=308, 307: number analyzed (Participants) | 308 | 307
  Basophils, Baseline, n=308, 307 | 0.021 (0.0147) | 0.021 (0.0148)
  Basophils, Week 4, n=299, 291: number analyzed (Participants) | 299 | 291
  Basophils, Week 4, n=299, 291 | 0.024 (0.0153) | 0.023 (0.0161)
  Basophils, Week 8, n=216, 294: number analyzed (Participants) | 216 | 294
  Basophils, Week 8, n=216, 294 | 0.023 (0.0188) | 0.022 (0.0155)
  Basophils, Week 12, n=293, 290: number analyzed (Participants) | 293 | 290
  Basophils, Week 12, n=293, 290 | 0.022 (0.0154) | 0.022 (0.0157)
  Basophils, Week 16, n=274, 292: number analyzed (Participants) | 274 | 292
  Basophils, Week 16, n=274, 292 | 0.022 (0.0147) | 0.022 (0.0140)
  Basophils, Week 20, n=273, 292: number analyzed (Participants) | 273 | 292
  Basophils, Week 20, n=273, 292 | 0.023 (0.0182) | 0.024 (0.0195)
  Basophils, Week 24, n=277, 292: number analyzed (Participants) | 277 | 292
  Basophils, Week 24, n=277, 292 | 0.023 (0.0139) | 0.024 (0.0133)
  Basophils, Week 28, n=266, 295: number analyzed (Participants) | 266 | 295
  Basophils, Week 28, n=266, 295 | 0.024 (0.0150) | 0.023 (0.0138)
  Basophils, Week 32, n=262, 283: number analyzed (Participants) | 262 | 283
  Basophils, Week 32, n=262, 283 | 0.025 (0.0171) | 0.024 (0.0159)
  Basophils, Week 36, n=260, 282: number analyzed (Participants) | 260 | 282
  Basophils, Week 36, n=260, 282 | 0.029 (0.0211) | 0.028 (0.0190)
  Basophils, Week 40, n=258, 280: number analyzed (Participants) | 258 | 280
  Basophils, Week 40, n=258, 280 | 0.035 (0.0266) | 0.031 (0.0206)
  Basophils, Week 44, n=258, 268: number analyzed (Participants) | 258 | 268
  Basophils, Week 44, n=258, 268 | 0.037 (0.0275) | 0.033 (0.0222)
  Basophils, Week 48, n=246, 274: number analyzed (Participants) | 246 | 274
  Basophils, Week 48, n=246, 274 | 0.040 (0.0253) | 0.039 (0.0249)
  Eosinophils, Baseline, n=308, 307: number analyzed (Participants) | 308 | 307
  Eosinophils, Baseline, n=308, 307 | 0.142 (0.1409) | 0.140 (0.1538)
  Eosinophils, Week 4, n=299, 291: number analyzed (Participants) | 299 | 291
  Eosinophils, Week 4, n=299, 291 | 0.168 (0.1587) | 0.145 (0.1422)
  Eosinophils, Week 8, n=216, 294: number analyzed (Participants) | 216 | 294
  Eosinophils, Week 8, n=216, 294 | 0.154 (0.1379) | 0.131 (0.1333)
  Eosinophils, Week 12, n=293, 290: number analyzed (Participants) | 293 | 290
  Eosinophils, Week 12, n=293, 290 | 0.142 (0.1172) | 0.132 (0.1471)
  Eosinophils, Week 16, n=274, 292: number analyzed (Participants) | 274 | 292
  Eosinophils, Week 16, n=274, 292 | 0.153 (0.1395) | 0.131 (0.1584)
  Eosinophils, Week 20, n=273, 292: number analyzed (Participants) | 273 | 292
  Eosinophils, Week 20, n=273, 292 | 0.152 (0.1480) | 0.116 (0.1094)
  Eosinophils, Week 24, n=277, 292: number analyzed (Participants) | 277 | 292
  Eosinophils, Week 24, n=277, 292 | 0.143 (0.1323) | 0.121 (0.1337)
  Eosinophils, Week 28, n=266, 295: number analyzed (Participants) | 266 | 295
  Eosinophils, Week 28, n=266, 295 | 0.144 (0.1266) | 0.129 (0.1320)
  Eosinophils, Week 32, n=262, 283: number analyzed (Participants) | 262 | 283
  Eosinophils, Week 32, n=262, 283 | 0.170 (0.1643) | 0.131 (0.1319)
  Eosinophils, Week 36, n=260, 282: number analyzed (Participants) | 260 | 282
  Eosinophils, Week 36, n=260, 282 | 0.150 (0.1403) | 0.132 (0.1162)
  Eosinophils, Week 40, n=258, 280: number analyzed (Participants) | 258 | 280
  Eosinophils, Week 40, n=258, 280 | 0.161 (0.1206) | 0.132 (0.1124)
  Eosinophils, Week 44, n=258, 268: number analyzed (Participants) | 258 | 268
  Eosinophils, Week 44, n=258, 268 | 0.175 (0.1471) | 0.136 (0.1126)
  Eosinophils, Week 48, n=246, 274: number analyzed (Participants) | 246 | 274
  Eosinophils, Week 48, n=246, 274 | 0.174 (0.1412) | 0.140 (0.1265)
  Leukocytes, Baseline, n=308, 307: number analyzed (Participants) | 308 | 307
  Leukocytes, Baseline, n=308, 307 | 5.87 (1.928) | 5.65 (1.897)
  Leukocytes, Week 4, n=300, 298: number analyzed (Participants) | 300 | 298
  Leukocytes, Week 4, n=300, 298 | 6.43 (2.154) | 5.81 (1.733)
  Leukocytes, Week 8, n=217, 301: number analyzed (Participants) | 217 | 301
  Leukocytes, Week 8, n=217, 301 | 6.14 (1.875) | 5.64 (1.663)
  Leukocytes, Week 12, n=294, 293: number analyzed (Participants) | 294 | 293
  Leukocytes, Week 12, n=294, 293 | 6.24 (1.876) | 5.77 (1.751)
  Leukocytes, Week 16, n=279, 295: number analyzed (Participants) | 279 | 295
  Leukocytes, Week 16, n=279, 295 | 6.27 (1.920) | 5.82 (1.756)
  Leukocytes, Week 20, n=276, 298: number analyzed (Participants) | 276 | 298
  Leukocytes, Week 20, n=276, 298 | 6.27 (1.947) | 5.70 (1.721)
  Leukocytes, Week 24, n=279, 294: number analyzed (Participants) | 279 | 294
  Leukocytes, Week 24, n=279, 294 | 6.18 (1.931) | 5.78 (1.756)
  Leukocytes, Week 28, n=268, 297: number analyzed (Participants) | 268 | 297
  Leukocytes, Week 28, n=268, 297 | 6.08 (1.949) | 5.73 (1.637)
  Leukocytes, Week 32, n=267, 288: number analyzed (Participants) | 267 | 288
  Leukocytes, Week 32, n=267, 288 | 6.30 (1.914) | 5.73 (1.666)
  Leukocytes, Week 36, n=264, 285: number analyzed (Participants) | 264 | 285
  Leukocytes, Week 36, n=264, 285 | 6.14 (1.831) | 5.80 (1.968)
  Leukocytes, Week 40, n=264, 286: number analyzed (Participants) | 264 | 286
  Leukocytes, Week 40, n=264, 286 | 6.24 (2.046) | 5.74 (1.713)
  Leukocytes, Week 44, n=269, 279: number analyzed (Participants) | 269 | 279
  Leukocytes, Week 44, n=269, 279 | 6.15 (1.884) | 5.66 (1.745)
  Leukocytes, Week 48, n=252, 282: number analyzed (Participants) | 252 | 282
  Leukocytes, Week 48, n=252, 282 | 6.01 (1.943) | 5.62 (1.679)
  Lymphocytes, Baseline, n=308, 307: number analyzed (Participants) | 308 | 307
  Lymphocytes, Baseline, n=308, 307 | 1.943 (0.6073) | 1.940 (0.6880)
  Lymphocytes, Week 4, n=299, 291: number analyzed (Participants) | 299 | 291
  Lymphocytes, Week 4, n=299, 291 | 2.127 (0.6942) | 2.059 (0.6929)
  Lymphocytes, Week 8, n=216, 294: number analyzed (Participants) | 216 | 294
  Lymphocytes, Week 8, n=216, 294 | 1.995 (0.6347) | 1.975 (0.6549)
  Lymphocytes, Week 12, n=293, 290: number analyzed (Participants) | 293 | 290
  Lymphocytes, Week 12, n=293, 290 | 1.984 (0.6428) | 2.026 (0.6996)
  Lymphocytes, Week 16, n=274, 292: number analyzed (Participants) | 274 | 292
  Lymphocytes, Week 16, n=274, 292 | 2.057 (0.6840) | 2.029 (0.6584)
  Lymphocytes, Week 20, n=273, 292: number analyzed (Participants) | 273 | 292
  Lymphocytes, Week 20, n=273, 292 | 2.035 (0.6140) | 2.030 (0.6906)
  Lymphocytes, Week 24, n=277, 292: number analyzed (Participants) | 277 | 292
  Lymphocytes, Week 24, n=277, 292 | 2.016 (0.6523) | 1.980 (0.6047)
  Lymphocytes, Week 28, n=266, 295: number analyzed (Participants) | 266 | 295
  Lymphocytes, Week 28, n=266, 295 | 2.049 (0.6960) | 2.016 (0.6476)
  Lymphocytes, Week 32, n=262, 283: number analyzed (Participants) | 262 | 283
  Lymphocytes, Week 32, n=262, 283 | 2.020 (0.6157) | 2.007 (0.6511)
  Lymphocytes, Week 36, n=260, 282: number analyzed (Participants) | 260 | 282
  Lymphocytes, Week 36, n=260, 282 | 1.960 (0.6009) | 1.984 (0.6444)
  Lymphocytes, Week 40, n=258, 280: number analyzed (Participants) | 258 | 280
  Lymphocytes, Week 40, n=258, 280 | 1.994 (0.6149) | 1.957 (0.6305)
  Lymphocytes, Week 44, n=258, 268: number analyzed (Participants) | 258 | 268
  Lymphocytes, Week 44, n=258, 268 | 2.016 (0.6457) | 1.970 (0.6219)
  Lymphocytes, Week 48, n=246, 274: number analyzed (Participants) | 246 | 274
  Lymphocytes, Week 48, n=246, 274 | 1.900 (0.5725) | 1.915 (0.6204)
  Neutrophils, Baseline, n=308, 307: number analyzed (Participants) | 308 | 307
  Neutrophils, Baseline, n=308, 307 | 3.437 (1.6106) | 3.209 (1.5748)
  Neutrophils, Week 4, n=299, 291: number analyzed (Participants) | 299 | 291
  Neutrophils, Week 4, n=299, 291 | 3.708 (1.8763) | 3.244 (1.3931)
  Neutrophils, Week 8, n=216, 294: number analyzed (Participants) | 216 | 294
  Neutrophils, Week 8, n=216, 294 | 3.597 (1.6128) | 3.190 (1.3370)
  Neutrophils, Week 12, n=293, 290: number analyzed (Participants) | 293 | 290
  Neutrophils, Week 12, n=293, 290 | 3.724 (1.5751) | 3.268 (1.4153)
  Neutrophils, Week 16, n=274, 292: number analyzed (Participants) | 274 | 292
  Neutrophils, Week 16, n=274, 292 | 3.670 (1.6777) | 3.308 (1.3870)
  Neutrophils, Week 20, n=273, 292: number analyzed (Participants) | 273 | 292
  Neutrophils, Week 20, n=273, 292 | 3.707 (1.6532) | 3.188 (1.3345)
  Neutrophils, Week 24, n=277, 292: number analyzed (Participants) | 277 | 292
  Neutrophils, Week 24, n=277, 292 | 3.613 (1.5978) | 3.289 (1.4381)
  Neutrophils, Week 28, n=266, 295: number analyzed (Participants) | 266 | 295
  Neutrophils, Week 28, n=266, 295 | 3.528 (1.5464) | 3.221 (1.2962)
  Neutrophils, Week 32, n=262, 283: number analyzed (Participants) | 262 | 283
  Neutrophils, Week 32, n=262, 283 | 3.704 (1.6196) | 3.228 (1.2909)
  Neutrophils, Week 36, n=260, 282: number analyzed (Participants) | 260 | 282
  Neutrophils, Week 36, n=260, 282 | 3.629 (1.5688) | 3.314 (1.6341)
  Neutrophils, Week 40, n=258, 280: number analyzed (Participants) | 258 | 280
  Neutrophils, Week 40, n=258, 280 | 3.688 (1.7685) | 3.280 (1.4190)
  Neutrophils, Week 44, n=258, 268: number analyzed (Participants) | 258 | 268
  Neutrophils, Week 44, n=258, 268 | 3.571 (1.5425) | 3.169 (1.4140)
  Neutrophils, Week 48, n=246, 274: number analyzed (Participants) | 246 | 274
  Neutrophils, Week 48, n=246, 274 | 3.450 (1.5649) | 3.172 (1.3627)
  Monocytes, Baseline, n=308, 307: number analyzed (Participants) | 308 | 307
  Monocytes, Baseline, n=308, 307 | 0.353 (0.1745) | 0.339 (0.1596)
  Monocytes, Week 4, n=299, 291: number analyzed (Participants) | 299 | 291
  Monocytes, Week 4, n=299, 291 | 0.404 (0.1951) | 0.367 (0.1694)
  Monocytes, Week 8, n=216, 294: number analyzed (Participants) | 216 | 294
  Monocytes, Week 8, n=216, 294 | 0.369 (0.1628) | 0.358 (0.1875)
  Monocytes, Week 12, n=293, 290: number analyzed (Participants) | 293 | 290
  Monocytes, Week 12, n=293, 290 | 0.375 (0.1563) | 0.342 (0.1693)
  Monocytes, Week 16, n=274, 292: number analyzed (Participants) | 274 | 292
  Monocytes, Week 16, n=274, 292 | 0.364 (0.1537) | 0.345 (0.1645)
  Monocytes, Week 20, n=273, 292: number analyzed (Participants) | 273 | 292
  Monocytes, Week 20, n=273, 292 | 0.356 (0.1526) | 0.342 (0.1632)
  Monocytes, Week 24, n=277, 292: number analyzed (Participants) | 277 | 292
  Monocytes, Week 24, n=277, 292 | 0.370 (0.1632) | 0.341 (0.1632)
  Monocytes, Week 28, n=266, 295: number analyzed (Participants) | 266 | 295
  Monocytes, Week 28, n=266, 295 | 0.354 (0.1631) | 0.333 (0.1592)
  Monocytes, Week 32, n=262, 283: number analyzed (Participants) | 262 | 283
  Monocytes, Week 32, n=262, 283 | 0.378 (0.1629) | 0.351 (0.1801)
  Monocytes, Week 36, n=260, 282: number analyzed (Participants) | 260 | 282
  Monocytes, Week 36, n=260, 282 | 0.376 (0.1593) | 0.366 (0.1824)
  Monocytes, Week 40, n=258, 280: number analyzed (Participants) | 258 | 280
  Monocytes, Week 40, n=258, 280 | 0.402 (0.1612) | 0.359 (0.1823)
  Monocytes, Week 44, n=258, 268: number analyzed (Participants) | 258 | 268
  Monocytes, Week 44, n=258, 268 | 0.409 (0.1643) | 0.388 (0.1795)
  Monocytes, Week 48, n=246, 274: number analyzed (Participants) | 246 | 274
  Monocytes, Week 48, n=246, 274 | 0.407 (0.1600) | 0.384 (0.1742)
  Platelets, Baseline, n=308, 308 | 231.1 (56.75) | 232.9 (59.28)
  Platelets, Week 4, n=300, 298: number analyzed (Participants) | 300 | 298
  Platelets, Week 4, n=300, 298 | 233.5 (55.09) | 238.1 (61.98)
  Platelets, Week 8, n=216, 298: number analyzed (Participants) | 216 | 298
  Platelets, Week 8, n=216, 298 | 227.4 (47.04) | 234.0 (61.84)
  Platelets, Week 12, n=294, 290: number analyzed (Participants) | 294 | 290
  Platelets, Week 12, n=294, 290 | 230.2 (57.32) | 237.8 (64.42)
  Platelets, Week 16, n=279, 294: number analyzed (Participants) | 279 | 294
  Platelets, Week 16, n=279, 294 | 226.1 (56.82) | 236.4 (61.63)
  Platelets, Week 20, n=274, 297: number analyzed (Participants) | 274 | 297
  Platelets, Week 20, n=274, 297 | 226.5 (58.11) | 237.7 (61.51)
  Platelets, Week 24, n=279, 292: number analyzed (Participants) | 279 | 292
  Platelets, Week 24, n=279, 292 | 224.9 (53.19) | 239.8 (64.11)
  Platelets, Week 28, n=268, 295: number analyzed (Participants) | 268 | 295
  Platelets, Week 28, n=268, 295 | 224.7 (54.15) | 239.0 (62.32)
  Platelets, Week 32, n=267, 289: number analyzed (Participants) | 267 | 289
  Platelets, Week 32, n=267, 289 | 226.5 (50.84) | 239.3 (59.53)
  Platelets, Week 36, n=267, 284: number analyzed (Participants) | 267 | 284
  Platelets, Week 36, n=267, 284 | 229.0 (53.90) | 242.9 (66.12)
  Platelets, Week 40, n=263, 288: number analyzed (Participants) | 263 | 288
  Platelets, Week 40, n=263, 288 | 230.1 (53.48) | 240.8 (61.92)
  Platelets, Week 44, n=270, 286: number analyzed (Participants) | 270 | 286
  Platelets, Week 44, n=270, 286 | 235.5 (55.80) | 241.4 (61.73)
  Platelets, Week 48, n=253, 281: number analyzed (Participants) | 253 | 281
  Platelets, Week 48, n=253, 281 | 230.5 (54.33) | 240.2 (62.95)

13. Secondary Outcome: Absolute Values for Hematology Parameters: Erythrocyte Mean Corpuscular Volume
Description: Blood samples were collected for the analysis of hematology parameter including erythrocyte mean corpuscular volume at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Femtoliters
  Baseline, n=308, 308 | 95.7 (7.97) | 96.6 (9.35)
  Week 4, n=300, 300: number analyzed (Participants) | 300 | 300
  Week 4, n=300, 300 | 94.6 (6.88) | 96.9 (9.31)
  Week 8, n=218, 301: number analyzed (Participants) | 218 | 301
  Week 8, n=218, 301 | 92.7 (5.76) | 96.8 (9.25)
  Week 12, n=294, 293: number analyzed (Participants) | 294 | 293
  Week 12, n=294, 293 | 91.7 (5.69) | 96.9 (9.34)
  Week 16, n=280, 296: number analyzed (Participants) | 280 | 296
  Week 16, n=280, 296 | 90.6 (5.48) | 96.8 (9.64)
  Week 20, n=276, 298: number analyzed (Participants) | 276 | 298
  Week 20, n=276, 298 | 90.3 (5.37) | 97.0 (9.63)
  Week 24, n=279, 294: number analyzed (Participants) | 279 | 294
  Week 24, n=279, 294 | 90.2 (5.44) | 96.9 (9.75)
  Week 28, n=268, 297: number analyzed (Participants) | 268 | 297
  Week 28, n=268, 297 | 90.2 (5.68) | 97.2 (9.77)
  Week 32, n=268, 291: number analyzed (Participants) | 268 | 291
  Week 32, n=268, 291 | 90.1 (5.55) | 96.7 (9.36)
  Week 36, n=267, 288: number analyzed (Participants) | 267 | 288
  Week 36, n=267, 288 | 89.8 (5.64) | 96.5 (9.08)
  Week 40, n=264, 289: number analyzed (Participants) | 264 | 289
  Week 40, n=264, 289 | 89.9 (5.57) | 96.5 (9.05)
  Week 44, n=273, 286: number analyzed (Participants) | 273 | 286
  Week 44, n=273, 286 | 89.9 (5.52) | 96.2 (9.08)
  Week 48, n=255, 284: number analyzed (Participants) | 255 | 284
  Week 48, n=255, 284 | 89.9 (5.58) | 96.2 (9.38)

14. Secondary Outcome: Absolute Values for Hematology Parameters: Erythrocytes
Description: Blood samples were collected for the analysis of hematology parameters including erythrocytes at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
10^12 cells per liter
  Baseline, n=308, 308 | 4.55 (0.563) | 4.49 (0.570)
  Week 4, n=300, 300: number analyzed (Participants) | 300 | 300
  Week 4, n=300, 300 | 4.59 (0.503) | 4.45 (0.567)
  Week 8, n=218, 301: number analyzed (Participants) | 218 | 301
  Week 8, n=218, 301 | 4.68 (0.479) | 4.49 (0.566)
  Week 12, n=294, 293: number analyzed (Participants) | 294 | 293
  Week 12, n=294, 293 | 4.79 (0.464) | 4.51 (0.580)
  Week 16, n=280, 296: number analyzed (Participants) | 280 | 296
  Week 16, n=280, 296 | 4.84 (0.475) | 4.48 (0.549)
  Week 20, n=276, 298: number analyzed (Participants) | 276 | 298
  Week 20, n=276, 298 | 4.86 (0.459) | 4.48 (0.586)
  Week 24, n=279, 294: number analyzed (Participants) | 279 | 294
  Week 24, n=279, 294 | 4.86 (0.471) | 4.48 (0.572)
  Week 28, n=268, 297: number analyzed (Participants) | 268 | 297
  Week 28, n=268, 297 | 4.85 (0.456) | 4.47 (0.565)
  Week 32, n=268, 291: number analyzed (Participants) | 268 | 291
  Week 32, n=268, 291 | 4.84 (0.452) | 4.48 (0.550)
  Week 36, n=267, 288: number analyzed (Participants) | 267 | 288
  Week 36, n=267, 288 | 4.81 (0.462) | 4.49 (0.561)
  Week 40, n=264, 289: number analyzed (Participants) | 264 | 289
  Week 40, n=264, 289 | 4.84 (0.456) | 4.49 (0.572)
  Week 44, n=273, 286: number analyzed (Participants) | 273 | 286
  Week 44, n=273, 286 | 4.86 (0.448) | 4.49 (0.572)
  Week 48, n=255, 284: number analyzed (Participants) | 255 | 284
  Week 48, n=255, 284 | 4.81 (0.448) | 4.50 (0.600)

15. Secondary Outcome: Absolute Values for Hematology Parameters: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter including hemoglobin at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Grams per liter
  Baseline, n=308, 308 | 142.2 (17.24) | 141.4 (16.29)
  Week 4, n=300, 300: number analyzed (Participants) | 300 | 300
  Week 4, n=300, 300 | 141.7 (16.30) | 140.5 (16.44)
  Week 8, n=218, 301: number analyzed (Participants) | 218 | 301
  Week 8, n=218, 301 | 141.5 (16.08) | 141.2 (16.51)
  Week 12, n=294, 293: number analyzed (Participants) | 294 | 293
  Week 12, n=294, 293 | 142.4 (15.90) | 141.6 (16.62)
  Week 16, n=280, 296: number analyzed (Participants) | 280 | 296
  Week 16, n=280, 296 | 142.5 (16.19) | 140.5 (15.81)
  Week 20, n=276, 298: number analyzed (Participants) | 276 | 298
  Week 20, n=276, 298 | 142.6 (15.52) | 141.2 (16.62)
  Week 24, n=279, 294: number analyzed (Participants) | 279 | 294
  Week 24, n=279, 294 | 143.3 (15.66) | 141.6 (16.18)
  Week 28, n=268, 297: number analyzed (Participants) | 268 | 297
  Week 28, n=268, 297 | 142.8 (16.05) | 140.9 (15.89)
  Week 32, n=268, 291: number analyzed (Participants) | 268 | 291
  Week 32, n=268, 291 | 143.0 (15.42) | 141.8 (15.81)
  Week 36, n=267, 288: number analyzed (Participants) | 267 | 288
  Week 36, n=267, 288 | 142.7 (16.31) | 142.3 (15.72)
  Week 40, n=264, 289: number analyzed (Participants) | 264 | 289
  Week 40, n=264, 289 | 143.5 (15.80) | 142.4 (15.90)
  Week 44, n=273, 286: number analyzed (Participants) | 273 | 286
  Week 44, n=273, 286 | 143.6 (15.66) | 142.1 (16.38)
  Week 48, n=255, 284: number analyzed (Participants) | 255 | 284
  Week 48, n=255, 284 | 142.7 (15.93) | 142.8 (16.34)

16. Secondary Outcome: Absolute Values for Hematology Parameters: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameters including hematocrit at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Proportion of red blood cells in blood
  Baseline, n=308, 308 | 0.4333 (0.04804) | 0.4305 (0.04454)
  Week 4, n=300, 300: number analyzed (Participants) | 300 | 300
  Week 4, n=300, 300 | 0.4325 (0.04570) | 0.4283 (0.04548)
  Week 8, n=218, 301: number analyzed (Participants) | 218 | 301
  Week 8, n=218, 301 | 0.4327 (0.04570) | 0.4310 (0.04580)
  Week 12, n=294, 293: number analyzed (Participants) | 294 | 293
  Week 12, n=294, 293 | 0.4379 (0.04483) | 0.4338 (0.04640)
  Week 16, n=280, 296: number analyzed (Participants) | 280 | 296
  Week 16, n=280, 296 | 0.4369 (0.04626) | 0.4304 (0.04418)
  Week 20, n=276, 298: number analyzed (Participants) | 276 | 298
  Week 20, n=276, 298 | 0.4378 (0.04476) | 0.4312 (0.04755)
  Week 24, n=279, 294: number analyzed (Participants) | 279 | 294
  Week 24, n=279, 294 | 0.4376 (0.04589) | 0.4312 (0.04595)
  Week 28, n=268, 297: number analyzed (Participants) | 268 | 297
  Week 28, n=268, 297 | 0.4364 (0.04607) | 0.4308 (0.04555)
  Week 32, n=268, 291: number analyzed (Participants) | 268 | 291
  Week 32, n=268, 291 | 0.4350 (0.04311) | 0.4299 (0.04431)
  Week 36, n=267, 288: number analyzed (Participants) | 267 | 288
  Week 36, n=267, 288 | 0.4311 (0.04462) | 0.4295 (0.04348)
  Week 40, n=264, 289: number analyzed (Participants) | 264 | 289
  Week 40, n=264, 289 | 0.4342 (0.04381) | 0.4300 (0.04449)
  Week 44, n=273, 286: number analyzed (Participants) | 273 | 286
  Week 44, n=273, 286 | 0.4357 (0.04288) | 0.4282 (0.04472)
  Week 48, n=255, 284: number analyzed (Participants) | 255 | 284
  Week 48, n=255, 284 | 0.4318 (0.04438) | 0.4286 (0.04465)

17. Secondary Outcome: Change From Baseline for Hematology Parameters: Basophil, Eosinophils, Leukocytes, Lymphocytes, Neutrophils, Monocytes, and Platelets
Description: Blood samples were collected for the analysis of hematology parameters including basophil, eosinophils, leukocytes, lymphocytes, neutrophils, monocytes, and platelets at indicated timepoints. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^9 cells per liters
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
10^9 cells per liters
  Basophils, Week 4, n=299, 290: number analyzed (Participants) | 299 | 290
  Basophils, Week 4, n=299, 290 | 0.003 (0.0202) | 0.003 (0.0185)
  Basophils, Week 8, n=216, 293: number analyzed (Participants) | 216 | 293
  Basophils, Week 8, n=216, 293 | 0.003 (0.0204) | 0.000 (0.0181)
  Basophils, Week 12, n=293, 289: number analyzed (Participants) | 293 | 289
  Basophils, Week 12, n=293, 289 | 0.002 (0.0205) | 0.001 (0.0197)
  Basophils, Week 16, n=274, 291: number analyzed (Participants) | 274 | 291
  Basophils, Week 16, n=274, 291 | 0.001 (0.0186) | 0.001 (0.0181)
  Basophils, Week 20, n=273, 291: number analyzed (Participants) | 273 | 291
  Basophils, Week 20, n=273, 291 | 0.002 (0.0225) | 0.002 (0.0212)
  Basophils, Week 24, n=277, 291: number analyzed (Participants) | 277 | 291
  Basophils, Week 24, n=277, 291 | 0.002 (0.0169) | 0.003 (0.0167)
  Basophils, Week 28, n=266, 294: number analyzed (Participants) | 266 | 294
  Basophils, Week 28, n=266, 294 | 0.003 (0.0200) | 0.002 (0.0181)
  Basophils, Week 32, n=262, 282: number analyzed (Participants) | 262 | 282
  Basophils, Week 32, n=262, 282 | 0.005 (0.0199) | 0.003 (0.0189)
  Basophils, Week 36, n=260, 281: number analyzed (Participants) | 260 | 281
  Basophils, Week 36, n=260, 281 | 0.009 (0.0231) | 0.007 (0.0217)
  Basophils, Week 40, n=258, 279: number analyzed (Participants) | 258 | 279
  Basophils, Week 40, n=258, 279 | 0.014 (0.0292) | 0.011 (0.0233)
  Basophils, Week 44, n=258, 267: number analyzed (Participants) | 258 | 267
  Basophils, Week 44, n=258, 267 | 0.017 (0.0283) | 0.012 (0.0239)
  Basophils, Week 48, n=246, 273: number analyzed (Participants) | 246 | 273
  Basophils, Week 48, n=246, 273 | 0.019 (0.0273) | 0.018 (0.0263)
  Eosinophils, Week 4, n=299, 290: number analyzed (Participants) | 299 | 290
  Eosinophils, Week 4, n=299, 290 | 0.026 (0.1394) | 0.009 (0.1409)
  Eosinophils, Week 8, n=216, 293: number analyzed (Participants) | 216 | 293
  Eosinophils, Week 8, n=216, 293 | 0.015 (0.1278) | -0.008 (0.1319)
  Eosinophils, Week 12, n=293, 289: number analyzed (Participants) | 293 | 289
  Eosinophils, Week 12, n=293, 289 | -0.003 (0.1155) | -0.010 (0.1533)
  Eosinophils, Week 16, n=274, 291: number analyzed (Participants) | 274 | 291
  Eosinophils, Week 16, n=274, 291 | 0.009 (0.1246) | -0.011 (0.1759)
  Eosinophils, Week 20, n=273, 291: number analyzed (Participants) | 273 | 291
  Eosinophils, Week 20, n=273, 291 | 0.009 (0.1410) | -0.027 (0.1352)
  Eosinophils, Week 24, n=277, 291: number analyzed (Participants) | 277 | 291
  Eosinophils, Week 24, n=277, 291 | 0.002 (0.1228) | -0.021 (0.1490)
  Eosinophils, Week 28, n=266, 294: number analyzed (Participants) | 266 | 294
  Eosinophils, Week 28, n=266, 294 | -0.002 (0.1298) | -0.011 (0.1387)
  Eosinophils, Week 32, n=262, 282: number analyzed (Participants) | 262 | 282
  Eosinophils, Week 32, n=262, 282 | 0.022 (0.1629) | -0.012 (0.1511)
  Eosinophils, Week 36, n=260, 281: number analyzed (Participants) | 260 | 281
  Eosinophils, Week 36, n=260, 281 | 0.002 (0.1413) | -0.012 (0.1382)
  Eosinophils, Week 40, n=258, 279: number analyzed (Participants) | 258 | 279
  Eosinophils, Week 40, n=258, 279 | 0.019 (0.1319) | -0.006 (0.1283)
  Eosinophils, Week 44, n=258, 267: number analyzed (Participants) | 258 | 267
  Eosinophils, Week 44, n=258, 267 | 0.032 (0.1388) | -0.004 (0.1061)
  Eosinophils, Week 48, n=246, 273: number analyzed (Participants) | 246 | 273
  Eosinophils, Week 48, n=246, 273 | 0.032 (0.1321) | 0.002 (0.1253)
  Leukocytes, Week 4, n=300, 297: number analyzed (Participants) | 300 | 297
  Leukocytes, Week 4, n=300, 297 | 0.54 (1.599) | 0.13 (1.544)
  Leukocytes, Week 8, n=217, 300: number analyzed (Participants) | 217 | 300
  Leukocytes, Week 8, n=217, 300 | 0.19 (1.579) | -0.02 (1.548)
  Leukocytes, Week 12, n=294, 292: number analyzed (Participants) | 294 | 292
  Leukocytes, Week 12, n=294, 292 | 0.35 (1.743) | 0.10 (1.571)
  Leukocytes, Week 16, n=279, 294: number analyzed (Participants) | 279 | 294
  Leukocytes, Week 16, n=279, 294 | 0.34 (1.653) | 0.17 (1.558)
  Leukocytes, Week 20, n=276, 297: number analyzed (Participants) | 276 | 297
  Leukocytes, Week 20, n=276, 297 | 0.46 (1.565) | 0.04 (1.529)
  Leukocytes, Week 24, n=279, 293: number analyzed (Participants) | 279 | 293
  Leukocytes, Week 24, n=279, 293 | 0.32 (1.720) | 0.10 (1.661)
  Leukocytes, Week 28, n=268, 296: number analyzed (Participants) | 268 | 296
  Leukocytes, Week 28, n=268, 296 | 0.25 (1.651) | 0.07 (1.471)
  Leukocytes, Week 32, n=267, 287: number analyzed (Participants) | 267 | 287
  Leukocytes, Week 32, n=267, 287 | 0.43 (1.602) | 0.07 (1.631)
  Leukocytes, Week 36, n=264, 284: number analyzed (Participants) | 264 | 284
  Leukocytes, Week 36, n=264, 284 | 0.33 (1.699) | 0.13 (1.821)
  Leukocytes, Week 40, n=264, 285: number analyzed (Participants) | 264 | 285
  Leukocytes, Week 40, n=264, 285 | 0.35 (1.808) | 0.12 (1.675)
  Leukocytes, Week 44, n=269, 278: number analyzed (Participants) | 269 | 278
  Leukocytes, Week 44, n=269, 278 | 0.22 (1.581) | -0.03 (1.561)
  Leukocytes, Week 48, n=252, 281: number analyzed (Participants) | 252 | 281
  Leukocytes, Week 48, n=252, 281 | 0.09 (1.646) | -0.06 (1.538)
  Lymphocytes, Week 4, n=299, 290: number analyzed (Participants) | 299 | 290
  Lymphocytes, Week 4, n=299, 290 | 0.174 (0.5185) | 0.128 (0.5618)
  Lymphocytes, Week 8, n=216, 293: number analyzed (Participants) | 216 | 293
  Lymphocytes, Week 8, n=216, 293 | 0.068 (0.5319) | 0.023 (0.5250)
  Lymphocytes, Week 12, n=293, 289: number analyzed (Participants) | 293 | 289
  Lymphocytes, Week 12, n=293, 289 | 0.033 (0.5073) | 0.079 (0.5844)
  Lymphocytes, Week 16, n=274, 291: number analyzed (Participants) | 274 | 291
  Lymphocytes, Week 16, n=274, 291 | 0.114 (0.5596) | 0.095 (0.5389)
  Lymphocytes, Week 20, n=273, 291: number analyzed (Participants) | 273 | 291
  Lymphocytes, Week 20, n=273, 291 | 0.071 (0.5274) | 0.086 (0.5411)
  Lymphocytes, Week 24, n=277, 291: number analyzed (Participants) | 277 | 291
  Lymphocytes, Week 24, n=277, 291 | 0.079 (0.5408) | 0.049 (0.4863)
  Lymphocytes, Week 28, n=266, 294: number analyzed (Participants) | 266 | 294
  Lymphocytes, Week 28, n=266, 294 | 0.101 (0.6133) | 0.069 (0.6005)
  Lymphocytes, Week 32, n=262, 282: number analyzed (Participants) | 262 | 282
  Lymphocytes, Week 32, n=262, 282 | 0.063 (0.5392) | 0.064 (0.5757)
  Lymphocytes, Week 36, n=260, 281: number analyzed (Participants) | 260 | 281
  Lymphocytes, Week 36, n=260, 281 | 0.008 (0.5333) | 0.036 (0.5525)
  Lymphocytes, Week 40, n=258, 279: number analyzed (Participants) | 258 | 279
  Lymphocytes, Week 40, n=258, 279 | 0.020 (0.5171) | 0.035 (0.5280)
  Lymphocytes, Week 44, n=258, 267: number analyzed (Participants) | 258 | 267
  Lymphocytes, Week 44, n=258, 267 | 0.045 (0.5430) | 0.045 (0.5472)
  Lymphocytes, Week 48, n=246, 273: number analyzed (Participants) | 246 | 273
  Lymphocytes, Week 48, n=246, 273 | -0.063 (0.5528) | -0.035 (0.5115)
  Neutrophils, Week 4, n=299, 290: number analyzed (Participants) | 299 | 290
  Neutrophils, Week 4, n=299, 290 | 0.258 (1.5445) | 0.004 (1.3601)
  Neutrophils, Week 8, n=216, 293: number analyzed (Participants) | 216 | 293
  Neutrophils, Week 8, n=216, 293 | 0.080 (1.4401) | -0.031 (1.3599)
  Neutrophils, Week 12, n=293, 289: number analyzed (Participants) | 293 | 289
  Neutrophils, Week 12, n=293, 289 | 0.283 (1.6227) | 0.028 (1.3884)
  Neutrophils, Week 16, n=274, 291: number analyzed (Participants) | 274 | 291
  Neutrophils, Week 16, n=274, 291 | 0.181 (1.5415) | 0.080 (1.4451)
  Neutrophils, Week 20, n=273, 291: number analyzed (Participants) | 273 | 291
  Neutrophils, Week 20, n=273, 291 | 0.341 (1.4475) | -0.019 (1.4228)
  Neutrophils, Week 24, n=277, 291: number analyzed (Participants) | 277 | 291
  Neutrophils, Week 24, n=277, 291 | 0.175 (1.5883) | 0.056 (1.5091)
  Neutrophils, Week 28, n=266, 294: number analyzed (Participants) | 266 | 294
  Neutrophils, Week 28, n=266, 294 | 0.129 (1.4052) | -0.001 (1.3377)
  Neutrophils, Week 32, n=262, 282: number analyzed (Participants) | 262 | 282
  Neutrophils, Week 32, n=262, 282 | 0.291 (1.6015) | 0.008 (1.4430)
  Neutrophils, Week 36, n=260, 281: number analyzed (Participants) | 260 | 281
  Neutrophils, Week 36, n=260, 281 | 0.289 (1.5702) | 0.077 (1.6758)
  Neutrophils, Week 40, n=258, 279: number analyzed (Participants) | 258 | 279
  Neutrophils, Week 40, n=258, 279 | 0.245 (1.6621) | 0.075 (1.5336)
  Neutrophils, Week 44, n=258, 267: number analyzed (Participants) | 258 | 267
  Neutrophils, Week 44, n=258, 267 | 0.063 (1.4874) | -0.105 (1.4587)
  Neutrophils, Week 48, n=246, 273: number analyzed (Participants) | 246 | 273
  Neutrophils, Week 48, n=246, 273 | 0.009 (1.5413) | -0.066 (1.3969)
  Monocytes, Week 4, n=299, 290: number analyzed (Participants) | 299 | 290
  Monocytes, Week 4, n=299, 290 | 0.049 (0.1663) | 0.030 (0.1270)
  Monocytes Week 8, n=216, 293: number analyzed (Participants) | 216 | 293
  Monocytes Week 8, n=216, 293 | 0.014 (0.1433) | 0.018 (0.1591)
  Monocytes, Week 12, n=293, 289: number analyzed (Participants) | 293 | 289
  Monocytes, Week 12, n=293, 289 | 0.018 (0.1553) | 0.001 (0.1367)
  Monocytes, Week 16, n=274, 291: number analyzed (Participants) | 274 | 291
  Monocytes, Week 16, n=274, 291 | 0.005 (0.1588) | 0.003 (0.1403)
  Monocytes, Week 20, n=273, 291: number analyzed (Participants) | 273 | 291
  Monocytes, Week 20, n=273, 291 | 0.003 (0.1527) | 0.004 (0.1328)
  Monocytes, Week 24, n=277, 291: number analyzed (Participants) | 277 | 291
  Monocytes, Week 24, n=277, 291 | 0.012 (0.1484) | 0.002 (0.1331)
  Monocytes, Week 28, n=266, 294: number analyzed (Participants) | 266 | 294
  Monocytes, Week 28, n=266, 294 | 0.001 (0.1548) | -0.004 (0.1343)
  Monocytes, Week 32, n=262, 282: number analyzed (Participants) | 262 | 282
  Monocytes, Week 32, n=262, 282 | 0.019 (0.1535) | 0.011 (0.1585)
  Monocytes, Week 36, n=260, 281: number analyzed (Participants) | 260 | 281
  Monocytes, Week 36, n=260, 281 | 0.016 (0.1501) | 0.024 (0.1551)
  Monocytes, Week 40, n=258, 279: number analyzed (Participants) | 258 | 279
  Monocytes, Week 40, n=258, 279 | 0.039 (0.1507) | 0.020 (0.1550)
  Monocytes, Week 44, n=258, 267: number analyzed (Participants) | 258 | 267
  Monocytes, Week 44, n=258, 267 | 0.045 (0.1673) | 0.045 (0.1539)
  Monocytes, Week 48, n=246, 273: number analyzed (Participants) | 246 | 273
  Monocytes, Week 48, n=246, 273 | 0.047 (0.1502) | 0.039 (0.1499)
  Platelets, Week 4, n=300, 298: number analyzed (Participants) | 300 | 298
  Platelets, Week 4, n=300, 298 | 1.8 (38.02) | 4.3 (36.15)
  Platelets, Week 8, n=216, 298: number analyzed (Participants) | 216 | 298
  Platelets, Week 8, n=216, 298 | -5.5 (31.98) | 0.7 (35.15)
  Platelets, Week 12, n=294, 290: number analyzed (Participants) | 294 | 290
  Platelets, Week 12, n=294, 290 | -0.8 (40.83) | 5.5 (36.76)
  Platelets, Week 16, n=279, 294: number analyzed (Participants) | 279 | 294
  Platelets, Week 16, n=279, 294 | -5.2 (40.67) | 4.3 (34.61)
  Platelets, Week 20, n=274, 297: number analyzed (Participants) | 274 | 297
  Platelets, Week 20, n=274, 297 | -3.7 (36.87) | 5.5 (38.86)
  Platelets, Week 24, n=279, 292: number analyzed (Participants) | 279 | 292
  Platelets, Week 24, n=279, 292 | -4.7 (35.22) | 6.7 (41.78)
  Platelets, Week 28, n=268, 295: number analyzed (Participants) | 268 | 295
  Platelets, Week 28, n=268, 295 | -5.3 (35.22) | 5.4 (38.41)
  Platelets, Week 32, n=267, 289: number analyzed (Participants) | 267 | 289
  Platelets, Week 32, n=267, 289 | -2.6 (36.51) | 6.5 (35.99)
  Platelets, Week 36, n=267, 284: number analyzed (Participants) | 267 | 284
  Platelets, Week 36, n=267, 284 | -1.2 (37.26) | 9.8 (44.52)
  Platelets, Week 40, n=263, 288: number analyzed (Participants) | 263 | 288
  Platelets, Week 40, n=263, 288 | 0.0 (40.74) | 9.7 (39.91)
  Platelets, Week 44, n=270, 286: number analyzed (Participants) | 270 | 286
  Platelets, Week 44, n=270, 286 | 4.5 (38.31) | 9.2 (42.82)
  Platelets, Week 48, n=253, 281: number analyzed (Participants) | 253 | 281
  Platelets, Week 48, n=253, 281 | 0.0 (38.63) | 10.4 (41.75)

18. Secondary Outcome: Change From Baseline for Hematology Parameters: Erythrocyte Mean Corpuscular Volume
Description: Blood samples were collected for the analysis of hematology parameter including erythrocyte mean corpuscular volume at indicated timepoints. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Femtoliters
  Week 4, n=300, 300: number analyzed (Participants) | 300 | 300
  Week 4, n=300, 300 | -1.1 (2.71) | 0.2 (1.82)
  Week 8, n=218, 301: number analyzed (Participants) | 218 | 301
  Week 8, n=218, 301 | -3.0 (4.30) | 0.1 (1.76)
  Week 12, n=294, 293: number analyzed (Participants) | 294 | 293
  Week 12, n=294, 293 | -3.9 (5.23) | 0.2 (2.08)
  Week 16, n=280, 296: number analyzed (Participants) | 280 | 296
  Week 16, n=280, 296 | -4.9 (5.86) | 0.2 (2.42)
  Week 20, n=276, 298: number analyzed (Participants) | 276 | 298
  Week 20, n=276, 298 | -5.3 (5.98) | 0.3 (2.88)
  Week 24, n=279, 294: number analyzed (Participants) | 279 | 294
  Week 24, n=279, 294 | -5.4 (5.97) | 0.3 (3.24)
  Week 28, n=268, 297: number analyzed (Participants) | 268 | 297
  Week 28, n=268, 297 | -5.5 (6.11) | 0.4 (3.46)
  Week 32, n=268, 291: number analyzed (Participants) | 268 | 291
  Week 32, n=268, 291 | -5.5 (6.10) | 0.1 (3.47)
  Week 36, n=267, 288: number analyzed (Participants) | 267 | 288
  Week 36, n=267, 288 | -5.8 (6.24) | -0.0 (3.69)
  Week 40, n=264, 289: number analyzed (Participants) | 264 | 289
  Week 40, n=264, 289 | -5.6 (6.21) | -0.1 (3.62)
  Week 44, n=273, 286: number analyzed (Participants) | 273 | 286
  Week 44, n=273, 286 | -5.8 (6.33) | -0.3 (3.68)
  Week 48, n=255, 284: number analyzed (Participants) | 255 | 284
  Week 48, n=255, 284 | -5.7 (6.76) | -0.4 (3.57)

19. Secondary Outcome: Change From Baseline for Hematology Parameters: Erythrocytes
Description: Blood samples were collected for the analysis of hematology parameters including erythrocytes at indicated timepoints. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
10^12 cells per liter
  Week 4, n=300, 300: number analyzed (Participants) | 300 | 300
  Week 4, n=300, 300 | 0.04 (0.255) | -0.03 (0.226)
  Week 8, n=218, 301: number analyzed (Participants) | 218 | 301
  Week 8, n=218, 301 | 0.14 (0.331) | -0.01 (0.249)
  Week 12, n=294, 293: number analyzed (Participants) | 294 | 293
  Week 12, n=294, 293 | 0.23 (0.374) | 0.01 (0.252)
  Week 16, n=280, 296: number analyzed (Participants) | 280 | 296
  Week 16, n=280, 296 | 0.28 (0.380) | -0.01 (0.256)
  Week 20, n=276, 298: number analyzed (Participants) | 276 | 298
  Week 20, n=276, 298 | 0.30 (0.408) | -0.01 (0.273)
  Week 24, n=279, 294: number analyzed (Participants) | 279 | 294
  Week 24, n=279, 294 | 0.32 (0.397) | -0.01 (0.246)
  Week 28, n=268, 297: number analyzed (Participants) | 268 | 297
  Week 28, n=268, 297 | 0.28 (0.386) | -0.01 (0.246)
  Week 32, n=268, 291: number analyzed (Participants) | 268 | 291
  Week 32, n=268, 291 | 0.29 (0.393) | -0.01 (0.261)
  Week 36, n=267, 288: number analyzed (Participants) | 267 | 288
  Week 36, n=267, 288 | 0.26 (0.401) | -0.01 (0.259)
  Week 40, n=264, 289: number analyzed (Participants) | 264 | 289
  Week 40, n=264, 289 | 0.27 (0.396) | -0.01 (0.260)
  Week 44, n=273, 286: number analyzed (Participants) | 273 | 286
  Week 44, n=273, 286 | 0.31 (0.391) | -0.01 (0.264)
  Week 48, n=255, 284: number analyzed (Participants) | 255 | 284
  Week 48, n=255, 284 | 0.25 (0.394) | -0.01 (0.262)

20. Secondary Outcome: Change From Baseline for Hematology Parameters: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameters including hematocrit at indicated timepoints. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Proportion of red blood cells in blood
  Week 4, n=300, 300: number analyzed (Participants) | 300 | 300
  Week 4, n=300, 300 | -0.0003 (0.02236) | -0.0023 (0.02194)
  Week 8, n=218, 301: number analyzed (Participants) | 218 | 301
  Week 8, n=218, 301 | 0.0007 (0.02613) | -0.0005 (0.02330)
  Week 12, n=294, 293: number analyzed (Participants) | 294 | 293
  Week 12, n=294, 293 | 0.0042 (0.02607) | 0.0020 (0.02408)
  Week 16, n=280, 296: number analyzed (Participants) | 280 | 296
  Week 16, n=280, 296 | 0.0038 (0.02509) | -0.0007 (0.02513)
  Week 20, n=276, 298: number analyzed (Participants) | 276 | 298
  Week 20, n=276, 298 | 0.0043 (0.02742) | 0.0002 (0.02613)
  Week 24, n=279, 294: number analyzed (Participants) | 279 | 294
  Week 24, n=279, 294 | 0.0052 (0.02790) | 0.0002 (0.02576)
  Week 28, n=268, 297: number analyzed (Participants) | 268 | 297
  Week 28, n=268, 297 | 0.0023 (0.02699) | 0.0002 (0.02603)
  Week 32, n=268, 291: number analyzed (Participants) | 268 | 291
  Week 32, n=268, 291 | 0.0022 (0.02872) | -0.0011 (0.02916)
  Week 36, n=267, 288: number analyzed (Participants) | 267 | 288
  Week 36, n=267, 288 | -0.0012 (0.02793) | -0.0011 (0.02797)
  Week 40, n=264, 289: number analyzed (Participants) | 264 | 289
  Week 40, n=264, 289 | -0.0001 (0.02741) | -0.0011 (0.02781)
  Week 44, n=273, 286: number analyzed (Participants) | 273 | 286
  Week 44, n=273, 286 | 0.0031 (0.02896) | -0.0025 (0.02814)
  Week 48, n=255, 284: number analyzed (Participants) | 255 | 284
  Week 48, n=255, 284 | -0.0021 (0.02717) | -0.0031 (0.02700)

21. Secondary Outcome: Change From Baseline for Hematology Parameters: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter including hemoglobin at indicated timepoints. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Grams per liter
  Week 4, n=300, 300: number analyzed (Participants) | 300 | 300
  Week 4, n=300, 300 | -0.4 (6.91) | -1.0 (6.73)
  Week 8, n=218, 301: number analyzed (Participants) | 218 | 301
  Week 8, n=218, 301 | -0.4 (8.18) | -0.6 (7.33)
  Week 12, n=294, 293: number analyzed (Participants) | 294 | 293
  Week 12, n=294, 293 | 0.0 (8.14) | -0.3 (7.52)
  Week 16, n=280, 296: number analyzed (Participants) | 280 | 296
  Week 16, n=280, 296 | 0.4 (8.22) | -1.2 (7.75)
  Week 20, n=276, 298: number analyzed (Participants) | 276 | 298
  Week 20, n=276, 298 | 0.3 (8.60) | -0.5 (8.55)
  Week 24, n=279, 294: number analyzed (Participants) | 279 | 294
  Week 24, n=279, 294 | 1.2 (8.78) | -0.0 (8.46)
  Week 28, n=268, 297: number analyzed (Participants) | 268 | 297
  Week 28, n=268, 297 | 0.3 (8.49) | -0.6 (8.68)
  Week 32, n=268, 291: number analyzed (Participants) | 268 | 291
  Week 32, n=268, 291 | 0.9 (8.94) | 0.2 (9.45)
  Week 36, n=267, 288: number analyzed (Participants) | 267 | 288
  Week 36, n=267, 288 | 0.7 (9.03) | 0.8 (9.32)
  Week 40, n=264, 289: number analyzed (Participants) | 264 | 289
  Week 40, n=264, 289 | 0.8 (8.96) | 0.7 (9.29)
  Week 44, n=273, 286: number analyzed (Participants) | 273 | 286
  Week 44, n=273, 286 | 1.7 (9.49) | 0.6 (9.53)
  Week 48, n=255, 284: number analyzed (Participants) | 255 | 284
  Week 48, n=255, 284 | 0.2 (9.26) | 0.9 (9.07)

22. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Over Time Including Week 48: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Creatinine Kinase (CK)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALT, ALP, AST and CK at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
International units per liter
  ALT, Baseline (Day 1), n=308, 308 | 23.8 (13.47) | 22.4 (12.90)
  ALT, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  ALT, Week 4, n=301, 303 | 24.4 (15.60) | 22.3 (11.10)
  ALT, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  ALT, Week 8, n=229, 303 | 24.0 (16.85) | 24.0 (29.86)
  ALT, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  ALT, Week 12, n=295, 299 | 29.0 (114.25) | 22.7 (13.48)
  ALT, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  ALT, Week 16, n=284, 298 | 23.7 (22.32) | 21.8 (11.31)
  ALT, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  ALT, Week 20, n=277, 302 | 23.1 (22.49) | 21.2 (10.50)
  ALT, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  ALT, Week 24, n=284, 299 | 26.3 (62.05) | 21.6 (12.64)
  ALT, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  ALT, Week 28, n=267, 296 | 21.1 (12.13) | 22.1 (14.62)
  ALT, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  ALT, Week 32, n=275, 294 | 21.8 (12.56) | 21.8 (12.09)
  ALT, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  ALT, Week 36, n=273, 292 | 23.2 (24.94) | 22.3 (12.17)
  ALT, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  ALT, Week 40, n=270, 293 | 24.5 (37.39) | 22.1 (12.78)
  ALT, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  ALT, Week 44, n=275, 293 | 21.6 (13.10) | 22.1 (13.67)
  ALT, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  ALT, Week 48, n=265, 292 | 21.8 (13.54) | 21.7 (11.08)
  ALP, Baseline (Day 1), n=308, 308 | 76.6 (28.20) | 77.5 (26.77)
  ALP, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  ALP, Week 4, n=301, 303 | 70.4 (22.75) | 75.7 (25.58)
  ALP, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  ALP, Week 8, n=229, 303 | 68.9 (21.98) | 78.8 (32.40)
  ALP, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  ALP, Week 12, n=295, 299 | 68.9 (24.79) | 78.6 (28.87)
  ALP, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  ALP, Week 16, n=284, 298 | 67.9 (19.76) | 77.3 (27.21)
  ALP, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  ALP, Week 20, n=277, 302 | 67.6 (18.72) | 76.7 (25.48)
  ALP, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  ALP, Week 24, n=284, 299 | 68.1 (19.15) | 77.5 (26.36)
  ALP, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  ALP, Week 28, n=267, 296 | 67.6 (18.89) | 77.2 (26.72)
  ALP, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  ALP, Week 32, n=275, 294 | 66.6 (19.14) | 75.8 (25.56)
  ALP, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  ALP, Week 36, n=273, 292 | 66.8 (20.68) | 76.4 (25.93)
  ALP, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  ALP, Week 40, n=270, 293 | 66.2 (17.58) | 76.2 (26.08)
  ALP, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  ALP, Week 44, n=275, 293 | 66.1 (18.34) | 76.8 (25.82)
  ALP, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  ALP, Week 48, n=265, 292 | 66.5 (18.84) | 77.1 (26.39)
  AST, Baseline (Day 1), n=308, 308 | 23.9 (11.31) | 22.5 (10.21)
  AST, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  AST, Week 4, n=301, 303 | 23.2 (11.77) | 22.7 (10.93)
  AST, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  AST, Week 8, n=229, 303 | 24.3 (19.49) | 22.5 (12.31)
  AST, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  AST, Week 12, n=295, 299 | 26.1 (64.69) | 23.2 (10.61)
  AST, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  AST, Week 16, n=284, 298 | 24.1 (18.20) | 22.5 (8.59)
  AST, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  AST, Week 20, n=277, 302 | 23.5 (15.23) | 22.0 (6.83)
  AST, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  AST, Week 24, n=284, 298 | 24.2 (22.89) | 22.5 (9.30)
  AST, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  AST, Week 28, n=267, 296 | 22.2 (8.72) | 22.9 (9.61)
  AST, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  AST, Week 32, n=275, 294 | 22.8 (13.71) | 23.2 (12.32)
  AST, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  AST, Week 36, n=273, 292 | 23.0 (11.27) | 22.6 (7.18)
  AST, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  AST, Week 40, n=270, 293 | 23.8 (14.96) | 22.5 (7.79)
  AST, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  AST, Week 44, n=275, 293 | 22.9 (14.82) | 22.6 (10.26)
  AST Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  AST Week 48, n=265, 292 | 22.9 (10.35) | 23.2 (9.30)
  CK, Baseline (Day 1), n=308, 308 | 196.6 (367.30) | 160.8 (367.57)
  CK, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  CK, Week 4, n=301, 303 | 192.9 (437.09) | 190.6 (472.57)
  CK, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  CK, Week 8, n=229, 303 | 275.9 (1064.72) | 145.4 (141.19)
  CK, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  CK, Week 12, n=295, 299 | 200.7 (484.08) | 177.0 (321.29)
  CK, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  CK, Week 16, n=284, 298 | 253.5 (849.45) | 167.5 (286.90)
  CK, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  CK, Week 20, n=277, 302 | 228.4 (570.80) | 144.5 (133.32)
  CK, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  CK, Week 24, n=284, 299 | 193.1 (444.27) | 161.2 (241.73)
  CK, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  CK, Week 28, n=267, 296 | 168.8 (163.54) | 182.7 (420.44)
  CK, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  CK, Week 32, n=275, 294 | 216.5 (593.10) | 195.9 (489.99)
  CK, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  CK, Week 36, n=273, 292 | 186.4 (325.64) | 150.7 (134.40)
  CK, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  CK, Week 40, n=270, 293 | 235.1 (624.03) | 160.7 (179.64)
  CK, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  CK, Week 44, n=275, 293 | 245.5 (1189.35) | 149.9 (148.23)
  CK, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  CK, Week 48, n=265, 292 | 198.8 (398.14) | 179.0 (331.51)

23. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter Over Time Including Week 48: Albumin
Description: Blood samples were collected for the analysis of clinical chemistry parameter-albumin at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Grams per liter
  Baseline (Day 1), n=308, 308 | 44.2 (3.12) | 44.3 (3.19)
  Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Week 4, n=301, 303 | 43.7 (2.88) | 43.8 (2.87)
  Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Week 8, n=229, 303 | 43.8 (3.06) | 43.7 (3.17)
  Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Week 12, n=295, 299 | 43.6 (2.99) | 43.9 (3.12)
  Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Week 16, n=284, 298 | 43.5 (2.77) | 43.5 (3.12)
  Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Week 20, n=277, 302 | 43.4 (2.72) | 43.5 (3.07)
  Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Week 24, n=284, 299 | 43.4 (2.74) | 43.5 (3.02)
  Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Week 28, n=267, 296 | 43.6 (2.85) | 43.3 (3.07)
  Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Week 32, n=275, 294 | 43.5 (2.83) | 43.4 (3.25)
  Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Week 36, n=273, 292 | 43.3 (2.82) | 43.4 (3.07)
  Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Week 40, n=270, 293 | 43.7 (2.72) | 43.4 (3.04)
  Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Week 44, n=275, 293 | 43.7 (2.78) | 43.5 (3.02)
  Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Week 48, n=265, 292 | 43.8 (2.74) | 44.0 (2.92)

24. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Over Time Including Week 48: Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters including bilirubin, creatinine and direct bilirubin at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Micromoles per liter
  Bilirubin, Baseline (Day 1), n=308, 308 | 9.9 (9.71) | 9.2 (6.39)
  Bilirubin, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Bilirubin, Week 4, n=301, 303 | 9.1 (3.98) | 8.9 (6.14)
  Bilirubin, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Bilirubin, Week 8, n=229, 303 | 9.3 (4.05) | 9.4 (9.06)
  Bilirubin, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Bilirubin, Week 12, n=295, 299 | 9.3 (4.45) | 9.3 (6.62)
  Bilirubin, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Bilirubin, Week 16, n=284, 298 | 10.0 (10.71) | 9.1 (6.28)
  Bilirubin, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Bilirubin, Week 20, n=277, 302 | 9.7 (4.28) | 9.3 (7.56)
  Bilirubin, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  Bilirubin, Week 24, n=284, 298 | 9.3 (3.90) | 9.4 (8.38)
  Bilirubin, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Bilirubin, Week 28, n=267, 296 | 9.8 (3.99) | 9.1 (7.05)
  Bilirubin, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Bilirubin, Week 32, n=275, 294 | 9.8 (4.36) | 9.3 (7.05)
  Bilirubin, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Bilirubin, Week 36, n=273, 292 | 9.3 (3.79) | 9.2 (7.34)
  Bilirubin, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Bilirubin, Week 40, n=270, 293 | 9.6 (4.07) | 9.5 (9.04)
  Bilirubin, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Bilirubin, Week 44, n=275, 293 | 9.6 (4.19) | 9.7 (8.49)
  Bilirubin, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Bilirubin, Week 48, n=265, 292 | 9.7 (4.24) | 9.5 (6.36)
  Direct bilirubin, Baseline (Day 1), n=308, 308 | 2.4 (1.35) | 2.2 (1.25)
  Direct bilirubin, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Direct bilirubin, Week 4, n=301, 303 | 2.3 (1.04) | 2.3 (1.27)
  Direct bilirubin, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Direct bilirubin, Week 8, n=229, 303 | 2.3 (1.08) | 2.4 (3.96)
  Direct bilirubin, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Direct bilirubin, Week 12, n=295, 299 | 2.2 (1.03) | 2.3 (1.30)
  Direct bilirubin, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Direct bilirubin, Week 16, n=284, 298 | 2.5 (4.98) | 2.1 (1.08)
  Direct bilirubin, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Direct bilirubin, Week 20, n=277, 302 | 2.2 (0.95) | 2.0 (1.31)
  Direct bilirubin, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  Direct bilirubin, Week 24, n=284, 298 | 2.2 (0.99) | 2.1 (1.26)
  Direct bilirubin, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Direct bilirubin, Week 28, n=267, 296 | 2.1 (0.94) | 2.0 (1.28)
  Direct bilirubin, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Direct bilirubin, Week 32, n=275, 294 | 2.1 (1.00) | 2.0 (1.22)
  Direct bilirubin, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Direct bilirubin, Week 36, n=273, 292 | 2.1 (1.11) | 2.1 (1.27)
  Direct bilirubin, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Direct bilirubin, Week 40, n=270, 293 | 2.1 (1.08) | 2.1 (1.37)
  Direct bilirubin, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Direct bilirubin, Week 44, n=275, 293 | 2.2 (0.95) | 2.2 (1.30)
  Direct bilirubin, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Direct bilirubin, Week 48, n=265, 292 | 2.2 (0.92) | 2.2 (1.23)
  Creatinine, Baseline (Day 1), n=308, 308 | 79.05 (16.380) | 77.83 (16.497)
  Creatinine, Week 4, n=301, 301: number analyzed (Participants) | 301 | 301
  Creatinine, Week 4, n=301, 301 | 80.17 (15.464) | 79.47 (16.284)
  Creatinine, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Creatinine, Week 8, n=229, 303 | 78.79 (16.122) | 79.22 (16.824)
  Creatinine, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Creatinine, Week 12, n=295, 299 | 78.65 (16.534) | 79.50 (17.191)
  Creatinine, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Creatinine, Week 16, n=284, 298 | 78.72 (15.606) | 79.51 (17.171)
  Creatinine, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Creatinine, Week 20, n=277, 302 | 79.75 (15.695) | 79.62 (16.909)
  Creatinine, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  Creatinine, Week 24, n=284, 298 | 80.15 (18.478) | 79.05 (16.673)
  Creatinine, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Creatinine, Week 28, n=267, 296 | 80.42 (16.335) | 79.35 (16.574)
  Creatinine, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Creatinine, Week 32, n=275, 294 | 79.65 (15.044) | 79.69 (16.634)
  Creatinine, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Creatinine, Week 36, n=273, 292 | 79.73 (15.994) | 79.34 (16.527)
  Creatinine, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Creatinine, Week 40, n=270, 293 | 80.28 (15.856) | 79.42 (16.856)
  Creatinine, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Creatinine, Week 44, n=275, 293 | 79.98 (15.775) | 79.16 (16.583)
  Creatinine, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Creatinine, Week 48, n=265, 292 | 80.77 (16.456) | 78.65 (16.204)

25. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters: Total Carbon-dioxide (CO2), Chloride, Glucose, Phosphate, Potassium, Sodium and Urea Over Time Including Week 48
Description: Blood samples were collected for the analysis of clinical chemistry parameters which includes total CO2, chloride, glucose, phosphate, potassium, sodium and urea at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Millimoles per liter
  CO2, Baseline (Day 1), n=308, 308 | 22.7 (2.33) | 22.6 (2.24)
  CO2, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  CO2, Week 4, n=301, 303 | 23.7 (2.49) | 23.3 (2.27)
  CO2, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  CO2, Week 8, n=229, 303 | 23.1 (2.17) | 23.2 (2.47)
  CO2, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  CO2, Week 12, n=295, 299 | 23.2 (2.14) | 23.0 (2.36)
  CO2, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  CO2, Week 16, n=284, 298 | 22.9 (2.16) | 23.0 (2.31)
  CO2, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  CO2, Week 20, n=277, 302 | 22.9 (2.16) | 22.9 (2.29)
  CO2, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  CO2, Week 24, n=284, 298 | 22.9 (2.31) | 22.8 (2.41)
  CO2, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  CO2, Week 28, n=267, 296 | 22.7 (2.42) | 22.7 (2.27)
  CO2, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  CO2, Week 32, n=275, 294 | 22.6 (2.15) | 22.8 (2.34)
  CO2, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  CO2, Week 36, n=273, 292 | 22.8 (2.19) | 23.0 (2.26)
  CO2, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  CO2, Week 40, n=270, 293 | 23.1 (2.27) | 23.0 (2.45)
  CO2, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  CO2, Week 44, n=275, 293 | 23.0 (2.19) | 23.2 (2.31)
  CO2, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  CO2, Week 48, n=265, 292 | 22.7 (2.29) | 22.9 (2.29)
  Chloride, Baseline (Day 1), n=308, 308 | 103.8 (2.03) | 103.8 (2.39)
  Chloride, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Chloride, Week 4, n=301, 303 | 104.3 (2.13) | 104.3 (2.22)
  Chloride, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Chloride, Week 8, n=229, 303 | 104.3 (2.26) | 104.2 (2.40)
  Chloride, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Chloride, Week 12, n=295, 299 | 104.2 (2.27) | 104.3 (2.24)
  Chloride, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Chloride, Week 16, n=284, 298 | 104.5 (2.21) | 104.5 (2.28)
  Chloride, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Chloride, Week 20, n=277, 302 | 104.7 (2.41) | 104.5 (2.38)
  Chloride, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Chloride, Week 24, n=284, 299 | 104.5 (2.36) | 104.7 (2.30)
  Chloride, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Chloride, Week 28, n=267, 296 | 104.8 (2.19) | 104.8 (2.36)
  Chloride, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Chloride, Week 32, n=275, 294 | 104.7 (2.50) | 104.7 (2.31)
  Chloride, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Chloride, Week 36, n=273, 292 | 104.8 (2.18) | 104.6 (2.36)
  Chloride, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Chloride, Week 40, n=270, 293 | 104.7 (2.22) | 104.6 (2.61)
  Chloride, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Chloride, Week 44, n=275, 293 | 104.6 (2.10) | 104.6 (2.27)
  Chloride, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Chloride, Week 48, n=265, 292 | 104.4 (2.38) | 104.1 (2.37)
  Glucose, Baseline (Day 1), n=301, 299: number analyzed (Participants) | 301 | 299
  Glucose, Baseline (Day 1), n=301, 299 | 5.00 (0.714) | 5.17 (0.988)
  Glucose, Week 4, n=216, 226: number analyzed (Participants) | 216 | 226
  Glucose, Week 4, n=216, 226 | 5.17 (0.747) | 5.42 (1.250)
  Glucose, Week 8, n=153, 218: number analyzed (Participants) | 153 | 218
  Glucose, Week 8, n=153, 218 | 5.16 (0.990) | 5.35 (1.037)
  Glucose, Week 12, n=206, 221: number analyzed (Participants) | 206 | 221
  Glucose, Week 12, n=206, 221 | 5.19 (0.965) | 5.35 (1.091)
  Glucose, Week 16, n=209, 216: number analyzed (Participants) | 209 | 216
  Glucose, Week 16, n=209, 216 | 5.22 (1.163) | 5.36 (1.317)
  Glucose, Week 20, n=194, 221: number analyzed (Participants) | 194 | 221
  Glucose, Week 20, n=194, 221 | 5.20 (0.736) | 5.37 (1.209)
  Glucose, Week 24, n=215, 229: number analyzed (Participants) | 215 | 229
  Glucose, Week 24, n=215, 229 | 5.24 (0.810) | 5.35 (0.840)
  Glucose, Week 28, n=190, 226: number analyzed (Participants) | 190 | 226
  Glucose, Week 28, n=190, 226 | 5.16 (0.697) | 5.36 (0.876)
  Glucose, Week 32, n=194, 219: number analyzed (Participants) | 194 | 219
  Glucose, Week 32, n=194, 219 | 5.33 (1.042) | 5.45 (1.102)
  Glucose, Week 36, n=191, 220: number analyzed (Participants) | 191 | 220
  Glucose, Week 36, n=191, 220 | 5.19 (0.777) | 5.40 (1.507)
  Glucose, Week 40, n=195, 218: number analyzed (Participants) | 195 | 218
  Glucose, Week 40, n=195, 218 | 5.30 (0.797) | 5.44 (1.227)
  Glucose, Week 44, n=193, 213: number analyzed (Participants) | 193 | 213
  Glucose, Week 44, n=193, 213 | 5.22 (0.887) | 5.44 (1.317)
  Glucose, Week 48, n=242, 277: number analyzed (Participants) | 242 | 277
  Glucose, Week 48, n=242, 277 | 5.08 (0.614) | 5.22 (0.963)
  Phosphate, Baseline (Day 1), n=308, 308 | 1.042 (0.1771) | 1.051 (0.1722)
  Phosphate, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Phosphate, Week 4, n=301, 303 | 1.110 (0.1793) | 1.066 (0.1773)
  Phosphate, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Phosphate, Week 8, n=229, 303 | 1.097 (0.1944) | 1.042 (0.1843)
  Phosphate, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Phosphate, Week 12, n=295, 299 | 1.080 (0.1872) | 1.062 (0.1922)
  Phosphate, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Phosphate, Week 16, n=284, 298 | 1.081 (0.1796) | 1.052 (0.1724)
  Phosphate, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Phosphate, Week 20, n=277, 302 | 1.073 (0.1746) | 1.061 (0.1873)
  Phosphate, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Phosphate, Week 24, n=284, 299 | 1.082 (0.1788) | 1.057 (0.1849)
  Phosphate, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Phosphate, Week 28, n=267, 296 | 1.072 (0.1714) | 1.053 (0.1741)
  Phosphate, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Phosphate, Week 32, n=275, 294 | 1.061 (0.1730) | 1.054 (0.1761)
  Phosphate, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Phosphate, Week 36, n=273, 292 | 1.052 (0.1700) | 1.049 (0.1798)
  Phosphate, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Phosphate, Week 40, n=270, 293 | 1.065 (0.1789) | 1.046 (0.1763)
  Phosphate, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Phosphate, Week 44, n=275, 293 | 1.066 (0.1798) | 1.052 (0.1902)
  Phosphate, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Phosphate, Week 48, n=265, 292 | 1.077 (0.1816) | 1.052 (0.1834)
  Potassium, Baseline (Day 1), n=308, 308 | 4.16 (0.281) | 4.17 (0.314)
  Potassium, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Potassium, Week 4, n=301, 303 | 4.21 (0.307) | 4.28 (0.352)
  Potassium, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Potassium, Week 8, n=229, 303 | 4.16 (0.296) | 4.22 (0.393)
  Potassium, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Potassium, Week 12, n=295, 299 | 4.19 (0.330) | 4.24 (0.332)
  Potassium, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Potassium, Week 16, n=284, 298 | 4.18 (0.316) | 4.23 (0.321)
  Potassium, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Potassium, Week 20, n=277, 302 | 4.19 (0.311) | 4.21 (0.320)
  Potassium, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  Potassium, Week 24, n=284, 298 | 4.18 (0.287) | 4.23 (0.337)
  Potassium, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Potassium, Week 28, n=267, 296 | 4.19 (0.346) | 4.24 (0.391)
  Potassium, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Potassium, Week 32, n=275, 294 | 4.18 (0.368) | 4.21 (0.341)
  Potassium, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Potassium, Week 36, n=273, 292 | 4.19 (0.326) | 4.23 (0.345)
  Potassium, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Potassium, Week 40, n=270, 293 | 4.20 (0.301) | 4.23 (0.322)
  Potassium, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Potassium, Week 44, n=275, 293 | 4.21 (0.323) | 4.23 (0.359)
  Potassium, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Potassium, Week 48, n=265, 292 | 4.15 (0.271) | 4.16 (0.331)
  Sodium, Baseline (Day 1), n=308, 308 | 139.0 (1.91) | 139.0 (1.76)
  Sodium, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Sodium, Week 4, n=301, 303 | 139.3 (1.70) | 139.1 (1.87)
  Sodium, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Sodium, Week 8, n=229, 303 | 139.1 (1.98) | 139.0 (1.80)
  Sodium, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Sodium, Week 12, n=295, 299 | 139.2 (1.84) | 139.2 (1.85)
  Sodium, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Sodium, Week 16, n=284, 298 | 139.1 (1.98) | 139.1 (1.96)
  Sodium, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Sodium, Week 20, n=277, 302 | 139.2 (1.87) | 139.3 (1.81)
  Sodium, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Sodium, Week 24, n=284, 299 | 139.3 (1.88) | 139.3 (1.96)
  Sodium, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Sodium, Week 28, n=267, 296 | 139.5 (1.77) | 139.2 (2.01)
  Sodium, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Sodium, Week 32, n=275, 294 | 139.3 (1.75) | 139.5 (1.84)
  Sodium, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Sodium, Week 36, n=273, 292 | 139.4 (1.79) | 139.5 (2.15)
  Sodium, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Sodium, Week 40, n=270, 293 | 139.4 (1.93) | 139.5 (1.97)
  Sodium, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Sodium, Week 44, n=275, 293 | 139.4 (1.80) | 139.5 (1.93)
  Sodium, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Sodium, Week 48, n=265, 292 | 139.4 (1.94) | 139.4 (1.83)
  Urea, Baseline (Day 1), n=308, 308 | 5.23 (1.546) | 5.22 (1.632)
  Urea, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Urea, Week 4, n=301, 303 | 5.24 (1.495) | 5.28 (1.549)
  Urea, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Urea, Week 8, n=229, 303 | 5.32 (1.640) | 5.22 (1.529)
  Urea, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Urea, Week 12, n=295, 299 | 5.38 (1.612) | 5.30 (1.649)
  Urea, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Urea, Week 16, n=284, 298 | 5.30 (1.662) | 5.41 (1.659)
  Urea, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Urea, Week 20, n=277, 302 | 5.37 (1.631) | 5.33 (1.662)
  Urea, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Urea, Week 24, n=284, 299 | 5.49 (1.749) | 5.36 (1.639)
  Urea, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Urea, Week 28, n=267, 296 | 5.39 (1.756) | 5.24 (1.527)
  Urea, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Urea, Week 32, n=275, 294 | 5.44 (1.624) | 5.29 (1.599)
  Urea, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Urea, Week 36, n=273, 292 | 5.26 (1.664) | 5.20 (1.485)
  Urea, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Urea, Week 40, n=270, 293 | 5.47 (1.593) | 5.30 (1.537)
  Urea, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Urea, Week 44, n=275, 293 | 5.37 (1.531) | 5.26 (1.524)
  Urea, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Urea, Week 48, n=265, 292 | 5.48 (1.648) | 5.21 (1.437)

26. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter Over Time Including Week 48: Lipase
Description: Blood samples were collected for the analysis of clinical chemistry parameter-lipase at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Units per liter
  Baseline, n=308, 308 | 30.5 (22.88) | 30.8 (19.12)
  Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Week 4, n=301, 303 | 35.3 (52.73) | 32.3 (23.30)
  Week 8, n=227, 303: number analyzed (Participants) | 227 | 303
  Week 8, n=227, 303 | 30.6 (22.70) | 31.9 (20.71)
  Week 12, n=294, 297: number analyzed (Participants) | 294 | 297
  Week 12, n=294, 297 | 33.2 (27.92) | 30.0 (18.06)
  Week 16, n=285, 299: number analyzed (Participants) | 285 | 299
  Week 16, n=285, 299 | 33.8 (30.49) | 33.9 (34.69)
  Week 20, n=278, 302: number analyzed (Participants) | 278 | 302
  Week 20, n=278, 302 | 31.0 (21.73) | 31.6 (28.88)
  Week 24, n=283, 299: number analyzed (Participants) | 283 | 299
  Week 24, n=283, 299 | 33.1 (24.09) | 33.8 (29.69)
  Week 28, n=267, 297: number analyzed (Participants) | 267 | 297
  Week 28, n=267, 297 | 32.9 (27.42) | 33.1 (19.69)
  Week 32, n=274, 294: number analyzed (Participants) | 274 | 294
  Week 32, n=274, 294 | 35.7 (60.63) | 33.8 (21.64)
  Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Week 36, n=273, 292 | 36.2 (51.58) | 31.6 (18.46)
  Week 40, n=269, 293: number analyzed (Participants) | 269 | 293
  Week 40, n=269, 293 | 35.7 (36.06) | 31.4 (15.80)
  Week 44, n=274, 293: number analyzed (Participants) | 274 | 293
  Week 44, n=274, 293 | 33.3 (26.29) | 33.3 (20.44)
  Week 48, n=264, 290: number analyzed (Participants) | 264 | 290
  Week 48, n=264, 290 | 34.3 (30.97) | 32.4 (20.40)

27. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter Over Time Including Week 48: Creatinine Clearance
Description: Blood samples were collected for the analysis of clinical chemistry parameter-creatinine clearance at indicated timepoints. Glomerular filtration rate (GFR) will be estimated by the central laboratory using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliter per minute per 1.73meter^2
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Milliliter per minute per 1.73meter^2
  Baseline, n=308, 308 | 100.5 (18.30) | 101.1 (17.72)
  Week 4, n=301, 301: number analyzed (Participants) | 301 | 301
  Week 4, n=301, 301 | 98.7 (17.26) | 98.9 (17.93)
  Week 8, n=227, 303: number analyzed (Participants) | 227 | 303
  Week 8, n=227, 303 | 100.1 (17.19) | 99.5 (17.59)
  Week 12, n=295, 297: number analyzed (Participants) | 295 | 297
  Week 12, n=295, 297 | 100.9 (17.72) | 99.2 (18.34)
  Week 16, n=284, 297: number analyzed (Participants) | 284 | 297
  Week 16, n=284, 297 | 100.5 (17.26) | 99.0 (18.32)
  Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Week 20, n=277, 302 | 99.4 (17.37) | 98.7 (17.73)
  Week 24, n=283, 298: number analyzed (Participants) | 283 | 298
  Week 24, n=283, 298 | 98.9 (17.04) | 98.9 (17.44)
  Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Week 28, n=267, 296 | 98.5 (17.66) | 99.0 (17.33)
  Week 32, n=274, 294: number analyzed (Participants) | 274 | 294
  Week 32, n=274, 294 | 99.1 (16.89) | 98.4 (17.54)
  Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Week 36, n=273, 292 | 99.0 (17.19) | 98.6 (16.85)
  Week 40, n=268, 293: number analyzed (Participants) | 268 | 293
  Week 40, n=268, 293 | 98.5 (17.32) | 98.5 (17.37)
  Week 44, n=274, 293: number analyzed (Participants) | 274 | 293
  Week 44, n=274, 293 | 98.2 (16.96) | 99.0 (17.39)
  Week 48, n=264, 291: number analyzed (Participants) | 264 | 291
  Week 48, n=264, 291 | 97.6 (16.97) | 99.3 (17.09)

28. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameters Over Time Including Week 48
Description: The dipstick test gives results in a semi-quantitative manner and results for urinalysis parameters (ketones, glucose, bilirubin, occult blood, nitrite and blood protein) can be read as positive, trace, 1+, 2+, 3+ and 4+ indicating proportional concentrations in the urine sample. The urine parameters were graded according to Division of AIDS (DAIDS) scale where Grade 1 indicates mild (trace to 1+), Grade 2 indicates moderate (2+) and Grade 3 indicates severe (3+ or higher). Only participants with abnormal findings for urinalysis at any visit has been presented.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48.
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants
  Urine bilirubin,Baseline (Day 1),Trace, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine bilirubin,Baseline (Day 1),Trace, n=303, 301 | 0 | 0
  Urine bilirubin, Baseline (Day 1), 1+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine bilirubin, Baseline (Day 1), 1+, n=303, 301 | 6 | 7
  Urine bilirubin, Baseline (Day 1), 2+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine bilirubin, Baseline (Day 1), 2+, n=303, 301 | 0 | 0
  Urine bilirubin, Baseline (Day 1), 3+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine bilirubin, Baseline (Day 1), 3+, n=303, 301 | 0 | 0
  Urine glucose, Baseline (Day 1), Trace, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine glucose, Baseline (Day 1), Trace, n=303, 301 | 1 | 1
  Urine glucose, Baseline (Day 1), 1+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine glucose, Baseline (Day 1), 1+, n=303, 301 | 0 | 1
  Urine glucose, Baseline (Day 1), 2+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine glucose, Baseline (Day 1), 2+, n=303, 301 | 0 | 0
  Urine glucose, Baseline (Day 1), 3+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine glucose, Baseline (Day 1), 3+, n=303, 301 | 0 | 1
  Urine ketones, Baseline (Day 1), Trace, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine ketones, Baseline (Day 1), Trace, n=303, 301 | 16 | 17
  Urine ketones, Baseline (Day 1), 1+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine ketones, Baseline (Day 1), 1+, n=303, 301 | 4 | 0
  Urine ketones, Baseline (Day 1), 2+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine ketones, Baseline (Day 1), 2+, n=303, 301 | 2 | 1
  Urine ketones, Baseline (Day 1), 3+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine ketones, Baseline (Day 1), 3+, n=303, 301 | 0 | 0
  Urine leukocyte esterase,Baseline,Trace,n=303,301: number analyzed (Participants) | 303 | 301
  Urine leukocyte esterase,Baseline,Trace,n=303,301 | 25 | 18
  Urine leukocyte esterase, Baseline, 1+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine leukocyte esterase, Baseline, 1+, n=303, 301 | 14 | 16
  Urine leukocyte esterase, Baseline, 2+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine leukocyte esterase, Baseline, 2+, n=303, 301 | 14 | 8
  Urine leukocyte esterase, Baseline, 3+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine leukocyte esterase, Baseline, 3+, n=303, 301 | 5 | 5
  Urine nitrite, Baseline, positive, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine nitrite, Baseline, positive, n=303, 301 | 11 | 11
  Urine occult blood, Baseline, Trace, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine occult blood, Baseline, Trace, n=303, 301 | 19 | 12
  Urine occult blood, Baseline, 1+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine occult blood, Baseline, 1+, n=303, 301 | 8 | 9
  Urine occult blood, Baseline, 2+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine occult blood, Baseline, 2+, n=303, 301 | 7 | 5
  Urine occult blood, Baseline, 3+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine occult blood, Baseline, 3+, n=303, 301 | 5 | 3
  Urine protein, Baseline, Trace, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine protein, Baseline, Trace, n=303, 301 | 14 | 20
  Urine protein, Baseline, 1+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine protein, Baseline, 1+, n=303, 301 | 6 | 12
  Urine protein, Baseline, 2+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine protein, Baseline, 2+, n=303, 301 | 0 | 1
  Urine protein, Baseline, 3+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine protein, Baseline, 3+, n=303, 301 | 0 | 0
  Urine protein, Baseline, 4+, n=303, 301: number analyzed (Participants) | 303 | 301
  Urine protein, Baseline, 4+, n=303, 301 | 0 | 0
  Urine bilirubin, Week 4, Trace, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine bilirubin, Week 4, Trace, n=303, 302 | 0 | 0
  Urine bilirubin, Week 4, 1+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine bilirubin, Week 4, 1+, n=303, 302 | 9 | 5
  Urine bilirubin, Week 4, 2+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine bilirubin, Week 4, 2+, n=303, 302 | 0 | 0
  Urine bilirubin, Week 4, 3+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine bilirubin, Week 4, 3+, n=303, 302 | 0 | 0
  Urine glucose, Week 4, Trace, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine glucose, Week 4, Trace, n=303, 302 | 3 | 2
  Urine glucose, Week 4, 1+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine glucose, Week 4, 1+, n=303, 302 | 1 | 2
  Urine glucose, Week 4, 2+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine glucose, Week 4, 2+, n=303, 302 | 2 | 0
  Urine glucose, Week 4, 3+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine glucose, Week 4, 3+, n=303, 302 | 0 | 1
  Urine ketones, Week 4, Trace, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine ketones, Week 4, Trace, n=303, 302 | 9 | 15
  Urine ketones, Week 4, 1+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine ketones, Week 4, 1+, n=303, 302 | 0 | 2
  Urine ketones, Week 4, 2+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine ketones, Week 4, 2+, n=303, 302 | 1 | 1
  Urine ketones, Week 4, 3+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine ketones, Week 4, 3+, n=303, 302 | 0 | 0
  Urine leukocyte esterase, Week 4, Trace,n=303, 302: number analyzed (Participants) | 303 | 302
  Urine leukocyte esterase, Week 4, Trace,n=303, 302 | 25 | 29
  Urine leukocyte esterase, Week 4, 1+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine leukocyte esterase, Week 4, 1+, n=303, 302 | 14 | 15
  Urine leukocyte esterase, Week 4, 2+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine leukocyte esterase, Week 4, 2+, n=303, 302 | 14 | 9
  Urine leukocyte esterase, Week 4, 3+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine leukocyte esterase, Week 4, 3+, n=303, 302 | 3 | 4
  Urine nitrite, Week 4, positive, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine nitrite, Week 4, positive, n=303, 302 | 10 | 12
  Urine occult blood, Week 4, Trace, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine occult blood, Week 4, Trace, n=303, 302 | 15 | 18
  Urine occult blood, Week 4, 1+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine occult blood, Week 4, 1+, n=303, 302 | 9 | 10
  Urine occult blood, Week 4, 2+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine occult blood, Week 4, 2+, n=303, 302 | 5 | 5
  Urine occult blood, Week 4, 3+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine occult blood, Week 4, 3+, n=303, 302 | 4 | 3
  Urine protein, Week 4, Trace, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine protein, Week 4, Trace, n=303, 302 | 10 | 13
  Urine protein, Week 4, 1+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine protein, Week 4, 1+, n=303, 302 | 8 | 7
  Urine protein, Week 4, 2+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine protein, Week 4, 2+, n=303, 302 | 2 | 4
  Urine protein, Week 4, 3+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine protein, Week 4, 3+, n=303, 302 | 0 | 0
  Urine protein, Week 4, 4+, n=303, 302: number analyzed (Participants) | 303 | 302
  Urine protein, Week 4, 4+, n=303, 302 | 0 | 0
  Urine bilirubin, Week 24, Trace, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine bilirubin, Week 24, Trace, n=279, 298 | 0 | 0
  Urine bilirubin, Week 24, 1+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine bilirubin, Week 24, 1+, n=279, 298 | 10 | 13
  Urine bilirubin, Week 24, 2+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine bilirubin, Week 24, 2+, n=279, 298 | 0 | 0
  Urine bilirubin, Week 24, 3+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine bilirubin, Week 24, 3+, n=279, 298 | 0 | 0
  Urine glucose, Week 24, Trace, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine glucose, Week 24, Trace, n=279, 298 | 0 | 1
  Urine glucose, Week 24, 1+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine glucose, Week 24, 1+, n=279, 298 | 2 | 0
  Urine glucose, Week 24, 2+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine glucose, Week 24, 2+, n=279, 298 | 0 | 1
  Urine glucose, Week 24, 3+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine glucose, Week 24, 3+, n=279, 298 | 1 | 1
  Urine ketones, Week 24, Trace, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine ketones, Week 24, Trace, n=279, 298 | 16 | 13
  Urine ketones, Week 24, 1+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine ketones, Week 24, 1+, n=279, 298 | 1 | 1
  Urine ketones, Week 24, 2+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine ketones, Week 24, 2+, n=279, 298 | 0 | 0
  Urine ketones, Week 24, 3+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine ketones, Week 24, 3+, n=279, 298 | 0 | 0
  Urine leukocyte esterase,Week 24, Trace, n=279,298: number analyzed (Participants) | 279 | 298
  Urine leukocyte esterase,Week 24, Trace, n=279,298 | 22 | 17
  Urine leukocyte esterase, Week 24, 1+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine leukocyte esterase, Week 24, 1+, n=279, 298 | 14 | 14
  Urine leukocyte esterase, Week 24, 2+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine leukocyte esterase, Week 24, 2+, n=279, 298 | 6 | 14
  Urine leukocyte esterase, Week 24, 3+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine leukocyte esterase, Week 24, 3+, n=279, 298 | 3 | 7
  Urine nitrite, Week 24, positive, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine nitrite, Week 24, positive, n=279, 298 | 9 | 10
  Urine occult blood, Week 24, Trace, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine occult blood, Week 24, Trace, n=279, 298 | 13 | 10
  Urine occult blood, Week 24, 1+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine occult blood, Week 24, 1+, n=279, 298 | 5 | 6
  Urine occult blood, Week 24, 2+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine occult blood, Week 24, 2+, n=279, 298 | 6 | 4
  Urine occult blood, Week 24, 3+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine occult blood, Week 24, 3+, n=279, 298 | 0 | 6
  Urine protein, Week 24, Trace, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine protein, Week 24, Trace, n=279, 298 | 10 | 21
  Urine protein, Week 24, 1+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine protein, Week 24, 1+, n=279, 298 | 4 | 12
  Urine protein, Week 24, 2+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine protein, Week 24, 2+, n=279, 298 | 1 | 3
  Urine protein, Week 24, 3+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine protein, Week 24, 3+, n=279, 298 | 0 | 0
  Urine protein, Week 24, 4+, n=279, 298: number analyzed (Participants) | 279 | 298
  Urine protein, Week 24, 4+, n=279, 298 | 0 | 0
  Urine bilirubin, Week 48, Trace, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine bilirubin, Week 48, Trace, n=279, 290 | 0 | 0
  Urine bilirubin, Week 48, 1+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine bilirubin, Week 48, 1+, n=279, 290 | 9 | 8
  Urine bilirubin, Week 48, 2+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine bilirubin, Week 48, 2+, n=279, 290 | 1 | 0
  Urine bilirubin, Week 48, 3+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine bilirubin, Week 48, 3+, n=279, 290 | 0 | 0
  Urine glucose, Week 48, Trace, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine glucose, Week 48, Trace, n=279, 290 | 0 | 1
  Urine glucose, Week 48, 1+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine glucose, Week 48, 1+, n=279, 290 | 0 | 2
  Urine glucose, Week 48, 2+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine glucose, Week 48, 2+, n=279, 290 | 1 | 0
  Urine glucose, Week 48, 3+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine glucose, Week 48, 3+, n=279, 290 | 0 | 2
  Urine ketones, Week 48, Trace, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine ketones, Week 48, Trace, n=279, 290 | 13 | 9
  Urine ketones, Week 48, 1+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine ketones, Week 48, 1+, n=279, 290 | 0 | 0
  Urine ketones, Week 48, 2+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine ketones, Week 48, 2+, n=279, 290 | 0 | 0
  Urine ketones, Week 48, 3+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine ketones, Week 48, 3+, n=279, 290 | 0 | 0
  Urine leukocyte esterase, Week 48, Trace,n=279,290: number analyzed (Participants) | 279 | 290
  Urine leukocyte esterase, Week 48, Trace,n=279,290 | 24 | 27
  Urine leukocyte esterase, Week 48, 1+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine leukocyte esterase, Week 48, 1+, n=279, 290 | 13 | 15
  Urine leukocyte esterase, Week 48, 2+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine leukocyte esterase, Week 48, 2+, n=279, 290 | 7 | 7
  Urine leukocyte esterase, Week 48, 3+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine leukocyte esterase, Week 48, 3+, n=279, 290 | 5 | 6
  Urine nitrite, Week 48, positive, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine nitrite, Week 48, positive, n=279, 290 | 10 | 6
  Urine occult blood, Week 48, Trace, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine occult blood, Week 48, Trace, n=279, 290 | 11 | 12
  Urine occult blood, Week 48, 1+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine occult blood, Week 48, 1+, n=279, 290 | 5 | 5
  Urine occult blood, Week 48, 2+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine occult blood, Week 48, 2+, n=279, 290 | 4 | 4
  Urine occult blood, Week 48, 3+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine occult blood, Week 48, 3+, n=279, 290 | 6 | 0
  Urine protein, Week 48, Trace, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine protein, Week 48, Trace, n=279, 290 | 10 | 15
  Urine protein, Week 48, 1+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine protein, Week 48, 1+, n=279, 290 | 4 | 6
  Urine protein, Week 48, 2+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine protein, Week 48, 2+, n=279, 290 | 3 | 3
  Urine protein, Week 48, 3+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine protein, Week 48, 3+, n=279, 290 | 0 | 0
  Urine protein, Week 48, 4+, n=279, 290: number analyzed (Participants) | 279 | 290
  Urine protein, Week 48, 4+, n=279, 290 | 0 | 1

29. Secondary Outcome: Number of Participants With Urine Potential of Hydrogen (pH) Over Time Including Week 48
Description: Urine samples were collected for analysis of urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0).
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants
  Baseline, pH=5, n=303, 301: number analyzed (Participants) | 303 | 301
  Baseline, pH=5, n=303, 301 | 44 | 42
  Baseline, pH=5.5, n=303, 301: number analyzed (Participants) | 303 | 301
  Baseline, pH=5.5, n=303, 301 | 78 | 80
  Baseline, pH=6, n=303, 301: number analyzed (Participants) | 303 | 301
  Baseline, pH=6, n=303, 301 | 85 | 72
  Baseline, pH=6.5, n=303, 301: number analyzed (Participants) | 303 | 301
  Baseline, pH=6.5, n=303, 301 | 47 | 45
  Baseline, pH=7, n=303, 301: number analyzed (Participants) | 303 | 301
  Baseline, pH=7, n=303, 301 | 32 | 34
  Baseline, pH=7.5, n=303, 301: number analyzed (Participants) | 303 | 301
  Baseline, pH=7.5, n=303, 301 | 12 | 19
  Baseline, pH=8, n=303, 301: number analyzed (Participants) | 303 | 301
  Baseline, pH=8, n=303, 301 | 3 | 7
  Baseline, pH=8.5, n=303, 301: number analyzed (Participants) | 303 | 301
  Baseline, pH=8.5, n=303, 301 | 0 | 1
  Baseline, pH>9.0, n=303, 301: number analyzed (Participants) | 303 | 301
  Baseline, pH>9.0, n=303, 301 | 2 | 1
  Week 4, pH=5, n=303, 302: number analyzed (Participants) | 303 | 302
  Week 4, pH=5, n=303, 302 | 41 | 53
  Week 4, pH=5.5, n=303, 302: number analyzed (Participants) | 303 | 302
  Week 4, pH=5.5, n=303, 302 | 78 | 93
  Week 4, pH=6, n=303, 302: number analyzed (Participants) | 303 | 302
  Week 4, pH=6, n=303, 302 | 73 | 67
  Week 4, pH=6.5, n=303, 302: number analyzed (Participants) | 303 | 302
  Week 4, pH=6.5, n=303, 302 | 49 | 41
  Week 4, pH=7, n=303, 302: number analyzed (Participants) | 303 | 302
  Week 4, pH=7, n=303, 302 | 38 | 28
  Week 4, pH=7.5, n=303, 302: number analyzed (Participants) | 303 | 302
  Week 4, pH=7.5, n=303, 302 | 12 | 14
  Week 4, pH=8, n=303, 302: number analyzed (Participants) | 303 | 302
  Week 4, pH=8, n=303, 302 | 8 | 3
  Week 4, pH=8.5, n=303, 302: number analyzed (Participants) | 303 | 302
  Week 4, pH=8.5, n=303, 302 | 3 | 2
  Week 4, pH>9.0, n=303, 302: number analyzed (Participants) | 303 | 302
  Week 4, pH>9.0, n=303, 302 | 1 | 1
  Week 24, pH=5, n=279, 298: number analyzed (Participants) | 279 | 298
  Week 24, pH=5, n=279, 298 | 23 | 26
  Week 24, pH=5.5, n=279, 298: number analyzed (Participants) | 279 | 298
  Week 24, pH=5.5, n=279, 298 | 85 | 96
  Week 24, pH=6, n=279, 298: number analyzed (Participants) | 279 | 298
  Week 24, pH=6, n=279, 298 | 66 | 67
  Week 24, pH=6.5, n=279, 298: number analyzed (Participants) | 279 | 298
  Week 24, pH=6.5, n=279, 298 | 44 | 52
  Week 24, pH=7, n=279, 298: number analyzed (Participants) | 279 | 298
  Week 24, pH=7, n=279, 298 | 32 | 31
  Week 24, pH=7.5, n=279, 298: number analyzed (Participants) | 279 | 298
  Week 24, pH=7.5, n=279, 298 | 16 | 15
  Week 24, pH=8, n=279, 298: number analyzed (Participants) | 279 | 298
  Week 24, pH=8, n=279, 298 | 7 | 8
  Week 24, pH=8.5, n=279, 298: number analyzed (Participants) | 279 | 298
  Week 24, pH=8.5, n=279, 298 | 2 | 2
  Week 24, pH>9.0, n=279, 298: number analyzed (Participants) | 279 | 298
  Week 24, pH>9.0, n=279, 298 | 4 | 1
  Week 48, pH=5, n=279, 290: number analyzed (Participants) | 279 | 290
  Week 48, pH=5, n=279, 290 | 45 | 43
  Week 48, pH=5.5, n=279, 290: number analyzed (Participants) | 279 | 290
  Week 48, pH=5.5, n=279, 290 | 69 | 83
  Week 48, pH=6, n=279, 290: number analyzed (Participants) | 279 | 290
  Week 48, pH=6, n=279, 290 | 61 | 58
  Week 48, pH=6.5, n=279, 290: number analyzed (Participants) | 279 | 290
  Week 48, pH=6.5, n=279, 290 | 47 | 48
  Week 48, pH=7, n=279, 290: number analyzed (Participants) | 279 | 290
  Week 48, pH=7, n=279, 290 | 31 | 30
  Week 48, pH=7.5, n=279, 290: number analyzed (Participants) | 279 | 290
  Week 48, pH=7.5, n=279, 290 | 17 | 17
  Week 48, pH=8, n=279, 290: number analyzed (Participants) | 279 | 290
  Week 48, pH=8, n=279, 290 | 6 | 5
  Week 48, pH=8.5, n=279, 290: number analyzed (Participants) | 279 | 290
  Week 48, pH=8.5, n=279, 290 | 0 | 4
  Week 48, pH>9.0, n=279, 290: number analyzed (Participants) | 279 | 290
  Week 48, pH>9.0, n=279, 290 | 3 | 2

30. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Over Time Including Week 48: ALT, ALP, AST and CK
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALT, ALP, AST and CK. Baseline values is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
International units per liter
  ALT, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  ALT, Week 4, n=301, 303 | 0.8 (13.98) | 0.1 (9.65)
  ALT, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  ALT, Week 8, n=229, 303 | 0.7 (15.35) | 1.6 (29.98)
  ALT, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  ALT, Week 12, n=295, 299 | 5.2 (113.34) | 0.4 (11.60)
  ALT, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  ALT, Week 16, n=284, 298 | -0.1 (21.80) | -0.6 (10.14)
  ALT, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  ALT, Week 20, n=277, 302 | -0.8 (22.62) | -1.1 (10.86)
  ALT, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  ALT, Week 24, n=284, 299 | 2.2 (61.65) | -0.6 (10.57)
  ALT, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  ALT, Week 28, n=267, 296 | -2.7 (11.14) | -0.2 (12.52)
  ALT, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  ALT, Week 32, n=275, 294 | -1.9 (14.44) | -0.5 (11.49)
  ALT, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  ALT, Week 36, n=273, 292 | -0.8 (23.51) | 0.1 (10.95)
  ALT, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  ALT, Week 40, n=270, 293 | 0.6 (36.29) | -0.2 (11.82)
  ALT, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  ALT, Week 44, n=275, 293 | -2.2 (13.97) | -0.2 (12.37)
  ALT, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  ALT, Week 48, n=265, 292 | -1.9 (13.43) | -0.6 (10.50)
  ALP, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  ALP, Week 4, n=301, 303 | -6.0 (12.74) | -2.2 (8.85)
  ALP, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  ALP, Week 8, n=229, 303 | -6.7 (16.59) | 1.1 (20.99)
  ALP, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  ALP, Week 12, n=295, 299 | -8.0 (20.87) | 0.9 (14.45)
  ALP, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  ALP, Week 16, n=284, 298 | -9.7 (19.47) | -0.5 (10.35)
  ALP, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  ALP, Week 20, n=277, 302 | -9.2 (19.05) | -1.0 (11.65)
  ALP, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  ALP, Week 24, n=284, 299 | -9.0 (19.02) | -0.1 (10.67)
  ALP, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  ALP, Week 28, n=267, 296 | -10.1 (19.08) | -0.2 (11.44)
  ALP, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  ALP, Week 32, n=275, 294 | -9.9 (19.10) | -1.7 (11.29)
  ALP, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  ALP, Week 36, n=273, 292 | -10.5 (20.41) | -1.1 (11.44)
  ALP, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  ALP, Week 40, n=270, 293 | -10.4 (20.71) | -1.1 (11.34)
  ALP, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  ALP, Week 44, n=275, 293 | -11.4 (20.64) | -0.7 (12.02)
  ALP, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  ALP, Week 48, n=265, 292 | -10.9 (23.27) | -0.3 (12.51)
  AST, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  AST, Week 4, n=301, 303 | -0.3 (12.52) | 0.2 (10.02)
  AST, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  AST, Week 8, n=229, 303 | 1.2 (19.73) | -0.1 (13.68)
  AST, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  AST, Week 12, n=295, 299 | 2.3 (65.03) | 0.6 (8.82)
  AST, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  AST, Week 16, n=284, 298 | 0.1 (18.49) | -0.1 (9.71)
  AST, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  AST, Week 20, n=277, 302 | -0.5 (17.02) | -0.6 (9.80)
  AST, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  AST, Week 24, n=284, 298 | 0.1 (24.12) | 0.0 (9.57)
  AST, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  AST, Week 28, n=267, 296 | -1.4 (8.77) | 0.3 (11.19)
  AST, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  AST, Week 32, n=275, 294 | -1.2 (16.08) | 0.6 (13.40)
  AST, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  AST, Week 36, n=273, 292 | -1.2 (12.95) | 0.1 (9.61)
  AST, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  AST, Week 40, n=270, 293 | -0.2 (17.27) | 0.0 (10.64)
  AST, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  AST, Week 44, n=275, 293 | -1.1 (16.51) | 0.1 (11.09)
  AST Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  AST Week 48, n=265, 292 | -1.0 (12.79) | 0.7 (10.75)
  CK, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  CK, Week 4, n=301, 303 | -0.1 (548.15) | 30.8 (435.12)
  CK, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  CK, Week 8, n=229, 303 | 98.2 (1076.99) | -16.5 (344.96)
  CK, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  CK, Week 12, n=295, 299 | 6.0 (585.45) | 14.9 (288.85)
  CK, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  CK, Week 16, n=284, 298 | 54.2 (882.23) | 5.8 (411.52)
  CK, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  CK, Week 20, n=277, 302 | 31.2 (653.11) | -16.7 (363.30)
  CK, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  CK, Week 24, n=284, 299 | -9.2 (538.95) | -0.7 (353.99)
  CK, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  CK, Week 28, n=267, 296 | -1.9 (213.98) | 20.8 (538.83)
  CK, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  CK, Week 32, n=275, 294 | 13.3 (699.60) | 34.0 (597.29)
  CK, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  CK, Week 36, n=273, 292 | -18.2 (476.64) | -10.8 (358.72)
  CK, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  CK, Week 40, n=270, 293 | 39.7 (704.18) | -0.3 (373.96)
  CK, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  CK, Week 44, n=275, 293 | 47.4 (1185.55) | -10.9 (350.64)
  CK, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  CK, Week 48, n=265, 292 | -0.6 (528.71) | 18.1 (463.49)

31. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter Over Time Including Week 48: Albumin
Description: Blood samples were collected for the analysis of clinical chemistry parameter-albumin. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Grams per liter
  Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Week 4, n=301, 303 | -0.5 (2.60) | -0.5 (2.49)
  Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Week 8, n=229, 303 | -0.3 (2.76) | -0.7 (2.70)
  Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Week 12, n=295, 299 | -0.6 (2.72) | -0.4 (2.63)
  Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Week 16, n=284, 298 | -0.6 (2.78) | -0.8 (2.70)
  Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Week 20, n=277, 302 | -0.8 (2.78) | -0.8 (2.56)
  Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Week 24, n=284, 299 | -0.7 (2.69) | -0.8 (2.59)
  Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Week 28, n=267, 296 | -0.7 (2.60) | -1.0 (2.47)
  Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Week 32, n=275, 294 | -0.6 (2.78) | -1.0 (2.56)
  Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Week 36, n=273, 292 | -0.9 (2.71) | -0.9 (2.65)
  Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Week 40, n=270, 293 | -0.5 (2.53) | -1.0 (2.61)
  Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Week 44, n=275, 293 | -0.4 (2.58) | -0.8 (2.47)
  Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Week 48, n=265, 292 | -0.4 (2.64) | -0.4 (2.55)

32. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Over Time Including Week 48: Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters including bilirubin, creatinine and direct bilirubin. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Micromoles per liter
  Bilirubin, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Bilirubin, Week 4, n=301, 303 | -0.8 (9.87) | -0.3 (4.17)
  Bilirubin, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Bilirubin, Week 8, n=229, 303 | -0.1 (6.92) | 0.1 (7.66)
  Bilirubin, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Bilirubin, Week 12, n=295, 299 | -0.6 (10.23) | 0.1 (4.56)
  Bilirubin, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Bilirubin, Week 16, n=284, 298 | 0.2 (14.00) | -0.2 (4.12)
  Bilirubin, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Bilirubin, Week 20, n=277, 302 | -0.2 (10.04) | 0.0 (6.10)
  Bilirubin, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  Bilirubin, Week 24, n=284, 298 | -0.6 (9.90) | 0.2 (5.90)
  Bilirubin, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Bilirubin, Week 28, n=267, 296 | 0.0 (10.46) | -0.1 (4.76)
  Bilirubin, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Bilirubin, Week 32, n=275, 294 | -0.1 (10.36) | 0.0 (4.94)
  Bilirubin, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Bilirubin, Week 36, n=273, 292 | -0.6 (10.39) | 0.1 (4.55)
  Bilirubin, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Bilirubin, Week 40, n=270, 293 | -0.3 (10.61) | 0.2 (6.28)
  Bilirubin, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Bilirubin, Week 44, n=275, 293 | -0.4 (10.11) | 0.4 (5.24)
  Bilirubin, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Bilirubin, Week 48, n=265, 292 | -0.3 (10.57) | 0.2 (3.91)
  Direct bilirubin, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Direct bilirubin, Week 4, n=301, 303 | -0.1 (1.48) | 0.1 (1.20)
  Direct bilirubin, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Direct bilirubin, Week 8, n=229, 303 | -0.1 (1.42) | 0.2 (3.96)
  Direct bilirubin, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Direct bilirubin, Week 12, n=295, 299 | -0.2 (1.61) | 0.1 (1.21)
  Direct bilirubin, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Direct bilirubin, Week 16, n=284, 298 | 0.1 (5.02) | -0.1 (1.12)
  Direct bilirubin, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Direct bilirubin, Week 20, n=277, 302 | -0.3 (1.52) | -0.2 (1.29)
  Direct bilirubin, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  Direct bilirubin, Week 24, n=284, 298 | -0.2 (1.55) | -0.1 (1.24)
  Direct bilirubin, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Direct bilirubin, Week 28, n=267, 296 | -0.3 (1.55) | -0.2 (1.29)
  Direct bilirubin, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Direct bilirubin, Week 32, n=275, 294 | -0.3 (1.61) | -0.2 (1.24)
  Direct bilirubin, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Direct bilirubin, Week 36, n=273, 292 | -0.3 (1.70) | -0.1 (1.20)
  Direct bilirubin, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Direct bilirubin, Week 40, n=270, 293 | -0.3 (1.68) | -0.2 (1.18)
  Direct bilirubin, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Direct bilirubin, Week 44, n=275, 293 | -0.2 (1.55) | -0.1 (1.19)
  Direct bilirubin, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Direct bilirubin, Week 48, n=265, 292 | -0.2 (1.54) | 0.0 (1.23)
  Creatinine, Week 4, n=301, 301: number analyzed (Participants) | 301 | 301
  Creatinine, Week 4, n=301, 301 | 1.15 (8.205) | 1.80 (8.022)
  Creatinine, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Creatinine, Week 8, n=229, 303 | -0.66 (9.042) | 1.23 (7.560)
  Creatinine, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Creatinine, Week 12, n=295, 299 | -0.38 (9.380) | 1.71 (7.638)
  Creatinine, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Creatinine, Week 16, n=284, 298 | -0.60 (9.225) | 1.62 (8.169)
  Creatinine, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Creatinine, Week 20, n=277, 302 | 0.53 (9.390) | 1.80 (8.454)
  Creatinine, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  Creatinine, Week 24, n=284, 298 | 0.90 (12.494) | 1.36 (8.038)
  Creatinine, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Creatinine, Week 28, n=267, 296 | 1.14 (10.998) | 1.59 (8.303)
  Creatinine, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Creatinine, Week 32, n=275, 294 | 0.33 (10.102) | 1.95 (8.331)
  Creatinine, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Creatinine, Week 36, n=273, 292 | 0.34 (10.585) | 1.62 (7.891)
  Creatinine, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Creatinine, Week 40, n=270, 293 | 0.88 (9.986) | 1.64 (8.318)
  Creatinine, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Creatinine, Week 44, n=275, 293 | 1.03 (11.253) | 1.40 (8.008)
  Creatinine, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Creatinine, Week 48, n=265, 292 | 1.59 (11.253) | 0.82 (7.846)

33. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Over Time Including Week 48
Description: Blood samples were collected for the analysis of clinical chemistry parameters which includes total CO2, chloride, glucose, phosphate, potassium, sodium and urea. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Millimoles per liter
  CO2, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  CO2, Week 4, n=301, 303 | 1.0 (2.53) | 0.7 (2.21)
  CO2, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  CO2, Week 8, n=229, 303 | 0.4 (2.31) | 0.6 (2.52)
  CO2, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  CO2, Week 12, n=295, 299 | 0.5 (2.42) | 0.3 (2.39)
  CO2, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  CO2, Week 16, n=284, 298 | 0.3 (2.42) | 0.5 (2.41)
  CO2, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  CO2, Week 20, n=277, 302 | 0.2 (2.26) | 0.3 (2.31)
  CO2, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  CO2, Week 24, n=284, 298 | 0.2 (2.46) | 0.2 (2.44)
  CO2, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  CO2, Week 28, n=267, 296 | 0.1 (2.47) | 0.1 (2.39)
  CO2, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  CO2, Week 32, n=275, 294 | 0.0 (2.37) | 0.2 (2.31)
  CO2, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  CO2, Week 36, n=273, 292 | 0.2 (2.37) | 0.3 (2.39)
  CO2, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  CO2, Week 40, n=270, 293 | 0.5 (2.49) | 0.4 (2.29)
  CO2, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  CO2, Week 44, n=275, 293 | 0.5 (2.34) | 0.5 (2.19)
  CO2, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  CO2, Week 48, n=265, 292 | 0.1 (2.41) | 0.2 (2.31)
  Chloride, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Chloride, Week 4, n=301, 303 | 0.4 (2.05) | 0.5 (2.13)
  Chloride, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Chloride, Week 8, n=229, 303 | 0.3 (2.12) | 0.5 (2.19)
  Chloride, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Chloride, Week 12, n=295, 299 | 0.4 (2.30) | 0.5 (2.25)
  Chloride, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Chloride, Week 16, n=284, 298 | 0.6 (2.41) | 0.8 (2.25)
  Chloride, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Chloride, Week 20, n=277, 302 | 0.8 (2.32) | 0.8 (2.38)
  Chloride, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Chloride, Week 24, n=284, 299 | 0.6 (2.48) | 0.9 (2.26)
  Chloride, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Chloride, Week 28, n=267, 296 | 0.9 (2.21) | 1.0 (2.55)
  Chloride, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Chloride, Week 32, n=275, 294 | 0.8 (2.41) | 0.9 (2.33)
  Chloride, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Chloride, Week 36, n=273, 292 | 0.9 (2.18) | 0.9 (2.48)
  Chloride, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Chloride, Week 40, n=270, 293 | 0.8 (2.24) | 0.8 (2.76)
  Chloride, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Chloride, Week 44, n=275, 293 | 0.7 (2.20) | 0.8 (2.28)
  Chloride, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Chloride, Week 48, n=265, 292 | 0.5 (2.36) | 0.3 (2.38)
  Glucose, Week 4, n=218, 226: number analyzed (Participants) | 218 | 226
  Glucose, Week 4, n=218, 226 | 0.17 (0.721) | 0.21 (0.900)
  Glucose, Week 8, n=151, 213: number analyzed (Participants) | 151 | 213
  Glucose, Week 8, n=151, 213 | 0.22 (0.841) | 0.22 (0.832)
  Glucose, Week 12, n=204, 216: number analyzed (Participants) | 204 | 216
  Glucose, Week 12, n=204, 216 | 0.19 (0.855) | 0.19 (0.974)
  Glucose, Week 16, n=207, 211: number analyzed (Participants) | 207 | 211
  Glucose, Week 16, n=207, 211 | 0.23 (1.050) | 0.27 (1.084)
  Glucose, Week 20, n=192, 216: number analyzed (Participants) | 192 | 216
  Glucose, Week 20, n=192, 216 | 0.19 (0.712) | 0.19 (0.961)
  Glucose, Week 24, n=212, 224: number analyzed (Participants) | 212 | 224
  Glucose, Week 24, n=212, 224 | 0.23 (0.710) | 0.16 (0.881)
  Glucose, Week 28, n=188, 225: number analyzed (Participants) | 188 | 225
  Glucose, Week 28, n=188, 225 | 0.17 (0.793) | 0.28 (0.903)
  Glucose, Week 32, n=192, 213: number analyzed (Participants) | 192 | 213
  Glucose, Week 32, n=192, 213 | 0.35 (0.956) | 0.27 (0.939)
  Glucose, Week 36, n=190, 215: number analyzed (Participants) | 190 | 215
  Glucose, Week 36, n=190, 215 | 0.18 (0.803) | 0.26 (1.070)
  Glucose, Week 40, n=193, 213: number analyzed (Participants) | 193 | 213
  Glucose, Week 40, n=193, 213 | 0.27 (0.833) | 0.25 (0.891)
  Glucose, Week 44, n=193, 213: number analyzed (Participants) | 193 | 213
  Glucose, Week 44, n=193, 213 | 0.23 (0.895) | 0.27 (0.898)
  Glucose, Week 48, n=238, 274: number analyzed (Participants) | 238 | 274
  Glucose, Week 48, n=238, 274 | 0.04 (0.693) | 0.02 (0.924)
  Phosphate, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Phosphate, Week 4, n=301, 303 | 0.066 (0.1666) | 0.015 (0.1595)
  Phosphate, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Phosphate, Week 8, n=229, 303 | 0.062 (0.1862) | -0.006 (0.1609)
  Phosphate, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Phosphate, Week 12, n=295, 299 | 0.041 (0.1978) | 0.013 (0.1742)
  Phosphate, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Phosphate, Week 16, n=284, 298 | 0.041 (0.2012) | 0.003 (0.1640)
  Phosphate, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Phosphate, Week 20, n=277, 302 | 0.035 (0.1871) | 0.010 (0.1839)
  Phosphate, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Phosphate, Week 24, n=284, 299 | 0.042 (0.1963) | 0.006 (0.1845)
  Phosphate, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Phosphate, Week 28, n=267, 296 | 0.037 (0.1822) | 0.004 (0.1823)
  Phosphate, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Phosphate, Week 32, n=275, 294 | 0.021 (0.1980) | 0.005 (0.1886)
  Phosphate, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Phosphate, Week 36, n=273, 292 | 0.011 (0.1846) | -0.002 (0.1855)
  Phosphate, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Phosphate, Week 40, n=270, 293 | 0.024 (0.2035) | -0.004 (0.1736)
  Phosphate, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Phosphate, Week 44, n=275, 293 | 0.027 (0.1982) | 0.004 (0.1811)
  Phosphate, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Phosphate, Week 48, n=265, 292 | 0.034 (0.2007) | 0.003 (0.1741)
  Potassium, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Potassium, Week 4, n=301, 303 | 0.05 (0.342) | 0.11 (0.375)
  Potassium, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Potassium, Week 8, n=229, 303 | 0.01 (0.311) | 0.06 (0.393)
  Potassium, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Potassium, Week 12, n=295, 299 | 0.04 (0.341) | 0.08 (0.356)
  Potassium, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Potassium, Week 16, n=284, 298 | 0.01 (0.341) | 0.06 (0.340)
  Potassium, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Potassium, Week 20, n=277, 302 | 0.04 (0.345) | 0.05 (0.359)
  Potassium, Week 24, n=284, 298: number analyzed (Participants) | 284 | 298
  Potassium, Week 24, n=284, 298 | 0.03 (0.325) | 0.07 (0.337)
  Potassium, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Potassium, Week 28, n=267, 296 | 0.04 (0.380) | 0.07 (0.389)
  Potassium, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Potassium, Week 32, n=275, 294 | 0.02 (0.390) | 0.05 (0.347)
  Potassium, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Potassium, Week 36, n=273, 292 | 0.03 (0.356) | 0.07 (0.359)
  Potassium, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Potassium, Week 40, n=270, 293 | 0.04 (0.344) | 0.07 (0.350)
  Potassium, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Potassium, Week 44, n=275, 293 | 0.06 (0.344) | 0.07 (0.372)
  Potassium, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Potassium, Week 48, n=265, 292 | -0.02 (0.299) | 0.00 (0.332)
  Sodium, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Sodium, Week 4, n=301, 303 | 0.3 (1.84) | 0.1 (1.99)
  Sodium, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Sodium, Week 8, n=229, 303 | 0.2 (1.99) | -0.1 (1.92)
  Sodium, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Sodium, Week 12, n=295, 299 | 0.2 (2.07) | 0.2 (1.91)
  Sodium, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Sodium, Week 16, n=284, 298 | 0.1 (2.18) | 0.1 (2.06)
  Sodium, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Sodium, Week 20, n=277, 302 | 0.3 (2.10) | 0.3 (1.95)
  Sodium, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Sodium, Week 24, n=284, 299 | 0.3 (2.07) | 0.2 (1.95)
  Sodium, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Sodium, Week 28, n=267, 296 | 0.5 (2.11) | 0.2 (2.24)
  Sodium, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Sodium, Week 32, n=275, 294 | 0.3 (2.05) | 0.4 (1.89)
  Sodium, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Sodium, Week 36, n=273, 292 | 0.5 (2.01) | 0.5 (2.19)
  Sodium, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Sodium, Week 40, n=270, 293 | 0.4 (2.02) | 0.5 (2.07)
  Sodium, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Sodium, Week 44, n=275, 293 | 0.5 (2.03) | 0.5 (2.05)
  Sodium, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Sodium, Week 48, n=265, 292 | 0.4 (2.20) | 0.3 (1.95)
  Urea, Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Urea, Week 4, n=301, 303 | 0.01 (1.369) | 0.08 (1.334)
  Urea, Week 8, n=229, 303: number analyzed (Participants) | 229 | 303
  Urea, Week 8, n=229, 303 | 0.07 (1.453) | 0.00 (1.363)
  Urea, Week 12, n=295, 299: number analyzed (Participants) | 295 | 299
  Urea, Week 12, n=295, 299 | 0.15 (1.409) | 0.09 (1.381)
  Urea, Week 16, n=284, 298: number analyzed (Participants) | 284 | 298
  Urea, Week 16, n=284, 298 | 0.08 (1.387) | 0.19 (1.496)
  Urea, Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Urea, Week 20, n=277, 302 | 0.15 (1.399) | 0.11 (1.461)
  Urea, Week 24, n=284, 299: number analyzed (Participants) | 284 | 299
  Urea, Week 24, n=284, 299 | 0.25 (1.420) | 0.15 (1.311)
  Urea, Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Urea, Week 28, n=267, 296 | 0.15 (1.524) | 0.00 (1.439)
  Urea, Week 32, n=275, 294: number analyzed (Participants) | 275 | 294
  Urea, Week 32, n=275, 294 | 0.20 (1.511) | 0.06 (1.415)
  Urea, Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Urea, Week 36, n=273, 292 | 0.06 (1.420) | -0.02 (1.386)
  Urea, Week 40, n=270, 293: number analyzed (Participants) | 270 | 293
  Urea, Week 40, n=270, 293 | 0.19 (1.400) | 0.09 (1.452)
  Urea, Week 44, n=275, 293: number analyzed (Participants) | 275 | 293
  Urea, Week 44, n=275, 293 | 0.13 (1.426) | 0.02 (1.467)
  Urea, Week 48, n=265, 292: number analyzed (Participants) | 265 | 292
  Urea, Week 48, n=265, 292 | 0.24 (1.465) | -0.01 (1.312)

34. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter Over Time Including Week 48: Lipase
Description: Blood samples were collected for the analysis of clinical chemistry parameter-lipase. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Units per liter
  Week 4, n=301, 303: number analyzed (Participants) | 301 | 303
  Week 4, n=301, 303 | 5.2 (41.42) | 1.5 (23.88)
  Week 8, n=227, 303: number analyzed (Participants) | 227 | 303
  Week 8, n=227, 303 | 1.2 (19.31) | 1.0 (17.96)
  Week 12, n=294, 297: number analyzed (Participants) | 294 | 297
  Week 12, n=294, 297 | 2.7 (25.12) | -0.8 (18.59)
  Week 16, n=285, 299: number analyzed (Participants) | 285 | 299
  Week 16, n=285, 299 | 2.6 (24.79) | 3.5 (31.03)
  Week 20, n=278, 302: number analyzed (Participants) | 278 | 302
  Week 20, n=278, 302 | 0.9 (15.65) | 0.8 (28.95)
  Week 24, n=283, 299: number analyzed (Participants) | 283 | 299
  Week 24, n=283, 299 | 2.1 (20.79) | 3.0 (23.85)
  Week 28, n=267, 297: number analyzed (Participants) | 267 | 297
  Week 28, n=267, 297 | 2.2 (24.93) | 2.3 (18.96)
  Week 32, n=274, 294: number analyzed (Participants) | 274 | 294
  Week 32, n=274, 294 | 5.2 (57.44) | 3.1 (21.31)
  Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Week 36, n=273, 292 | 5.1 (49.92) | 0.7 (17.39)
  Week 40, n=269, 293: number analyzed (Participants) | 269 | 293
  Week 40, n=269, 293 | 5.1 (33.58) | 0.5 (17.60)
  Week 44, n=274, 293: number analyzed (Participants) | 274 | 293
  Week 44, n=274, 293 | 2.0 (22.57) | 2.3 (21.13)
  Week 48, n=264, 290: number analyzed (Participants) | 264 | 290
  Week 48, n=264, 290 | 3.0 (28.26) | 1.5 (19.00)

35. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter Over Time Including Week 48: Creatinine Clearance.
Description: Blood samples were collected for the analysis of clinical chemistry parameter-creatinine clearance. GFR will be estimated by the central laboratory using the CKD-EPI. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliters per minute per 1.73meter^2
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Milliliters per minute per 1.73meter^2
  Week 4, n=301, 301: number analyzed (Participants) | 301 | 301
  Week 4, n=301, 301 | -1.8 (9.51) | -2.3 (9.18)
  Week 8, n=227, 303: number analyzed (Participants) | 227 | 303
  Week 8, n=227, 303 | 0.4 (9.88) | -1.5 (8.06)
  Week 12, n=295, 297: number analyzed (Participants) | 295 | 297
  Week 12, n=295, 297 | 0.3 (10.28) | -1.9 (8.02)
  Week 16, n=284, 297: number analyzed (Participants) | 284 | 297
  Week 16, n=284, 297 | 0.4 (10.63) | -1.9 (8.69)
  Week 20, n=277, 302: number analyzed (Participants) | 277 | 302
  Week 20, n=277, 302 | -1.0 (10.37) | -2.4 (8.55)
  Week 24, n=283, 298: number analyzed (Participants) | 283 | 298
  Week 24, n=283, 298 | -1.0 (10.52) | -2.3 (8.76)
  Week 28, n=267, 296: number analyzed (Participants) | 267 | 296
  Week 28, n=267, 296 | -1.8 (11.47) | -2.4 (8.93)
  Week 32, n=274, 294: number analyzed (Participants) | 274 | 294
  Week 32, n=274, 294 | -1.2 (11.11) | -3.0 (8.94)
  Week 36, n=273, 292: number analyzed (Participants) | 273 | 292
  Week 36, n=273, 292 | -1.2 (11.26) | -2.6 (8.52)
  Week 40, n=268, 293: number analyzed (Participants) | 268 | 293
  Week 40, n=268, 293 | -1.7 (10.70) | -2.7 (9.10)
  Week 44, n=274, 293: number analyzed (Participants) | 274 | 293
  Week 44, n=274, 293 | -2.1 (10.45) | -2.3 (8.74)
  Week 48, n=264, 291: number analyzed (Participants) | 264 | 291
  Week 48, n=264, 291 | -2.5 (11.80) | -1.9 (8.50)

36. Secondary Outcome: Change From Baseline Values for Fasting Lipid Panel Over Time Including Week 48
Description: Blood samples were collected for the analysis of fasting lipid parameters- total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Millimoles per liter
  Total cholesterol, Week 48, n=231, 242: number analyzed (Participants) | 231 | 242
  Total cholesterol, Week 48, n=231, 242 | 0.08 (0.688) | -0.04 (0.665)
  HDL cholesterol, Week 48, n=231, 242: number analyzed (Participants) | 231 | 242
  HDL cholesterol, Week 48, n=231, 242 | 0.040 (0.2702) | 0.002 (0.2682)
  LDL cholesterol, Week 48, n=224, 238: number analyzed (Participants) | 224 | 238
  LDL cholesterol, Week 48, n=224, 238 | 0.098 (0.6105) | -0.017 (0.5314)
  Triglycerides, Week 48, n=231, 242: number analyzed (Participants) | 231 | 242
  Triglycerides, Week 48, n=231, 242 | -0.159 (0.8670) | -0.033 (0.7844)

37. Secondary Outcome: Change From Baseline Values in Urine Albumin/Creatinine Ratio and Urine Protein/Creatinine Ratio Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine albumin/creatinine ratio and urine protein/creatinine ratio.Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per mole
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Grams per mole
  Urine albumin/creatinine ratio, Week 4,n=210, 221: number analyzed (Participants) | 210 | 221
  Urine albumin/creatinine ratio, Week 4,n=210, 221 | 0.32 (3.948) | 0.06 (6.383)
  Urine albumin/creatinine ratio, Week 24,n=198, 208: number analyzed (Participants) | 198 | 208
  Urine albumin/creatinine ratio, Week 24,n=198, 208 | -0.08 (3.360) | -0.11 (8.552)
  Urine albumin/creatinine ratio, Week 48,n=191, 197: number analyzed (Participants) | 191 | 197
  Urine albumin/creatinine ratio, Week 48,n=191, 197 | 0.15 (6.049) | -0.14 (5.286)
  Urine protein/creatinine, Week 4, n=234, 236: number analyzed (Participants) | 234 | 236
  Urine protein/creatinine, Week 4, n=234, 236 | -0.66 (11.803) | 1.85 (31.997)
  Urine protein/creatinine, Week 24, n=208, 232: number analyzed (Participants) | 208 | 232
  Urine protein/creatinine, Week 24, n=208, 232 | -2.49 (8.028) | 1.67 (20.505)
  Urine protein/creatinine, Week 48, n=206, 225: number analyzed (Participants) | 206 | 225
  Urine protein/creatinine, Week 48, n=206, 225 | -1.72 (9.551) | 6.70 (112.353)

38. Secondary Outcome: Change From Baseline Values in Urine Creatinine Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine creatinine. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Micromoles per liter
  Week 4, n=304, 302: number analyzed (Participants) | 304 | 302
  Week 4, n=304, 302 | -543.9 (8693.94) | -305.5 (8787.62)
  Week 24, n=282, 297: number analyzed (Participants) | 282 | 297
  Week 24, n=282, 297 | -341.8 (9286.26) | -270.4 (8437.76)
  Week 48, n=282, 291: number analyzed (Participants) | 282 | 291
  Week 48, n=282, 291 | -342.9 (8965.01) | -521.6 (7873.28)

39. Secondary Outcome: Change From Baseline Values in Urine Phosphate Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine phosphate. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Millimoles per liter
  Week 4, n=302, 300: number analyzed (Participants) | 302 | 300
  Week 4, n=302, 300 | -0.460 (15.2707) | 1.483 (15.0378)
  Week 24, n=281, 294: number analyzed (Participants) | 281 | 294
  Week 24, n=281, 294 | 0.286 (16.1887) | 0.640 (14.4201)
  Week 48, n=280, 291: number analyzed (Participants) | 280 | 291
  Week 48, n=280, 291 | -0.369 (14.2441) | 1.254 (15.6532)

40. Secondary Outcome: Change From Baseline Values in Urine Retinol Binding Protein Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine retinol binding protein. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Week 48
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 275 | 284
Nanomoles per liter | -1.8913 (14.10125) | 1.4289 (15.70559)

41. Secondary Outcome: Change From Baseline Values in Urine Specific Gravity Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The dipstick test gives results in a semi-quantitative manner. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value. The urine specific gravity was measured as the ratio of urine density compared with water density.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Ratio of urine density to water density
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Ratio of urine density to water density
  Week 4, n=298, 295: number analyzed (Participants) | 298 | 295
  Week 4, n=298, 295 | -0.0009 (0.00800) | -0.0000 (0.00785)
  Week 24, n=274, 291: number analyzed (Participants) | 274 | 291
  Week 24, n=274, 291 | -0.0008 (0.00784) | -0.0000 (0.00770)
  Week 48, n=274, 283: number analyzed (Participants) | 274 | 283
  Week 48, n=274, 283 | -0.0009 (0.00772) | -0.0002 (0.00768)

42. Secondary Outcome: Change From Baseline Values in Urine pH Over Time Including Week 48
Description: Urine samples were collected for analysis of urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0). The dipstick test gives results in a semi-quantitative manner. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
pH
  Week 4, n=298, 295: number analyzed (Participants) | 298 | 295
  Week 4, n=298, 295 | 0.08 (0.886) | -0.13 (0.935)
  Week 24, n=274, 291: number analyzed (Participants) | 274 | 291
  Week 24, n=274, 291 | 0.18 (1.021) | 0.01 (0.870)
  Week 48, n=274, 283: number analyzed (Participants) | 274 | 283
  Week 48, n=274, 283 | 0.09 (1.036) | -0.02 (0.951)

43. Secondary Outcome: Number of Participants Who Discontinued or Withdrawn Due to AEs Over Time Including Week 48
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Time Frame: Up to Week 48
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants | 13 | 5

44. Secondary Outcome: Percentage Change From Baseline in Fasting Lipids Overtime Including Week 48
Description: Blood samples were collected at Baseline and at Week 48 to assess fasting lipids which included total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Percentage change from Baseline is calculated as: value at Week 48 minus Baseline value divided by Baseline value multiplied by 100.
Time Frame: Baseline (Day 1) and at Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Percent change
  Cholesterol, Week 48, Overall, n=231, 242: number analyzed (Participants) | 231 | 242
  Cholesterol, Week 48, Overall, n=231, 242 | 3.25 (15.563) | 0.13 (13.379)
  HDL cholesterol, Week 48, Overall, n=231, 242: number analyzed (Participants) | 231 | 242
  HDL cholesterol, Week 48, Overall, n=231, 242 | 5.059 (20.5368) | 2.132 (18.0473)
  LDL cholesterol, Week 48, Overall, n=224, 238: number analyzed (Participants) | 224 | 238
  LDL cholesterol, Week 48, Overall, n=224, 238 | 6.762 (31.7209) | 1.029 (19.4719)
  Triglycerides, Week 48, Overall, n=231, 242: number analyzed (Participants) | 231 | 242
  Triglycerides, Week 48, Overall, n=231, 242 | 0.708 (43.5160) | 8.203 (51.7632)

45. Secondary Outcome: Number of Participants With Phenotypic Resistance Through Week 48
Description: Plasma samples were collected and analyzed from participants who met confirmed virologic withdrawal criteria.The CVF population comprised of all participants in ITT-E population who met CVF criteria.Phenotypic Resistance data for following drugs:CAB,dolutegravir(DTG),elvitegravir(EVG), raltegravir(RAL),delavirdine(DLV),efavirenz(EFV),etravirine(ETR),nevirapine(NVP),RPV,lamivudine(3TC),abacavir(ABC),emtricitabine(FTC),tenofovir(TDF),zidovudine(ZDV),stavudine(d4T),didanosine(ddI), atazanavir(ATV),darunavir(DRV),fosamprenavir(FPV),indinavir(IDV),lopinavir(LPV),nelfinavir(NFV),rito-navir(RTV),saquinavir(SQV) and tipranavir(TPV) in participants meeting CVF criteria is presented.Phenotypic resistance, partially sensitive, and Sensitive were defined based on fold change(FC) value from Monogram as:resistance(FC>clinical higher cutoff/biologic cutoff),partially sensitive(FC <=clinical higher cutoff and > clinical lower cutoff),sensitive(FC <= clinical lower cutoff/biologic cutoff).
Time Frame: At the time of CVF
Population: CVF Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 3 | 4
Participants
  INI, CAB, resistant, n=3, 4 | 1 | 0
  INI, CAB, sensitive, n=3, 4 | 2 | 4
  INI, DTG, resistant, n=3, 4 | 0 | 0
  INI, DTG, partially sensitive, n=3, 4 | 0 | 0
  INI, DTG, sensitive, n=3, 4 | 3 | 4
  INI, EVG, resistant, n=3, 4 | 1 | 0
  INI, EVG, sensitive, n=3, 4 | 2 | 4
  INI, RAL, resistant, n=3, 4 | 1 | 0
  INI, RAL, sensitive, n=3, 4 | 2 | 4
  NNRTI, DLV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, DLV, resistant, n=3, 3 | 2 | 0
  NNRTI, DLV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, DLV, sensitive, n=3, 3 | 1 | 3
  NNRTI, EFV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, EFV, resistant, n=3, 3 | 2 | 0
  NNRTI, EFV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, EFV, sensitive, n=3, 3 | 1 | 3
  NNRTI, ETR, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, ETR, resistant, n=3, 3 | 0 | 0
  NNRTI, ETR, partially sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, ETR, partially sensitive, n=3, 3 | 2 | 0
  NNRTI, ETR, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, ETR, sensitive, n=3, 3 | 1 | 3
  NNRTI, NVP, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, NVP, resistant, n=3, 3 | 2 | 0
  NNRTI, NVP, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, NVP, sensitive, n=3, 3 | 1 | 3
  NNRTI, RPV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, RPV, resistant, n=3, 3 | 3 | 0
  NNRTI, RPV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NNRTI, RPV, sensitive, n=3, 3 | 0 | 3
  NRTI, 3TC, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, 3TC, resistant, n=3, 3 | 0 | 1
  NRTI, 3TC, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, 3TC, sensitive, n=3, 3 | 3 | 2
  NRTI, ABC, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, ABC, resistant, n=3, 3 | 0 | 0
  NRTI, ABC, partially sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, ABC, partially sensitive, n=3, 3 | 0 | 0
  NRTI, ABC, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, ABC, sensitive, n=3, 3 | 3 | 3
  NRTI, FTC, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, FTC, resistant, n=3, 3 | 0 | 1
  NRTI, FTC, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, FTC, sensitive, n=3, 3 | 3 | 2
  NRTI, TDF, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, TDF, resistant, n=3, 3 | 0 | 0
  NRTI, TDF, partially sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, TDF, partially sensitive, n=3, 3 | 0 | 0
  NRTI, TDF, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, TDF, sensitive, n=3, 3 | 3 | 3
  NRTI, ZDV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, ZDV, resistant, n=3, 3 | 1 | 0
  NRTI, ZDV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, ZDV, sensitive, n=3, 3 | 2 | 3
  NRTI, d4T, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, d4T, resistant, n=3, 3 | 0 | 0
  NRTI, d4T, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, d4T, sensitive, n=3, 3 | 3 | 3
  NRTI, ddI, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, ddI, resistant, n=3, 3 | 0 | 0
  NRTI, ddI, partially sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, ddI, partially sensitive, n=3, 3 | 0 | 0
  NRTI, ddI, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  NRTI, ddI, sensitive, n=3, 3 | 3 | 3
  PI, ATV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, ATV, resistant, n=3, 3 | 0 | 0
  PI, ATV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, ATV, sensitive, n=3, 3 | 3 | 3
  PI, DRV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, DRV, resistant, n=3, 3 | 0 | 0
  PI, DRV, partially sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, DRV, partially sensitive, n=3, 3 | 0 | 0
  PI, DRV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, DRV, sensitive, n=3, 3 | 3 | 3
  PI, FPV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, FPV, resistant, n=3, 3 | 0 | 0
  PI, FPV, partially sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, FPV, partially sensitive, n=3, 3 | 0 | 0
  PI, FPV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, FPV, sensitive, n=3, 3 | 3 | 3
  PI, IDV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, IDV, resistant, n=3, 3 | 0 | 0
  PI, IDV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, IDV, sensitive, n=3, 3 | 3 | 3
  PI, LPV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, LPV, resistant, n=3, 3 | 0 | 0
  PI, LPV, partially sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, LPV, partially sensitive, n=3, 3 | 0 | 0
  PI, LPV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, LPV, sensitive, n=3, 3 | 3 | 3
  PI, NFV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, NFV, resistant, n=3, 3 | 0 | 0
  PI, NFV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, NFV, sensitive, n=3, 3 | 3 | 3
  PI, RTV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, RTV, resistant, n=3, 3 | 0 | 0
  PI, RTV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, RTV, sensitive, n=3, 3 | 3 | 3
  PI, SQV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, SQV, resistant, n=3, 3 | 0 | 0
  PI, SQV, partially sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, SQV, partially sensitive, n=3, 3 | 0 | 0
  PI, SQV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, SQV, sensitive, n=3, 3 | 3 | 3
  PI, TPV, resistant, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, TPV, resistant, n=3, 3 | 0 | 0
  PI, TPV, partially sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, TPV, partially sensitive, n=3, 3 | 0 | 0
  PI, TPV, sensitive, n=3, 3: number analyzed (Participants) | 3 | 3
  PI, TPV, sensitive, n=3, 3 | 3 | 3

46. Secondary Outcome: Number of Participants With Genotypic Resistance Through Week 48
Description: Plasma samples were collected and analyzed from participants who met confirmed virologic withdrawal criteria. Genotypic Resistance data for the following drugs: DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV, DRV, FPV, IDV, LPV, NFV, RTV, SQV and TPV in participants meeting CVF criteria has been presented.
Time Frame: At the time of CVF
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 3 | 4
Participants
  INI, DTG, resistant | 0 | 0
  INI, DTG, resistance possible | 0 | 0
  INI, DTG, sensitive | 3 | 4
  INI, EVG, resistant | 1 | 0
  INI, EVG, resistance possible | 0 | 0
  INI, EVG, sensitive | 2 | 4
  INI, RAL, resistant | 1 | 0
  INI, RAL, resistance possible | 0 | 0
  INI, RAL, sensitive | 2 | 4
  NNRTI, DLV, resistant | 0 | 0
  NNRTI, DLV, resistance possible | 0 | 0
  NNRTI, DLV, sensitive | 3 | 4
  NNRTI, EFV, resistant | 1 | 1
  NNRTI, EFV, resistance possible | 0 | 0
  NNRTI, EFV, sensitive | 2 | 3
  NNRTI, ETR, resistant | 0 | 0
  NNRTI, ETR, resistance possible | 2 | 0
  NNRTI, ETR, sensitive | 1 | 4
  NNRTI, NVP, resistant | 1 | 1
  NNRTI, NVP, resistance possible | 0 | 0
  NNRTI, NVP, sensitive | 2 | 3
  NNRTI, RPV, resistant | 3 | 1
  NNRTI, RPV, resistance possible | 0 | 0
  NNRTI, RPV, sensitive | 0 | 3
  NRTI, 3TC, resistant | 0 | 2
  NNRTI, 3TC, resistance possible | 0 | 0
  NRTI, 3TC, sensitive | 3 | 2
  NRTI, ABC, resistant | 0 | 0
  NRTI, ABC, resistance possible | 0 | 0
  NRTI, ABC, sensitive | 3 | 4
  NRTI, FTC, resistant | 0 | 2
  NRTI, FTC, resistance possible | 0 | 0
  NRTI, FTC, sensitive | 3 | 2
  NRTI, TDF, resistant | 0 | 0
  NRTI, TDF, resistance possible | 0 | 0
  NRTI, TDF, sensitive | 3 | 4
  NRTI, ZDV, resistant | 0 | 0
  NRTI, ZDV, resistance possible | 0 | 0
  NRTI, ZDV, sensitive | 3 | 4
  NRTI, d4T, resistant | 0 | 0
  NRTI, d4T, resistance possible | 0 | 0
  NRTI, d4T, sensitive | 3 | 4
  NRTI, ddI, resistant | 0 | 0
  NRTI, ddI, resistance possible | 0 | 2
  NRTI, ddI, sensitive | 3 | 2
  PI, ATV, resistant | 1 | 0
  PI, ATV, resistance possible | 0 | 0
  PI, ATV, sensitive | 2 | 4
  PI, ATV/r, resistant | 0 | 0
  PI, ATV/r, resistance possible | 1 | 0
  PI, ATV/r, sensitive | 2 | 4
  PI, DRV/r, resistant | 0 | 0
  PI, DRV/r, resistance possible | 0 | 0
  PI, DRV/r, sensitive | 3 | 4
  PI, FPV/r, resistant | 0 | 0
  PI, FPV/r, resistance possible | 0 | 0
  PI, FPV/r, sensitive | 3 | 4
  PI, IDV/r, resistant | 0 | 0
  PI, IDV/r, resistance possible | 0 | 0
  PI, IDV/r, sensitive | 3 | 4
  PI, LPV/r, resistant | 0 | 0
  PI, LPV/r, resistance possible | 0 | 0
  PI, LPV/r, sensitive | 3 | 4
  PI, NFV, resistant | 1 | 0
  PI, NFV, resistance possible | 0 | 0
  PI, NFV, sensitive | 2 | 4
  PI, RTV, resistant | 0 | 0
  PI, RTV, resistance possible | 0 | 0
  PI, RTV, sensitive | 3 | 4
  PI, SQV/r, resistant | 0 | 0
  PI, SQV/r, resistance possible | 0 | 0
  PI, SQV/r, sensitive | 3 | 4
  PI, TPV/r, resistant | 0 | 0
  PI, TPV/r, resistance possible | 0 | 0
  PI, TPV/r, sensitive | 3 | 4

47. Secondary Outcome: Number of Participants With AEs by Using Baseline Third Agent Treatment Class Overtime Including Week 48
Description: as for outcome 43
Time Frame: Up to Week 48
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants
  Any AE, INI, n=102, 99: number analyzed (Participants) | 102 | 99
  Any AE, INI, n=102, 99 | 99 | 68
  Any AE, NNRTI, n=155, 155: number analyzed (Participants) | 155 | 155
  Any AE, NNRTI, n=155, 155 | 148 | 116
  Any AE, PI, n=51, 54: number analyzed (Participants) | 51 | 54
  Any AE, PI, n=51, 54 | 47 | 36

48. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: ALT, ALP, AST and CK
Description: Blood samples were collected for the analysis of clinical chemistry parameters to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI).
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
International units per liter
  PI, ALT, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, ALT, Baseline, n=51, 54 | 19.3 (11.23) | 18.7 (9.13)
  PI, ALT, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, ALT, Week 4, n=51, 53 | 28.7 (20.12) | 19.8 (12.29)
  PI, ALT, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, ALT, Week 8, n=34, 53 | 25.8 (19.28) | 19.6 (10.43)
  PI, ALT, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, ALT, Week 12, n=50, 52 | 24.7 (17.09) | 20.1 (14.19)
  PI, ALT, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, ALT, Week 16, n=48, 53 | 26.3 (19.89) | 20.0 (12.04)
  PI, ALT, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, ALT, Week 20, n=46, 53 | 24.9 (18.46) | 19.0 (9.52)
  PI, ALT, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, ALT, Week 24, n=47, 53 | 24.1 (13.75) | 19.1 (10.02)
  PI, ALT, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, ALT, Week 28, n=42, 53 | 22.0 (12.42) | 19.4 (10.45)
  PI, ALT, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, ALT, Week 32, n=45, 51 | 22.7 (15.18) | 18.8 (8.18)
  PI, ALT, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, ALT, Week 36, n=44, 50 | 22.3 (15.09) | 20.7 (13.18)
  PI, ALT, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, ALT, Week 40, n=42, 51 | 24.9 (19.63) | 19.5 (13.46)
  PI, ALT, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, ALT, Week 44, n=47, 51 | 23.2 (17.05) | 19.3 (14.23)
  PI, ALT, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, ALT, Week 48, n=43, 50 | 22.5 (13.28) | 19.0 (8.52)
  INI, ALT, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, ALT, Baseline, n=102, 99 | 24.8 (15.23) | 21.2 (10.93)
  INI, ALT, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, ALT, Week 4, n=99, 97 | 26.5 (18.35) | 21.7 (10.09)
  INI, ALT, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, ALT, Week 8, n=73, 98 | 28.4 (22.77) | 26.8 (49.37)
  INI, ALT, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, ALT, Week 12, n=99, 95 | 23.8 (14.21) | 22.9 (16.05)
  INI, ALT, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, ALT, Week 16, n=93, 96 | 23.2 (13.62) | 21.2 (11.24)
  INI, ALT, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, ALT, Week 20, n=93, 97 | 23.0 (15.29) | 20.7 (9.83)
  INI, ALT, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, ALT, Week 24, n=94, 95 | 25.7 (20.09) | 21.0 (13.40)
  INI, ALT, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, ALT, Week 28, n=89, 93 | 21.5 (13.06) | 20.9 (14.10)
  INI, ALT, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, ALT, Week 32, n=93, 95 | 22.5 (10.95) | 21.1 (12.32)
  INI, ALT, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, ALT, Week 36, n=94, 95 | 26.5 (38.41) | 20.5 (9.38)
  INI, ALT, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, ALT, Week 40, n=90, 95 | 30.2 (61.80) | 20.6 (9.20)
  INI, ALT, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, ALT, Week 44, n=91, 94 | 23.2 (15.03) | 20.7 (10.01)
  INI, ALT, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, ALT, Week 48, n=91, 95 | 24.4 (17.58) | 20.3 (9.79)
  NNRTI, ALT, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, ALT, Baseline, n=155, 155 | 24.6 (12.67) | 24.4 (14.74)
  NNRTI, ALT, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, ALT, Week 4, n=151, 153 | 21.6 (10.72) | 23.7 (11.16)
  NNRTI, ALT, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, ALT, Week 8, n=122, 152 | 20.8 (10.13) | 23.7 (12.94)
  NNRTI, ALT, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, ALT, Week 12, n=146, 152 | 33.9 (161.81) | 23.6 (11.27)
  NNRTI, ALT, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, ALT, Week 16, n=143, 149 | 23.2 (27.18) | 22.8 (11.06)
  NNRTI, ALT, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, ALT, Week 20, n=138, 152 | 22.6 (27.36) | 22.3 (11.15)
  NNRTI, ALT, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, ALT, Week 24, n=143, 151 | 27.4 (85.70) | 22.9 (12.88)
  NNRTI, ALT, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, ALT, Week 28, n=136, 150 | 20.6 (11.45) | 23.8 (16.00)
  NNRTI, ALT, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, ALT, Week 32, n=137, 148 | 21.1 (12.69) | 23.4 (12.86)
  NNRTI, ALT, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, ALT, Week 36, n=135, 147 | 21.2 (12.38) | 24.1 (13.19)
  NNRTI, ALT, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, ALT, Week 40, n=138, 147 | 20.8 (10.63) | 23.9 (14.24)
  NNRTI, ALT, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, ALT, Week 44, n=137, 148 | 20.0 (9.61) | 23.9 (15.22)
  NNRTI, ALT, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, ALT, Week 48, n=131, 147 | 19.8 (9.62) | 23.5 (12.32)
  PI, ALP, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, ALP, Baseline, n=51, 54 | 73.8 (24.90) | 70.2 (19.56)
  PI, ALP, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, ALP, Week 4, n=51, 53 | 70.4 (20.03) | 67.7 (19.24)
  PI, ALP, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, ALP, Week 8, n=34, 53 | 72.4 (34.86) | 70.9 (23.18)
  PI, ALP, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, ALP, Week 12, n=50, 52 | 68.2 (17.49) | 71.6 (23.60)
  PI, ALP, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, ALP, Week 16, n=48, 53 | 66.9 (15.70) | 71.2 (21.50)
  PI, ALP, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, ALP, Week 20, n=46, 53 | 67.7 (16.36) | 70.8 (20.96)
  PI, ALP, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, ALP, Week 24, n=47, 53 | 67.6 (16.14) | 70.3 (19.23)
  PI, ALP, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, ALP, Week 28, n=42, 53 | 67.3 (17.71) | 73.7 (21.89)
  PI, ALP, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, ALP, Week 32, n=45, 51 | 63.8 (16.09) | 69.8 (21.44)
  PI, ALP, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, ALP, Week 36, n=44, 50 | 64.3 (16.50) | 71.7 (23.57)
  PI, ALP, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, ALP, Week 40, n=42, 51 | 65.5 (13.63) | 68.5 (19.55)
  PI, ALP, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, ALP, Week 44, n=47, 51 | 63.0 (15.76) | 69.1 (20.67)
  PI, ALP, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, ALP, Week 48, n=43, 50 | 63.6 (14.22) | 69.9 (18.94)
  INI, ALP, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, ALP, Baseline, n=102, 99 | 66.3 (17.31) | 64.9 (19.05)
  INI, ALP, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, ALP, Week 4, n=99, 97 | 65.9 (17.25) | 64.4 (18.77)
  INI, ALP, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, ALP, Week 8, n=73, 98 | 64.0 (16.21) | 69.7 (38.92)
  INI, ALP, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, ALP, Week 12, n=99, 95 | 64.7 (16.33) | 67.7 (27.73)
  INI, ALP, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, ALP, Week 16, n=93, 96 | 65.3 (17.01) | 64.4 (20.89)
  INI, ALP, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, ALP, Week 20, n=93, 97 | 64.9 (16.80) | 64.2 (19.58)
  INI, ALP, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, ALP, Week 24, n=94, 95 | 65.0 (17.08) | 64.4 (19.46)
  INI, ALP, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, ALP, Week 28, n=89, 93 | 65.0 (15.81) | 63.3 (18.76)
  INI, ALP, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, ALP, Week 32, n=93, 95 | 64.4 (16.12) | 62.3 (17.96)
  INI, ALP, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, ALP, Week 36, n=94, 95 | 64.3 (18.15) | 62.2 (18.12)
  INI, ALP, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, ALP, Week 40, n=90, 95 | 65.1 (17.07) | 62.2 (18.22)
  INI, ALP, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, ALP, Week 44, n=91, 94 | 64.0 (16.71) | 64.1 (19.31)
  INI, ALP, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, ALP, Week 48, n=91, 95 | 65.1 (15.98) | 63.0 (18.76)
  NNRTI, ALP, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, ALP, Baseline, n=155, 155 | 84.4 (32.47) | 88.1 (28.83)
  NNRTI, ALP, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, ALP, Week 4, n=151, 153 | 73.4 (26.16) | 85.6 (27.39)
  NNRTI, ALP, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, ALP, Week 8, n=122, 152 | 70.9 (20.00) | 87.4 (28.15)
  NNRTI, ALP, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, ALP, Week 12, n=146, 152 | 72.0 (30.68) | 87.8 (28.30)
  NNRTI, ALP, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, ALP, Week 16, n=143, 149 | 69.9 (22.37) | 87.7 (28.55)
  NNRTI, ALP, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, ALP, Week 20, n=138, 152 | 69.3 (20.51) | 86.7 (26.18)
  NNRTI, ALP, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, ALP, Week 24, n=143, 151 | 70.2 (21.08) | 88.3 (27.77)
  NNRTI, ALP, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, ALP, Week 28, n=136, 150 | 69.3 (20.91) | 87.0 (28.40)
  NNRTI, ALP, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, ALP, Week 32, n=137, 148 | 69.1 (21.60) | 86.5 (26.32)
  NNRTI, ALP, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, ALP, Week 36, n=135, 147 | 69.3 (23.22) | 87.1 (26.24)
  NNRTI, ALP, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, ALP, Week 40, n=138, 147 | 67.1 (18.98) | 87.8 (27.07)
  NNRTI, ALP, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, ALP, Week 44, n=137, 148 | 68.4 (19.94) | 87.5 (26.53)
  NNRTI, ALP, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, ALP, Week 48, n=131, 147 | 68.5 (21.69) | 88.6 (27.61)
  PI, AST, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, AST, Baseline, n=51, 54 | 19.7 (6.97) | 20.1 (5.66)
  PI, AST, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, AST, Week 4, n=51, 53 | 23.5 (9.76) | 22.5 (17.53)
  PI, AST, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, AST, Week 8, n=34, 53 | 23.4 (11.04) | 20.0 (5.24)
  PI, AST, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, AST, Week 12, n=50, 52 | 22.5 (11.60) | 21.8 (9.63)
  PI, AST, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, AST, Week 16, n=48, 53 | 23.7 (15.77) | 22.0 (10.39)
  PI, AST, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, AST, Week 20, n=46, 53 | 24.1 (20.53) | 20.6 (6.35)
  PI, AST, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, AST, Week 24, n=47, 53 | 21.5 (7.02) | 21.7 (11.65)
  PI, AST, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, AST, Week 28, n=42, 53 | 22.9 (9.20) | 22.0 (8.47)
  PI, AST, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, AST, Week 32, n=45, 51 | 23.0 (13.51) | 20.3 (5.57)
  PI, AST, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, AST, Week 36, n=44, 50 | 21.5 (7.88) | 21.8 (7.04)
  PI, AST, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, AST, Week 40, n=42, 51 | 25.1 (23.51) | 20.5 (7.55)
  PI, AST, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, AST, Week 44, n=47, 51 | 21.6 (8.80) | 21.4 (13.16)
  PI, AST, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, AST, Week 48, n=43, 50 | 21.6 (7.59) | 22.2 (8.85)
  INI, AST, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, AST, Baseline, n=102, 99 | 24.5 (13.03) | 22.2 (13.13)
  INI, AST, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, AST, Week 4, n=99, 97 | 24.5 (13.22) | 22.0 (10.41)
  INI, AST, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, AST, Week 8, n=73, 98 | 26.8 (25.34) | 23.6 (19.30)
  INI, AST, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, AST, Week 12, n=99, 95 | 23.2 (10.47) | 23.2 (13.10)
  INI, AST, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, AST, Week 16, n=93, 96 | 22.5 (8.78) | 22.5 (9.96)
  INI, AST, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, AST, Week 20, n=93, 97 | 22.8 (10.11) | 21.4 (6.12)
  INI, AST, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, AST, Week 24, n=94, 95 | 24.4 (12.42) | 22.0 (9.44)
  INI, AST, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, AST, Week 28, n=89, 93 | 21.3 (7.14) | 21.6 (8.49)
  INI, AST, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, AST, Week 32, n=93, 95 | 22.2 (7.77) | 21.6 (7.87)
  INI, AST, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, AST, Week 36, n=94, 95 | 23.9 (15.06) | 21.1 (5.43)
  INI, AST, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, AST, Week 40, n=90, 95 | 25.4 (18.01) | 21.8 (7.30)
  INI, AST, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, AST, Week 44, n=91, 94 | 25.6 (23.29) | 21.4 (6.51)
  INI, AST, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, AST, Week 48, n=91, 95 | 24.9 (13.88) | 22.4 (9.70)
  NNRTI, AST, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, AST, Baseline, n=155, 155 | 24.8 (10.99) | 23.6 (9.16)
  NNRTI, AST, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, AST, Week 4, n=151, 153 | 22.2 (11.35) | 23.2 (7.95)
  NNRTI, AST, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, AST, Week 8, n=122, 152 | 23.0 (17.16) | 22.8 (7.19)
  NNRTI, AST, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, AST, Week 12, n=146, 152 | 29.4 (91.34) | 23.6 (9.12)
  NNRTI, AST, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, AST, Week 16, n=143, 149 | 25.3 (22.91) | 22.6 (6.80)
  NNRTI, AST, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, AST, Week 20, n=138, 152 | 23.8 (16.12) | 22.9 (7.33)
  NNRTI, AST, Week 24, n=143, 150: number analyzed (Participants) | 143 | 150
  NNRTI, AST, Week 24, n=143, 150 | 25.1 (30.40) | 23.1 (8.25)
  NNRTI, AST, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, AST, Week 28, n=136, 150 | 22.6 (9.49) | 24.0 (10.53)
  NNRTI, AST, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, AST, Week 32, n=137, 148 | 23.2 (16.69) | 25.1 (15.63)
  NNRTI, AST, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, AST, Week 36, n=135, 147 | 22.8 (8.90) | 23.9 (7.99)
  NNRTI, AST, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, AST, Week 40, n=138, 147 | 22.3 (7.66) | 23.7 (8.01)
  NNRTI, AST, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, AST, Week 44, n=137, 148 | 21.7 (7.11) | 23.8 (10.98)
  NNRTI, AST, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, AST, Week 48, n=131, 147 | 22.0 (7.86) | 24.2 (9.16)
  PI, CK, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, CK, Baseline, n=51, 54 | 121.3 (173.52) | 111.8 (66.03)
  PI, CK, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, CK, Week 4, n=51, 53 | 130.0 (94.61) | 244.2 (908.06)
  PI, CK, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, CK, Week 8, n=34, 53 | 157.7 (174.37) | 134.2 (179.01)
  PI, CK, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, CK, Week 12, n=50, 52 | 124.2 (71.36) | 168.8 (406.86)
  PI, CK, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, CK, Week 16, n=48, 53 | 142.3 (197.96) | 127.0 (82.59)
  PI, CK, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, CK, Week 20, n=46, 53 | 227.9 (689.65) | 117.5 (76.83)
  PI, CK, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, CK, Week 24, n=47, 53 | 120.8 (72.63) | 128.9 (85.38)
  PI, CK, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, CK, Week 28, n=42, 53 | 185.9 (237.49) | 124.2 (96.15)
  PI, CK, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, CK, Week 32, n=45, 51 | 282.5 (959.49) | 110.1 (58.84)
  PI, CK, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, CK, Week 36, n=44, 50 | 115.5 (81.36) | 130.9 (95.59)
  PI, CK, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, CK, Week 40, n=42, 51 | 319.4 (1169.15) | 109.9 (53.99)
  PI, CK, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, CK, Week 44, n=47, 51 | 117.2 (74.25) | 114.4 (62.44)
  PI, CK, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, CK, Week 48, n=43, 50 | 123.5 (90.77) | 183.1 (485.07)
  INI, CK, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, CK, Baseline, n=102, 99 | 257.9 (565.99) | 214.3 (627.94)
  INI, CK, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, CK, Week 4, n=99, 97 | 225.9 (484.50) | 193.6 (415.15)
  INI, CK, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, CK, Week 8, n=73, 98 | 306.8 (791.76) | 158.0 (164.72)
  INI, CK, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, CK, Week 12, n=99, 95 | 242.5 (649.06) | 195.3 (383.74)
  INI, CK, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, CK, Week 16, n=93, 96 | 198.6 (335.16) | 216.4 (422.21)
  INI, CK, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, CK, Week 20, n=93, 97 | 200.9 (301.61) | 158.8 (156.94)
  INI, CK, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, CK, Week 24, n=94, 95 | 202.1 (276.49) | 178.8 (356.60)
  INI, CK, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, CK, Week 28, n=89, 93 | 151.1 (128.42) | 192.6 (463.71)
  INI, CK, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, CK, Week 32, n=93, 95 | 182.2 (202.28) | 175.1 (256.84)
  INI, CK, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, CK, Week 36, n=94, 95 | 190.7 (268.67) | 153.8 (151.29)
  INI, CK, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, CK, Week 40, n=90, 95 | 286.9 (705.76) | 178.2 (200.25)
  INI, CK, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, CK, Week 44, n=91, 94 | 457.7 (2054.68) | 153.6 (139.48)
  INI, CK, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, CK, Week 48, n=91, 95 | 278.9 (651.96) | 188.7 (339.93)
  NNRTI, CK, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, CK, Baseline, n=155, 155 | 180.9 (210.84) | 143.8 (118.05)
  NNRTI, CK, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, CK, Week 4, n=151, 153 | 192.5 (472.95) | 170.1 (226.58)
  NNRTI, CK, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, CK, Week 8, n=122, 152 | 290.4 (1322.89) | 141.1 (106.01)
  NNRTI, CK, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, CK, Week 12, n=146, 152 | 198.5 (430.65) | 168.5 (236.30)
  NNRTI, CK, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, CK, Week 16, n=143, 149 | 326.5 (1157.93) | 150.4 (214.31)
  NNRTI, CK, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, CK, Week 20, n=138, 152 | 247.2 (661.97) | 144.9 (131.72)
  NNRTI, CK, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, CK, Week 24, n=143, 151 | 210.9 (582.66) | 161.5 (182.51)
  NNRTI, CK, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, CK, Week 28, n=136, 150 | 175.0 (156.46) | 197.3 (460.97)
  NNRTI, CK, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, CK, Week 32, n=137, 148 | 218.0 (617.20) | 238.8 (656.12)
  NNRTI, CK, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, CK, Week 36, n=135, 147 | 206.4 (401.19) | 155.5 (134.30)
  NNRTI, CK, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, CK, Week 40, n=138, 147 | 175.6 (156.39) | 166.9 (191.28)
  NNRTI, CK, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, CK, Week 44, n=137, 148 | 148.6 (94.67) | 159.7 (171.66)
  NNRTI, CK, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, CK, Week 48, n=131, 147 | 167.8 (132.83) | 171.3 (256.04)

49. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: Albumin
Description: Blood samples were collected for the analysis of clinical chemistry parameter: albumin to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI).
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Grams per Liter
  PI, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Baseline, n=51, 54 | 43.9 (3.22) | 44.2 (3.36)
  PI, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Week 4, n=51, 53 | 44.1 (2.90) | 43.9 (2.92)
  PI, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Week 8, n=34, 53 | 44.6 (3.36) | 44.1 (3.32)
  PI, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Week 12, n=50, 52 | 43.7 (3.25) | 43.8 (3.56)
  PI, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Week 16, n=48, 53 | 43.8 (3.19) | 43.4 (3.36)
  PI, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Week 20, n=46, 53 | 43.6 (2.70) | 43.3 (3.57)
  PI, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Week 24, n=47, 53 | 43.5 (2.80) | 43.3 (3.09)
  PI, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Week 28, n=42, 53 | 43.5 (2.74) | 42.8 (3.43)
  PI, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Week 32, n=45, 51 | 43.2 (2.85) | 43.7 (3.31)
  PI, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Week 36, n=44, 50 | 43.5 (2.87) | 43.4 (3.02)
  PI, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Week 40, n=42, 51 | 44.2 (2.64) | 43.9 (3.11)
  PI, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Week 44, n=47, 51 | 43.6 (2.58) | 43.9 (3.03)
  PI, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Week 48, n=43, 50 | 43.9 (2.97) | 44.5 (2.44)
  INI, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Baseline, n=102, 99 | 44.3 (3.08) | 44.9 (3.21)
  INI, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Week 4, n=99, 97 | 43.9 (2.91) | 43.8 (2.57)
  INI, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Week 8, n=73, 98 | 43.7 (3.07) | 43.9 (3.10)
  INI, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Week 12, n=99, 95 | 44.1 (3.01) | 44.3 (2.62)
  INI, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Week 16, n=93, 96 | 43.9 (2.77) | 43.7 (2.76)
  INI, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Week 20, n=93, 97 | 43.6 (2.70) | 44.1 (2.87)
  INI, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 24, n=94, 95 | 43.4 (3.03) | 43.9 (3.00)
  INI, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Week 28, n=89, 93 | 44.0 (2.97) | 43.9 (2.87)
  INI, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Week 32, n=93, 95 | 44.1 (2.87) | 43.7 (2.89)
  INI, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 36, n=94, 95 | 43.6 (2.74) | 43.7 (2.60)
  INI, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Week 40, n=90, 95 | 44.1 (2.79) | 43.6 (2.70)
  INI, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Week 44, n=91, 94 | 43.6 (2.96) | 43.8 (2.83)
  INI, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Week 48, n=91, 95 | 44.3 (2.58) | 44.3 (2.73)
  NNRTI, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Baseline, n=155, 155 | 44.1 (3.11) | 44.0 (3.10)
  NNRTI, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Week 4, n=151, 153 | 43.4 (2.83) | 43.7 (3.04)
  NNRTI, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Week 8, n=122, 152 | 43.6 (2.96) | 43.4 (3.16)
  NNRTI, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Week 12, n=146, 152 | 43.3 (2.86) | 43.7 (3.25)
  NNRTI, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Week 16, n=143, 149 | 43.3 (2.61) | 43.3 (3.27)
  NNRTI, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Week 20, n=138, 152 | 43.1 (2.75) | 43.2 (2.98)
  NNRTI, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Week 24, n=143, 151 | 43.4 (2.54) | 43.4 (3.01)
  NNRTI, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Week 28, n=136, 150 | 43.3 (2.78) | 43.2 (3.03)
  NNRTI, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Week 32, n=137, 148 | 43.2 (2.74) | 43.1 (3.43)
  NNRTI, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Week 36, n=135, 147 | 43.0 (2.86) | 43.3 (3.37)
  NNRTI, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Week 40, n=138, 147 | 43.3 (2.66) | 43.1 (3.20)
  NNRTI, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Week 44, n=137, 148 | 43.7 (2.74) | 43.2 (3.13)
  NNRTI, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Week 48, n=131, 147 | 43.4 (2.73) | 43.6 (3.14)

50. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameter: bilirubin, direct bilirubin and creatinine to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI).
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Micromoles per liter
  PI, Bilirubin, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Bilirubin, Baseline, n=51, 54 | 18.3 (20.54) | 13.9 (11.07)
  PI, Bilirubin, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Bilirubin, Week 4, n=51, 53 | 9.3 (3.81) | 14.4 (10.37)
  PI, Bilirubin, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Bilirubin, Week 8, n=34, 53 | 8.9 (3.45) | 14.2 (10.79)
  PI, Bilirubin, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Bilirubin, Week 12, n=50, 52 | 8.1 (3.44) | 15.6 (11.70)
  PI, Bilirubin, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Bilirubin, Week 16, n=48, 53 | 8.7 (3.95) | 14.7 (10.78)
  PI, Bilirubin, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Bilirubin, Week 20, n=46, 53 | 9.3 (3.60) | 15.6 (14.96)
  PI, Bilirubin, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Bilirubin, Week 24, n=47, 53 | 9.5 (3.42) | 16.8 (16.15)
  PI, Bilirubin, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Bilirubin, Week 28, n=42, 53 | 9.4 (4.29) | 15.0 (12.75)
  PI, Bilirubin, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Bilirubin, Week 32, n=45, 51 | 9.7 (3.66) | 17.1 (12.45)
  PI, Bilirubin, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Bilirubin, Week 36, n=44, 50 | 8.3 (3.17) | 16.0 (14.09)
  PI, Bilirubin, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Bilirubin, Week 40, n=42, 51 | 9.2 (3.51) | 17.9 (18.08)
  PI, Bilirubin, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Bilirubin, Week 44, n=47, 51 | 9.5 (3.41) | 18.1 (16.62)
  PI, Bilirubin, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Bilirubin, Week 48, n=43, 50 | 9.3 (3.77) | 16.7 (10.73)
  INI, Bilirubin, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Bilirubin, Baseline, n=102, 99 | 9.4 (3.94) | 9.7 (5.07)
  INI, Bilirubin, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Bilirubin, Week 4, n=99, 97 | 9.5 (3.88) | 9.0 (4.77)
  INI, Bilirubin, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Bilirubin, Week 8, n=73, 98 | 10.1 (4.29) | 10.7 (12.28)
  INI, Bilirubin, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Bilirubin, Week 12, n=99, 95 | 9.9 (4.50) | 9.2 (3.91)
  INI, Bilirubin, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Bilirubin, Week 16, n=93, 96 | 9.8 (4.29) | 9.6 (3.80)
  INI, Bilirubin, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Bilirubin, Week 20, n=93, 97 | 10.1 (4.05) | 9.3 (3.60)
  INI, Bilirubin, Week 24, n=94, 94: number analyzed (Participants) | 94 | 94
  INI, Bilirubin, Week 24, n=94, 94 | 9.4 (4.11) | 9.1 (3.81)
  INI, Bilirubin, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Bilirubin, Week 28, n=89, 93 | 10.3 (3.53) | 9.5 (4.67)
  INI, Bilirubin, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Bilirubin, Week 32, n=93, 95 | 9.9 (4.42) | 8.8 (3.32)
  INI, Bilirubin, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Bilirubin, Week 36, n=94, 95 | 9.8 (4.09) | 9.1 (3.76)
  INI, Bilirubin, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Bilirubin, Week 40, n=90, 95 | 9.9 (4.12) | 8.9 (3.63)
  INI, Bilirubin, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Bilirubin, Week 44, n=91, 94 | 10.1 (4.75) | 9.0 (3.40)
  INI, Bilirubin, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Bilirubin, Week 48, n=91, 95 | 10.3 (4.37) | 8.9 (3.76)
  NNRTI, Bilirubin, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Bilirubin, Baseline, n=155, 155 | 7.4 (3.30) | 7.2 (3.30)
  NNRTI, Bilirubin, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Bilirubin, Week 4, n=151, 153 | 8.7 (4.10) | 6.9 (2.98)
  NNRTI, Bilirubin, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Bilirubin, Week 8, n=122, 152 | 8.9 (4.01) | 6.8 (3.40)
  NNRTI, Bilirubin, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Bilirubin, Week 12, n=146, 152 | 9.3 (4.66) | 7.1 (3.50)
  NNRTI, Bilirubin, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Bilirubin, Week 16, n=143, 149 | 10.5 (14.51) | 6.8 (3.52)
  NNRTI, Bilirubin, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Bilirubin, Week 20, n=138, 152 | 9.6 (4.63) | 7.1 (3.15)
  NNRTI, Bilirubin, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Bilirubin, Week 24, n=143, 151 | 9.1 (3.93) | 6.9 (3.75)
  NNRTI, Bilirubin, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Bilirubin, Week 28, n=136, 150 | 9.7 (4.17) | 6.9 (3.29)
  NNRTI, Bilirubin, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Bilirubin, Week 32, n=137, 148 | 9.7 (4.55) | 6.9 (3.52)
  NNRTI, Bilirubin, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Bilirubin, Week 36, n=135, 147 | 9.3 (3.72) | 7.0 (3.33)
  NNRTI, Bilirubin, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Bilirubin, Week 40, n=138, 147 | 9.6 (4.21) | 7.0 (3.43)
  NNRTI, Bilirubin, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Bilirubin, Week 44, n=137, 148 | 9.4 (4.03) | 7.1 (3.25)
  NNRTI, Bilirubin, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Bilirubin, Week 48, n=131, 147 | 9.4 (4.28) | 7.3 (3.19)
  PI, Direct bilirubin, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Direct bilirubin, Baseline, n=51, 54 | 3.6 (2.13) | 2.9 (1.68)
  PI, Direct bilirubin, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Direct bilirubin, Week 4, n=51, 53 | 2.4 (1.20) | 3.3 (1.67)
  PI, Direct bilirubin, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Direct bilirubin, Week 8, n=34, 53 | 2.3 (1.12) | 2.8 (1.68)
  PI, Direct bilirubin, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Direct bilirubin, Week 12, n=50, 52 | 1.9 (0.80) | 3.2 (1.95)
  PI, direct bilirubin, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, direct bilirubin, Week 16, n=48, 53 | 2.0 (0.87) | 2.9 (1.45)
  PI, Direct bilirubin, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Direct bilirubin, Week 20, n=46, 53 | 2.2 (0.79) | 2.9 (2.17)
  PI, Direct bilirubin, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Direct bilirubin, Week 24, n=47, 53 | 2.2 (0.75) | 3.1 (2.02)
  PI, Direct bilirubin, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Direct bilirubin, Week 28, n=42, 53 | 2.1 (1.08) | 2.7 (1.84)
  PI, Direct bilirubin, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Direct bilirubin, Week 32, n=45, 51 | 2.2 (0.88) | 3.1 (1.84)
  PI, Direct bilirubin, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Direct bilirubin, Week 36, n=44, 50 | 1.9 (0.80) | 3.1 (1.95)
  PI, Direct bilirubin, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Direct bilirubin, Week 40, n=42, 51 | 2.0 (0.77) | 3.2 (2.05)
  PI, Direct bilirubin, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Direct bilirubin, Week 44, n=47, 51 | 2.1 (0.83) | 3.3 (1.99)
  PI, Direct bilirubin, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Direct bilirubin, Week 48, n=43, 50 | 2.3 (0.93) | 3.2 (1.71)
  INI, Direct bilirubin, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Direct bilirubin, Baseline, n=102, 99 | 2.4 (0.96) | 2.3 (1.16)
  INI, Direct bilirubin, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Direct bilirubin, Week 4, n=99, 97 | 2.4 (0.90) | 2.3 (1.18)
  INI, Direct bilirubin, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Direct bilirubin, Week 8, n=73, 98 | 2.4 (1.02) | 3.0 (6.70)
  INI, Direct bilirubin, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Direct bilirubin, Week 12, n=99, 95 | 2.3 (0.98) | 2.3 (1.06)
  INI, Direct bilirubin, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Direct bilirubin, Week 16, n=93, 96 | 2.3 (1.03) | 2.1 (0.87)
  INI, Direct bilirubin, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Direct bilirubin, Week 20, n=93, 97 | 2.2 (0.85) | 2.1 (0.89)
  INI, Direct bilirubin, Week 24, n=94, 94: number analyzed (Participants) | 94 | 94
  INI, Direct bilirubin, Week 24, n=94, 94 | 2.2 (1.02) | 2.0 (0.78)
  INI, Direct bilirubin, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Direct bilirubin, Week 28, n=89, 93 | 2.2 (0.74) | 2.1 (1.12)
  INI, Direct bilirubin, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Direct bilirubin, Week 32, n=93, 95 | 2.2 (0.94) | 1.9 (0.77)
  INI, Direct bilirubin, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Direct bilirubin, Week 36, n=94, 95 | 2.2 (1.25) | 2.0 (0.97)
  INI, Direct bilirubin, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Direct bilirubin, Week 40, n=90, 95 | 2.2 (1.06) | 2.0 (1.11)
  INI, Direct bilirubin. Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Direct bilirubin. Week 44, n=91, 94 | 2.3 (0.99) | 2.1 (0.95)
  INI, Direct bilirubin, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Direct bilirubin, Week 48, n=91, 95 | 2.3 (0.82) | 2.2 (1.00)
  NNRTI, Direct bilirubin, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Direct bilirubin, Baseline, n=155, 155 | 2.1 (1.00) | 1.9 (1.00)
  NNRTI, Direct bilirubin, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Direct bilirubin, Week 4, n=151, 153 | 2.2 (1.06) | 2.0 (0.96)
  NNRTI, Direct bilirubin, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Direct bilirubin, Week 8, n=122, 152 | 2.2 (1.10) | 1.9 (0.97)
  NNRTI, Direct bilirubin, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Direct bilirubin, Week 12, n=146, 152 | 2.2 (1.12) | 1.9 (0.98)
  NNRTI, Direct bilirubin, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Direct bilirubin, Week 16, n=143, 149 | 2.7 (6.95) | 1.9 (0.90)
  NNRTI, Direct bilirubin, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Direct bilirubin, Week 20, n=138, 152 | 2.2 (1.07) | 1.7 (0.97)
  NNRTI, Week 24, Direct bilirubin, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Week 24, Direct bilirubin, n=143, 151 | 2.1 (1.04) | 1.8 (0.95)
  NNRTI, Direct bilirubin, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Direct bilirubin, Week 28, n=136, 150 | 2.1 (1.01) | 1.7 (1.01)
  NNRTI, Direct bilirubin, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Direct bilirubin, Week 32, n=137, 148 | 2.1 (1.08) | 1.7 (0.94)
  NNRTI, Direct bilirubin, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Direct bilirubin, Week 36, n=135, 147 | 2.1 (1.10) | 1.7 (0.94)
  NNRTI, Direct bilirubin, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Direct bilirubin, Week 40, n=138, 147 | 2.1 (1.18) | 1.7 (1.00)
  NNRTI, Direct bilirubin, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Direct bilirubin, Week 44, n=137, 148 | 2.1 (0.96) | 1.8 (0.91)
  NNRTI, Direct bilirubin, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Direct bilirubin, Week 48, n=131, 147 | 2.2 (0.98) | 1.9 (0.96)
  PI, Creatinine, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Creatinine, Baseline, n=51, 54 | 71.41 (12.315) | 70.20 (13.391)
  PI, Creatinine, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Creatinine, Week 4, n=51, 53 | 72.87 (11.632) | 72.53 (14.574)
  PI, Creatinine, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Creatinine, Week 8, n=34, 53 | 71.66 (13.012) | 71.54 (14.362)
  PI, Creatinine, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Creatinine, Week 12, n=50, 52 | 70.05 (11.609) | 73.22 (14.968)
  PI, Creatinine, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Creatinine, Week 16, n=48, 53 | 71.05 (11.778) | 73.25 (15.740)
  PI, Creatinine, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Creatinine, Week 20, n=46, 53 | 73.40 (12.191) | 75.37 (15.799)
  PI, Creatinine, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Creatinine, Week 24, n=47, 53 | 72.75 (11.654) | 72.84 (14.549)
  PI, Creatinine, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Creatinine, Week 28, n=42, 53 | 75.18 (13.118) | 73.42 (14.738)
  PI, Creatinine, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Creatinine, Week 32, n=45, 51 | 74.59 (13.730) | 73.93 (15.399)
  PI, Creatinine, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Creatinine, Week 36, n=44, 50 | 74.41 (12.217) | 72.37 (14.570)
  PI, Creatinine, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Creatinine, Week 40, n=42, 51 | 74.31 (11.749) | 73.73 (15.726)
  PI, Creatinine, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Creatinine, Week 44, n=47, 51 | 75.38 (13.405) | 73.00 (14.885)
  PI, Creatinine, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Creatinine, Week 48, n=43, 50 | 76.95 (13.021) | 72.21 (15.031)
  INI, Creatinine, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Creatinine, Baseline, n=102, 99 | 88.16 (16.835) | 86.34 (17.320)
  INI, Creatinine, Week 4, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Creatinine, Week 4, n=99, 95 | 86.39 (14.472) | 87.66 (16.208)
  INI, Creatinine, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Creatinine, Week 8, n=73, 98 | 85.52 (15.851) | 88.11 (17.308)
  INI, Creatinine, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Creatinine, Week 12, n=99, 95 | 85.53 (17.539) | 89.36 (17.923)
  INI, Creatinine, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Creatinine, Week 16, n=93, 96 | 84.99 (15.429) | 86.85 (17.320)
  INI, Creatinine, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Creatinine, Week 20, n=93, 97 | 85.01 (14.695) | 87.06 (16.987)
  INI, Creatinine, Week 24, n=94, 94: number analyzed (Participants) | 94 | 94
  INI, Creatinine, Week 24, n=94, 94 | 84.21 (15.039) | 87.02 (16.777)
  INI, Creatinine, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Creatinine, Week 28, n=89, 93 | 84.84 (15.670) | 87.41 (17.065)
  INI, Creatinine, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Creatinine, Week 32, n=93, 95 | 85.42 (15.349) | 86.91 (15.628)
  INI, Creatinine, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Creatinine, Week 36, n=94, 95 | 84.49 (15.189) | 87.20 (15.835)
  INI, Creatinine, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Creatinine, Week 40, n=90, 95 | 85.92 (14.651) | 87.70 (17.119)
  INI, Creatinine, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Creatinine, Week 44, n=91, 94 | 84.66 (15.701) | 87.08 (16.694)
  INI, Creatinine, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Creatinine, Week 48, n=91, 95 | 85.27 (15.683) | 86.64 (15.958)
  NNRTI, Creatinine, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Creatinine, Baseline, n=155, 155 | 75.57 (14.604) | 75.06 (14.671)
  NNRTI, Creatinine, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Creatinine, Week 4, n=151, 153 | 78.57 (15.814) | 76.79 (14.908)
  NNRTI, Creatinine, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Creatinine, Week 8, n=122, 152 | 76.75 (15.759) | 76.17 (14.876)
  NNRTI, Creatinine, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Creatinine, Week 12, n=146, 152 | 76.93 (15.495) | 75.50 (14.723)
  NNRTI, Creatinine, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Creatinine, Week 16, n=143, 149 | 77.22 (15.406) | 77.00 (16.025)
  NNRTI, Creatinine, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Creatinine, Week 20, n=138, 152 | 78.32 (16.372) | 76.36 (15.744)
  NNRTI, Creatinine, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Creatinine, Week 24, n=143, 151 | 79.92 (21.430) | 76.26 (15.534)
  NNRTI, Creatinine, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Creatinine, Week 28, n=136, 150 | 79.13 (17.039) | 76.45 (15.060)
  NNRTI, Creatinine, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Creatinine, Week 32, n=137, 148 | 77.40 (14.117) | 77.05 (16.200)
  NNRTI, Creatinine, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Creatinine, Week 36, n=135, 147 | 78.15 (16.839) | 76.64 (15.734)
  NNRTI, Creatinine, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Creatinine, Week 40, n=138, 147 | 78.42 (16.662) | 76.04 (15.083)
  NNRTI, Creatinine, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Creatinine, Week 44, n=137, 148 | 78.45 (15.909) | 76.25 (15.257)
  NNRTI, Creatinine, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Creatinine, Week 48, n=131, 147 | 78.91 (17.389) | 75.67 (14.794)

51. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: Creatinine Clearance
Description: Blood samples were collected for the analysis of clinical chemistry parameter: creatinine clearance to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). GFR will be estimated by the central laboratory using the CKD-EPI.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliters per minute per 1.73meter^2
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Milliliters per minute per 1.73meter^2
  PI, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Baseline, n=51, 54 | 105.2 (15.67) | 104.9 (15.22)
  PI, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Week 4, n=51, 53 | 103.0 (15.59) | 102.1 (15.68)
  PI, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Week 8, n=34, 53 | 104.3 (14.52) | 103.5 (15.61)
  PI, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Week 12, n=50, 52 | 107.1 (14.95) | 101.1 (15.94)
  PI, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Week 16, n=48, 53 | 105.4 (15.88) | 101.8 (15.99)
  PI, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Week 20, n=46, 53 | 102.9 (17.17) | 99.8 (16.53)
  PI, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Week 24, n=47, 53 | 103.3 (14.64) | 101.0 (15.54)
  PI, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Week 28, n=42, 53 | 100.6 (16.62) | 100.8 (14.58)
  PI, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Week 32, n=45, 51 | 101.0 (17.38) | 100.4 (16.04)
  PI, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Week 36, n=44, 50 | 100.7 (16.68) | 101.7 (14.42)
  PI, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Week 40, n=42, 51 | 100.2 (14.54) | 100.3 (15.51)
  PI, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Week 44, n=47, 51 | 99.8 (18.00) | 101.0 (15.31)
  PI, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Week 48, n=43, 50 | 98.8 (17.31) | 102.2 (15.45)
  INI, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Baseline, n=102, 99 | 92.3 (17.62) | 94.9 (18.82)
  INI, Week 4, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Week 4, n=99, 95 | 93.4 (15.07) | 93.1 (18.22)
  INI, Week 8, n=72, 98: number analyzed (Participants) | 72 | 98
  INI, Week 8, n=72, 98 | 94.4 (17.05) | 93.0 (18.12)
  INI, Week 12, n=99, 93: number analyzed (Participants) | 99 | 93
  INI, Week 12, n=99, 93 | 94.5 (16.82) | 91.6 (18.81)
  INI, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Week 16, n=93, 96 | 94.9 (16.02) | 94.4 (18.30)
  INI, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Week 20, n=93, 97 | 95.3 (15.97) | 93.3 (17.48)
  INI, Week 24, n=94, 94: number analyzed (Participants) | 94 | 94
  INI, Week 24, n=94, 94 | 95.6 (15.88) | 93.1 (17.21)
  INI, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Week 28, n=89, 93 | 95.4 (17.00) | 93.6 (17.89)
  INI, Week 32, n=92, 95: number analyzed (Participants) | 92 | 95
  INI, Week 32, n=92, 95 | 94.8 (17.16) | 93.1 (16.94)
  INI, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 36, n=94, 95 | 95.6 (15.81) | 92.7 (15.65)
  INI, Week 40, n=89, 95: number analyzed (Participants) | 89 | 95
  INI, Week 40, n=89, 95 | 94.8 (16.32) | 92.9 (18.15)
  INI, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Week 44, n=91, 94 | 94.8 (15.64) | 93.4 (17.94)
  INI, Week 48, n=90, 94: number analyzed (Participants) | 90 | 94
  INI, Week 48, n=90, 94 | 95.4 (16.20) | 93.5 (17.00)
  NNRTI, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Baseline, n=155, 155 | 104.4 (17.78) | 103.7 (16.85)
  NNRTI, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Week 4, n=151, 153 | 100.8 (18.35) | 101.5 (17.72)
  NNRTI, Week 8, n=121, 152: number analyzed (Participants) | 121 | 152
  NNRTI, Week 8, n=121, 152 | 102.3 (17.23) | 102.2 (16.85)
  NNRTI, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Week 12, n=146, 152 | 103.1 (18.02) | 103.2 (17.47)
  NNRTI, Week 16, n=143, 148: number analyzed (Participants) | 143 | 148
  NNRTI, Week 16, n=143, 148 | 102.5 (17.66) | 101.0 (18.66)
  NNRTI, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Week 20, n=138, 152 | 101.0 (17.94) | 101.8 (17.61)
  NNRTI, Week 24, n=142, 151: number analyzed (Participants) | 142 | 151
  NNRTI, Week 24, n=142, 151 | 99.6 (18.18) | 101.7 (17.43)
  NNRTI, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Week 28, n=136, 150 | 99.9 (18.23) | 101.7 (17.20)
  NNRTI, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Week 32, n=137, 148 | 101.3 (16.10) | 101.0 (17.79)
  NNRTI, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Week 36, n=135, 147 | 100.8 (18.02) | 101.4 (17.46)
  NNRTI, Week 40, n=137, 147: number analyzed (Participants) | 137 | 147
  NNRTI, Week 40, n=137, 147 | 100.5 (18.40) | 101.6 (16.68)
  NNRTI, Week 44, n=136, 148: number analyzed (Participants) | 136 | 148
  NNRTI, Week 44, n=136, 148 | 99.9 (17.23) | 101.8 (16.96)
  NNRTI, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Week 48, n=131, 147 | 98.7 (17.35) | 102.1 (16.83)

52. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: Lipase
Description: Blood samples were collected for the analysis of clinical chemistry parameter: lipase to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI).
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Units per liter
  PI, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Baseline, n=51, 54 | 27.6 (21.69) | 33.0 (22.44)
  PI, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Week 4, n=51, 53 | 25.5 (14.41) | 34.4 (20.77)
  PI, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Week 8, n=34, 53 | 23.4 (10.96) | 35.7 (28.85)
  PI, Week 12, n=49, 52: number analyzed (Participants) | 49 | 52
  PI, Week 12, n=49, 52 | 26.4 (12.00) | 31.2 (15.31)
  PI, Week 16, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Week 16, n=47, 53 | 28.1 (13.01) | 34.6 (18.14)
  PI, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Week 20, n=46, 53 | 25.8 (11.37) | 32.7 (16.37)
  PI, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Week 24, n=47, 53 | 25.8 (11.74) | 30.5 (15.48)
  PI, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Week 28, n=42, 53 | 26.4 (10.86) | 33.4 (15.92)
  PI, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Week 32, n=45, 51 | 26.9 (12.18) | 36.2 (24.23)
  PI, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Week 36, n=44, 50 | 27.1 (13.69) | 32.7 (17.14)
  PI, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Week 40, n=42, 51 | 30.5 (19.78) | 32.0 (15.16)
  PI, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Week 44, n=47, 51 | 27.1 (10.70) | 35.2 (18.59)
  PI, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Week 48, n=43, 50 | 26.3 (12.02) | 32.7 (15.62)
  INI, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Baseline, n=102, 99 | 29.3 (20.90) | 28.2 (16.64)
  INI, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Week 4, n=99, 97 | 36.8 (43.46) | 32.1 (31.31)
  INI, Week 8, n=72, 98: number analyzed (Participants) | 72 | 98
  INI, Week 8, n=72, 98 | 28.8 (16.80) | 27.7 (12.72)
  INI, Week 12, n=99, 93: number analyzed (Participants) | 99 | 93
  INI, Week 12, n=99, 93 | 33.1 (20.98) | 29.8 (23.81)
  INI, Week 16, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Week 16, n=93, 97 | 34.4 (33.09) | 28.9 (14.77)
  INI, Week 20, n=94, 97: number analyzed (Participants) | 94 | 97
  INI, Week 20, n=94, 97 | 32.0 (28.19) | 29.1 (16.34)
  INI, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 24, n=94, 95 | 32.0 (19.15) | 30.1 (21.56)
  INI, Week 28, n=89, 94: number analyzed (Participants) | 89 | 94
  INI, Week 28, n=89, 94 | 35.1 (38.32) | 32.8 (24.85)
  INI, Week 32, n=92, 95: number analyzed (Participants) | 92 | 95
  INI, Week 32, n=92, 95 | 32.6 (23.00) | 32.7 (21.75)
  INI, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 36, n=94, 95 | 35.0 (32.32) | 27.6 (12.20)
  INI, Week 40, n=89, 95: number analyzed (Participants) | 89 | 95
  INI, Week 40, n=89, 95 | 33.8 (20.14) | 29.6 (14.21)
  INI, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Week 44, n=91, 94 | 34.6 (34.66) | 32.8 (22.45)
  INI, Week 48, n=90, 94: number analyzed (Participants) | 90 | 94
  INI, Week 48, n=90, 94 | 35.1 (36.88) | 31.6 (23.18)
  NNRTI, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Baseline, n=155, 155 | 32.1 (24.46) | 31.8 (19.30)
  NNRTI, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Week 4, n=151, 153 | 37.6 (64.95) | 31.7 (17.60)
  NNRTI, Week 8, n=121, 152: number analyzed (Participants) | 121 | 152
  NNRTI, Week 8, n=121, 152 | 33.8 (27.26) | 33.4 (21.17)
  NNRTI, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Week 12, n=146, 152 | 35.6 (34.76) | 29.7 (14.64)
  NNRTI, Week 16, n=145, 149: number analyzed (Participants) | 145 | 149
  NNRTI, Week 16, n=145, 149 | 35.3 (32.66) | 36.8 (46.27)
  NNRTI, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Week 20, n=138, 152 | 32.0 (19.03) | 32.9 (37.34)
  NNRTI, Week 24, n=142, 151: number analyzed (Participants) | 142 | 151
  NNRTI, Week 24, n=142, 151 | 36.2 (29.08) | 37.2 (36.77)
  NNRTI, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Week 28, n=136, 150 | 33.4 (21.71) | 33.1 (17.20)
  NNRTI, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Week 32, n=137, 148 | 40.6 (83.20) | 33.6 (20.70)
  NNRTI, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Week 36, n=135, 147 | 39.9 (67.63) | 33.9 (21.66)
  NNRTI, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Week 40, n=138, 147 | 38.6 (46.34) | 32.3 (16.96)
  NNRTI, Week 44, n=136, 148: number analyzed (Participants) | 136 | 148
  NNRTI, Week 44, n=136, 148 | 34.5 (23.27) | 32.9 (19.81)
  NNRTI, Week 48, n=131, 146: number analyzed (Participants) | 131 | 146
  NNRTI, Week 48, n=131, 146 | 36.3 (30.60) | 32.8 (20.04)

53. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48
Description: Blood samples were collected for the analysis of clinical chemistry parameters: CO2, chloride, glucose, phosphate, potassium, sodium and urea to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI).
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Millimoles per liter
  PI, CO2, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, CO2, Baseline, n=51, 54 | 22.3 (2.53) | 22.7 (2.17)
  PI, CO2, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, CO2, Week 4, n=51, 53 | 23.6 (2.37) | 23.4 (2.28)
  PI, CO2, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, CO2, Week 8, n=34, 53 | 23.0 (1.95) | 23.0 (2.53)
  PI, CO2, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, CO2, Week 12, n=50, 52 | 22.9 (2.14) | 22.9 (2.41)
  PI, CO2, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, CO2, Week 16, n=48, 53 | 23.0 (2.07) | 22.9 (2.32)
  PI, CO2, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, CO2, Week 20, n=46, 53 | 23.1 (2.04) | 22.7 (2.59)
  PI, CO2, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, CO2, Week 24, n=47, 53 | 22.7 (1.95) | 22.8 (2.62)
  PI, CO2, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, CO2, Week 28, n=42, 53 | 22.7 (2.31) | 22.5 (2.48)
  PI, CO2, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, CO2, Week 32, n=45, 51 | 22.6 (2.22) | 22.6 (2.84)
  PI, CO2, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, CO2, Week 36, n=44, 50 | 22.6 (2.21) | 22.4 (2.36)
  PI, CO2, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, CO2, Week 40, n=42, 51 | 22.8 (2.24) | 23.1 (2.37)
  PI, CO2, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, CO2, Week 44, n=47, 51 | 22.9 (1.94) | 23.1 (2.37)
  PI, CO2, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, CO2, Week 48, n=43, 50 | 23.0 (2.01) | 22.7 (2.19)
  INI, CO2, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, CO2, Baseline, n=102, 99 | 22.8 (2.09) | 22.9 (2.08)
  INI, CO2, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, CO2, Week 4, n=99, 97 | 23.7 (2.36) | 23.7 (2.28)
  INI, CO2, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, CO2, Week 8, n=73, 98 | 23.0 (2.10) | 23.6 (2.20)
  INI, CO2, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, CO2, Week 12, n=99, 95 | 23.2 (2.07) | 23.3 (2.26)
  INI, CO2, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, CO2, Week 16, n=93, 96 | 22.8 (2.10) | 23.5 (2.39)
  INI, CO2, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, CO2, Week 20, n=93, 97 | 22.8 (2.11) | 23.6 (2.14)
  INI, CO2, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, CO2, Week 24, n=94, 95 | 22.8 (2.22) | 23.1 (2.21)
  INI, CO2, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, CO2, Week 28, n=89, 93 | 22.5 (2.21) | 23.1 (2.14)
  INI, CO2, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, CO2, Week 32, n=93, 95 | 22.8 (2.17) | 23.0 (2.09)
  INI, CO2, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, CO2, Week 36, n=94, 95 | 22.8 (1.90) | 23.5 (2.12)
  INI, CO2, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, CO2, Week 40, n=90, 95 | 23.1 (2.07) | 23.2 (2.09)
  INI, CO2, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, CO2, Week 44, n=91, 94 | 23.1 (2.08) | 23.7 (2.11)
  INI, CO2, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, CO2, Week 48, n=91, 95 | 22.9 (1.97) | 23.3 (2.32)
  NNRTI, CO2, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, CO2, Baseline, n=155, 155 | 22.7 (2.41) | 22.3 (2.35)
  NNRTI, CO2, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, CO2, Week 4, n=151, 153 | 23.7 (2.63) | 23.0 (2.24)
  NNRTI, CO2, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, CO2, Week 8, n=122, 152 | 23.2 (2.28) | 23.1 (2.61)
  NNRTI, CO2, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, CO2, Week 12, n=146, 152 | 23.2 (2.18) | 22.8 (2.39)
  NNRTI, CO2, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, CO2, Week 16, n=143, 149 | 23.0 (2.24) | 22.8 (2.23)
  NNRTI, CO2, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, CO2, Week 20, n=138, 152 | 22.9 (2.24) | 22.5 (2.20)
  NNRTI, CO2, Week 24, n=143, 150: number analyzed (Participants) | 143 | 150
  NNRTI, CO2, Week 24, n=143, 150 | 23.0 (2.49) | 22.7 (2.45)
  NNRTI, CO2, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, CO2, Week 28, n=136, 150 | 22.8 (2.58) | 22.6 (2.27)
  NNRTI, CO2, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, CO2, Week 32, n=137, 148 | 22.5 (2.11) | 22.7 (2.29)
  NNRTI, CO2, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, CO2, Week 36, n=135, 147 | 22.8 (2.38) | 22.8 (2.27)
  NNRTI, CO2, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, CO2, Week 40, n=138, 147 | 23.1 (2.40) | 22.8 (2.68)
  NNRTI, CO2, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, CO2, Week 44, n=137, 148 | 23.0 (2.35) | 22.8 (2.38)
  NNRTI, CO2, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, CO2, Week 48, n=131, 147 | 22.5 (2.55) | 22.6 (2.29)
  PI, Chloride, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Chloride, Baseline, n=51, 54 | 104.0 (1.46) | 103.5 (2.61)
  PI, Chloride, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Chloride, Week 4, n=51, 53 | 104.5 (1.80) | 104.0 (2.10)
  PI, Chloride, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Chloride, Week 8, n=34, 53 | 104.4 (2.35) | 104.2 (2.28)
  PI, Chloride, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Chloride, Week 12, n=50, 52 | 104.4 (2.02) | 104.3 (2.13)
  PI, Chloride, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Chloride, Week 16, n=48, 53 | 104.4 (2.08) | 104.5 (2.10)
  PI, Chloride, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Chloride, Week 20, n=46, 53 | 104.8 (1.98) | 104.2 (1.97)
  PI, Chloride, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Chloride, Week 24, n=47, 53 | 105.1 (1.85) | 104.7 (2.02)
  PI, Chloride, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Chloride, Week 28, n=42, 53 | 105.3 (1.88) | 104.6 (2.47)
  PI, Chloride, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Chloride, Week 32, n=45, 51 | 105.0 (2.32) | 104.4 (1.92)
  PI, Chloride, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Chloride, Week 36, n=44, 50 | 105.0 (2.17) | 104.4 (2.27)
  PI, Chloride, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Chloride, Week 40, n=42, 51 | 105.2 (2.27) | 104.5 (2.31)
  PI, Chloride, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Chloride, Week 44, n=47, 51 | 105.1 (1.84) | 104.5 (1.88)
  PI, Chloride, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Chloride, Week 48, n=43, 50 | 104.4 (1.72) | 104.3 (1.88)
  INI, Chloride, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Chloride, Baseline, n=102, 99 | 103.6 (2.03) | 103.5 (2.26)
  INI, Chloride, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Chloride, Week 4, n=99, 97 | 104.0 (2.17) | 104.0 (2.15)
  INI, Chloride, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Chloride, Week 8, n=73, 98 | 104.1 (2.16) | 103.5 (2.58)
  INI, Chloride, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Chloride, Week 12, n=99, 95 | 104.1 (2.31) | 104.0 (2.32)
  INI, Chloride, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Chloride, Week 16, n=93, 96 | 104.7 (2.05) | 104.2 (2.26)
  INI, Chloride, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Chloride, Week 20, n=93, 97 | 104.8 (2.39) | 103.8 (2.36)
  INI, Chloride, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Chloride, Week 24, n=94, 95 | 104.3 (2.30) | 104.1 (2.50)
  INI, Chloride, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Chloride, Week 28, n=89, 93 | 104.7 (1.92) | 104.0 (2.16)
  INI, Chloride, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Chloride, Week 32, n=93, 95 | 104.5 (2.33) | 104.2 (2.47)
  INI, Chloride, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Chloride, Week 36, n=94, 95 | 104.6 (2.04) | 104.1 (2.40)
  INI, Chloride, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Chloride, Week 40, n=90, 95 | 104.4 (1.94) | 103.9 (2.48)
  INI, Chloride, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Chloride, Week 44, n=91, 94 | 104.5 (2.12) | 104.0 (2.27)
  INI, Chloride, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Chloride, Week 48, n=91, 95 | 104.2 (2.43) | 103.2 (2.26)
  NNRTI, Chloride, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Chloride, Baseline, n=155, 155 | 103.9 (2.18) | 104.0 (2.37)
  NNRTI, Chloride, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Chloride, Week 4, n=151, 153 | 104.3 (2.21) | 104.6 (2.29)
  NNRTI, Chloride, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Chloride, Week 8, n=122, 152 | 104.4 (2.31) | 104.7 (2.22)
  NNRTI, Chloride, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Chloride, Week 12, n=146, 152 | 104.3 (2.33) | 104.5 (2.23)
  NNRTI, Chloride, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Chloride, Week 16, n=143, 149 | 104.4 (2.37) | 104.8 (2.34)
  NNRTI, Chloride, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Chloride, Week 20, n=138, 152 | 104.6 (2.55) | 105.1 (2.38)
  NNRTI, Chloride, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Chloride, Week 24, n=143, 151 | 104.4 (2.52) | 105.1 (2.18)
  NNRTI, Chloride, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Chloride, Week 28, n=136, 150 | 104.7 (2.41) | 105.3 (2.31)
  NNRTI, Chloride, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Chloride, Week 32, n=137, 148 | 104.7 (2.68) | 105.1 (2.26)
  NNRTI, Chloride, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Chloride, Week 36, n=135, 147 | 105.0 (2.28) | 105.1 (2.30)
  NNRTI, Chloride, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Chloride, Week 40, n=138, 147 | 104.7 (2.36) | 105.0 (2.70)
  NNRTI, Chloride, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Chloride, Week 44, n=137, 148 | 104.6 (2.17) | 105.0 (2.32)
  NNRTI, Chloride, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Chloride, Week 48, n=131, 147 | 104.6 (2.54) | 104.5 (2.46)
  PI, Glucose, Baseline, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Glucose, Baseline, n=51, 53 | 5.11 (0.878) | 5.03 (0.505)
  PI, Glucose, Week 4, n=43, 43: number analyzed (Participants) | 43 | 43
  PI, Glucose, Week 4, n=43, 43 | 5.06 (0.481) | 5.29 (0.452)
  PI, Glucose, Week 8, n=25, 41: number analyzed (Participants) | 25 | 41
  PI, Glucose, Week 8, n=25, 41 | 5.11 (0.456) | 5.18 (0.462)
  PI, Glucose, Week 12, n=40, 43: number analyzed (Participants) | 40 | 43
  PI, Glucose, Week 12, n=40, 43 | 5.21 (0.533) | 5.25 (0.535)
  PI, Glucose, Week 16, n=39, 44: number analyzed (Participants) | 39 | 44
  PI, Glucose, Week 16, n=39, 44 | 5.24 (0.800) | 5.26 (0.614)
  PI, Glucose, Week 20, n=35, 42: number analyzed (Participants) | 35 | 42
  PI, Glucose, Week 20, n=35, 42 | 5.11 (0.580) | 5.29 (0.718)
  PI, Glucose, Week 24, n=38, 43: number analyzed (Participants) | 38 | 43
  PI, Glucose, Week 24, n=38, 43 | 5.31 (0.526) | 5.29 (0.747)
  PI, Glucose, Week 28, n=32, 43: number analyzed (Participants) | 32 | 43
  PI, Glucose, Week 28, n=32, 43 | 5.16 (0.651) | 5.12 (0.512)
  PI, Glucose, Week 32, n=36, 42: number analyzed (Participants) | 36 | 42
  PI, Glucose, Week 32, n=36, 42 | 5.37 (0.700) | 5.31 (0.643)
  PI, Glucose, Week 36, n=35, 42: number analyzed (Participants) | 35 | 42
  PI, Glucose, Week 36, n=35, 42 | 5.13 (0.525) | 5.23 (0.513)
  PI, Glucose, Week 40, n=34, 41: number analyzed (Participants) | 34 | 41
  PI, Glucose, Week 40, n=34, 41 | 5.31 (0.464) | 5.17 (0.555)
  PI, Glucose, Week 44, n=40, 40: number analyzed (Participants) | 40 | 40
  PI, Glucose, Week 44, n=40, 40 | 5.13 (0.681) | 5.20 (0.408)
  PI, Glucose, Week 48, n=39, 48: number analyzed (Participants) | 39 | 48
  PI, Glucose, Week 48, n=39, 48 | 5.16 (0.647) | 5.18 (0.661)
  INI, Glucose, Baseline, n=98, 96: number analyzed (Participants) | 98 | 96
  INI, Glucose, Baseline, n=98, 96 | 5.06 (0.638) | 5.25 (0.801)
  INI, Glucose, Week 4, n=55, 54: number analyzed (Participants) | 55 | 54
  INI, Glucose, Week 4, n=55, 54 | 5.39 (0.771) | 5.37 (1.043)
  INI, Glucose, Week 8, n=36, 58: number analyzed (Participants) | 36 | 58
  INI, Glucose, Week 8, n=36, 58 | 5.16 (0.584) | 5.49 (1.307)
  INI, Glucose, Week 12, n=53, 56: number analyzed (Participants) | 53 | 56
  INI, Glucose, Week 12, n=53, 56 | 5.50 (1.317) | 5.51 (1.414)
  INI, Glucose, Week 16, n=54, 53: number analyzed (Participants) | 54 | 53
  INI, Glucose, Week 16, n=54, 53 | 5.41 (1.727) | 5.25 (0.624)
  INI, Glucose, Week 20, n=52, 58: number analyzed (Participants) | 52 | 58
  INI, Glucose, Week 20, n=52, 58 | 5.36 (0.674) | 5.21 (0.793)
  INI, Glucose, Week 24, n=61, 62: number analyzed (Participants) | 61 | 62
  INI, Glucose, Week 24, n=61, 62 | 5.34 (0.660) | 5.36 (0.753)
  INI, Glucose, Week 28, n=53, 63: number analyzed (Participants) | 53 | 63
  INI, Glucose, Week 28, n=53, 63 | 5.32 (0.817) | 5.45 (0.940)
  INI, Glucose, Week 32, n=54, 56: number analyzed (Participants) | 54 | 56
  INI, Glucose, Week 32, n=54, 56 | 5.57 (1.260) | 5.52 (0.839)
  INI, Glucose, Week 36, n=53, 58: number analyzed (Participants) | 53 | 58
  INI, Glucose, Week 36, n=53, 58 | 5.46 (0.697) | 5.34 (1.142)
  INI, Glucose, Week 40, n=59, 63: number analyzed (Participants) | 59 | 63
  INI, Glucose, Week 40, n=59, 63 | 5.53 (0.931) | 5.46 (0.765)
  INI, Glucose, Week 44, n=54, 57: number analyzed (Participants) | 54 | 57
  INI, Glucose, Week 44, n=54, 57 | 5.40 (1.020) | 5.43 (0.637)
  INI, Glucose, Week 48, n=84, 91: number analyzed (Participants) | 84 | 91
  INI, Glucose, Week 48, n=84, 91 | 5.16 (0.549) | 5.24 (0.752)
  NNRTI, Glucose, Baseline, n=152, 150: number analyzed (Participants) | 152 | 150
  NNRTI, Glucose, Baseline, n=152, 150 | 4.93 (0.697) | 5.17 (1.201)
  NNRTI, Glucose, Week 4, n=118, 129: number analyzed (Participants) | 118 | 129
  NNRTI, Glucose, Week 4, n=118, 129 | 5.11 (0.798) | 5.48 (1.490)
  NNRTI, Glucose, Week 8, n=92, 119: number analyzed (Participants) | 92 | 119
  NNRTI, Glucose, Week 8, n=92, 119 | 5.17 (1.204) | 5.35 (1.030)
  NNRTI, Glucose, Week 12, n=113, 122: number analyzed (Participants) | 113 | 122
  NNRTI, Glucose, Week 12, n=113, 122 | 5.04 (0.856) | 5.30 (1.067)
  NNRTI, Glucose, Week 16, n=116, 119: number analyzed (Participants) | 116 | 119
  NNRTI, Glucose, Week 16, n=116, 119 | 5.12 (0.914) | 5.45 (1.683)
  NNRTI, Glucose, Week 20, n=107, 121: number analyzed (Participants) | 107 | 121
  NNRTI, Glucose, Week 20, n=107, 121 | 5.16 (0.802) | 5.48 (1.476)
  NNRTI, Glucose, Week 24, n=116, 124: number analyzed (Participants) | 116 | 124
  NNRTI, Glucose, Week 24, n=116, 124 | 5.16 (0.944) | 5.36 (0.914)
  NNRTI, Glucose, Week 28, n=105, 120: number analyzed (Participants) | 105 | 120
  NNRTI, Glucose, Week 28, n=105, 120 | 5.08 (0.635) | 5.40 (0.934)
  NNRTI, Glucose, Week 32, n=104, 121: number analyzed (Participants) | 104 | 121
  NNRTI, Glucose, Week 32, n=104, 121 | 5.18 (1.000) | 5.47 (1.316)
  NNRTI, Glucose, Week 36, n=103, 120: number analyzed (Participants) | 103 | 120
  NNRTI, Glucose, Week 36, n=103, 120 | 5.07 (0.856) | 5.49 (1.857)
  NNRTI, Glucose, Week 40, n=102, 114: number analyzed (Participants) | 102 | 114
  NNRTI, Glucose, Week 40, n=102, 114 | 5.16 (0.776) | 5.53 (1.558)
  NNRTI, Glucose, Week 44, n=99, 116: number analyzed (Participants) | 99 | 116
  NNRTI, Glucose, Week 44, n=99, 116 | 5.15 (0.877) | 5.53 (1.708)
  NNRTI, Glucose, Week 48, n=119, 138: number analyzed (Participants) | 119 | 138
  NNRTI, Glucose, Week 48, n=119, 138 | 5.01 (0.640) | 5.23 (1.160)
  PI, Phosphate, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Phosphate, Baseline, n=51, 54 | 1.048 (0.1523) | 1.060 (0.1719)
  PI, Phosphate, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Phosphate, Week 4, n=51, 53 | 1.116 (0.1648) | 1.069 (0.1647)
  PI, Phosphate, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Phosphate, Week 8, n=34, 53 | 1.119 (0.1891) | 1.041 (0.1664)
  PI, Phosphate, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Phosphate, Week 12, n=50, 52 | 1.073 (0.1788) | 1.064 (0.1872)
  PI, Phosphate, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Phosphate, Week 16, n=48, 53 | 1.111 (0.2006) | 1.051 (0.1849)
  PI, Phosphate, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Phosphate, Week 20, n=46, 53 | 1.119 (0.1689) | 1.076 (0.2187)
  PI, Phosphate, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Phosphate, Week 24, n=47, 53 | 1.086 (0.1647) | 1.077 (0.1631)
  PI, Phosphate, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Phosphate, Week 28, n=42, 53 | 1.085 (0.1803) | 1.076 (0.1970)
  PI, Phosphate, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Phosphate, Week 32, n=45, 51 | 1.109 (0.1869) | 1.081 (0.1769)
  PI, Phosphate, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Phosphate, Week 36, n=44, 50 | 1.084 (0.1659) | 1.058 (0.1830)
  PI, Phosphate, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Phosphate, Week 40, n=42, 51 | 1.067 (0.2020) | 1.053 (0.1932)
  PI, Phosphate, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Phosphate, Week 44, n=47, 51 | 1.084 (0.1785) | 1.063 (0.2227)
  PI, Phosphate, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Phosphate, Week 48, n=43, 50 | 1.095 (0.1636) | 1.070 (0.1804)
  INI, Phosphate, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Phosphate, Baseline, n=102, 99 | 1.045 (0.1687) | 1.063 (0.1700)
  INI, Phosphate, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Phosphate, Week 4, n=99, 97 | 1.080 (0.1725) | 1.082 (0.1857)
  INI, Phosphate, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Phosphate, Week 8, n=73, 98 | 1.086 (0.1901) | 1.071 (0.2001)
  INI, Phosphate, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Phosphate, Week 12, n=99, 95 | 1.068 (0.1970) | 1.078 (0.1823)
  INI, Phosphate, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Phosphate, Week 16, n=93, 96 | 1.063 (0.1623) | 1.061 (0.1702)
  INI, Phosphate, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Phosphate, Week 20, n=93, 97 | 1.046 (0.1717) | 1.091 (0.1757)
  INI, Phosphate, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Phosphate, Week 24, n=94, 95 | 1.066 (0.1661) | 1.052 (0.1921)
  INI, Phosphate, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Phosphate, Week 28, n=89, 93 | 1.060 (0.1602) | 1.065 (0.1835)
  INI, Phosphate, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Phosphate, Week 32, n=93, 95 | 1.045 (0.1649) | 1.045 (0.1569)
  INI, Phosphate, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Phosphate, Week 36, n=94, 95 | 1.032 (0.1572) | 1.059 (0.1800)
  INI, Phosphate, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Phosphate, Week 40, n=90, 95 | 1.054 (0.1838) | 1.062 (0.1731)
  INI, Phosphate, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Phosphate, Week 44, n=91, 94 | 1.043 (0.1805) | 1.066 (0.2029)
  INI, Phosphate, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Phosphate, Week 48, n=91, 95 | 1.072 (0.1721) | 1.066 (0.1918)
  NNRTI, Phosphate, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Phosphate, Baseline, n=155, 155 | 1.038 (0.1905) | 1.040 (0.1741)
  NNRTI, Phosphate, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Phosphate, Week 4, n=151, 153 | 1.128 (0.1867) | 1.056 (0.1764)
  NNRTI, Phosphate, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Phosphate, Week 8, n=122, 152 | 1.097 (0.1994) | 1.024 (0.1784)
  NNRTI, Phosphate, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Phosphate, Week 12, n=146, 152 | 1.091 (0.1838) | 1.051 (0.2002)
  NNRTI, Phosphate, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Phosphate, Week 16, n=143, 149 | 1.082 (0.1827) | 1.046 (0.1700)
  NNRTI, Phosphate, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Phosphate, Week 20, n=138, 152 | 1.076 (0.1763) | 1.037 (0.1806)
  NNRTI, Phosphate, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Phosphate, Week 24, n=143, 151 | 1.091 (0.1914) | 1.052 (0.1882)
  NNRTI, Phosphate, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Phosphate, Week 28, n=136, 150 | 1.076 (0.1764) | 1.038 (0.1585)
  NNRTI, Phosphate, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Phosphate, Week 32, n=137, 148 | 1.057 (0.1722) | 1.050 (0.1874)
  NNRTI, Phosphate, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Phosphate, Week 36, n=135, 147 | 1.055 (0.1790) | 1.039 (0.1793)
  NNRTI, Phosphate, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Phosphate, Week 40, n=138, 147 | 1.071 (0.1689) | 1.033 (0.1724)
  NNRTI, Phosphate, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Phosphate, Week 44, n=137, 148 | 1.076 (0.1795) | 1.040 (0.1693)
  NNRTI, Phosphate, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Phosphate, Week 48, n=131, 147 | 1.075 (0.1941) | 1.037 (0.1789)
  PI, Potassium, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Potassium, Baseline, n=51, 54 | 4.13 (0.288) | 4.10 (0.308)
  PI, Potassium, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Potassium, Week 4, n=51, 53 | 4.25 (0.355) | 4.31 (0.395)
  PI, Potassium, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Potassium, Week 8, n=34, 53 | 4.18 (0.283) | 4.19 (0.331)
  PI, Potassium, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Potassium, Week 12, n=50, 52 | 4.25 (0.335) | 4.31 (0.364)
  PI, Potassium, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Potassium, Week 16, n=48, 53 | 4.16 (0.322) | 4.30 (0.359)
  PI, Potassium, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Potassium, Week 20, n=46, 53 | 4.18 (0.291) | 4.29 (0.314)
  PI, Potassium, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Potassium, Week 24, n=47, 53 | 4.15 (0.335) | 4.30 (0.379)
  PI, Potassium, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Potassium, Week 28, n=42, 53 | 4.21 (0.342) | 4.26 (0.348)
  PI, Potassium, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Potassium, Week 32, n=45, 51 | 4.15 (0.326) | 4.31 (0.367)
  PI, Potassium, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Potassium, Week 36, n=44, 50 | 4.25 (0.345) | 4.26 (0.378)
  PI, Potassium, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Potassium, Week 40, n=42, 51 | 4.23 (0.293) | 4.26 (0.363)
  PI, Potassium, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Potassium, Week 44, n=47, 51 | 4.24 (0.348) | 4.32 (0.375)
  PI, Potassium, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Potassium, Week 48, n=43, 50 | 4.15 (0.292) | 4.12 (0.320)
  INI, Potassium, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Potassium, Baseline, n=102, 99 | 4.17 (0.245) | 4.18 (0.289)
  INI, Potassium, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Potassium, Week 4, n=99, 97 | 4.20 (0.311) | 4.26 (0.359)
  INI, Potassium, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Potassium, Week 8, n=73, 98 | 4.14 (0.306) | 4.24 (0.462)
  INI, Potassium, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Potassium, Week 12, n=99, 95 | 4.19 (0.340) | 4.18 (0.291)
  INI, Potassium, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Potassium, Week 16, n=93, 96 | 4.15 (0.317) | 4.19 (0.297)
  INI, Potassium, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Potassium, Week 20, n=93, 97 | 4.20 (0.299) | 4.18 (0.289)
  INI, Potassium, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Potassium, Week 24, n=94, 95 | 4.19 (0.304) | 4.21 (0.304)
  INI, Potassium,Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Potassium,Week 28, n=89, 93 | 4.19 (0.412) | 4.22 (0.341)
  INI, Potassium, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Potassium, Week 32, n=93, 95 | 4.20 (0.358) | 4.19 (0.307)
  INI, Potassium, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Potassium, Week 36, n=94, 95 | 4.19 (0.365) | 4.23 (0.332)
  INI, Potassium, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Potassium, Week 40, n=90, 95 | 4.18 (0.332) | 4.19 (0.297)
  INI, Potassium, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Potassium, Week 44, n=91, 94 | 4.18 (0.309) | 4.17 (0.314)
  INI, Potassium, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Potassium, Week 48, n=91, 95 | 4.15 (0.266) | 4.16 (0.305)
  NNRTI, Potassium, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Potassium, Baseline, n=155, 155 | 4.16 (0.302) | 4.18 (0.331)
  NNRTI, Potassium, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Potassium, Week 4, n=151, 153 | 4.21 (0.287) | 4.28 (0.333)
  NNRTI, Potassium, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Potassium, Week 8, n=122, 152 | 4.17 (0.295) | 4.23 (0.366)
  NNRTI, Potassium, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Potassium, Week 12, n=146, 152 | 4.18 (0.322) | 4.26 (0.341)
  NNRTI, Potassium, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Potassium, Week 16, n=143, 149 | 4.20 (0.313) | 4.23 (0.320)
  NNRTI, Potassium,Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Potassium,Week 20, n=138, 152 | 4.20 (0.326) | 4.21 (0.337)
  NNRTI, Potassium, Week 24, n=143, 150: number analyzed (Participants) | 143 | 150
  NNRTI, Potassium, Week 24, n=143, 150 | 4.19 (0.259) | 4.22 (0.341)
  NNRTI, Potassium, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Potassium, Week 28, n=136, 150 | 4.18 (0.301) | 4.25 (0.434)
  NNRTI, Potassium, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Potassium, Week 32, n=137, 148 | 4.17 (0.388) | 4.20 (0.349)
  NNRTI, Potassium, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Potassium, Week 36, n=135, 147 | 4.17 (0.289) | 4.22 (0.343)
  NNRTI, Potassium, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Potassium, Week 40, n=138, 147 | 4.20 (0.283) | 4.26 (0.321)
  NNRTI, Potassium, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Potassium, Week 44, n=137, 148 | 4.23 (0.324) | 4.24 (0.374)
  NNRTI, Potassium, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Potassium, Week 48, n=131, 147 | 4.14 (0.271) | 4.17 (0.352)
  PI, Sodium, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Sodium, Baseline, n=51, 54 | 138.9 (2.15) | 138.7 (2.10)
  PI, Sodium, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Sodium, Week 4, n=51, 53 | 139.3 (1.64) | 139.0 (2.08)
  PI, Sodium, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Sodium, Week 8, n=34, 53 | 139.6 (2.10) | 139.0 (1.95)
  PI, Sodium, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Sodium, Week 12, n=50, 52 | 139.3 (1.76) | 139.4 (2.03)
  PI, Sodium, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Sodium, Week 16, n=48, 53 | 139.4 (2.18) | 139.0 (1.75)
  PI, Sodium, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Sodium, Week 20, n=46, 53 | 139.6 (1.71) | 139.1 (1.97)
  PI, Sodium, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Sodium, Week 24, n=47, 53 | 139.4 (2.08) | 139.1 (2.07)
  PI, Sodium, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Sodium, Week 28, n=42, 53 | 140.3 (1.59) | 139.5 (2.49)
  PI, Sodium, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Sodium, Week 32, n=45, 51 | 139.4 (2.14) | 139.3 (2.28)
  PI, Sodium, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Sodium, Week 36, n=44, 50 | 139.7 (1.63) | 139.4 (2.32)
  PI, Sodium, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Sodium, Week 40, n=42, 51 | 139.8 (1.94) | 139.4 (1.93)
  PI, Sodium, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Sodium, Week 44, n=47, 51 | 139.7 (1.78) | 139.4 (2.09)
  PI, Sodium, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Sodium, Week 48, n=43, 50 | 139.8 (1.86) | 139.6 (1.90)
  INI, Sodium, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Sodium, Baseline, n=102, 99 | 138.8 (1.62) | 139.0 (1.67)
  INI, Sodium, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Sodium, Week 4, n=99, 97 | 139.2 (1.58) | 139.1 (1.72)
  INI, Sodium, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Sodium, Week 8, n=73, 98 | 138.8 (2.00) | 138.8 (1.79)
  INI, Sodium, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Sodium, Week 12, n=99, 95 | 139.1 (1.97) | 139.0 (1.88)
  INI, Sodium, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Sodium, Week 16, n=93, 96 | 139.1 (1.87) | 139.4 (1.89)
  INI, Sodium, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Sodium, Week 20, n=93, 97 | 139.4 (1.92) | 139.2 (1.67)
  INI, Sodium, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Sodium, Week 24, n=94, 95 | 139.3 (1.86) | 139.1 (1.91)
  INI, Sodium, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Sodium, Week 28, n=89, 93 | 139.4 (1.65) | 138.8 (1.67)
  INI, Sodium, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Sodium, Week 32, n=93, 95 | 139.4 (1.63) | 139.2 (1.68)
  INI, Sodium, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Sodium, Week 36, n=94, 95 | 139.2 (1.84) | 139.4 (1.99)
  INI, Sodium, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Sodium, Week 40, n=90, 95 | 139.3 (2.01) | 139.3 (1.83)
  INI, Sodium, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Sodium, Week 44, n=91, 94 | 139.3 (1.67) | 139.4 (1.88)
  INI, Sodium, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Sodium, Week 48, n=91, 95 | 139.3 (1.98) | 139.0 (1.76)
  NNRTI, Sodium, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Sodium, Baseline, n=155, 155 | 139.1 (2.00) | 139.2 (1.68)
  NNRTI, Sodium, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Sodium, Week 4, n=151, 153 | 139.4 (1.79) | 139.2 (1.90)
  NNRTI, Sodium, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Sodium, Week 8, n=122, 152 | 139.1 (1.91) | 139.2 (1.76)
  NNRTI, Sodium, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Sodium, Week 12, n=146, 152 | 139.2 (1.78) | 139.2 (1.77)
  NNRTI, Sodium, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Sodium, Week 16, n=143, 149 | 139.0 (1.99) | 139.0 (2.06)
  NNRTI, Sodium, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Sodium, Week 20, n=138, 152 | 139.0 (1.87) | 139.5 (1.83)
  NNRTI, Sodium, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Sodium, Week 24, n=143, 151 | 139.2 (1.83) | 139.4 (1.94)
  NNRTI, Sodium, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Sodium, Week 28, n=136, 150 | 139.3 (1.84) | 139.4 (1.99)
  NNRTI, Sodium, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Sodium, Week 32, n=137, 148 | 139.2 (1.68) | 139.7 (1.75)
  NNRTI, Sodium, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Sodium, Week 36, n=135, 147 | 139.4 (1.80) | 139.7 (2.19)
  NNRTI, Sodium, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Sodium, Week 40, n=138, 147 | 139.4 (1.87) | 139.7 (2.06)
  NNRTI, Sodium, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Sodium, Week 44, n=137, 148 | 139.5 (1.88) | 139.7 (1.92)
  NNRTI, Sodium, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Sodium, Week 48, n=131, 147 | 139.4 (1.93) | 139.5 (1.82)
  PI, Urea, Baseline, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, Urea, Baseline, n=51, 54 | 4.97 (1.409) | 4.89 (1.316)
  PI, Urea, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Urea, Week 4, n=51, 53 | 4.99 (1.210) | 4.91 (1.455)
  PI, Urea, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Urea, Week 8, n=34, 53 | 5.10 (1.353) | 4.88 (1.447)
  PI, Urea, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Urea, Week 12, n=50, 52 | 5.03 (1.368) | 4.85 (1.480)
  PI, Urea, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Urea, Week 16, n=48, 53 | 5.20 (1.295) | 5.09 (1.754)
  PI, Urea, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Urea, Week 20, n=46, 53 | 5.18 (1.216) | 5.07 (1.535)
  PI, Urea, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Urea, Week 24, n=47, 53 | 5.44 (1.587) | 5.00 (1.414)
  PI, Urea, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Urea, Week 28, n=42, 53 | 5.21 (1.358) | 4.90 (1.530)
  PI, Urea, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Urea, Week 32, n=45, 51 | 5.13 (1.135) | 5.09 (1.482)
  PI, Urea, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Urea, Week 36, n=44, 50 | 4.99 (1.310) | 4.78 (1.411)
  PI, Urea, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Urea, Week 40, n=42, 51 | 5.35 (1.227) | 5.30 (1.758)
  PI, Urea, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Urea, Week 44, n=47, 51 | 5.38 (1.483) | 5.10 (1.517)
  PI, Urea, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Urea, Week 48, n=43, 50 | 5.22 (1.469) | 5.11 (1.489)
  INI, Urea, Baseline, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, Urea, Baseline, n=102, 99 | 5.76 (1.528) | 5.61 (1.894)
  INI, Urea, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Urea, Week 4, n=99, 97 | 5.63 (1.471) | 5.77 (1.676)
  INI, Urea, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Urea, Week 8, n=73, 98 | 5.80 (1.617) | 5.60 (1.607)
  INI, Urea, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Urea, Week 12, n=99, 95 | 5.81 (1.536) | 5.83 (1.724)
  INI, Urea, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Urea, Week 16, n=93, 96 | 5.76 (1.577) | 5.70 (1.574)
  INI, Urea, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Urea, Week 20, n=93, 97 | 5.75 (1.640) | 5.76 (1.580)
  INI, Urea, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Urea, Week 24, n=94, 95 | 5.84 (1.578) | 5.72 (1.774)
  INI, Urea, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Urea, Week 28, n=89, 93 | 5.76 (1.593) | 5.65 (1.435)
  INI, Urea, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Urea, Week 32, n=93, 95 | 5.67 (1.537) | 5.63 (1.477)
  INI, Urea, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Urea, Week 36, n=94, 95 | 5.67 (1.670) | 5.53 (1.456)
  INI, Urea, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Urea, Week 40, n=90, 95 | 5.81 (1.669) | 5.66 (1.593)
  INI, Urea, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Urea, Week 44, n=91, 94 | 5.59 (1.607) | 5.46 (1.368)
  INI, Urea, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Urea, Week 48, n=91, 95 | 5.83 (1.654) | 5.50 (1.468)
  NNRTI, Urea, Baseline, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, Urea, Baseline, n=155, 155 | 4.96 (1.519) | 5.10 (1.510)
  NNRTI, Urea, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Urea, Week 4, n=151, 153 | 5.08 (1.556) | 5.09 (1.426)
  NNRTI, Urea, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Urea, Week 8, n=122, 152 | 5.09 (1.675) | 5.10 (1.465)
  NNRTI, Urea, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Urea, Week 12, n=146, 152 | 5.20 (1.684) | 5.13 (1.583)
  NNRTI, Urea, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Urea, Week 16, n=143, 149 | 5.03 (1.768) | 5.34 (1.660)
  NNRTI, Urea, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Urea, Week 20, n=138, 152 | 5.18 (1.709) | 5.15 (1.713)
  NNRTI, Urea, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Urea, Week 24, n=143, 151 | 5.29 (1.878) | 5.26 (1.591)
  NNRTI, Urea, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Urea, Week 28, n=136, 150 | 5.20 (1.931) | 5.10 (1.537)
  NNRTI, Urea, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Urea, Week 32, n=137, 148 | 5.38 (1.796) | 5.14 (1.687)
  NNRTI, Urea, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Urea, Week 36, n=135, 147 | 5.07 (1.719) | 5.13 (1.493)
  NNRTI, Urea, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Urea, Week 40, n=138, 147 | 5.30 (1.616) | 5.07 (1.377)
  NNRTI, Urea, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Urea, Week 44, n=137, 148 | 5.23 (1.489) | 5.18 (1.613)
  NNRTI, Urea, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Urea, Week 48, n=131, 147 | 5.32 (1.671) | 5.06 (1.380)

54. Secondary Outcome: Absolute Values for Fasting Lipid Panel Using Baseline Third Agent Treatment Class Overtime Including Week 48
Description: Blood samples were collected for the analysis of fasting lipid panel: triglycerides, total cholesterol, HDL cholesterol and LDL cholesterol to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI).
Time Frame: Baseline (Day 1) and at Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Millimoles per liter
  PI, Triglycerides, Baseline, n=46, 50: number analyzed (Participants) | 46 | 50
  PI, Triglycerides, Baseline, n=46, 50 | 1.951 (1.8801) | 1.894 (1.4058)
  PI, Triglycerides, Week 48, n=40, 45: number analyzed (Participants) | 40 | 45
  PI, Triglycerides, Week 48, n=40, 45 | 1.309 (0.7647) | 1.772 (1.1828)
  INI, Triglycerides, Baseline, n=82, 84: number analyzed (Participants) | 82 | 84
  INI, Triglycerides, Baseline, n=82, 84 | 1.470 (1.0152) | 1.426 (0.8720)
  INI, Triglycerides, Week 48, n=72, 77: number analyzed (Participants) | 72 | 77
  INI, Triglycerides, Week 48, n=72, 77 | 1.405 (0.9068) | 1.307 (0.7427)
  NNRTI, Triglycerides, Baseline, n=136, 140: number analyzed (Participants) | 136 | 140
  NNRTI, Triglycerides, Baseline, n=136, 140 | 1.322 (0.7986) | 1.506 (1.4388)
  NNRTI, Triglycerides, Week 48, n=119, 120: number analyzed (Participants) | 119 | 120
  NNRTI, Triglycerides, Week 48, n=119, 120 | 1.305 (0.8771) | 1.316 (0.7914)
  PI, Cholesterol, Baseline, n=46, 50: number analyzed (Participants) | 46 | 50
  PI, Cholesterol, Baseline, n=46, 50 | 4.98 (0.960) | 5.14 (1.152)
  PI, Cholesterol, Week 48, n=40, 45: number analyzed (Participants) | 40 | 45
  PI, Cholesterol, Week 48, n=40, 45 | 5.07 (0.775) | 5.16 (1.130)
  INI, Cholesterol, Baseline, n=82, 84: number analyzed (Participants) | 82 | 84
  INI, Cholesterol, Baseline, n=82, 84 | 4.81 (1.077) | 5.01 (1.080)
  INI, Cholesterol, Week 48, n=72, 77: number analyzed (Participants) | 72 | 77
  INI, Cholesterol, Week 48, n=72, 77 | 4.90 (0.881) | 4.87 (0.997)
  NNRTI, Cholesterol, Baseline, n=136, 140: number analyzed (Participants) | 136 | 140
  NNRTI, Cholesterol, Baseline, n=136, 140 | 4.87 (0.958) | 4.98 (1.007)
  NNRTI, Cholesterol, Week 48, n=119, 120: number analyzed (Participants) | 119 | 120
  NNRTI, Cholesterol, Week 48, n=119, 120 | 4.93 (0.904) | 4.91 (1.007)
  PI, HDL cholesterol, Baseline, n=46, 50: number analyzed (Participants) | 46 | 50
  PI, HDL cholesterol, Baseline, n=46, 50 | 1.389 (0.4943) | 1.537 (0.6096)
  PI, HDL cholesterol, Week 48, n=40, 45: number analyzed (Participants) | 40 | 45
  PI, HDL cholesterol, Week 48, n=40, 45 | 1.505 (0.5459) | 1.550 (0.5950)
  INI, HDL cholesterol, Baseline, n=82, 84: number analyzed (Participants) | 82 | 84
  INI, HDL cholesterol, Baseline, n=82, 84 | 1.257 (0.3450) | 1.383 (0.3890)
  INI, HDL cholesterol, Week 48, n=72, 77: number analyzed (Participants) | 72 | 77
  INI, HDL cholesterol, Week 48, n=72, 77 | 1.288 (0.3664) | 1.323 (0.3588)
  NNRTI, HDL cholesterol, Baseline, n=136, 140: number analyzed (Participants) | 136 | 140
  NNRTI, HDL cholesterol, Baseline, n=136, 140 | 1.449 (0.4756) | 1.405 (0.4401)
  NNRTI, HDL cholesterol, Week 48, n=119, 120: number analyzed (Participants) | 119 | 120
  NNRTI, HDL cholesterol, Week 48, n=119, 120 | 1.442 (0.4413) | 1.471 (0.4226)
  PI, LDL cholesterol, Baseline, n=43, 48: number analyzed (Participants) | 43 | 48
  PI, LDL cholesterol, Baseline, n=43, 48 | 2.734 (0.7891) | 2.743 (0.7948)
  PI, LDL cholesterol, Week 48, n=37, 43: number analyzed (Participants) | 37 | 43
  PI, LDL cholesterol, Week 48, n=37, 43 | 2.944 (0.7175) | 2.784 (0.8477)
  INI, LDL cholesterol, Basline, n=81, 83: number analyzed (Participants) | 81 | 83
  INI, LDL cholesterol, Basline, n=81, 83 | 2.881 (0.9196) | 2.946 (0.8614)
  INI, LDL cholesterol, Week 48, n=71, 76: number analyzed (Participants) | 71 | 76
  INI, LDL cholesterol, Week 48, n=71, 76 | 2.975 (0.8787) | 2.939 (0.8591)
  NNRTI, LDL cholesterol, Baseline, n=134, 137: number analyzed (Participants) | 134 | 137
  NNRTI, LDL cholesterol, Baseline, n=134, 137 | 2.834 (0.8442) | 2.901 (0.8714)
  NNRTI, LDL cholesterol, Week 48, n=116, 119: number analyzed (Participants) | 116 | 119
  NNRTI, LDL cholesterol, Week 48, n=116, 119 | 2.900 (0.8415) | 2.834 (0.8763)

55. Secondary Outcome: Number of Participants Discontinued or Withdrawn Due to AEs When Baseline Third Agent Treatment Class Was Used Over Time Including Week 48
Description: as for outcome 43
Time Frame: Up to Week 48
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants
  PI | 2 | 2
  INI | 6 | 0
  NNRTI | 5 | 3

56. Secondary Outcome: Plasma Trough Concentration (Ctrough) for CAB LA Evaluable
Description: Blood samples will be collected at indicated time points for pharmacokinetic (PK) analysis of CAB LA. PK population includes all participants who received CAB and / or RPV and underwent PK sampling during the study, and provided CAB and /or RPV plasma concentration data.
Time Frame: Pre-dose at Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: PK population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Groups:
- CAB LA: Participants received IM injections of CAB LA 400 mg every four weeks through Week 52.
Arm/Group | CAB LA
Number analyzed (Participants) | 308
Micrograms per milliliter
  Pre-dose, Week 8, n=252: number analyzed (Participants) | 252
  Pre-dose, Week 8, n=252 | 1.2277 [1.1293 to 1.3346]
  Pre-dose, Week 12, n=261: number analyzed (Participants) | 261
  Pre-dose, Week 12, n=261 | 1.6925 [1.6005 to 1.7897]
  Pre-dose, Week 16, n=248: number analyzed (Participants) | 248
  Pre-dose, Week 16, n=248 | 1.9533 [1.8492 to 2.0632]
  Pre-dose, Week 20, n=233: number analyzed (Participants) | 233
  Pre-dose, Week 20, n=233 | 2.1036 [1.9924 to 2.2209]
  Pre-dose, Week 24, n=234: number analyzed (Participants) | 234
  Pre-dose, Week 24, n=234 | 2.2537 [2.1177 to 2.3984]
  Pre-dose, Week 28, n=232: number analyzed (Participants) | 232
  Pre-dose, Week 28, n=232 | 2.4300 [2.3093 to 2.5569]
  Pre-dose, Week 32, n=219: number analyzed (Participants) | 219
  Pre-dose, Week 32, n=219 | 2.4483 [2.3321 to 2.5703]
  Pre-dose, Week 36, n=209: number analyzed (Participants) | 209
  Pre-dose, Week 36, n=209 | 2.4681 [2.3377 to 2.6057]
  Pre-dose, Week 40, n=209: number analyzed (Participants) | 209
  Pre-dose, Week 40, n=209 | 2.5126 [2.3477 to 2.6890]
  Pre-dose, Week 44, n=221: number analyzed (Participants) | 221
  Pre-dose, Week 44, n=221 | 2.7748 [2.6323 to 2.9250]
  Pre-dose, Week 48, n=217: number analyzed (Participants) | 217
  Pre-dose, Week 48, n=217 | 2.8378 [2.6763 to 3.0090]

57. Secondary Outcome: Ctrough for RPV LA Evaluable
Description: Blood samples will be collected at indicated time points for PK analysis of RPV LA.
Time Frame: Pre-dose at Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 56
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter
Groups:
- RPV LA: Participants received IM injections of RPV LA 600 mg every four weeks through Week 52.
Arm/Group | RPV LA
Number analyzed (Participants) | 308
Nanograms per milliliter
  Pre-dose, Week 8, n=251: number analyzed (Participants) | 251
  Pre-dose, Week 8, n=251 | 38.58 [35.96 to 41.39]
  Pre-dose, Week 12, n=261: number analyzed (Participants) | 261
  Pre-dose, Week 12, n=261 | 47.00 [44.50 to 49.64]
  Pre-dose, Week 16, n=247: number analyzed (Participants) | 247
  Pre-dose, Week 16, n=247 | 53.87 [50.92 to 56.98]
  Pre-dose, Week 20, n=233: number analyzed (Participants) | 233
  Pre-dose, Week 20, n=233 | 54.14 [51.13 to 57.34]
  Pre-dose, Week 24, n=231: number analyzed (Participants) | 231
  Pre-dose, Week 24, n=231 | 61.26 [57.80 to 64.93]
  Pre-dose, Week 28, n=232: number analyzed (Participants) | 232
  Pre-dose, Week 28, n=232 | 66.53 [62.87 to 70.40]
  Pre-dose, Week 32, n=218: number analyzed (Participants) | 218
  Pre-dose, Week 32, n=218 | 70.93 [66.97 to 75.11]
  Pre-dose, Week 36, n=209: number analyzed (Participants) | 209
  Pre-dose, Week 36, n=209 | 73.00 [68.54 to 77.75]
  Pre-dose, Week 40, n=208: number analyzed (Participants) | 208
  Pre-dose, Week 40, n=208 | 76.24 [71.71 to 81.07]
  Pre-dose, Week 44, n=223: number analyzed (Participants) | 223
  Pre-dose, Week 44, n=223 | 83.65 [78.94 to 88.63]
  Pre-dose, Week 48, n=216: number analyzed (Participants) | 216
  Pre-dose, Week 48, n=216 | 90.28 [84.92 to 95.98]

58. Secondary Outcome: Area Under the Curve (AUC) for CAB LA
Description: AUC values are Bayesian PK parameter estimates obtained from a population PK meta-analysis of the data collected from studies 201585 and 201584 # NCT02938520. Blood samples from the current study 201585 were collected at indicated time points to analyze concentration in plasma for CAB LA.
Time Frame: Pre-dose at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48; 1 Week post-dose at Weeks 5 and 41
Population: PK population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours*microgram per milliliter
Arm/Group | CAB LA
Number analyzed (Participants) | 303
Hours*microgram per milliliter | 2324.29 [2249.850 to 2401.187]

59. Secondary Outcome: AUC for RPV LA
Description: AUC values are Bayesian PK parameter estimates obtained from a population PK meta-analysis of the data collected from studies 201585 and 201584 # NCT02938520. Blood samples from the current study 201585 were collected at indicated time points to analyze concentration in plasma for RPV LA.
Time Frame: Pre-dose at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48; 1 Week post-dose at Weeks 5 and 41
Population: PK population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours*nanogram per milliliter
Groups:
- RPV LA: Participants received IM injections of RPV LA 900 mg every four weeks through Week 52.
Arm/Group | RPV LA
Number analyzed (Participants) | 303
Hours*nanogram per milliliter | 67119.84 [64426.092 to 69926.208]

60. Secondary Outcome: Maximum Concentration (Cmax) in Plasma for CAB LA Evaluable at Week 41
Description: Blood samples will be collected at indicated time points for PK analysis of CAB LA.
Time Frame: Week 41- 1 Week post dose
Population: PK population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | CAB LA
Number analyzed (Participants) | 251
Micrograms per milliliter | 3.3862 [3.1804 to 3.6054]

61. Secondary Outcome: Cmax in Plasma for RPV LA Evaluable at Week 41
Description: Blood samples will be collected at indicated time points for PK analysis of RPV LA.
Time Frame: Week 41- 1 Week post dose
Population: PK population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | RPV LA
Number analyzed (Participants) | 251
Nanograms per milliliter | 110.36 [103.28 to 117.93]

62. Secondary Outcome: Percentage of Participants With a Virologic Failure Using Snapshot Algorithm by Baseline Third Agent
Description: Percentage of participants with virologic failure endpoint as per FDA snapshot algorithm at Week 48 was assessed based on the non-inferior antiviral activity of switching IM CAB LA+RPV LA every 4 weeks compared to continuation of current ART regimen over 48 weeks in HIV-1 infected ART-experienced participants. The HIV-RNA >=50 copies/mL per snapshot algorithm was determined using a Cochran-Mantel Haenszel test stratified by baseline third agent class: INI, NNRTI, or PI.
Time Frame: Week 48
Population: ITT-E population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Percentage of participants
  PI, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, n=51, 54 | 2.0 | 0
  INI, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, n=102, 99 | 0 | 2.0
  NNRTI, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, n=155, 155 | 2.6 | 0.6

63. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50copies/mL Using Snapshot Algorithm by Baseline Third Agent
Description: Percentage of participants with HIV-1 RNA < 50copies/mL endpoint as per FDA snapshot algorithm at Week 48 was assessed based on the non-inferior antiviral activity of switching IM CAB LA+RPV LA every 4 weeks compared to continuation of current ART regimen over 48 weeks in HIV-1 infected ART-experienced participants. The HIV-RNA <50 copies/mL per snapshot algorithm was determined using a Cochran-Mantel Haenszel test stratified by baseline third agent class: INI, NNRTI, or PI.
Time Frame: Week 48
Population: as for outcome 62
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Percentage of participants
  PI, n=51, 54: number analyzed (Participants) | 51 | 54
  PI, n=51, 54 | 92 | 94
  INI, n=102, 99: number analyzed (Participants) | 102 | 99
  INI, n=102, 99 | 94 | 96
  NNRTI, n=155, 155: number analyzed (Participants) | 155 | 155
  NNRTI, n=155, 155 | 92 | 95

64. Secondary Outcome: Number of Participants With Severity of Adverse Events by Baseline Third Agents
Description: Severity of AEs were defined as per The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table). Severity grades for AEs were as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (Potentially life-threatening) and Grade 5 were all deaths related to an AE.
Time Frame: Up to Week 48
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Participants
  PI, Grade 1 | 22 | 20
  PI, Grade 2 | 20 | 11
  PI, Grade 3 | 4 | 4
  PI, Grade 4 | 1 | 0
  PI, Grade 5 | 0 | 1
  INI, Grade 1 | 40 | 40
  INI, Grade 2 | 50 | 23
  INI, Grade 3 | 8 | 3
  INI, Grade 4 | 1 | 2
  INI, Grade 5 | 0 | 0
  NNRTI, Grade 1 | 39 | 55
  NNRTI, Grade 2 | 88 | 47
  NNRTI, Grade 3 | 15 | 12
  NNRTI, Grade 4 | 6 | 2
  NNRTI, Grade 5 | 0 | 0

65. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: ALT, ALP, AST and CK
Description: Blood samples were collected for the analysis of clinical chemistry parameters: ALT, ALP, AST and CK to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
International units per liter
  PI, ALT, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, ALT, Week 4, n=51, 53 | 9.4 (17.93) | 1.1 (9.99)
  PI, ALT, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, ALT, Week 8, n=34, 53 | 7.9 (17.19) | 0.9 (7.20)
  PI, ALT, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, ALT, Week 12, n=50, 52 | 5.3 (17.31) | 1.4 (9.76)
  PI, ALT, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, ALT, Week 16, n=48, 53 | 6.5 (20.92) | 1.4 (8.75)
  PI, ALT, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, ALT, Week 20, n=46, 53 | 4.9 (18.06) | 0.3 (7.34)
  PI, ALT, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, ALT, Week 24, n=47, 53 | 4.1 (14.42) | 0.5 (7.30)
  PI, ALT, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, ALT, Week 28, n=42, 53 | 2.6 (11.47) | 0.8 (7.46)
  PI, ALT, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, ALT, Week 32, n=45, 51 | 3.5 (14.88) | 0.5 (7.36)
  PI, ALT, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, ALT, Week 36, n=44, 50 | 3.3 (13.55) | 2.0 (9.78)
  PI, ALT, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, ALT, Week 40, n=42, 51 | 5.4 (17.81) | 1.1 (10.52)
  PI, ALT, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, ALT, Week 44, n=47, 51 | 4.0 (15.83) | 0.9 (11.97)
  PI, ALT, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, ALT, Week 48, n=43, 50 | 2.9 (10.69) | 0.5 (8.04)
  INI, ALT, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, ALT, Week 4, n=99, 97 | 1.7 (15.15) | 0.7 (7.20)
  INI, ALT, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, ALT, Week 8, n=73, 98 | 3.3 (18.20) | 5.4 (50.20)
  INI, ALT, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, ALT, Week 12, n=99, 95 | -1.0 (12.48) | 1.7 (10.63)
  INI, ALT, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, ALT, Week 16, n=93, 96 | -1.8 (12.27) | -0.1 (8.58)
  INI, ALT, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, ALT, Week 20, n=93, 97 | -1.9 (13.60) | -0.5 (9.38)
  INI, ALT, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, ALT, Week 24, n=94, 95 | 0.6 (17.33) | 0.1 (9.95)
  INI, ALT, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, ALT, Week 28, n=89, 93 | -2.4 (9.70) | -0.4 (12.31)
  INI, ALT, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, ALT, Week 32, n=93, 95 | -1.8 (12.87) | -0.3 (7.79)
  INI, ALT, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, ALT, Week 36, n=94, 95 | 1.5 (35.82) | -0.4 (8.79)
  INI, ALT, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, ALT, Week 40, n=90, 95 | 5.0 (59.10) | -0.6 (9.62)
  INI, ALT, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, ALT, Week 44, n=91, 94 | -1.6 (13.90) | -0.4 (7.91)
  INI, ALT, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, ALT, Week 48, n=91, 95 | -0.2 (15.17) | -0.8 (7.41)
  NNRTI, ALT, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, ALT, Week 4, n=151, 153 | -2.6 (9.82) | -0.7 (10.80)
  NNRTI, ALT, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, ALT, Week 8, n=122, 152 | -2.9 (11.62) | -0.8 (12.06)
  NNRTI, ALT, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, ALT, Week 12, n=146, 152 | 9.5 (160.61) | -0.8 (12.66)
  NNRTI, ALT, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, ALT, Week 16, n=143, 149 | -1.3 (26.21) | -1.6 (11.39)
  NNRTI, ALT, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, ALT, Week 20, n=138, 152 | -2.0 (28.04) | -2.0 (12.61)
  NNRTI, ALT, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, ALT, Week 24, n=143, 151 | 2.6 (85.48) | -1.3 (11.85)
  NNRTI, ALT, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, ALT, Week 28, n=136, 150 | -4.5 (11.46) | -0.5 (14.03)
  NNRTI, ALT, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, ALT, Week 32, n=137, 148 | -3.8 (14.93) | -0.9 (14.33)
  NNRTI, ALT, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, ALT, Week 36, n=135, 147 | -3.8 (12.44) | -0.1 (12.48)
  NNRTI, ALT, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, ALT, Week 40, n=138, 147 | -3.8 (13.48) | -0.4 (13.47)
  NNRTI, ALT, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, ALT, Week 44, n=137, 148 | -4.7 (12.67) | -0.4 (14.67)
  NNRTI, ALT, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, ALT, Week 48, n=131, 147 | -4.6 (12.38) | -0.9 (12.75)
  PI, ALP, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, ALP, Week 4, n=51, 53 | -3.5 (11.63) | -2.9 (8.07)
  PI, ALP, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, ALP, Week 8, n=34, 53 | -2.1 (24.59) | 0.2 (11.37)
  PI, ALP, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, ALP, Week 12, n=50, 52 | -5.7 (14.40) | 0.9 (10.22)
  PI, ALP, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, ALP, Week 16, n=48, 53 | -7.3 (17.09) | 0.6 (8.68)
  PI, ALP, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, ALP, Week 20, n=46, 53 | -6.8 (16.71) | 0.1 (10.70)
  PI, ALP, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, ALP, Week 24, n=47, 53 | -7.5 (17.90) | -0.4 (7.67)
  PI, ALP, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, ALP, Week 28, n=42, 53 | -7.3 (17.23) | 3.0 (9.69)
  PI, ALP, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, ALP, Week 32, n=45, 51 | -9.3 (16.47) | -0.7 (8.50)
  PI, ALP, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, ALP, Week 36, n=44, 50 | -10.2 (18.52) | 0.6 (13.52)
  PI, ALP, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, ALP, Week 40, n=42, 51 | -8.7 (17.37) | -1.4 (8.79)
  PI, ALP, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, ALP, Week 44, n=47, 51 | -11.5 (17.49) | -0.9 (9.05)
  PI, ALP, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, ALP, Week 48, n=43, 50 | -8.0 (16.05) | -0.2 (9.08)
  INI, ALP, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, ALP, Week 4, n=99, 97 | -0.5 (10.59) | -0.9 (7.92)
  INI, ALP, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, ALP, Week 8, n=73, 98 | -1.8 (8.55) | 4.9 (33.17)
  INI, ALP, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, ALP, Week 12, n=99, 95 | -1.6 (8.57) | 3.5 (19.97)
  INI, ALP, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, ALP, Week 16, n=93, 96 | -1.7 (10.53) | -0.2 (10.93)
  INI, ALP, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, ALP, Week 20, n=93, 97 | -2.0 (10.23) | -0.4 (7.93)
  INI, ALP, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, ALP, Week 24, n=94, 95 | -1.4 (10.23) | -0.6 (8.25)
  INI, ALP, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, ALP, Week 28, n=89, 93 | -2.1 (10.83) | -0.8 (8.80)
  INI, ALP, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, ALP, Week 32, n=93, 95 | -1.6 (11.08) | -2.0 (8.23)
  INI, ALP, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, ALP, Week 36, n=94, 95 | -2.4 (12.03) | -2.2 (9.41)
  INI, ALP, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, ALP, Week 40, n=90, 95 | -0.9 (13.77) | -1.9 (9.33)
  INI, ALP, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, ALP, Week 44, n=91, 94 | -2.6 (13.69) | -0.4 (11.60)
  INI, ALP, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, ALP, Week 48, n=91, 95 | -1.9 (13.29) | -1.2 (10.26)
  NNRTI, ALP, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, ALP, Week 4, n=151, 153 | -10.4 (12.81) | -2.7 (9.60)
  NNRTI, ALP, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, ALP, Week 8, n=122, 152 | -10.9 (16.50) | -1.0 (10.77)
  NNRTI, ALP, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, ALP, Week 12, n=146, 152 | -13.0 (26.62) | -0.7 (11.04)
  NNRTI, ALP, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, ALP, Week 16, n=143, 149 | -15.7 (22.52) | -1.0 (10.54)
  NNRTI, ALP, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, ALP, Week 20, n=138, 152 | -14.9 (22.35) | -1.8 (13.77)
  NNRTI, ALP, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, ALP, Week 24, n=143, 151 | -14.5 (21.88) | 0.4 (12.75)
  NNRTI, ALP, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, ALP, Week 28, n=136, 150 | -16.2 (21.66) | -1.0 (13.18)
  NNRTI, ALP, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, ALP, Week 32, n=137, 148 | -15.8 (21.98) | -1.8 (13.63)
  NNRTI, ALP, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, ALP, Week 36, n=135, 147 | -16.1 (23.60) | -1.0 (11.86)
  NNRTI, ALP, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, ALP, Week 40, n=138, 147 | -17.2 (22.83) | -0.4 (13.19)
  NNRTI, ALP, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, ALP, Week 44, n=137, 148 | -17.3 (23.32) | -0.8 (13.20)
  NNRTI, ALP, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, ALP, Week 48, n=131, 147 | -18.0 (27.97) | 0.2 (14.69)
  PI, AST, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, AST, Week 4, n=51, 53 | 3.8 (9.18) | 2.3 (16.78)
  PI, AST, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, AST, Week 8, n=34, 53 | 5.1 (8.35) | -0.1 (4.60)
  PI, AST, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, AST, Week 12, n=50, 52 | 2.7 (11.49) | 1.7 (7.21)
  PI, AST, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, AST, Week 16, n=48, 53 | 3.9 (16.81) | 1.8 (10.69)
  PI, AST, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, AST, Week 20, n=46, 53 | 4.1 (20.85) | 0.5 (4.29)
  PI, AST, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, AST, Week 24, n=47, 53 | 1.5 (7.76) | 1.6 (9.93)
  PI, AST, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, AST, Week 28, n=42, 53 | 2.9 (8.86) | 1.9 (7.45)
  PI, AST, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, AST, Week 32, n=45, 51 | 3.1 (14.13) | 0.6 (4.93)
  PI, AST, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, AST, Week 36, n=44, 50 | 1.7 (8.04) | 1.9 (6.24)
  PI, AST, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, AST, Week 40, n=42, 51 | 5.7 (24.61) | 0.5 (6.05)
  PI, AST, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, AST, Week 44, n=47, 51 | 1.7 (9.71) | 1.4 (11.60)
  PI, AST, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, AST, Week 48, n=43, 50 | 1.7 (7.09) | 2.1 (8.74)
  INI, AST, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, AST, Week 4, n=99, 97 | 0.0 (15.36) | -0.1 (6.29)
  INI, AST, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, AST, Week 8, n=73, 98 | 3.3 (25.01) | 1.2 (21.48)
  INI, AST, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, AST, Week 12, n=99, 95 | -1.3 (14.22) | 0.8 (7.35)
  INI, AST, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, AST, Week 16, n=93, 96 | -2.1 (12.73) | 0.1 (10.96)
  INI, AST, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, AST, Week 20, n=93, 97 | -1.7 (13.77) | -0.9 (12.67)
  INI, AST, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, AST, Week 24, n=94, 95 | -0.4 (14.88) | -0.2 (10.40)
  INI, AST, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, AST, Week 28, n=89, 93 | -1.4 (7.74) | -0.9 (13.48)
  INI, AST, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, AST, Week 32, n=93, 95 | -2.1 (13.06) | -0.8 (10.01)
  INI, AST, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, AST, Week 36, n=94, 95 | -0.7 (17.34) | -1.1 (11.70)
  INI, AST, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, AST, Week 40, n=90, 95 | 1.0 (20.11) | -0.4 (13.96)
  INI, AST, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, AST, Week 44, n=91, 94 | 1.0 (24.54) | -0.7 (10.69)
  INI, AST, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, AST, Week 48, n=91, 95 | 0.4 (16.57) | 0.2 (11.91)
  NNRTI, AST, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, AST, Week 4, n=151, 153 | -1.9 (11.09) | -0.5 (8.73)
  NNRTI, AST, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, AST, Week 8, n=122, 152 | -1.3 (18.14) | -0.9 (8.31)
  NNRTI, AST, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, AST, Week 12, n=146, 152 | 4.7 (91.54) | 0.0 (10.08)
  NNRTI, AST, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, AST, Week 16, n=143, 149 | 0.3 (21.80) | -1.0 (8.37)
  NNRTI, AST, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, AST, Week 20, n=138, 152 | -1.2 (17.47) | -0.7 (9.09)
  NNRTI, AST, Week 24, n=143, 150: number analyzed (Participants) | 143 | 150
  NNRTI, AST, Week 24, n=143, 150 | -0.1 (31.53) | -0.4 (8.87)
  NNRTI, AST, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, AST, Week 28, n=136, 150 | -2.8 (9.02) | 0.4 (10.70)
  NNRTI, AST, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, AST, Week 32, n=137, 148 | -2.0 (18.27) | 1.5 (16.84)
  NNRTI, AST, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, AST, Week 36, n=135, 147 | -2.5 (10.33) | 0.2 (9.00)
  NNRTI, AST, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, AST, Week 40, n=138, 147 | -2.7 (11.14) | 0.1 (9.40)
  NNRTI, AST, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, AST, Week 44, n=137, 148 | -3.4 (10.38) | 0.1 (11.20)
  NNRTI, AST, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, AST, Week 48, n=131, 147 | -2.9 (10.87) | 0.5 (10.60)
  PI, CK, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, CK, Week 4, n=51, 53 | 8.6 (182.21) | 133.5 (907.82)
  PI, CK, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, CK, Week 8, n=34, 53 | 67.9 (176.14) | 23.5 (174.40)
  PI, CK, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, CK, Week 12, n=50, 52 | 3.1 (162.71) | 57.9 (406.52)
  PI, CK, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, CK, Week 16, n=48, 53 | 19.4 (253.86) | 16.3 (66.34)
  PI, CK, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, CK, Week 20, n=46, 53 | 103.6 (696.54) | 6.8 (72.86)
  PI, CK, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, CK, Week 24, n=47, 53 | -3.0 (181.03) | 18.2 (86.69)
  PI, CK, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, CK, Week 28, n=42, 53 | 60.3 (299.83) | 13.5 (93.14)
  PI, CK, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, CK, Week 32, n=45, 51 | 157.1 (988.65) | 1.5 (64.94)
  PI, CK, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, CK, Week 36, n=44, 50 | -9.0 (191.25) | 22.3 (62.09)
  PI, CK, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, CK, Week 40, n=42, 51 | 193.7 (1188.89) | 0.3 (48.24)
  PI, CK, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, CK, Week 44, n=47, 51 | -6.3 (185.69) | 4.8 (62.91)
  PI, CK, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, CK, Week 48, n=43, 50 | -1.0 (158.33) | 72.9 (478.94)
  INI, CK, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, CK, Week 4, n=99, 97 | -32.7 (717.86) | -17.9 (260.84)
  INI, CK, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, CK, Week 8, n=73, 98 | 95.6 (801.75) | -58.0 (577.11)
  INI, CK, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, CK, Week 12, n=99, 95 | -16.1 (852.44) | -23.9 (304.61)
  INI, CK, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, CK, Week 16, n=93, 96 | -59.5 (629.54) | -1.9 (686.38)
  INI, CK, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, CK, Week 20, n=93, 97 | -55.7 (623.92) | -58.1 (622.84)
  INI, CK, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, CK, Week 24, n=94, 95 | -63.1 (549.02) | -40.7 (588.24)
  INI, CK Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, CK Week 28, n=89, 93 | -17.4 (224.35) | -27.4 (759.07)
  INI, CK, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, CK, Week 32, n=93, 95 | -82.8 (587.51) | -42.1 (637.00)
  INI, CK, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, CK, Week 36, n=94, 95 | -76.1 (602.03) | -60.9 (603.48)
  INI, CK, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, CK, Week 40, n=90, 95 | 40.3 (864.00) | -36.2 (609.80)
  INI, CK, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, CK, Week 44, n=91, 94 | 199.8 (2043.35) | -60.2 (576.84)
  INI, CK, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, CK, Week 48, n=91, 95 | 20.5 (861.55) | -25.0 (653.03)
  NNRTI, CK, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, CK, Week 4, n=151, 153 | 18.2 (502.12) | 26.0 (214.58)
  NNRTI, CK, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, CK, Week 8, n=122, 152 | 108.2 (1339.52) | -3.6 (108.28)
  NNRTI, CK, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, CK, Week 12, n=146, 152 | 21.9 (440.81) | 24.5 (222.26)
  NNRTI, CK, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, CK, Week 16, n=143, 149 | 139.9 (1121.08) | 7.0 (189.21)
  NNRTI, CK, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, CK, Week 20, n=138, 152 | 65.5 (656.11) | 1.6 (114.05)
  NNRTI, CK, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, CK, Week 24, n=143, 151 | 24.1 (606.47) | 17.7 (167.38)
  NNRTI, CK, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, CK, Week 28, n=136, 150 | -10.9 (169.29) | 53.2 (462.07)
  NNRTI, CK, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, CK, Week 32, n=137, 148 | 31.3 (650.27) | 94.0 (665.17)
  NNRTI, CK, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, CK, Week 36, n=135, 147 | 19.0 (440.56) | 10.3 (135.08)
  NNRTI, CK, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, CK, Week 40, n=138, 147 | -7.7 (237.00) | 22.6 (195.23)
  NNRTI, CK, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, CK, Week 44, n=137, 148 | -35.4 (183.15) | 14.9 (173.39)
  NNRTI, CK, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, CK, Week 48, n=131, 147 | -15.1 (212.52) | 27.3 (272.59)

66. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: Albumin
Description: Blood samples were collected for the analysis of clinical chemistry parameter: albumin to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Grams per Liter
  PI, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Week 4, n=51, 53 | 0.2 (2.21) | -0.2 (2.41)
  PI, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Week 8, n=34, 53 | 0.7 (2.73) | -0.1 (2.74)
  PI, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Week 12, n=50, 52 | -0.2 (2.67) | -0.3 (2.81)
  PI, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Week 16, n=48, 53 | -0.2 (2.77) | -0.8 (2.72)
  PI, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Week 20, n=46, 53 | -0.4 (2.35) | -0.8 (2.82)
  PI, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Week 24, n=47, 53 | -0.6 (2.24) | -0.8 (2.40)
  PI, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Week 28, n=42, 53 | -0.6 (2.26) | -1.4 (2.08)
  PI, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Week 32, n=45, 51 | -0.7 (2.39) | -0.5 (2.42)
  PI, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Week 36, n=44, 50 | -0.6 (2.44) | -0.9 (2.48)
  PI, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Week 40, n=42, 51 | -0.1 (2.72) | -0.5 (2.37)
  PI, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Week 44, n=47, 51 | -0.5 (2.15) | -0.5 (2.60)
  PI, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Week 48, n=43, 50 | -0.3 (2.74) | -0.1 (2.44)
  INI, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Week 4, n=99, 97 | -0.4 (2.56) | -0.9 (2.62)
  INI, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Week 8, n=73, 98 | -0.5 (2.59) | -1.0 (2.89)
  INI, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Week 12, n=99, 95 | -0.3 (2.92) | -0.5 (2.59)
  INI, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Week 16, n=93, 96 | -0.5 (2.78) | -1.1 (2.80)
  INI, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Week 20, n=93, 97 | -0.7 (2.71) | -0.7 (2.77)
  INI, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 24, n=94, 95 | -0.8 (2.86) | -1.0 (2.74)
  INI, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Week 28, n=89, 93 | -0.3 (2.55) | -1.1 (2.87)
  INI, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Week 32, n=93, 95 | -0.2 (2.70) | -1.3 (2.77)
  INI, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 36, n=94, 95 | -0.8 (2.67) | -1.1 (2.54)
  INI, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Week 40, n=90, 95 | -0.3 (2.40) | -1.3 (2.84)
  INI, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Week 44, n=91, 94 | -0.5 (2.77) | -1.0 (2.76)
  INI, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Week 48, n=91, 95 | -0.1 (2.69) | -0.5 (2.69)
  NNRTI, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Week 4, n=151, 153 | -0.8 (2.70) | -0.3 (2.42)
  NNRTI, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Week 8, n=122, 152 | -0.4 (2.83) | -0.6 (2.53)
  NNRTI, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Week 12, n=146, 152 | -0.8 (2.59) | -0.3 (2.61)
  NNRTI, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Week 16, n=143, 149 | -0.8 (2.79) | -0.7 (2.63)
  NNRTI, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Week 20, n=138, 152 | -0.9 (2.96) | -0.9 (2.33)
  NNRTI, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Week 24, n=143, 151 | -0.7 (2.73) | -0.7 (2.57)
  NNRTI, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Week 28, n=136, 150 | -0.9 (2.72) | -0.9 (2.34)
  NNRTI, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Week 32, n=137, 148 | -0.9 (2.94) | -1.0 (2.45)
  NNRTI, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Week 36, n=135, 147 | -1.0 (2.83) | -0.8 (2.79)
  NNRTI, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Week 40, n=138, 147 | -0.7 (2.54) | -1.0 (2.52)
  NNRTI, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Week 44, n=137, 148 | -0.3 (2.60) | -0.8 (2.22)
  NNRTI, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Week 48, n=131, 147 | -0.6 (2.57) | -0.5 (2.49)

67. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameter: bilirubin, direct bilirubin and creatinine to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Micromoles per liter
  PI, Bilirubin, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Bilirubin, Week 4, n=51, 53 | -9.0 (20.62) | 0.3 (6.95)
  PI, Bilirubin, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Bilirubin, Week 8, n=34, 53 | -6.6 (13.76) | 0.1 (5.76)
  PI, Bilirubin, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Bilirubin, Week 12, n=50, 52 | -10.2 (20.18) | 1.7 (7.11)
  PI, Bilirubin, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Bilirubin, Week 16, n=48, 53 | -10.0 (20.13) | 0.6 (6.42)
  PI, Bilirubin, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Bilirubin, Week 20, n=46, 53 | -9.2 (20.21) | 1.5 (12.45)
  PI, Bilirubin, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Bilirubin, Week 24, n=47, 53 | -9.6 (20.64) | 2.7 (11.87)
  PI, Bilirubin, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Bilirubin, Week 28, n=42, 53 | -10.0 (22.42) | 0.9 (7.70)
  PI, Bilirubin, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Bilirubin, Week 32, n=45, 51 | -8.9 (21.34) | 2.7 (8.64)
  PI, Bilirubin, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Bilirubin, Week 36, n=44, 50 | -10.5 (21.75) | 2.6 (7.35)
  PI, Bilirubin, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Bilirubin, Week 40, n=42, 51 | -11.0 (22.20) | 3.5 (12.74)
  PI, Bilirubin, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Bilirubin, Week 44, n=47, 51 | -9.6 (20.32) | 3.7 (9.10)
  PI, Bilirubin, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Bilirubin, Week 48, n=43, 50 | -10.7 (21.77) | 2.3 (5.23)
  INI, Bilirubin, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Bilirubin, Week 4, n=99, 97 | 0.2 (3.92) | -0.7 (3.93)
  INI, Bilirubin, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Bilirubin, Week 8, n=73, 98 | 0.4 (3.96) | 0.9 (12.43)
  INI, Bilirubin, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Bilirubin, Week 12, n=99, 95 | 0.6 (4.41) | -0.5 (4.69)
  INI, Bilirubin, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Bilirubin, Week 16, n=93, 96 | 0.6 (4.30) | -0.2 (4.35)
  INI, Bilirubin, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Bilirubin, Week 20, n=93, 97 | 0.9 (4.08) | -0.5 (4.32)
  INI, Bilirubin, Week 24, n=94, 94: number analyzed (Participants) | 94 | 94
  INI, Bilirubin, Week 24, n=94, 94 | 0.2 (3.72) | -0.5 (3.88)
  INI, Bilirubin, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Bilirubin, Week 28, n=89, 93 | 1.1 (3.58) | -0.4 (4.85)
  INI, Bilirubin, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Bilirubin, Week 32, n=93, 95 | 0.7 (4.67) | -1.1 (4.54)
  INI, Bilirubin, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Bilirubin, Week 36, n=94, 95 | 0.5 (4.07) | -0.6 (4.62)
  INI, Bilirubin, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Bilirubin, Week 40, n=90, 95 | 0.6 (4.28) | -1.0 (4.26)
  INI, Bilirubin, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Bilirubin, Week 44, n=91, 94 | 0.9 (4.34) | -0.7 (4.72)
  INI, Bilirubin, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Bilirubin, Week 48, n=91, 95 | 1.1 (3.72) | -0.9 (3.96)
  NNRTI, Bilirubin, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Bilirubin, Week 4, n=151, 153 | 1.4 (3.87) | -0.4 (2.85)
  NNRTI, Bilirubin, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Bilirubin, Week 8, n=122, 152 | 1.4 (3.84) | -0.4 (2.43)
  NNRTI, Bilirubin, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Bilirubin, Week 12, n=146, 152 | 2.0 (4.69) | -0.2 (3.01)
  NNRTI, Bilirubin, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Bilirubin, Week 16, n=143, 149 | 3.3 (14.12) | -0.5 (2.66)
  NNRTI, Bilirubin, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Bilirubin, Week 20, n=138, 152 | 2.1 (4.90) | -0.1 (2.81)
  NNRTI, Bilirubin, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Bilirubin, Week 24, n=143, 151 | 1.8 (3.91) | -0.3 (2.84)
  NNRTI, Bilirubin, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Bilirubin, Week 28, n=136, 150 | 2.4 (4.11) | -0.4 (3.04)
  NNRTI, Bilirubin, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Bilirubin, Week 32, n=137, 148 | 2.2 (4.76) | -0.3 (2.57)
  NNRTI, Bilirubin, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Bilirubin, Week 36, n=135, 147 | 1.8 (4.14) | -0.2 (2.61)
  NNRTI, Bilirubin, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Bilirubin, Week 40, n=138, 147 | 2.2 (4.43) | -0.2 (2.61)
  NNRTI, Bilirubin, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Bilirubin, Week 44, n=137, 148 | 2.0 (4.15) | -0.1 (2.72)
  NNRTI, Bilirubin, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Bilirubin, Week 48, n=131, 147 | 2.2 (4.59) | 0.1 (2.98)
  PI, Direct bilirubin, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Direct bilirubin, Week 4, n=51, 53 | -1.2 (2.34) | 0.3 (1.40)
  PI, Direct bilirubin, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Direct bilirubin, Week 8, n=34, 53 | -0.9 (2.16) | -0.1 (1.44)
  PI, Direct bilirubin, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Direct bilirubin, Week 12, n=50, 52 | -1.6 (2.16) | 0.3 (1.39)
  PI, direct bilirubin, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, direct bilirubin, Week 16, n=48, 53 | -1.7 (2.12) | 0.0 (1.30)
  PI, Direct bilirubin, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Direct bilirubin, Week 20, n=46, 53 | -1.5 (2.27) | 0.0 (1.86)
  PI, Direct bilirubin, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Direct bilirubin, Week 24, n=47, 53 | -1.4 (2.27) | 0.2 (1.72)
  PI, Direct bilirubin, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Direct bilirubin, Week 28, n=42, 53 | -1.6 (2.43) | -0.3 (1.52)
  PI, Direct bilirubin, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Direct bilirubin, Week 32, n=45, 51 | -1.4 (2.48) | 0.2 (1.74)
  PI, Direct bilirubin, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Direct bilirubin, Week 36, n=44, 50 | -1.8 (2.29) | 0.2 (1.49)
  PI, Direct bilirubin, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Direct bilirubin, Week 40, n=42, 51 | -1.8 (2.29) | 0.2 (1.43)
  PI, Direct bilirubin, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Direct bilirubin, Week 44, n=47, 51 | -1.5 (2.22) | 0.3 (1.52)
  PI, Direct bilirubin, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Direct bilirubin, Week 48, n=43, 50 | -1.5 (2.35) | 0.2 (1.36)
  INI, Direct bilirubin, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Direct bilirubin, Week 4, n=99, 97 | 0.0 (1.11) | 0.0 (1.19)
  INI, Direct bilirubin, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Direct bilirubin, Week 8, n=73, 98 | 0.0 (1.13) | 0.7 (6.76)
  INI, Direct bilirubin, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Direct bilirubin, Week 12, n=99, 95 | 0.0 (1.14) | 0.0 (1.29)
  INI, Direct bilirubin, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Direct bilirubin, Week 16, n=93, 96 | 0.0 (1.14) | -0.3 (1.06)
  INI, Direct bilirubin, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Direct bilirubin, Week 20, n=93, 97 | -0.2 (0.96) | -0.2 (1.23)
  INI, Direct bilirubin, Week 24, n=94, 94: number analyzed (Participants) | 94 | 94
  INI, Direct bilirubin, Week 24, n=94, 94 | -0.1 (1.07) | -0.3 (1.16)
  INI, Direct bilirubin, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Direct bilirubin, Week 28, n=89, 93 | -0.1 (0.97) | -0.2 (1.30)
  INI, Direct bilirubin, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Direct bilirubin, Week 32, n=93, 95 | -0.2 (1.24) | -0.4 (1.15)
  INI, Direct bilirubin, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Direct bilirubin, Week 36, n=94, 95 | -0.2 (1.33) | -0.3 (1.18)
  INI, Direct bilirubin, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Direct bilirubin, Week 40, n=90, 95 | -0.1 (1.10) | -0.4 (1.24)
  INI, Direct bilirubin. Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Direct bilirubin. Week 44, n=91, 94 | 0.0 (1.14) | -0.3 (1.11)
  INI, Direct bilirubin, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Direct bilirubin, Week 48, n=91, 95 | 0.0 (1.01) | -0.1 (1.28)
  NNRTI, Direct bilirubin, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Direct bilirubin, Week 4, n=151, 153 | 0.1 (1.14) | 0.1 (1.12)
  NNRTI, Direct bilirubin, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Direct bilirubin, Week 8, n=122, 152 | 0.1 (1.24) | 0.0 (1.03)
  NNRTI, Direct bilirubin, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Direct bilirubin, Week 12, n=146, 152 | 0.2 (1.38) | 0.0 (1.08)
  NNRTI, Direct bilirubin, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Direct bilirubin, Week 16, n=143, 149 | 0.7 (6.82) | -0.1 (1.09)
  NNRTI, Direct bilirubin, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Direct bilirubin, Week 20, n=138, 152 | 0.1 (1.32) | -0.2 (1.08)
  NNRTI, Direct bilirubin, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Direct bilirubin, Week 24, n=143, 151 | 0.1 (1.34) | -0.1 (1.06)
  NNRTI, Direct bilirubin, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Direct bilirubin, Week 28, n=136, 150 | 0.1 (1.29) | -0.2 (1.19)
  NNRTI, Direct bilirubin, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Direct bilirubin, Week 32, n=137, 148 | 0.0 (1.31) | -0.2 (1.06)
  NNRTI, Direct bilirubin, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Direct bilirubin, Week 36, n=135, 147 | 0.0 (1.47) | -0.2 (1.09)
  NNRTI, Direct bilirubin, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Direct bilirubin, Week 40, n=138, 147 | 0.0 (1.55) | -0.2 (1.01)
  NNRTI, Direct bilirubin, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Direct bilirubin, Week 44, n=137, 148 | 0.1 (1.28) | -0.1 (1.08)
  NNRTI, Direct bilirubin, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Direct bilirubin, Week 48, n=131, 147 | 0.1 (1.27) | 0.0 (1.16)
  PI, Creatinine, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Creatinine, Week 4, n=51, 53 | 1.46 (7.726) | 2.16 (6.737)
  PI, Creatinine, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Creatinine, Week 8, n=34, 53 | 0.87 (7.777) | 1.17 (5.605)
  PI, Creatinine, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Creatinine, Week 12, n=50, 52 | -1.66 (8.971) | 3.01 (5.406)
  PI, Creatinine, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Creatinine, Week 16, n=48, 53 | -0.90 (8.658) | 2.88 (5.918)
  PI, Creatinine, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Creatinine, Week 20, n=46, 53 | 1.63 (8.709) | 5.00 (9.336)
  PI, Creatinine, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Creatinine, Week 24, n=47, 53 | 0.48 (7.143) | 2.47 (6.821)
  PI, Creatinine, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Creatinine, Week 28, n=42, 53 | 3.06 (9.741) | 3.05 (6.908)
  PI, Creatinine, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Creatinine, Week 32, n=45, 51 | 2.29 (10.124) | 3.79 (6.540)
  PI, Creatinine, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Creatinine, Week 36, n=44, 50 | 2.20 (7.347) | 2.36 (6.291)
  PI, Creatinine, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Creatinine, Week 40, n=42, 51 | 1.10 (9.155) | 3.46 (6.166)
  PI, Creatinine, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Creatinine, Week 44, n=47, 51 | 3.01 (8.981) | 2.73 (6.169)
  PI, Creatinine, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Creatinine, Week 48, n=43, 50 | 4.41 (10.009) | 1.86 (5.575)
  INI, Creatinine, Week 4, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Creatinine, Week 4, n=99, 95 | -1.61 (8.848) | 1.64 (10.592)
  INI, Creatinine, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Creatinine, Week 8, n=73, 98 | -3.93 (10.030) | 1.56 (9.444)
  INI, Creatinine, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Creatinine, Week 12, n=99, 95 | -2.47 (10.973) | 3.03 (10.203)
  INI, Creatinine, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Creatinine, Week 16, n=93, 96 | -3.93 (9.000) | 0.36 (8.651)
  INI, Creatinine, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Creatinine, Week 20, n=93, 97 | -3.73 (9.101) | 0.86 (9.608)
  INI, Creatinine, Week 24, n=94, 94: number analyzed (Participants) | 94 | 94
  INI, Creatinine, Week 24, n=94, 94 | -4.25 (8.281) | 0.87 (10.493)
  INI, Creatinine, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Creatinine, Week 28, n=89, 93 | -3.54 (10.713) | 0.92 (10.086)
  INI, Creatinine, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Creatinine, Week 32, n=93, 95 | -3.48 (10.591) | 0.86 (9.754)
  INI, Creatinine, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Creatinine, Week 36, n=94, 95 | -4.31 (10.360) | 1.34 (9.369)
  INI, Creatinine, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Creatinine, Week 40, n=90, 95 | -3.08 (9.913) | 1.66 (10.272)
  INI, Creatinine, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Creatinine, Week 44, n=91, 94 | -3.33 (9.165) | 0.98 (10.443)
  INI, Creatinine, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Creatinine, Week 48, n=91, 95 | -2.99 (9.442) | 0.47 (9.602)
  NNRTI, Creatinine, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Creatinine, Week 4, n=151, 153 | 2.86 (7.456) | 1.77 (6.484)
  NNRTI, Creatinine, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Creatinine, Week 8, n=122, 152 | 0.86 (8.263) | 1.05 (6.790)
  NNRTI, Creatinine, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Creatinine, Week 12, n=146, 152 | 1.47 (7.928) | 0.44 (6.096)
  NNRTI, Creatinine, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Creatinine, Week 16, n=143, 149 | 1.67 (8.934) | 1.98 (8.475)
  NNRTI, Creatinine, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Creatinine, Week 20, n=138, 152 | 3.04 (8.836) | 1.27 (7.023)
  NNRTI, Creatinine, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Creatinine, Week 24, n=143, 151 | 4.42 (14.819) | 1.28 (6.553)
  NNRTI, Creatinine, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Creatinine, Week 28, n=136, 150 | 3.61 (10.627) | 1.50 (7.483)
  NNRTI, Creatinine, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Creatinine, Week 32, n=137, 148 | 2.26 (9.033) | 2.01 (7.811)
  NNRTI, Creatinine, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Creatinine, Week 36, n=135, 147 | 2.98 (10.596) | 1.54 (7.354)
  NNRTI, Creatinine, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Creatinine, Week 40, n=138, 147 | 3.39 (9.496) | 0.99 (7.471)
  NNRTI, Creatinine, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Creatinine, Week 44, n=137, 148 | 3.24 (8.892) | 1.21 (6.686)
  NNRTI, Creatinine, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Creatinine, Week 48, n=131, 147 | 3.84 (11.860) | 0.69 (7.241)

68. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: Creatinine Clearance
Description: Blood samples were collected for the analysis of clinical chemistry parameter: creatinine clearance to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). GFR will be estimated by the central laboratory using the CKD-EPI. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliters per minute per 1.73meter^2
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Milliliters per minute per 1.73meter^2
  PI, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Week 4, n=51, 53 | -2.2 (9.77) | -2.8 (8.02)
  PI, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Week 8, n=34, 53 | -1.1 (10.19) | -1.3 (6.58)
  PI, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Week 12, n=50, 52 | 2.2 (11.04) | -3.7 (6.99)
  PI, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Week 16, n=48, 53 | 0.9 (11.02) | -3.1 (7.63)
  PI, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Week 20, n=46, 53 | -2.2 (10.80) | -5.0 (9.26)
  PI, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Week 24, n=47, 53 | -1.0 (8.60) | -3.8 (8.51)
  PI, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Week 28, n=42, 53 | -4.2 (11.82) | -4.0 (8.46)
  PI, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Week 32, n=45, 51 | -3.2 (12.30) | -5.2 (7.56)
  PI, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Week 36, n=44, 50 | -3.8 (8.68) | -3.6 (8.08)
  PI, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Week 40, n=42, 51 | -2.4 (10.71) | -4.9 (7.25)
  PI, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Week 44, n=47, 51 | -4.5 (10.63) | -4.2 (7.58)
  PI, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Week 48, n=43, 50 | -5.6 (12.22) | -3.1 (6.54)
  INI, Week 4, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Week 4, n=99, 95 | 1.0 (9.51) | -2.0 (11.28)
  INI, Week 8, n=72, 98: number analyzed (Participants) | 72 | 98
  INI, Week 8, n=72, 98 | 3.9 (9.84) | -1.9 (9.28)
  INI, Week 12, n=99, 93: number analyzed (Participants) | 99 | 93
  INI, Week 12, n=99, 93 | 2.1 (11.32) | -3.1 (9.60)
  INI, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Week 16, n=93, 96 | 3.6 (9.71) | -0.7 (8.59)
  INI, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Week 20, n=93, 97 | 3.5 (9.77) | -1.7 (9.58)
  INI, Week 24, n=94, 94: number analyzed (Participants) | 94 | 94
  INI, Week 24, n=94, 94 | 3.9 (9.26) | -1.8 (10.38)
  INI, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Week 28, n=89, 93 | 3.1 (11.02) | -1.6 (9.55)
  INI, Week 32, n=92, 95: number analyzed (Participants) | 92 | 95
  INI, Week 32, n=92, 95 | 3.0 (10.40) | -2.0 (9.69)
  INI, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 36, n=94, 95 | 3.7 (11.19) | -2.3 (9.30)
  INI, Week 40, n=89, 95: number analyzed (Participants) | 89 | 95
  INI, Week 40, n=89, 95 | 2.7 (10.45) | -2.6 (10.14)
  INI, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Week 44, n=91, 94 | 2.6 (9.88) | -1.6 (10.90)
  INI, Week 48, n=90, 94: number analyzed (Participants) | 90 | 94
  INI, Week 48, n=90, 94 | 3.0 (9.74) | -1.6 (9.73)
  NNRTI, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Week 4, n=151, 153 | -3.4 (9.06) | -2.3 (8.10)
  NNRTI, Week 8, n=121, 152: number analyzed (Participants) | 121 | 152
  NNRTI, Week 8, n=121, 152 | -1.1 (9.35) | -1.3 (7.72)
  NNRTI, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Week 12, n=146, 152 | -1.7 (8.90) | -0.5 (7.03)
  NNRTI, Week 16, n=143, 148: number analyzed (Participants) | 143 | 148
  NNRTI, Week 16, n=143, 148 | -1.8 (10.60) | -2.3 (9.06)
  NNRTI, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Week 20, n=138, 152 | -3.7 (9.64) | -1.9 (7.41)
  NNRTI, Week 24, n=142, 151: number analyzed (Participants) | 142 | 151
  NNRTI, Week 24, n=142, 151 | -4.3 (10.67) | -2.0 (7.67)
  NNRTI, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Week 28, n=136, 150 | -4.3 (10.68) | -2.4 (8.67)
  NNRTI, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Week 32, n=137, 148 | -3.3 (10.42) | -2.8 (8.80)
  NNRTI, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Week 36, n=135, 147 | -3.8 (10.97) | -2.5 (8.16)
  NNRTI, Week 40, n=137, 147: number analyzed (Participants) | 137 | 147
  NNRTI, Week 40, n=137, 147 | -4.4 (9.97) | -2.0 (8.90)
  NNRTI, Week 44, n=136, 148: number analyzed (Participants) | 136 | 148
  NNRTI, Week 44, n=136, 148 | -4.4 (9.75) | -2.0 (7.45)
  NNRTI, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Week 48, n=131, 147 | -5.2 (11.72) | -1.6 (8.25)

69. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48: Lipase
Description: Blood samples were collected for the analysis of clinical chemistry parameter: lipase to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Units per liter
  PI, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Week 4, n=51, 53 | -2.2 (16.83) | 1.2 (19.34)
  PI, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Week 8, n=34, 53 | -2.6 (6.71) | 2.5 (25.36)
  PI, Week 12, n=49, 52: number analyzed (Participants) | 49 | 52
  PI, Week 12, n=49, 52 | -1.4 (17.24) | -2.2 (15.95)
  PI, Week 16, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Week 16, n=47, 53 | -0.5 (18.71) | 1.4 (17.40)
  PI, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Week 20, n=46, 53 | -2.5 (17.90) | -0.6 (17.49)
  PI, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Week 24, n=47, 53 | -2.0 (16.61) | -2.7 (16.30)
  PI, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Week 28, n=42, 53 | -0.7 (18.60) | 0.2 (16.18)
  PI, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Week 32, n=45, 51 | -2.2 (19.27) | 2.5 (18.35)
  PI, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Week 36, n=44, 50 | -0.8 (17.96) | -1.2 (18.18)
  PI, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Week 40, n=42, 51 | 2.2 (26.77) | -1.8 (19.40)
  PI, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Week 44, n=47, 51 | -1.2 (18.28) | 1.4 (17.94)
  PI, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Week 48, n=43, 50 | -1.5 (19.38) | -1.3 (15.73)
  INI, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Week 4, n=99, 97 | 8.1 (34.32) | 3.8 (30.44)
  INI, Week 8, n=72, 98: number analyzed (Participants) | 72 | 98
  INI, Week 8, n=72, 98 | 0.7 (9.79) | -0.5 (14.46)
  INI, Week 12, n=99, 93: number analyzed (Participants) | 99 | 93
  INI, Week 12, n=99, 93 | 4.3 (17.70) | 1.8 (21.29)
  INI, Week 16, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Week 16, n=93, 97 | 4.4 (22.42) | 0.6 (16.13)
  INI, Week 20, n=94, 97: number analyzed (Participants) | 94 | 97
  INI, Week 20, n=94, 97 | 2.5 (17.23) | 0.9 (17.07)
  INI, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 24, n=94, 95 | 2.2 (15.17) | 2.2 (18.91)
  INI, Week 28, n=89, 94: number analyzed (Participants) | 89 | 94
  INI, Week 28, n=89, 94 | 5.6 (28.06) | 5.1 (24.20)
  INI, Week 32, n=92, 95: number analyzed (Participants) | 92 | 95
  INI, Week 32, n=92, 95 | 3.2 (18.68) | 5.4 (22.79)
  INI, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Week 36, n=94, 95 | 5.2 (21.04) | 0.1 (13.82)
  INI, Week 40, n=89, 95: number analyzed (Participants) | 89 | 95
  INI, Week 40, n=89, 95 | 3.5 (11.71) | 1.7 (16.60)
  INI, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Week 44, n=91, 94 | 4.3 (21.59) | 4.8 (23.54)
  INI, Week 48, n=90, 94: number analyzed (Participants) | 90 | 94
  INI, Week 48, n=90, 94 | 5.0 (24.95) | 3.9 (23.48)
  NNRTI, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Week 4, n=151, 153 | 5.7 (50.44) | 0.1 (20.35)
  NNRTI, Week 8, n=121, 152: number analyzed (Participants) | 121 | 152
  NNRTI, Week 8, n=121, 152 | 2.6 (25.04) | 1.5 (16.94)
  NNRTI, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Week 12, n=146, 152 | 3.0 (30.94) | -1.9 (17.59)
  NNRTI, Week 16, n=145, 149: number analyzed (Participants) | 145 | 149
  NNRTI, Week 16, n=145, 149 | 2.5 (27.82) | 6.1 (40.62)
  NNRTI, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Week 20, n=138, 152 | 0.9 (13.53) | 1.3 (37.14)
  NNRTI, Week 24, n=142, 151: number analyzed (Participants) | 142 | 151
  NNRTI, Week 24, n=142, 151 | 3.4 (24.81) | 5.4 (28.22)
  NNRTI, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Week 28, n=136, 150 | 0.8 (24.38) | 1.2 (15.79)
  NNRTI, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Week 32, n=137, 148 | 9.1 (78.96) | 1.9 (21.30)
  NNRTI, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Week 36, n=135, 147 | 6.9 (68.07) | 1.7 (19.14)
  NNRTI, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Week 40, n=138, 147 | 7.1 (43.53) | 0.5 (17.62)
  NNRTI, Week 44, n=136, 148: number analyzed (Participants) | 136 | 148
  NNRTI, Week 44, n=136, 148 | 1.6 (24.46) | 1.1 (20.52)
  NNRTI, Week 48, n=131, 146: number analyzed (Participants) | 131 | 146
  NNRTI, Week 48, n=131, 146 | 3.1 (32.54) | 0.9 (16.60)

70. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Using Baseline Third Agent Treatment Class Overtime Including Week 48
Description: Blood samples were collected for the analysis of clinical chemistry parameters: CO2, chloride, glucose, phosphate, potassium, sodium and urea to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Millimoles per liter
  PI, CO2, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, CO2, Week 4, n=51, 53 | 1.3 (2.63) | 0.7 (2.34)
  PI, CO2, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, CO2, Week 8, n=34, 53 | 0.4 (2.36) | 0.3 (2.65)
  PI, CO2, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, CO2, Week 12, n=50, 52 | 0.7 (2.84) | 0.2 (2.23)
  PI, CO2, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, CO2, Week 16, n=48, 53 | 0.8 (2.60) | 0.2 (2.32)
  PI, CO2, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, CO2, Week 20, n=46, 53 | 0.9 (2.53) | 0.0 (2.26)
  PI, CO2, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, CO2, Week 24, n=47, 53 | 0.4 (2.23) | 0.1 (1.94)
  PI, CO2, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, CO2, Week 28, n=42, 53 | 0.6 (2.54) | -0.2 (2.37)
  PI, CO2, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, CO2, Week 32, n=45, 51 | 0.5 (2.35) | -0.2 (2.36)
  PI, CO2, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, CO2, Week 36, n=44, 50 | 0.5 (2.38) | -0.4 (1.98)
  PI, CO2, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, CO2, Week 40, n=42, 51 | 0.5 (2.10) | 0.3 (2.26)
  PI, CO2, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, CO2, Week 44, n=47, 51 | 0.7 (2.29) | 0.3 (2.18)
  PI, CO2, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, CO2, Week 48, n=43, 50 | 0.9 (2.69) | -0.1 (1.87)
  INI, CO2, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, CO2, Week 4, n=99, 97 | 1.0 (2.37) | 0.8 (2.21)
  INI, CO2, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, CO2, Week 8, n=73, 98 | 0.5 (2.29) | 0.6 (2.46)
  INI, CO2, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, CO2, Week 12, n=99, 95 | 0.4 (2.27) | 0.3 (2.31)
  INI, CO2, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, CO2, Week 16, n=93, 96 | 0.1 (2.56) | 0.6 (2.53)
  INI, CO2, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, CO2, Week 20, n=93, 97 | 0.1 (2.07) | 0.7 (2.25)
  INI, CO2, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, CO2, Week 24, n=94, 95 | 0.1 (2.32) | 0.2 (2.49)
  INI, CO2, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, CO2, Week 28, n=89, 93 | -0.3 (2.30) | 0.2 (2.41)
  INI, CO2, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, CO2, Week 32, n=93, 95 | 0.2 (2.33) | 0.1 (2.34)
  INI, CO2, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, CO2, Week 36, n=94, 95 | 0.0 (2.36) | 0.5 (2.58)
  INI, CO2, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, CO2, Week 40, n=90, 95 | 0.5 (2.43) | 0.3 (2.18)
  INI, CO2, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, CO2, Week 44, n=91, 94 | 0.5 (2.36) | 0.7 (2.45)
  INI, CO2, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, CO2, Week 48, n=91, 95 | 0.1 (2.12) | 0.3 (2.53)
  NNRTI, CO2, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, CO2, Week 4, n=151, 153 | 0.9 (2.60) | 0.7 (2.18)
  NNRTI, CO2, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, CO2, Week 8, n=122, 152 | 0.4 (2.32) | 0.8 (2.52)
  NNRTI, CO2, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, CO2, Week 12, n=146, 152 | 0.5 (2.38) | 0.4 (2.51)
  NNRTI, CO2, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, CO2, Week 16, n=143, 149 | 0.3 (2.25) | 0.5 (2.37)
  NNRTI, CO2, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, CO2, Week 20, n=138, 152 | 0.1 (2.27) | 0.2 (2.35)
  NNRTI, CO2, Week 24, n=143, 150: number analyzed (Participants) | 143 | 150
  NNRTI, CO2, Week 24, n=143, 150 | 0.3 (2.63) | 0.3 (2.57)
  NNRTI, CO2, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, CO2, Week 28, n=136, 150 | 0.1 (2.54) | 0.2 (2.40)
  NNRTI, CO2, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, CO2, Week 32, n=137, 148 | -0.2 (2.39) | 0.4 (2.27)
  NNRTI, CO2, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, CO2, Week 36, n=135, 147 | 0.1 (2.38) | 0.5 (2.37)
  NNRTI, CO2, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, CO2, Week 40, n=138, 147 | 0.4 (2.64) | 0.5 (2.38)
  NNRTI, CO2, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, CO2, Week 44, n=137, 148 | 0.4 (2.35) | 0.5 (2.01)
  NNRTI, CO2, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, CO2, Week 48, n=131, 147 | -0.1 (2.47) | 0.3 (2.30)
  PI, Chloride, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Chloride, Week 4, n=51, 53 | 0.5 (1.80) | 0.5 (2.34)
  PI, Chloride, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Chloride, Week 8, n=34, 53 | 0.2 (2.59) | 0.7 (2.42)
  PI, Chloride, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Chloride, Week 12, n=50, 52 | 0.5 (2.39) | 0.8 (2.20)
  PI, Chloride, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Chloride, Week 16, n=48, 53 | 0.5 (2.46) | 1.0 (2.31)
  PI, Chloride, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Chloride, Week 20, n=46, 53 | 0.8 (2.20) | 0.7 (2.30)
  PI, Chloride, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Chloride, Week 24, n=47, 53 | 1.1 (2.07) | 1.3 (2.36)
  PI, Chloride, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Chloride, Week 28, n=42, 53 | 1.5 (2.19) | 1.2 (3.06)
  PI, Chloride, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Chloride, Week 32, n=45, 51 | 0.9 (2.43) | 0.9 (2.60)
  PI, Chloride, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Chloride, Week 36, n=44, 50 | 1.0 (2.28) | 1.0 (3.00)
  PI, Chloride, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Chloride, Week 40, n=42, 51 | 1.3 (2.35) | 1.1 (2.60)
  PI, Chloride, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Chloride, Week 44, n=47, 51 | 1.1 (2.21) | 1.1 (2.57)
  PI, Chloride, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Chloride, Week 48, n=43, 50 | 0.5 (2.10) | 0.9 (2.29)
  INI, Chloride, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Chloride, Week 4, n=99, 97 | 0.3 (2.02) | 0.5 (1.96)
  INI, Chloride, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Chloride, Week 8, n=73, 98 | 0.2 (2.02) | 0.1 (2.42)
  INI, Chloride, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Chloride, Week 12, n=99, 95 | 0.4 (2.53) | 0.5 (2.27)
  INI, Chloride, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Chloride, Week 16, n=93, 96 | 0.9 (2.45) | 0.7 (2.32)
  INI, Chloride, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Chloride, Week 20, n=93, 97 | 1.0 (2.44) | 0.2 (2.31)
  INI, Chloride, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Chloride, Week 24, n=94, 95 | 0.6 (2.46) | 0.5 (2.19)
  INI, Chloride, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Chloride, Week 28, n=89, 93 | 0.8 (1.92) | 0.3 (2.37)
  INI, Chloride, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Chloride, Week 32, n=93, 95 | 0.7 (2.39) | 0.7 (2.45)
  INI, Chloride, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Chloride, Week 36, n=94, 95 | 0.8 (2.20) | 0.5 (2.32)
  INI, Chloride, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Chloride, Week 40, n=90, 95 | 0.7 (2.24) | 0.4 (2.69)
  INI, Chloride, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Chloride, Week 44, n=91, 94 | 0.7 (2.38) | 0.5 (2.41)
  INI, Chloride, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Chloride, Week 48, n=91, 95 | 0.4 (2.37) | -0.3 (2.36)
  NNRTI, Chloride, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Chloride, Week 4, n=151, 153 | 0.4 (2.15) | 0.6 (2.17)
  NNRTI, Chloride, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Chloride, Week 8, n=122, 152 | 0.4 (2.05) | 0.7 (1.91)
  NNRTI, Chloride, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Chloride, Week 12, n=146, 152 | 0.4 (2.12) | 0.5 (2.27)
  NNRTI, Chloride, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Chloride, Week 16, n=143, 149 | 0.5 (2.37) | 0.8 (2.20)
  NNRTI, Chloride, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Chloride, Week 20, n=138, 152 | 0.7 (2.27) | 1.1 (2.40)
  NNRTI, Chloride, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Chloride, Week 24, n=143, 151 | 0.5 (2.60) | 1.1 (2.24)
  NNRTI, Chloride, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Chloride, Week 28, n=136, 150 | 0.8 (2.38) | 1.3 (2.39)
  NNRTI, Chloride, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Chloride, Week 32, n=137, 148 | 0.8 (2.44) | 1.1 (2.15)
  NNRTI, Chloride, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Chloride, Week 36, n=135, 147 | 1.0 (2.15) | 1.1 (2.37)
  NNRTI, Chloride, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Chloride, Week 40, n=138, 147 | 0.6 (2.20) | 1.0 (2.84)
  NNRTI, Chloride, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Chloride, Week 44, n=137, 148 | 0.6 (2.07) | 1.0 (2.08)
  NNRTI, Chloride, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Chloride, Week 48, n=131, 147 | 0.6 (2.45) | 0.5 (2.36)
  PI, Glucose, Week 4, n=43, 43: number analyzed (Participants) | 43 | 43
  PI, Glucose, Week 4, n=43, 43 | -0.08 (0.922) | 0.32 (0.401)
  PI, Glucose, Week 8, n=25, 41: number analyzed (Participants) | 25 | 41
  PI, Glucose, Week 8, n=25, 41 | 0.17 (0.513) | 0.22 (0.466)
  PI, Glucose, Week 12, n=40, 42: number analyzed (Participants) | 40 | 42
  PI, Glucose, Week 12, n=40, 42 | 0.03 (0.925) | 0.27 (0.494)
  PI, Glucose, Week 16, n=39, 43: number analyzed (Participants) | 39 | 43
  PI, Glucose, Week 16, n=39, 43 | 0.11 (1.163) | 0.28 (0.704)
  PI, Glucose, Week 20, n=35, 41: number analyzed (Participants) | 35 | 41
  PI, Glucose, Week 20, n=35, 41 | -0.07 (1.058) | 0.30 (0.799)
  PI, Glucose, Week 24, n=38, 42: number analyzed (Participants) | 38 | 42
  PI, Glucose, Week 24, n=38, 42 | 0.11 (0.705) | 0.32 (0.636)
  PI, Glucose, Week 28, n=32, 43: number analyzed (Participants) | 32 | 43
  PI, Glucose, Week 28, n=32, 43 | -0.03 (1.342) | 0.16 (0.441)
  PI, Glucose, Week 32, n=36, 41: number analyzed (Participants) | 36 | 41
  PI, Glucose, Week 32, n=36, 41 | 0.23 (1.148) | 0.29 (0.600)
  PI, Glucose, Week 36, n=35, 41: number analyzed (Participants) | 35 | 41
  PI, Glucose, Week 36, n=35, 41 | -0.01 (1.014) | 0.22 (0.483)
  PI, Glucose, Week 40, n=34, 40: number analyzed (Participants) | 34 | 40
  PI, Glucose, Week 40, n=34, 40 | 0.11 (1.035) | 0.18 (0.497)
  PI, Glucose, Week 44, n=40, 40: number analyzed (Participants) | 40 | 40
  PI, Glucose, Week 44, n=40, 40 | 0.01 (1.008) | 0.20 (0.278)
  PI, Glucose, Week 48, n=39, 48: number analyzed (Participants) | 39 | 48
  PI, Glucose, Week 48, n=39, 48 | -0.01 (0.977) | 0.11 (0.663)
  INI, Glucose, Week 4, n=55, 52: number analyzed (Participants) | 55 | 52
  INI, Glucose, Week 4, n=55, 52 | 0.30 (0.613) | 0.07 (0.774)
  INI, Glucose, Week 8, n=36, 57: number analyzed (Participants) | 36 | 57
  INI, Glucose, Week 8, n=36, 57 | 0.12 (0.595) | 0.21 (1.083)
  INI, Glucose, Week 12, n=52, 55: number analyzed (Participants) | 52 | 55
  INI, Glucose, Week 12, n=52, 55 | 0.36 (0.996) | 0.30 (1.357)
  INI, Glucose, Week 16, n=53, 52: number analyzed (Participants) | 53 | 52
  INI, Glucose, Week 16, n=53, 52 | 0.35 (1.437) | 0.13 (0.557)
  INI, Glucose, Week 20, n=51, 57: number analyzed (Participants) | 51 | 57
  INI, Glucose, Week 20, n=51, 57 | 0.25 (0.515) | -0.06 (0.676)
  INI, Glucose, Week 24, n=59, 61: number analyzed (Participants) | 59 | 61
  INI, Glucose, Week 24, n=59, 61 | 0.24 (0.596) | 0.04 (0.652)
  INI, Glucose, Week 28, n=52, 62: number analyzed (Participants) | 52 | 62
  INI, Glucose, Week 28, n=52, 62 | 0.17 (0.681) | 0.33 (0.763)
  INI, Glucose, Week 32, n=53, 55: number analyzed (Participants) | 53 | 55
  INI, Glucose, Week 32, n=53, 55 | 0.48 (1.071) | 0.32 (0.876)
  INI, Glucose, Week 36, n=53, 57: number analyzed (Participants) | 53 | 57
  INI, Glucose, Week 36, n=53, 57 | 0.34 (0.642) | 0.19 (1.063)
  INI, Glucose, Week 40, n=59, 62: number analyzed (Participants) | 59 | 62
  INI, Glucose, Week 40, n=59, 62 | 0.36 (0.922) | 0.14 (0.566)
  INI, Glucose, Week 44, n=54, 57: number analyzed (Participants) | 54 | 57
  INI, Glucose, Week 44, n=54, 57 | 0.33 (0.971) | 0.16 (0.626)
  INI, Glucose, Week 48, n=81, 90: number analyzed (Participants) | 81 | 90
  INI, Glucose, Week 48, n=81, 90 | 0.04 (0.577) | -0.03 (0.796)
  NNRTI, Glucose, Week 4, n=116, 124: number analyzed (Participants) | 116 | 124
  NNRTI, Glucose, Week 4, n=116, 124 | 0.20 (0.666) | 0.24 (1.055)
  NNRTI, Glucose, Week 8, n=90, 116: number analyzed (Participants) | 90 | 116
  NNRTI, Glucose, Week 8, n=90, 116 | 0.27 (0.987) | 0.23 (0.795)
  NNRTI, Glucose, Week 12, n=112, 119: number analyzed (Participants) | 112 | 119
  NNRTI, Glucose, Week 12, n=112, 119 | 0.16 (0.746) | 0.11 (0.887)
  NNRTI, Glucose, Week 16, n=115, 116: number analyzed (Participants) | 115 | 116
  NNRTI, Glucose, Week 16, n=115, 116 | 0.22 (0.767) | 0.33 (1.347)
  NNRTI, Glucose, Week 20, n=106, 118: number analyzed (Participants) | 106 | 118
  NNRTI, Glucose, Week 20, n=106, 118 | 0.25 (0.636) | 0.28 (1.104)
  NNRTI, Glucose, Week 24, n=115, 121: number analyzed (Participants) | 115 | 121
  NNRTI, Glucose, Week 24, n=115, 121 | 0.27 (0.763) | 0.16 (1.037)
  NNRTI, Glucose, Week 28, n=104, 120: number analyzed (Participants) | 104 | 120
  NNRTI, Glucose, Week 28, n=104, 120 | 0.23 (0.596) | 0.30 (1.077)
  NNRTI, Glucose, Week 32, n=103, 117: number analyzed (Participants) | 103 | 117
  NNRTI, Glucose, Week 32, n=103, 117 | 0.32 (0.811) | 0.24 (1.062)
  NNRTI, Glucose, Week 36, n=102, 117: number analyzed (Participants) | 102 | 117
  NNRTI, Glucose, Week 36, n=102, 117 | 0.17 (0.789) | 0.31 (1.217)
  NNRTI, Glucose, Week 40, n=100, 111: number analyzed (Participants) | 100 | 111
  NNRTI, Glucose, Week 40, n=100, 111 | 0.27 (0.692) | 0.33 (1.118)
  NNRTI, Glucose, Week 44, n=99, 116: number analyzed (Participants) | 99 | 116
  NNRTI, Glucose, Week 44, n=99, 116 | 0.26 (0.793) | 0.35 (1.121)
  NNRTI, Glucose, Week 48, n=118, 136: number analyzed (Participants) | 118 | 136
  NNRTI, Glucose, Week 48, n=118, 136 | 0.06 (0.659) | 0.02 (1.074)
  PI, Phosphate, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Phosphate, Week 4, n=51, 53 | 0.068 (0.1513) | 0.009 (0.1682)
  PI, Phosphate, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Phosphate, Week 8, n=34, 53 | 0.076 (0.2023) | -0.019 (0.1752)
  PI, Phosphate, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Phosphate, Week 12, n=50, 52 | 0.025 (0.1794) | 0.007 (0.1524)
  PI, Phosphate, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Phosphate, Week 16, n=48, 53 | 0.056 (0.2028) | -0.008 (0.1610)
  PI, Phosphate, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Phosphate, Week 20, n=46, 53 | 0.069 (0.1864) | 0.017 (0.1924)
  PI, Phosphate, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Phosphate, Week 24, n=47, 53 | 0.037 (0.1971) | 0.018 (0.1735)
  PI, Phosphate, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Phosphate, Week 28, n=42, 53 | 0.035 (0.2140) | 0.017 (0.1971)
  PI, Phosphate, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Phosphate, Week 32, n=45, 51 | 0.053 (0.2191) | 0.032 (0.1545)
  PI, Phosphate, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Phosphate, Week 36, n=44, 50 | 0.032 (0.1818) | -0.001 (0.1828)
  PI, Phosphate, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Phosphate, Week 40, n=42, 51 | 0.027 (0.2392) | 0.001 (0.1657)
  PI, Phosphate, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Phosphate, Week 44, n=47, 51 | 0.033 (0.2107) | 0.011 (0.1736)
  PI, Phosphate, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Phosphate, Week 48, n=43, 50 | 0.048 (0.1994) | 0.017 (0.1387)
  INI, Phosphate, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Phosphate, Week 4, n=99, 97 | 0.036 (0.1518) | 0.017 (0.1588)
  INI, Phosphate, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Phosphate, Week 8, n=73, 98 | 0.056 (0.1532) | 0.010 (0.1676)
  INI, Phosphate, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Phosphate, Week 12, n=99, 95 | 0.024 (0.2108) | 0.017 (0.1808)
  INI, Phosphate, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Phosphate, Week 16, n=93, 96 | 0.031 (0.1895) | 0.001 (0.1708)
  INI, Phosphate, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Phosphate, Week 20, n=93, 97 | 0.012 (0.1764) | 0.025 (0.1823)
  INI, Phosphate, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Phosphate, Week 24, n=94, 95 | 0.031 (0.1501) | -0.011 (0.1785)
  INI, Phosphate, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Phosphate, Week 28, n=89, 93 | 0.032 (0.1628) | 0.006 (0.1806)
  INI, Phosphate, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Phosphate, Week 32, n=93, 95 | 0.012 (0.1751) | -0.017 (0.1827)
  INI, Phosphate, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Phosphate, Week 36, n=94, 95 | -0.002 (0.1496) | -0.001 (0.1979)
  INI, Phosphate, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Phosphate, Week 40, n=90, 95 | 0.018 (0.1766) | -0.002 (0.1721)
  INI, Phosphate, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Phosphate, Week 44, n=91, 94 | 0.005 (0.1695) | 0.005 (0.1977)
  INI, Phosphate, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Phosphate, Week 48, n=91, 95 | 0.028 (0.1684) | 0.002 (0.2072)
  NNRTI, Phosphate, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Phosphate, Week 4, n=151, 153 | 0.085 (0.1785) | 0.016 (0.1580)
  NNRTI, Phosphate, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Phosphate, Week 8, n=122, 152 | 0.061 (0.2002) | -0.012 (0.1515)
  NNRTI, Phosphate, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Phosphate, Week 12, n=146, 152 | 0.057 (0.1946) | 0.012 (0.1780)
  NNRTI, Phosphate, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Phosphate, Week 16, n=143, 149 | 0.043 (0.2088) | 0.008 (0.1613)
  NNRTI, Phosphate, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Phosphate, Week 20, n=138, 152 | 0.039 (0.1935) | -0.002 (0.1823)
  NNRTI, Phosphate, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Phosphate, Week 24, n=143, 151 | 0.050 (0.2220) | 0.012 (0.1923)
  NNRTI, Phosphate, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Phosphate, Week 28, n=136, 150 | 0.040 (0.1850) | -0.003 (0.1789)
  NNRTI, Phosphate, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Phosphate, Week 32, n=137, 148 | 0.018 (0.2056) | 0.011 (0.2020)
  NNRTI, Phosphate, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Phosphate, Week 36, n=135, 147 | 0.014 (0.2069) | -0.002 (0.1794)
  NNRTI, Phosphate, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Phosphate, Week 40, n=138, 147 | 0.026 (0.2095) | -0.006 (0.1783)
  NNRTI, Phosphate, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Phosphate, Week 44, n=137, 148 | 0.041 (0.2112) | 0.000 (0.1735)
  NNRTI, Phosphate, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Phosphate, Week 48, n=131, 147 | 0.034 (0.2220) | -0.001 (0.1619)
  PI, Potassium, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Potassium, Week 4, n=51, 53 | 0.12 (0.369) | 0.20 (0.447)
  PI, Potassium, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Potassium, Week 8, n=34, 53 | 0.05 (0.245) | 0.08 (0.307)
  PI, Potassium, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Potassium, Week 12, n=50, 52 | 0.12 (0.353) | 0.19 (0.388)
  PI, Potassium, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Potassium, Week 16, n=48, 53 | 0.02 (0.343) | 0.19 (0.398)
  PI, Potassium, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Potassium, Week 20, n=46, 53 | 0.05 (0.338) | 0.18 (0.420)
  PI, Potassium, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Potassium, Week 24, n=47, 53 | 0.01 (0.354) | 0.19 (0.384)
  PI, Potassium, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Potassium, Week 28, n=42, 53 | 0.09 (0.338) | 0.15 (0.342)
  PI, Potassium, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Potassium, Week 32, n=45, 51 | 0.02 (0.356) | 0.19 (0.408)
  PI, Potassium, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Potassium, Week 36, n=44, 50 | 0.12 (0.363) | 0.14 (0.371)
  PI, Potassium, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Potassium, Week 40, n=42, 51 | 0.09 (0.348) | 0.15 (0.394)
  PI, Potassium, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Potassium, Week 44, n=47, 51 | 0.10 (0.409) | 0.21 (0.433)
  PI, Potassium, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Potassium, Week 48, n=43, 50 | 0.02 (0.359) | 0.01 (0.409)
  INI, Potassium, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Potassium, Week 4, n=99, 97 | 0.03 (0.308) | 0.08 (0.335)
  INI, Potassium, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Potassium, Week 8, n=73, 98 | -0.02 (0.282) | 0.06 (0.483)
  INI, Potassium, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Potassium, Week 12, n=99, 95 | 0.02 (0.316) | 0.01 (0.329)
  INI, Potassium, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Potassium, Week 16, n=93, 96 | -0.01 (0.286) | 0.01 (0.319)
  INI, Potassium, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Potassium, Week 20, n=93, 97 | 0.03 (0.333) | 0.00 (0.313)
  INI, Potassium, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Potassium, Week 24, n=94, 95 | 0.02 (0.304) | 0.04 (0.315)
  INI, Potassium,Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Potassium,Week 28, n=89, 93 | 0.02 (0.422) | 0.03 (0.372)
  INI, Potassium, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Potassium, Week 32, n=93, 95 | 0.02 (0.322) | 0.01 (0.289)
  INI, Potassium, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Potassium, Week 36, n=94, 95 | 0.01 (0.345) | 0.05 (0.349)
  INI, Potassium, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Potassium, Week 40, n=90, 95 | 0.01 (0.288) | 0.01 (0.329)
  INI, Potassium, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Potassium, Week 44, n=91, 94 | 0.01 (0.265) | 0.00 (0.327)
  INI, Potassium, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Potassium, Week 48, n=91, 95 | -0.03 (0.249) | -0.01 (0.292)
  NNRTI, Potassium, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Potassium, Week 4, n=151, 153 | 0.05 (0.354) | 0.10 (0.368)
  NNRTI, Potassium, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Potassium, Week 8, n=122, 152 | 0.02 (0.342) | 0.05 (0.355)
  NNRTI, Potassium, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Potassium, Week 12, n=146, 152 | 0.02 (0.351) | 0.08 (0.353)
  NNRTI, Potassium, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Potassium, Week 16, n=143, 149 | 0.03 (0.373) | 0.05 (0.320)
  NNRTI, Potassium,Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Potassium,Week 20, n=138, 152 | 0.04 (0.358) | 0.03 (0.355)
  NNRTI, Potassium, Week 24, n=143, 150: number analyzed (Participants) | 143 | 150
  NNRTI, Potassium, Week 24, n=143, 150 | 0.04 (0.329) | 0.04 (0.324)
  NNRTI, Potassium, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Potassium, Week 28, n=136, 150 | 0.03 (0.364) | 0.08 (0.412)
  NNRTI, Potassium, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Potassium, Week 32, n=137, 148 | 0.01 (0.442) | 0.02 (0.348)
  NNRTI, Potassium, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Potassium, Week 36, n=135, 147 | 0.02 (0.359) | 0.05 (0.360)
  NNRTI, Potassium, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Potassium, Week 40, n=138, 147 | 0.05 (0.375) | 0.08 (0.342)
  NNRTI, Potassium, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Potassium, Week 44, n=137, 148 | 0.08 (0.364) | 0.07 (0.366)
  NNRTI, Potassium, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Potassium, Week 48, n=131, 147 | -0.02 (0.311) | 0.00 (0.329)
  PI, Sodium, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Sodium, Week 4, n=51, 53 | 0.4 (1.93) | 0.3 (2.11)
  PI, Sodium, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Sodium, Week 8, n=34, 53 | 0.9 (2.21) | 0.3 (2.25)
  PI, Sodium, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Sodium, Week 12, n=50, 52 | 0.5 (2.09) | 0.7 (1.97)
  PI, Sodium, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Sodium, Week 16, n=48, 53 | 0.5 (2.30) | 0.3 (2.24)
  PI, Sodium, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Sodium, Week 20, n=46, 53 | 0.6 (2.15) | 0.4 (2.12)
  PI, Sodium, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Sodium, Week 24, n=47, 53 | 0.5 (2.33) | 0.4 (2.30)
  PI, Sodium, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Sodium, Week 28, n=42, 53 | 1.3 (2.06) | 0.8 (2.75)
  PI, Sodium, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Sodium, Week 32, n=45, 51 | 0.5 (2.47) | 0.5 (2.26)
  PI, Sodium, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Sodium, Week 36, n=44, 50 | 0.8 (2.21) | 0.6 (2.63)
  PI, Sodium, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Sodium, Week 40, n=42, 51 | 0.8 (2.20) | 0.7 (2.03)
  PI, Sodium, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Sodium, Week 44, n=47, 51 | 0.8 (2.10) | 0.7 (2.49)
  PI, Sodium, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Sodium, Week 48, n=43, 50 | 0.9 (1.98) | 0.8 (1.95)
  INI, Sodium, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Sodium, Week 4, n=99, 97 | 0.3 (1.62) | 0.0 (1.97)
  INI, Sodium, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Sodium, Week 8, n=73, 98 | 0.1 (1.98) | -0.3 (1.87)
  INI, Sodium, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Sodium, Week 12, n=99, 95 | 0.3 (2.11) | 0.0 (1.69)
  INI, Sodium, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Sodium, Week 16, n=93, 96 | 0.3 (1.95) | 0.4 (1.97)
  INI, Sodium, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Sodium, Week 20, n=93, 97 | 0.5 (1.94) | 0.1 (1.86)
  INI, Sodium, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Sodium, Week 24, n=94, 95 | 0.5 (1.79) | 0.0 (1.73)
  INI, Sodium, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Sodium, Week 28, n=89, 93 | 0.5 (1.74) | -0.3 (1.93)
  INI, Sodium, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Sodium, Week 32, n=93, 95 | 0.5 (1.87) | 0.2 (1.75)
  INI, Sodium, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Sodium, Week 36, n=94, 95 | 0.4 (1.86) | 0.3 (1.88)
  INI, Sodium, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Sodium, Week 40, n=90, 95 | 0.5 (1.91) | 0.2 (2.01)
  INI, Sodium, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Sodium, Week 44, n=91, 94 | 0.5 (1.77) | 0.3 (1.93)
  INI, Sodium, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Sodium, Week 48, n=91, 95 | 0.4 (2.00) | -0.1 (1.85)
  NNRTI, Sodium, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Sodium, Week 4, n=151, 153 | 0.2 (1.95) | 0.1 (1.98)
  NNRTI, Sodium, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Sodium, Week 8, n=122, 152 | 0.2 (1.91) | 0.0 (1.82)
  NNRTI, Sodium, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Sodium, Week 12, n=146, 152 | 0.1 (2.04) | 0.1 (2.01)
  NNRTI, Sodium, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Sodium, Week 16, n=143, 149 | -0.1 (2.28) | -0.2 (2.04)
  NNRTI, Sodium, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Sodium, Week 20, n=138, 152 | -0.1 (2.14) | 0.3 (1.95)
  NNRTI, Sodium, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Sodium, Week 24, n=143, 151 | 0.1 (2.14) | 0.3 (1.95)
  NNRTI, Sodium, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Sodium, Week 28, n=136, 150 | 0.3 (2.29) | 0.2 (2.18)
  NNRTI, Sodium, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Sodium, Week 32, n=137, 148 | 0.1 (2.01) | 0.5 (1.84)
  NNRTI, Sodium, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Sodium, Week 36, n=135, 147 | 0.4 (2.05) | 0.5 (2.22)
  NNRTI, Sodium, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Sodium, Week 40, n=138, 147 | 0.3 (2.04) | 0.5 (2.12)
  NNRTI, Sodium, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Sodium, Week 44, n=137, 148 | 0.5 (2.17) | 0.5 (1.96)
  NNRTI, Sodium, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Sodium, Week 48, n=131, 147 | 0.3 (2.39) | 0.4 (1.97)
  PI, Urea, Week 4, n=51, 53: number analyzed (Participants) | 51 | 53
  PI, Urea, Week 4, n=51, 53 | 0.02 (1.449) | 0.01 (1.124)
  PI, Urea, Week 8, n=34, 53: number analyzed (Participants) | 34 | 53
  PI, Urea, Week 8, n=34, 53 | 0.21 (1.142) | -0.02 (1.205)
  PI, Urea, Week 12, n=50, 52: number analyzed (Participants) | 50 | 52
  PI, Urea, Week 12, n=50, 52 | 0.04 (1.446) | -0.01 (1.312)
  PI, Urea, Week 16, n=48, 53: number analyzed (Participants) | 48 | 53
  PI, Urea, Week 16, n=48, 53 | 0.25 (1.309) | 0.20 (1.377)
  PI, Urea, Week 20, n=46, 53: number analyzed (Participants) | 46 | 53
  PI, Urea, Week 20, n=46, 53 | 0.18 (1.425) | 0.17 (1.275)
  PI, Urea, Week 24, n=47, 53: number analyzed (Participants) | 47 | 53
  PI, Urea, Week 24, n=47, 53 | 0.41 (1.248) | 0.10 (1.182)
  PI, Urea, Week 28, n=42, 53: number analyzed (Participants) | 42 | 53
  PI, Urea, Week 28, n=42, 53 | 0.18 (1.352) | 0.00 (1.236)
  PI, Urea, Week 32, n=45, 51: number analyzed (Participants) | 45 | 51
  PI, Urea, Week 32, n=45, 51 | 0.12 (1.567) | 0.16 (1.210)
  PI, Urea, Week 36, n=44, 50: number analyzed (Participants) | 44 | 50
  PI, Urea, Week 36, n=44, 50 | 0.01 (1.449) | -0.13 (1.190)
  PI, Urea, Week 40, n=42, 51: number analyzed (Participants) | 42 | 51
  PI, Urea, Week 40, n=42, 51 | 0.17 (1.291) | 0.33 (1.714)
  PI, Urea, Week 44, n=47, 51: number analyzed (Participants) | 47 | 51
  PI, Urea, Week 44, n=47, 51 | 0.36 (1.258) | 0.13 (1.276)
  PI, Urea, Week 48, n=43, 50: number analyzed (Participants) | 43 | 50
  PI, Urea, Week 48, n=43, 50 | 0.10 (1.303) | 0.13 (1.305)
  INI, Urea, Week 4, n=99, 97: number analyzed (Participants) | 99 | 97
  INI, Urea, Week 4, n=99, 97 | -0.14 (1.477) | 0.19 (1.635)
  INI, Urea, Week 8, n=73, 98: number analyzed (Participants) | 73 | 98
  INI, Urea, Week 8, n=73, 98 | -0.14 (1.799) | 0.01 (1.601)
  INI, Urea, Week 12, n=99, 95: number analyzed (Participants) | 99 | 95
  INI, Urea, Week 12, n=99, 95 | 0.05 (1.554) | 0.21 (1.481)
  INI, Urea, Week 16, n=93, 96: number analyzed (Participants) | 93 | 96
  INI, Urea, Week 16, n=93, 96 | 0.01 (1.402) | 0.05 (1.375)
  INI, Urea, Week 20, n=93, 97: number analyzed (Participants) | 93 | 97
  INI, Urea, Week 20, n=93, 97 | 0.01 (1.531) | 0.15 (1.495)
  INI, Urea, Week 24, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Urea, Week 24, n=94, 95 | 0.04 (1.367) | 0.12 (1.441)
  INI, Urea, Week 28, n=89, 93: number analyzed (Participants) | 89 | 93
  INI, Urea, Week 28, n=89, 93 | 0.01 (1.570) | -0.02 (1.579)
  INI, Urea, Week 32, n=93, 95: number analyzed (Participants) | 93 | 95
  INI, Urea, Week 32, n=93, 95 | -0.09 (1.592) | 0.01 (1.522)
  INI, Urea, Week 36, n=94, 95: number analyzed (Participants) | 94 | 95
  INI, Urea, Week 36, n=94, 95 | -0.10 (1.514) | -0.05 (1.478)
  INI, Urea, Week 40, n=90, 95: number analyzed (Participants) | 90 | 95
  INI, Urea, Week 40, n=90, 95 | 0.01 (1.519) | 0.12 (1.469)
  INI, Urea, Week 44, n=91, 94: number analyzed (Participants) | 91 | 94
  INI, Urea, Week 44, n=91, 94 | -0.16 (1.583) | -0.19 (1.721)
  INI, Urea, Week 48, n=91, 95: number analyzed (Participants) | 91 | 95
  INI, Urea, Week 48, n=91, 95 | 0.11 (1.633) | -0.05 (1.304)
  NNRTI, Urea, Week 4, n=151, 153: number analyzed (Participants) | 151 | 153
  NNRTI, Urea, Week 4, n=151, 153 | 0.10 (1.265) | 0.04 (1.185)
  NNRTI, Urea, Week 8, n=122, 152: number analyzed (Participants) | 122 | 152
  NNRTI, Urea, Week 8, n=122, 152 | 0.16 (1.286) | 0.01 (1.252)
  NNRTI, Urea, Week 12, n=146, 152: number analyzed (Participants) | 146 | 152
  NNRTI, Urea, Week 12, n=146, 152 | 0.26 (1.290) | 0.06 (1.344)
  NNRTI, Urea, Week 16, n=143, 149: number analyzed (Participants) | 143 | 149
  NNRTI, Urea, Week 16, n=143, 149 | 0.07 (1.407) | 0.28 (1.609)
  NNRTI, Urea, Week 20, n=138, 152: number analyzed (Participants) | 138 | 152
  NNRTI, Urea, Week 20, n=138, 152 | 0.25 (1.296) | 0.07 (1.507)
  NNRTI, Urea, Week 24, n=143, 151: number analyzed (Participants) | 143 | 151
  NNRTI, Urea, Week 24, n=143, 151 | 0.33 (1.499) | 0.18 (1.276)
  NNRTI, Urea, Week 28, n=136, 150: number analyzed (Participants) | 136 | 150
  NNRTI, Urea, Week 28, n=136, 150 | 0.22 (1.549) | 0.02 (1.422)
  NNRTI, Urea, Week 32, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Urea, Week 32, n=137, 148 | 0.41 (1.410) | 0.06 (1.416)
  NNRTI, Urea, Week 36, n=135, 147: number analyzed (Participants) | 135 | 147
  NNRTI, Urea, Week 36, n=135, 147 | 0.19 (1.339) | 0.04 (1.392)
  NNRTI, Urea, Week 40, n=138, 147: number analyzed (Participants) | 138 | 147
  NNRTI, Urea, Week 40, n=138, 147 | 0.32 (1.347) | -0.01 (1.339)
  NNRTI, Urea, Week 44, n=137, 148: number analyzed (Participants) | 137 | 148
  NNRTI, Urea, Week 44, n=137, 148 | 0.25 (1.346) | 0.10 (1.344)
  NNRTI, Urea, Week 48, n=131, 147: number analyzed (Participants) | 131 | 147
  NNRTI, Urea, Week 48, n=131, 147 | 0.37 (1.389) | -0.02 (1.325)

71. Secondary Outcome: Change From Baseline Values for Fasting Lipid Panel Using Baseline Third Agent Treatment Class Overtime Including Week 48
Description: Blood samples were collected for the analysis of fasting lipid panel: triglycerides, total cholesterol, HDL cholesterol and LDL cholesterol to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Millimoles per liter
  PI, Triglycerides, Week 48, n=40, 45: number analyzed (Participants) | 40 | 45
  PI, Triglycerides, Week 48, n=40, 45 | -0.733 (1.5612) | 0.060 (0.9960)
  INI, Triglycerides, Week 48, n=72, 77: number analyzed (Participants) | 72 | 77
  INI, Triglycerides, Week 48, n=72, 77 | -0.078 (0.4964) | -0.117 (0.8052)
  NNRTI, Triglycerides, Week 48, n=119, 120: number analyzed (Participants) | 119 | 120
  NNRTI, Triglycerides, Week 48, n=119, 120 | -0.015 (0.6121) | -0.014 (0.6761)
  PI, Cholesterol, Week 48, n=40, 45: number analyzed (Participants) | 40 | 45
  PI, Cholesterol, Week 48, n=40, 45 | -0.06 (0.629) | 0.06 (0.744)
  INI, Cholesterol, Week 48, n=72, 77: number analyzed (Participants) | 72 | 77
  INI, Cholesterol, Week 48, n=72, 77 | 0.18 (0.614) | -0.12 (0.674)
  NNRTI, Cholesterol, Week 48, n=119, 120: number analyzed (Participants) | 119 | 120
  NNRTI, Cholesterol, Week 48, n=119, 120 | 0.06 (0.743) | -0.02 (0.626)
  PI, HDL cholesterol, Week 48, n=40, 45: number analyzed (Participants) | 40 | 45
  PI, HDL cholesterol, Week 48, n=40, 45 | 0.130 (0.2272) | 0.001 (0.3429)
  INI, HDL cholesterol, Week 48, n=72, 77: number analyzed (Participants) | 72 | 77
  INI, HDL cholesterol, Week 48, n=72, 77 | 0.074 (0.2339) | -0.038 (0.2308)
  NNRTI, HDL cholesterol, Week 48, n=119, 120: number analyzed (Participants) | 119 | 120
  NNRTI, HDL cholesterol, Week 48, n=119, 120 | -0.011 (0.2936) | 0.028 (0.2577)
  PI, LDL cholesterol, Week 48, n=37, 43: number analyzed (Participants) | 37 | 43
  PI, LDL cholesterol, Week 48, n=37, 43 | 0.075 (0.5774) | 0.043 (0.5545)
  INI, LDL cholesterol, Week 48, n=71, 76: number analyzed (Participants) | 71 | 76
  INI, LDL cholesterol, Week 48, n=71, 76 | 0.144 (0.4840) | -0.015 (0.5333)
  NNRTI, LDL cholesterol, Week 48, n=116, 119: number analyzed (Participants) | 116 | 119
  NNRTI, LDL cholesterol, Week 48, n=116, 119 | 0.078 (0.6885) | -0.040 (0.5246)

72. Secondary Outcome: Number of Participants With Genotypic Resistance Using Baseline Third Agent Through Week 48
Description: Plasma samples were collected from participants who met confirmed virologic withdrawal criteria to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). Genotypic Resistance data for the following drugs: DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV, DRV, FPV, IDV, LPV, NFV, RTV, SQV and TPV in participants meeting CVF criteria has been presented.
Time Frame: At the time of CVF
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 3 | 4
Participants
  PI, INI, DTG, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, DTG, resistant, n=1, 0 | 0 | 0
  PI, INI, DTG, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, DTG, resistance possible, n=1, 0 | 0 | 0
  PI, INI, DTG, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, DTG, sensitive, n=1, 0 | 1 | 0
  PI, INI, EVG, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, EVG, resistant, n=1, 0 | 0 | 0
  PI, INI, EVG, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, EVG, resistance possible, n=1, 0 | 0 | 0
  PI, INI, EVG, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, EVG, sensitive, n=1, 0 | 1 | 0
  PI, INI, RAL, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, RAL, resistant, n=1, 0 | 0 | 0
  PI, INI, RAL, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, RAL, resistance possible, n=1, 0 | 0 | 0
  PI, INI, RAL, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, RAL, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, DLV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, DLV, resistant, n=1, 0 | 0 | 0
  PI, NNRTI, DLV, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, DLV, resistance possible, n=1, 0 | 0 | 0
  PI, NNRTI, DLV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, DLV, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, EFV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, EFV, resistant, n=1, 0 | 0 | 0
  PI, NNRTI, EFV, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, EFV, resistance possible, n=1, 0 | 0 | 0
  PI, NNRTI, EFV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, EFV, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, ETR, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, ETR, resistant, n=1, 0 | 0 | 0
  PI, NNRTI, ETR, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, ETR, resistance possible, n=1, 0 | 0 | 0
  PI, NNRTI, ETR, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, ETR, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, NVP, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, NVP, resistant, n=1, 0 | 0 | 0
  PI, NNRTI, NVP, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, NVP, resistance possible, n=1, 0 | 0 | 0
  PI, NNRTI, NVP, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, NVP, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, RPV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, RPV, resistant, n=1, 0 | 1 | 0
  PI, NNRTI, RPV, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, RPV, resistance possible, n=1, 0 | 0 | 0
  PI, NNRTI, RPV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, RPV, sensitive, n=1, 0 | 0 | 0
  PI, NRTI, 3TC, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, 3TC, resistant, n=1, 0 | 0 | 0
  PI, NNRTI, 3TC, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, 3TC, resistance possible, n=1, 0 | 0 | 0
  PI, NRTI, 3TC, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, 3TC, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, ABC, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ABC, resistant, n=1, 0 | 0 | 0
  PI, NRTI, ABC, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ABC, resistance possible, n=1, 0 | 0 | 0
  PI, NRTI, ABC, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ABC, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, FTC, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, FTC, resistant, n=1, 0 | 0 | 0
  PI, NRTI, FTC, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, FTC, resistance possible, n=1, 0 | 0 | 0
  PI, NRTI, FTC, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, FTC, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, TDF, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, TDF, resistant, n=1, 0 | 0 | 0
  PI, NRTI, TDF, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, TDF, resistance possible, n=1, 0 | 0 | 0
  PI, NRTI, TDF, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, TDF, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, ZDV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ZDV, resistant, n=1, 0 | 0 | 0
  PI, NRTI, ZDV, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ZDV, resistance possible, n=1, 0 | 0 | 0
  PI, NRTI, ZDV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ZDV, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, d4T, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, d4T, resistant, n=1, 0 | 0 | 0
  PI, NRTI, d4T, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, d4T, resistance possible, n=1, 0 | 0 | 0
  PI, NRTI, d4T, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, d4T, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, ddI, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ddI, resistant, n=1, 0 | 0 | 0
  PI, NRTI, ddI, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ddI, resistance possible, n=1, 0 | 0 | 0
  PI, NRTI, ddI, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ddI, sensitive, n=1, 0 | 1 | 0
  PI, PI, ATV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, ATV, resistant, n=1, 0 | 0 | 0
  PI, PI, ATV, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, ATV, resistance possible, n=1, 0 | 0 | 0
  PI, PI, ATV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, ATV, sensitive, n=1, 0 | 1 | 0
  PI, PI, ATV/r, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, ATV/r, resistant, n=1, 0 | 0 | 0
  PI, PI, ATV/r, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, ATV/r, resistance possible, n=1, 0 | 0 | 0
  PI, PI, ATV/r, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, ATV/r, sensitive, n=1, 0 | 1 | 0
  PI, PI, DRV/r, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, DRV/r, resistant, n=1, 0 | 0 | 0
  PI, PI, DRV/r, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, DRV/r, resistance possible, n=1, 0 | 0 | 0
  PI, PI, DRV/r, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, DRV/r, sensitive, n=1, 0 | 1 | 0
  PI, PI, FPV/r, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, FPV/r, resistant, n=1, 0 | 0 | 0
  PI, PI, FPV/r, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, FPV/r, resistance possible, n=1, 0 | 0 | 0
  PI, PI, FPV/r, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, FPV/r, sensitive, n=1, 0 | 1 | 0
  PI, PI, IDV/r, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, IDV/r, resistant, n=1, 0 | 0 | 0
  PI, PI, IDV/r, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, IDV/r, resistance possible, n=1, 0 | 0 | 0
  PI, PI, IDV/r, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, IDV/r, sensitive, n=1, 0 | 1 | 0
  PI, PI, LPV/r, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, LPV/r, resistant, n=1, 0 | 0 | 0
  PI, PI, LPV/r, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, LPV/r, resistance possible, n=1, 0 | 0 | 0
  PI, PI, LPV/r, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, LPV/r, sensitive, n=1, 0 | 1 | 0
  PI, PI, NFV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, NFV, resistant, n=1, 0 | 0 | 0
  PI, PI, NFV, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, NFV, resistance possible, n=1, 0 | 0 | 0
  PI, PI, NFV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, NFV, sensitive, n=1, 0 | 1 | 0
  PI, PI, RTV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, RTV, resistant, n=1, 0 | 0 | 0
  PI, PI, RTV, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, RTV, resistance possible, n=1, 0 | 0 | 0
  PI, PI, RTV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, RTV, sensitive, n=1, 0 | 1 | 0
  PI, PI, SQV/r, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, SQV/r, resistant, n=1, 0 | 0 | 0
  PI, PI, SQV/r, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, SQV/r, resistance possible, n=1, 0 | 0 | 0
  PI, PI, SQV/r, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, SQV/r, sensitive, n=1, 0 | 1 | 0
  PI, PI, TPV/r, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, TPV/r, resistant, n=1, 0 | 0 | 0
  PI, PI, TPV/r, resistance possible, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, TPV/r, resistance possible, n=1, 0 | 0 | 0
  PI, PI, TPV/r, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, TPV/r, sensitive, n=1, 0 | 1 | 0
  INI, INI, DTG, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, DTG, resistant, n=0, 3 | 0 | 0
  INI, INI, DTG, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, DTG, resistance possible, n=0, 3 | 0 | 0
  INI, INI, DTG, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, DTG, sensitive, n=0, 3 | 0 | 3
  INI, INI, EVG, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, EVG, resistant, n=0, 3 | 0 | 0
  INI, INI, EVG, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, EVG, resistance possible, n=0, 3 | 0 | 0
  INI, INI, EVG, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, EVG, sensitive, n=0, 3 | 0 | 3
  INI, INI, RAL, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, RAL, resistant, n=0, 3 | 0 | 0
  INI, INI, RAL, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, RAL, resistance possible, n=0, 3 | 0 | 0
  INI, INI, RAL, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, RAL, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, DLV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, DLV, resistant, n=0, 3 | 0 | 0
  INI, INI, DLV, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, DLV, resistance possible, n=0, 3 | 0 | 0
  INI, NNRTI, DLV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, DLV, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, EFV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, EFV, resistant, n=0, 3 | 0 | 0
  INI, INI, EFV, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, EFV, resistance possible, n=0, 3 | 0 | 0
  INI, NNRTI, EFV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, EFV, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, ETR, resistant,, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, ETR, resistant,, n=0, 3 | 0 | 0
  INI, NNRTI, ETR, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, ETR, resistance possible, n=0, 3 | 0 | 0
  INI, NNRTI, ETR, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, ETR, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, NVP, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, NVP, resistant, n=0, 3 | 0 | 0
  INI, NNRTI, NVP, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, NVP, resistance possible, n=0, 3 | 0 | 0
  INI, NNRTI, NVP, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, NVP, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, RPV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, RPV, resistant, n=0, 3 | 0 | 1
  INI, NNRTI, RPV, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, RPV, resistance possible, n=0, 3 | 0 | 0
  INI, NNRTI, RPV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, RPV, sensitive, n=0, 3 | 0 | 2
  INI, NRTI, 3TC, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, 3TC, resistant, n=0, 3 | 0 | 1
  INI, NNRTI, 3TC, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, 3TC, resistance possible, n=0, 3 | 0 | 0
  INI, NRTI, 3TC, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, 3TC, sensitive, n=0, 3 | 0 | 2
  INI, NRTI, ABC, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ABC, resistant, n=0, 3 | 0 | 0
  INI, NRTI, ABC, resistance possible,, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ABC, resistance possible,, n=0, 3 | 0 | 0
  INI, NRTI, ABC, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ABC, sensitive, n=0, 3 | 0 | 3
  INI, NRTI, FTC, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, FTC, resistant, n=0, 3 | 0 | 1
  INI, NRTI, FTC, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, FTC, resistance possible, n=0, 3 | 0 | 0
  INI, NRTI, FTC, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, FTC, sensitive, n=0, 3 | 0 | 2
  INI, NRTI, TDF, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, TDF, resistant, n=0, 3 | 0 | 0
  INI, NRTI, TDF, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, TDF, resistance possible, n=0, 3 | 0 | 0
  INI, NRTI, TDF, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, TDF, sensitive, n=0, 3 | 0 | 3
  INI, NRTI, ZDV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ZDV, resistant, n=0, 3 | 0 | 0
  INI, NRTI, ZDV, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ZDV, resistance possible, n=0, 3 | 0 | 0
  INI, NRTI, ZDV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ZDV, sensitive, n=0, 3 | 0 | 3
  INI, NRTI, d4T, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, d4T, resistant, n=0, 3 | 0 | 0
  INI, NRTI, d4T, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, d4T, resistance possible, n=0, 3 | 0 | 0
  INI, NRTI, d4T, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, d4T, sensitive, n=0, 3 | 0 | 3
  INI, NRTI, ddI, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ddI, resistant, n=0, 3 | 0 | 0
  INI, NRTI, ddI, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ddI, resistance possible, n=0, 3 | 0 | 1
  INI, NRTI, ddI, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ddI, sensitive, n=0, 3 | 0 | 2
  INI, PI, ATV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, ATV, resistant, n=0, 3 | 0 | 0
  INI, PI, ATV, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, ATV, resistance possible, n=0, 3 | 0 | 0
  INI, PI, ATV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, ATV, sensitive, n=0, 3 | 0 | 3
  INI, PI, ATV/r, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, ATV/r, n=0, 3 | 0 | 0
  INI, PI, ATV/r, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, ATV/r, resistance possible, n=0, 3 | 0 | 0
  INI, PI, ATV/r, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, ATV/r, sensitive, n=0, 3 | 0 | 3
  INI, PI, DRV/r, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, DRV/r, resistant, n=0, 3 | 0 | 0
  INI, PI, DRV/r, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, DRV/r, resistance possible, n=0, 3 | 0 | 0
  INI, PI, DRV/r, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, DRV/r, sensitive, n=0, 3 | 0 | 3
  INI, PI, FPV/r, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, FPV/r, resistant, n=0, 3 | 0 | 0
  INI, PI, FPV/r, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, FPV/r, resistance possible, n=0, 3 | 0 | 0
  INI, PI, FPV/r, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, FPV/r, sensitive, n=0, 3 | 0 | 3
  INI, PI, IDV/r, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, IDV/r, resistant, n=0, 3 | 0 | 0
  INI, PI, IDV/r, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, IDV/r, resistance possible, n=0, 3 | 0 | 0
  INI, PI, IDV/r, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, IDV/r, sensitive, n=0, 3 | 0 | 3
  INI, PI, LPV/r, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, LPV/r, resistant, n=0, 3 | 0 | 0
  INI, PI, LPV/r, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, LPV/r, resistance possible, n=0, 3 | 0 | 0
  INI, PI, LPV/r, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, LPV/r, sensitive, n=0, 3 | 0 | 3
  INI, PI, NFV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, NFV, resistant, n=0, 3 | 0 | 0
  INI, PI, NFV, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, NFV, resistance possible, n=0, 3 | 0 | 0
  INI, PI, NFV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, NFV, sensitive, n=0, 3 | 0 | 3
  INI, PI, RTV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, RTV, resistant, n=0, 3 | 0 | 0
  INI, PI, RTV, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, RTV, resistance possible, n=0, 3 | 0 | 0
  INI, PI, RTV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, RTV, sensitive, n=0, 3 | 0 | 3
  INI, PI, SQV/r, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, SQV/r, resistant, n=0, 3 | 0 | 0
  INI, PI, SQV/r, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, SQV/r, resistance possible, n=0, 3 | 0 | 0
  INI, PI, SQV/r, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, SQV/r, sensitive, n=0, 3 | 0 | 3
  INI, PI, TPV/r, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, TPV/r, resistant, n=0, 3 | 0 | 0
  INI, PI, TPV/r, resistance possible, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, TPV/r, resistance possible, n=0, 3 | 0 | 0
  INI, PI, TPV/r, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, TPV/r, sensitive, n=0, 3 | 0 | 3
  NNRTI, INI, DTG, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, DTG, resistant, n=2, 1 | 0 | 0
  NNRTI, INI, DTG, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, DTG, resistance possible, n=2, 1 | 0 | 0
  NNRTI, INI, DTG, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, DTG, sensitive, n=2, 1 | 2 | 1
  NNRTI, INI, EVG, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, EVG, resistant, n=2, 1 | 1 | 0
  NNRTI, INI, EVG, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, EVG, resistance possible, n=2, 1 | 0 | 0
  NNRTI, INI, EVG, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, EVG, sensitive, n=2, 1 | 1 | 1
  NNRTI, INI, RAL, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, RAL, resistant, n=2, 1 | 1 | 0
  NNRTI, INI, RAL, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, RAL, resistance possible, n=2, 1 | 0 | 0
  NNRTI, INI, RAL, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, RAL, sensitive, n=2, 1 | 1 | 1
  NNRTI, NNRTI, DLV, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, DLV, resistant, n=2, 1 | 0 | 0
  NNRTI, INI, DLV, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, DLV, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NNRTI, DLV, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, DLV, sensitive, n=2, 1 | 2 | 1
  NNRTI, NNRTI, EFV, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, EFV, resistant, n=2, 1 | 1 | 1
  NNRTI, INI, EFV, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, EFV, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NNRTI, EFV, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, EFV, sensitive, n=2, 1 | 1 | 0
  NNRTI, NNRTI, ETR, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, ETR, resistant, n=2, 1 | 0 | 0
  NNRTI, NNRTI, ETR, resistance possible,n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, ETR, resistance possible,n=2, 1 | 2 | 0
  NNRTI, NNRTI, ETR, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, ETR, sensitive, n=2, 1 | 0 | 1
  NNRTI, NNRTI, NVP, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, NVP, resistant, n=2, 1 | 1 | 1
  NNRTI, NNRTI, NVP, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, NVP, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NNRTI, NVP, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, NVP, sensitive, n=2, 1 | 1 | 0
  NNRTI, NNRTI, RPV, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, RPV, resistant, n=2, 1 | 2 | 0
  NNRTI, NNRTI, RPV, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, RPV, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NNRTI, RPV, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, RPV, sensitive, n=2, 1 | 0 | 1
  NNRTI, NRTI, 3TC, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, 3TC, resistant, n=2, 1 | 0 | 1
  NNRTI, NNRTI, 3TC, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NNRTI, 3TC, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NRTI, 3TC, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, 3TC, sensitive, n=2, 1 | 2 | 0
  NNRTI, NRTI, ABC, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, ABC, resistant, n=2, 1 | 0 | 0
  NNRTI, NRTI, ABC, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, ABC, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NRTI, ABC, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, ABC, sensitive, n=2, 1 | 2 | 1
  NNRTI, NRTI, FTC, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, FTC, resistant, n=2, 1 | 0 | 1
  NNRTI, NRTI, FTC, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, FTC, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NRTI, FTC, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, FTC, sensitive, n=2, 1 | 2 | 0
  NNRTI, NRTI, TDF, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, TDF, resistant, n=2, 1 | 0 | 0
  NNRTI, NRTI, TDF, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, TDF, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NRTI, TDF, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, TDF, sensitive, n=2, 1 | 2 | 1
  NNRTI, NRTI, ZDV, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, ZDV, resistant, n=2, 1 | 0 | 0
  NNRTI, NRTI, ZDV, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, ZDV, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NRTI, ZDV, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, ZDV, sensitive, n=2, 1 | 2 | 1
  NNRTI, NRTI, d4T, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, d4T, resistant, n=2, 1 | 0 | 0
  NNRTI, NRTI, d4T, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, d4T, resistance possible, n=2, 1 | 0 | 0
  NNRTI, NRTI, d4T, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, d4T, sensitive, n=2, 1 | 2 | 1
  NNRTI, NRTI, ddI, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, ddI, resistant, n=2, 1 | 0 | 0
  NNRTI, NRTI, ddI, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, ddI, resistance possible, n=2, 1 | 0 | 1
  NNRTI, NRTI, ddI, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, NRTI, ddI, sensitive, n=2, 1 | 2 | 0
  NNRTI, PI, ATV, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, ATV, resistant, n=2, 1 | 1 | 0
  NNRTI, PI, ATV, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, ATV, resistance possible, n=2, 1 | 0 | 0
  NNRTI, PI, ATV, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, ATV, sensitive, n=2, 1 | 1 | 1
  NNRTI, PI, ATV/r, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, ATV/r, resistant, n=2, 1 | 0 | 0
  NNRTI, PI, ATV/r, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, ATV/r, resistance possible, n=2, 1 | 1 | 0
  NNRTI, PI, ATV/r, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, ATV/r, sensitive, n=2, 1 | 1 | 1
  NNRTI, PI, DRV/r, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, DRV/r, resistant, n=2, 1 | 0 | 0
  NNRTI, PI, DRV/r, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, DRV/r, resistance possible, n=2, 1 | 0 | 0
  NNRTI, PI, DRV/r, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, DRV/r, sensitive, n=2, 1 | 2 | 1
  NNRTI, PI, FPV/r, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, FPV/r, resistant, n=2, 1 | 0 | 0
  NNRTI, PI, FPV/r, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, FPV/r, resistance possible, n=2, 1 | 0 | 0
  NNRTI, PI, FPV/r, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, FPV/r, sensitive, n=2, 1 | 2 | 1
  NNRTI, PI, IDV/r, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, IDV/r, resistant, n=2, 1 | 0 | 0
  NNRTI, PI, IDV/r, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, IDV/r, resistance possible, n=2, 1 | 0 | 0
  NNRTI, PI, IDV/r, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, IDV/r, sensitive, n=2, 1 | 2 | 1
  NNRTI, PI, LPV/r, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, LPV/r, resistant, n=2, 1 | 0 | 0
  NNRTI, PI, LPV/r, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, LPV/r, resistance possible, n=2, 1 | 0 | 0
  NNRTI, PI, LPV/r, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, LPV/r, sensitive, n=2, 1 | 2 | 1
  NNRTI, PI, NFV, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, NFV, resistant, n=2, 1 | 1 | 0
  NNRTI, PI, NFV, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, NFV, resistance possible, n=2, 1 | 0 | 0
  NNRTI, PI, NFV, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, NFV, sensitive, n=2, 1 | 1 | 1
  NNRTI, PI, RTV, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, RTV, resistant, n=2, 1 | 0 | 0
  NNRTI, PI, RTV, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, RTV, resistance possible, n=2, 1 | 0 | 0
  NNRTI, PI, RTV, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, RTV, sensitive, n=2, 1 | 2 | 1
  NNRTI, PI, SQV/r, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, SQV/r, resistant, n=2, 1 | 0 | 0
  NNRTI, PI, SQV/r, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, SQV/r, resistance possible, n=2, 1 | 0 | 0
  NNRTI, PI, SQV/r, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, SQV/r, sensitive, n=2, 1 | 2 | 1
  NNRTI, PI, TPV/r, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, TPV/r, resistant, n=2, 1 | 0 | 0
  NNRTI, PI, TPV/r, resistance possible, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, TPV/r, resistance possible, n=2, 1 | 0 | 0
  NNRTI, PI, TPV/r, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, PI, TPV/r, sensitive, n=2, 1 | 2 | 1

73. Secondary Outcome: Number of Participants With Phenotypic Resistance Using Baseline Third Agent Through Week 48
Description: Plasma samples were collected from participants who met confirmed virologic withdrawal criteria to assess the impact of Baseline third agent treatment class (PI, NNRTI and INI). Phenotypic Resistance data for the following drugs: CAB, DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV, DRV, FPV, IDV, LPV, NFV, RTV, SQV and TPV in participants meeting CVF criteria has been presented. Phenotypic resistance, partially sensitive, and Sensitive were defined based on FC value from Monogram as: resistance (FC>clinical higher cutoff/biologic cutoff), partially sensitive (FC <=clinical higher cutoff and > clinical lower cutoff), sensitive (FC <= clinical lower cutoff/biologic cutoff).
Time Frame: At the time of CVF
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 3 | 4
Participants
  PI, INI, CAB, resistant , n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, CAB, resistant , n=1, 0 | 0 | 0
  PI, INI, CAB, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, CAB, sensitive, n=1, 0 | 1 | 0
  PI, INI, DTG, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, DTG, resistant, n=1, 0 | 0 | 0
  PI, INI, DTG, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, DTG, partially sensitive, n=1, 0 | 0 | 0
  PI, INI, DTG, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, DTG, sensitive, n=1, 0 | 1 | 0
  PI, INI, EVG, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, EVG, resistant, n=1, 0 | 0 | 0
  PI, INI, EVG, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, EVG, sensitive, n=1, 0 | 1 | 0
  PI, INI, RAL, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, RAL, resistant, n=1, 0 | 0 | 0
  PI, INI, RAL, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, INI, RAL, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, DLV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, DLV, resistant, n=1, 0 | 0 | 0
  PI, NNRTI, DLV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, DLV, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, EFV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, EFV, resistant, n=1, 0 | 0 | 0
  PI, NNRTI, EFV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, EFV, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, ETR, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, ETR, resistant, n=1, 0 | 0 | 0
  PI, NNRTI, ETR, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, ETR, partially sensitive, n=1, 0 | 0 | 0
  PI, NNRTI, ETR, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, ETR, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, NVP, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, NVP, resistant, n=1, 0 | 0 | 0
  PI, NNRTI, NVP, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, NVP, sensitive, n=1, 0 | 1 | 0
  PI, NNRTI, RPV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, RPV, resistant, n=1, 0 | 1 | 0
  PI, NNRTI, RPV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NNRTI, RPV, sensitive, n=1, 0 | 0 | 0
  PI, NRTI, 3TC, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, 3TC, resistant, n=1, 0 | 0 | 0
  PI, NRTI, 3TC, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, 3TC, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, ABC, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ABC, resistant, n=1, 0 | 0 | 0
  PI, NRTI, ABC, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ABC, partially sensitive, n=1, 0 | 0 | 0
  PI, NRTI, ABC, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ABC, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, FTC, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, FTC, resistant, n=1, 0 | 0 | 0
  PI, NRTI, FTC, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, FTC, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, TDF, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, TDF, resistant, n=1, 0 | 0 | 0
  PI, NRTI, TDF, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, TDF, partially sensitive, n=1, 0 | 0 | 0
  PI, NRTI, TDF, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, TDF, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, ZDV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ZDV, resistant, n=1, 0 | 0 | 0
  PI, NRTI, ZDV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ZDV, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, d4T, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, d4T, resistant, n=1, 0 | 0 | 0
  PI, NRTI, d4T, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, d4T, sensitive, n=1, 0 | 1 | 0
  PI, NRTI, ddI, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ddI, resistant, n=1, 0 | 0 | 0
  PI, NRTI, ddI, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ddI, partially sensitive, n=1, 0 | 0 | 0
  PI, NRTI, ddI, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, NRTI, ddI, sensitive, n=1, 0 | 1 | 0
  PI, PI, ATV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, ATV, resistant, n=1, 0 | 0 | 0
  PI, PI, ATV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, ATV, sensitive, n=1, 0 | 1 | 0
  PI, PI, DRV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, DRV, resistant, n=1, 0 | 0 | 0
  PI, PI, DRV, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, DRV, partially sensitive, n=1, 0 | 0 | 0
  PI, PI, DRV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, DRV, sensitive, n=1, 0 | 1 | 0
  PI, PI, FPV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, FPV, resistant, n=1, 0 | 0 | 0
  PI, PI, FPV, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, FPV, partially sensitive, n=1, 0 | 0 | 0
  PI, PI, FPV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, FPV, sensitive, n=1, 0 | 1 | 0
  PI, PI, IDV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, IDV, resistant, n=1, 0 | 0 | 0
  PI, PI, IDV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, IDV, sensitive, n=1, 0 | 1 | 0
  PI, PI, LPV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, LPV, resistant, n=1, 0 | 0 | 0
  PI, PI, LPV, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, LPV, partially sensitive, n=1, 0 | 0 | 0
  PI, PI, LPV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, LPV, sensitive, n=1, 0 | 1 | 0
  PI, PI, NFV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, NFV, resistant, n=1, 0 | 0 | 0
  PI, PI, NFV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, NFV, sensitive, n=1, 0 | 1 | 0
  PI, PI, RTV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, RTV, resistant, n=1, 0 | 0 | 0
  PI, PI, RTV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, RTV, sensitive, n=1, 0 | 1 | 0
  PI, PI, SQV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, SQV, resistant, n=1, 0 | 0 | 0
  PI, PI, SQV, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, SQV, partially sensitive, n=1, 0 | 0 | 0
  PI, PI, SQV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, SQV, sensitive, n=1, 0 | 1 | 0
  PI, PI, TPV, resistant, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, TPV, resistant, n=1, 0 | 0 | 0
  PI, PI, TPV, partially sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, TPV, partially sensitive, n=1, 0 | 0 | 0
  PI, PI, TPV, sensitive, n=1, 0: number analyzed (Participants) | 1 | 0
  PI, PI, TPV, sensitive, n=1, 0 | 1 | 0
  INI, INI, CAB, resistant , n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, CAB, resistant , n=0, 3 | 0 | 0
  INI, INI, CAB, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, CAB, sensitive, n=0, 3 | 0 | 3
  INI, INI, DTG, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, DTG, resistant, n=0, 3 | 0 | 0
  INI, INI, DTG, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, DTG, partially sensitive, n=0, 3 | 0 | 0
  INI, INI, DTG, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, DTG, sensitive, n=0, 3 | 0 | 3
  INI, INI, EVG, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, EVG, resistant, n=0, 3 | 0 | 0
  INI, INI, EVG, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, EVG, sensitive, n=0, 3 | 0 | 3
  INI, INI, RAL, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, RAL, resistant, n=0, 3 | 0 | 0
  INI, INI, RAL, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, INI, RAL, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, DLV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, DLV, resistant, n=0, 3 | 0 | 0
  INI, NNRTI, DLV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, DLV, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, EFV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, EFV, resistant, n=0, 3 | 0 | 0
  INI, NNRTI, EFV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, EFV, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, ETR, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, ETR, resistant, n=0, 3 | 0 | 0
  INI, NNRTI, ETR, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, ETR, partially sensitive, n=0, 3 | 0 | 0
  INI, NNRTI, ETR, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, ETR, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, NVP, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, NVP, resistant, n=0, 3 | 0 | 0
  INI, NNRTI, NVP, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, NVP, sensitive, n=0, 3 | 0 | 3
  INI, NNRTI, RPV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, RPV, resistant, n=0, 3 | 0 | 0
  INI, NNRTI, RPV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NNRTI, RPV, sensitive, n=0, 3 | 0 | 3
  INI, NRTI, 3TC, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, 3TC, resistant, n=0, 3 | 0 | 1
  INI, NRTI, 3TC, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, 3TC, sensitive, n=0, 3 | 0 | 2
  INI, NRTI, ABC, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ABC, resistant, n=0, 3 | 0 | 0
  INI, NRTI, ABC, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ABC, partially sensitive, n=0, 3 | 0 | 0
  INI, NRTI, ABC, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ABC, sensitive, n=0, 3 | 0 | 3
  INI, NRTI, FTC, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, FTC, resistant, n=0, 3 | 0 | 1
  INI, NRTI, FTC, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, FTC, sensitive, n=0, 3 | 0 | 2
  INI, NRTI, TDF, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, TDF, resistant, n=0, 3 | 0 | 0
  INI, NRTI, TDF, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, TDF, partially sensitive, n=0, 3 | 0 | 0
  INI, NRTI, TDF, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, TDF, sensitive, n=0, 3 | 0 | 3
  INI, NRTI, ZDV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ZDV, resistant, n=0, 3 | 0 | 0
  INI, NRTI, ZDV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ZDV, sensitive, n=0, 3 | 0 | 3
  INI, NRTI, d4T, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, d4T, resistant, n=0, 3 | 0 | 0
  INI, NRTI, d4T, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, d4T, sensitive, n=0, 3 | 0 | 3
  INI, NRTI, ddI, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ddI, resistant, n=0, 3 | 0 | 0
  INI, NRTI, ddI, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ddI, partially sensitive, n=0, 3 | 0 | 0
  INI, NRTI, ddI, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, NRTI, ddI, sensitive, n=0, 3 | 0 | 3
  INI, PI, ATV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, ATV, resistant, n=0, 3 | 0 | 0
  INI, PI, ATV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, ATV, sensitive, n=0, 3 | 0 | 3
  INI, PI, DRV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, DRV, resistant, n=0, 3 | 0 | 0
  INI, PI, DRV, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, DRV, partially sensitive, n=0, 3 | 0 | 0
  INI, PI, DRV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, DRV, sensitive, n=0, 3 | 0 | 3
  INI, PI, FPV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, FPV, resistant, n=0, 3 | 0 | 0
  INI, PI, FPV, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, FPV, partially sensitive, n=0, 3 | 0 | 0
  INI, PI, FPV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, FPV, sensitive, n=0, 3 | 0 | 3
  INI, PI, IDV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, IDV, resistant, n=0, 3 | 0 | 0
  INI, PI, IDV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, IDV, sensitive, n=0, 3 | 0 | 3
  INI, PI, LPV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, LPV, resistant, n=0, 3 | 0 | 0
  INI, PI, LPV, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, LPV, partially sensitive, n=0, 3 | 0 | 0
  INI, PI, LPV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, LPV, sensitive, n=0, 3 | 0 | 3
  INI, PI, NFV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, NFV, resistant, n=0, 3 | 0 | 0
  INI, PI, NFV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, NFV, sensitive, n=0, 3 | 0 | 3
  INI, PI, RTV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, RTV, resistant, n=0, 3 | 0 | 0
  INI, PI, RTV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, RTV, sensitive, n=0, 3 | 0 | 3
  INI, PI, SQV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, SQV, resistant, n=0, 3 | 0 | 0
  INI, PI, SQV, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, SQV, partially sensitive, n=0, 3 | 0 | 0
  INI, PI, SQV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, SQV, sensitive, n=0, 3 | 0 | 3
  INI, PI, TPV, resistant, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, TPV, resistant, n=0, 3 | 0 | 0
  INI, PI, TPV, partially sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, TPV, partially sensitive, n=0, 3 | 0 | 0
  INI, PI, TPV, sensitive, n=0, 3: number analyzed (Participants) | 0 | 3
  INI, PI, TPV, sensitive, n=0, 3 | 0 | 3
  NNRTI, INI, CAB, resistant , n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, CAB, resistant , n=2, 1 | 1 | 0
  NNRTI, INI, CAB, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, CAB, sensitive, n=2, 1 | 1 | 1
  NNRTI, INI, DTG, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, DTG, resistant, n=2, 1 | 0 | 0
  NNRTI, INI, DTG, partially sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, DTG, partially sensitive, n=2, 1 | 0 | 0
  NNRTI, INI, DTG, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, DTG, sensitive, n=2, 1 | 2 | 1
  NNRTI, INI, EVG, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, EVG, resistant, n=2, 1 | 1 | 0
  NNRTI, INI, EVG, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, EVG, sensitive, n=2, 1 | 1 | 1
  NNRTI, INI, RAL, resistant, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, RAL, resistant, n=2, 1 | 1 | 0
  NNRTI, INI, RAL, sensitive, n=2, 1: number analyzed (Participants) | 2 | 1
  NNRTI, INI, RAL, sensitive, n=2, 1 | 1 | 1
  NNRTI, NNRTI, DLV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, DLV, resistant, n=2, 0 | 2 | 0
  NNRTI, NNRTI, DLV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, DLV, sensitive, n=2, 0 | 0 | 0
  NNRTI, NNRTI, EFV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, EFV, resistant, n=2, 0 | 2 | 0
  NNRTI, NNRTI, EFV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, EFV, sensitive, n=2, 0 | 0 | 0
  NNRTI, NNRTI, ETR, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, ETR, resistant, n=2, 0 | 0 | 0
  NNRTI, NNRTI, ETR, partially sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, ETR, partially sensitive, n=2, 0 | 2 | 0
  NNRTI, NNRTI, ETR, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, ETR, sensitive, n=2, 0 | 0 | 0
  NNRTI, NNRTI, NVP, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, NVP, resistant, n=2, 0 | 2 | 0
  NNRTI, NNRTI, NVP, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, NVP, sensitive, n=2, 0 | 0 | 0
  NNRTI, NNRTI, RPV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, RPV, resistant, n=2, 0 | 2 | 0
  NNRTI, NNRTI, RPV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NNRTI, RPV, sensitive, n=2, 0 | 0 | 0
  NNRTI, NRTI, 3TC, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, 3TC, resistant, n=2, 0 | 0 | 0
  NNRTI, NRTI, 3TC, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, 3TC, sensitive, n=2, 0 | 2 | 0
  NNRTI, NRTI, ABC, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, ABC, resistant, n=2, 0 | 0 | 0
  NNRTI, NRTI, ABC, partially sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, ABC, partially sensitive, n=2, 0 | 0 | 0
  NNRTI, NRTI, ABC, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, ABC, sensitive, n=2, 0 | 2 | 0
  NNRTI, NRTI, FTC, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, FTC, resistant, n=2, 0 | 0 | 0
  NNRTI, NRTI, FTC, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, FTC, sensitive, n=2, 0 | 2 | 0
  NNRTI, NRTI, TDF, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, TDF, resistant, n=2, 0 | 0 | 0
  NNRTI, NRTI, TDF, partially sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, TDF, partially sensitive, n=2, 0 | 0 | 0
  NNRTI, NRTI, TDF, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, TDF, sensitive, n=2, 0 | 2 | 0
  NNRTI, NRTI, ZDV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, ZDV, resistant, n=2, 0 | 1 | 0
  NNRTI, NRTI, ZDV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, ZDV, sensitive, n=2, 0 | 1 | 0
  NNRTI, NRTI, d4T, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, d4T, resistant, n=2, 0 | 0 | 0
  NNRTI, NRTI, d4T, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, d4T, sensitive, n=2, 0 | 2 | 0
  NNRTI, NRTI, ddI, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, ddI, resistant, n=2, 0 | 0 | 0
  NNRTI, NRTI, ddI, partially sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, ddI, partially sensitive, n=2, 0 | 0 | 0
  NNRTI, NRTI, ddI, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, NRTI, ddI, sensitive, n=2, 0 | 2 | 0
  NNRTI, PI, ATV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, ATV, resistant, n=2, 0 | 0 | 0
  NNRTI, PI, ATV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, ATV, sensitive, n=2, 0 | 2 | 0
  NNRTI, PI, DRV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, DRV, resistant, n=2, 0 | 0 | 0
  NNRTI, PI, DRV, partially sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, DRV, partially sensitive, n=2, 0 | 0 | 0
  NNRTI, PI, DRV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, DRV, sensitive, n=2, 0 | 2 | 0
  NNRTI, PI, FPV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, FPV, resistant, n=2, 0 | 0 | 0
  NNRTI, PI, FPV, partially sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, FPV, partially sensitive, n=2, 0 | 0 | 0
  NNRTI, PI, FPV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, FPV, sensitive, n=2, 0 | 2 | 0
  NNRTI, PI, IDV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, IDV, resistant, n=2, 0 | 0 | 0
  NNRTI, PI, IDV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, IDV, sensitive, n=2, 0 | 2 | 0
  NNRTI, PI, LPV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, LPV, resistant, n=2, 0 | 0 | 0
  NNRTI, PI, LPV, partially sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, LPV, partially sensitive, n=2, 0 | 0 | 0
  NNRTI, PI, LPV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, LPV, sensitive, n=2, 0 | 2 | 0
  NNRTI, PI, NFV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, NFV, resistant, n=2, 0 | 0 | 0
  NNRTI, PI, NFV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, NFV, sensitive, n=2, 0 | 2 | 0
  NNRTI, PI, RTV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, RTV, resistant, n=2, 0 | 0 | 0
  NNRTI, PI, RTV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, RTV, sensitive, n=2, 0 | 2 | 0
  NNRTI, PI, SQV, resistant, n=2,0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, SQV, resistant, n=2,0 | 0 | 0
  NNRTI, PI, SQV, partially sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, SQV, partially sensitive, n=2, 0 | 0 | 0
  NNRTI, PI, SQV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, SQV, sensitive, n=2, 0 | 2 | 0
  NNRTI, PI, TPV, resistant, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, TPV, resistant, n=2, 0 | 0 | 0
  NNRTI, PI, TPV, partially sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, TPV, partially sensitive, n=2, 0 | 0 | 0
  NNRTI, PI, TPV, sensitive, n=2, 0: number analyzed (Participants) | 2 | 0
  NNRTI, PI, TPV, sensitive, n=2, 0 | 2 | 0

74. Secondary Outcome: Change From Week 5 in Dimension Scores Using Percerption of Injection Questionnaire (PIN)-Last Observation Carried Forward (LOCF) in Q4W Arm
Description: The PIN questionnaire explores the bother of pain at the injection site and injection site reactions (ISR), anxiety before and after injection, willingness to receive an HIV injectable treatment the following visit and satisfaction with the mode of treatment administration of individuals receiving injection and perceptions of individuals associated with receiving injections.This measure contains 21 items that measure pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside of a clinical trial.Scores range from 1 to 5, and questions are phrased in such a way as to ensure that 1 always equated with the most favourable perception of vaccination, and 5 the most unfavourable.Dimension scores include bother from ISR, leg movement, sleep and acceptability.The score of a domain is calculated as the mean of all items with the domain.Higher scores represent worse perception of injection. LOCFwas used as primary method of analysis
Time Frame: Week 5 and at Weeks 41 and 48
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | CAB LA+RPV LA (Q4W)
Number analyzed (Participants) | 296
Scores on the scale
  Bother of ISRs, Week 41 | -0.21 (0.532)
  Bother of ISRs, Week 48 | -0.21 (0.524)
  Leg movement, Week 41 | -0.52 (0.903)
  Leg movement, Week 48 | -0.59 (0.950)
  Sleep, Week 41 | -0.56 (0.877)
  Sleep, Week 48 | -0.56 (0.937)
  Acceptance, Week 41 | -0.49 (1.094)
  Acceptance, Week 48 | -0.54 (1.080)

75. Secondary Outcome: Percentage of Participants With Extremely or Very Acceptable Pain and Local Reaction: Acceptability Score on PIN Questionnaire in Q4W Arm
Description: The PIN questionnaire explores the bother of pain at the injection site and injection site reactions(ISR), anxiety before and after injection, willingness to receive an HIV injectable treatment the following visit and satisfaction with the mode of treatment administration of individuals receiving injection and perceptions of individuals associated with receiving injections.This measure contains 21 items that measure pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside of a clinical trial.Scores range from 1 to 5, and questions are phrased in such a way as to ensure that 1 always equated with the most favourable perception of vaccination, and 5 the most unfavourable.Dimension scores include bother from ISR, leg movement, sleep and acceptability.The score of a domain is calculated as the mean of all items with the domain.Higher scores represent worse perception of injection. LOCF was used as primary method of analysis
Time Frame: Weeks 5, 41 and 48
Population: as for outcome 62
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA+RPV LA (Q4W)
Number analyzed (Participants) | 308
Percentage of participants
  Local reaction, Week 5, total, n=296: number analyzed (Participants) | 296
  Local reaction, Week 5, total, n=296 | 141
  Local reaction,Week 5, very acceptable, n=296: number analyzed (Participants) | 296
  Local reaction,Week 5, very acceptable, n=296 | 77
  Local reaction, Week 5, moderate, n=296: number analyzed (Participants) | 296
  Local reaction, Week 5, moderate, n=296 | 54
  Local reaction, Week 5, little, n=296: number analyzed (Participants) | 296
  Local reaction, Week 5, little, n=296 | 15
  Local reaction, Week 5, not at all, n=296: number analyzed (Participants) | 296
  Local reaction, Week 5, not at all, n=296 | 9
  Pain, Week 5, total, n=296: number analyzed (Participants) | 296
  Pain, Week 5, total, n=296 | 86
  Pain, Week 5, very acceptable, n=296: number analyzed (Participants) | 296
  Pain, Week 5, very acceptable, n=296 | 103
  Pain, Week 5, moderate, n=296: number analyzed (Participants) | 296
  Pain, Week 5, moderate, n=296 | 59
  Pain, Week 5, little, n=296: number analyzed (Participants) | 296
  Pain, Week 5, little, n=296 | 29
  Pain, Week 5, not at all, n=296: number analyzed (Participants) | 296
  Pain, Week 5, not at all, n=296 | 19
  Local reaction, Week 41, total, n=300: number analyzed (Participants) | 300
  Local reaction, Week 41, total, n=300 | 188
  Local reaction, Week 41, very acceptable, n=300: number analyzed (Participants) | 300
  Local reaction, Week 41, very acceptable, n=300 | 77
  Local reaction, Week 41, moderate, n=300: number analyzed (Participants) | 300
  Local reaction, Week 41, moderate, n=300 | 24
  Local reaction, Week 41, little, n=300: number analyzed (Participants) | 300
  Local reaction, Week 41, little, n=300 | 6
  Local reaction, Week 41, not at all, n=300: number analyzed (Participants) | 300
  Local reaction, Week 41, not at all, n=300 | 5
  Pain, Week 41, total, n=300: number analyzed (Participants) | 300
  Pain, Week 41, total, n=300 | 166
  Pain, Week 41, very acceptable, n=300: number analyzed (Participants) | 300
  Pain, Week 41, very acceptable, n=300 | 85
  Pain, Week 41, moderate, n=300: number analyzed (Participants) | 300
  Pain, Week 41, moderate, n=300 | 31
  Pain, Week 41, little, n=300: number analyzed (Participants) | 300
  Pain, Week 41, little, n=300 | 12
  Pain, Week 41, not at all, n=300: number analyzed (Participants) | 300
  Pain, Week 41, not at all, n=300 | 6
  Local reaction, week 48, total, n=303: number analyzed (Participants) | 303
  Local reaction, week 48, total, n=303 | 202
  Local reaction, Week 48, very acceptable, n=303: number analyzed (Participants) | 303
  Local reaction, Week 48, very acceptable, n=303 | 69
  Local reaction, Week 48, moderate, n=303: number analyzed (Participants) | 303
  Local reaction, Week 48, moderate, n=303 | 21
  Local reaction, Week 48, little, n=303: number analyzed (Participants) | 303
  Local reaction, Week 48, little, n=303 | 8
  Local reaction, Week 48, not at all, n=303: number analyzed (Participants) | 303
  Local reaction, Week 48, not at all, n=303 | 3
  Pain, Week 48, total, n=303: number analyzed (Participants) | 303
  Pain, Week 48, total, n=303 | 168
  Pain, Week 48, very acceptable, n=303: number analyzed (Participants) | 303
  Pain, Week 48, very acceptable, n=303 | 95
  Pain, Week 48, moderate, n=303: number analyzed (Participants) | 303
  Pain, Week 48, moderate, n=303 | 26
  Pain, Week 48, little, n=303: number analyzed (Participants) | 303
  Pain, Week 48, little, n=303 | 11
  Pain, Week 48, not at all, n=303: number analyzed (Participants) | 303
  Pain, Week 48, not at all, n=303 | 3

76. Secondary Outcome: Change From Baseline in Life Satisfaction (LISAT) Using HIV/AIDs-targeted Quality of Life (HATQoL) Questionnaire
Description: The HATQoL questionnaire was used to assess the health related QoL (HRQoL). It comprises of three dimensions: LISAT, medication worries (MEDWO) and disclosure worries (DISWO). The total imputed value score for LISAT is calculated on a 0-100 scale using the formula: LISAT 100=[100 divided by (20 minus 4)]*(LISAT minus 4). A response of 5 in LISAT score shows satisfaction all of the time and 1 as none of the time. The higher the score, the greater satisfaction to life and the less worry. The transformed dimension score for each domain was summarized and analyzed. LOCF was used as primary method of analysis. Measure type was considered as mean for adjusted mean and dispersion measure as 95% confidence interval (CI).Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 62
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Scores on a scale
  Week 24, n=292, 291: number analyzed (Participants) | 292 | 291
  Week 24, n=292, 291 | 1.0 [-0.6 to 2.6] | 1.1 [-0.5 to 2.7]
  Week 48, n=292, 297: number analyzed (Participants) | 292 | 297
  Week 48, n=292, 297 | 1.1 [-0.6 to 2.8] | 0.1 [-1.6 to 1.7]
Statistical Analysis 1: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.944, ANCOVA; Adjusted difference = -0.1, 95% CI 2-sided [-2.4 to 2.2] — Treatment comparison at Week 24 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 2: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.385, ANCOVA; Adjusted difference = 1.0, 95% CI 2-sided [-1.3 to 3.4] — Treatment comparison at Week 48 for the groups CAB LA+ RPV LA and current ART is presented

77. Secondary Outcome: Change From Baseline in HIV Medication, MEDWO Using HATQoL
Description: The HATQoL questionnaire was used to assess the health related QoL (HRQoL). It comprises of three dimensions: LISAT, medication worries (MEDWO) and disclosure worries (DISWO). The total imputed value score for MEDWO is calculated on a 0-100 scale using the formula: MEDWO 100=[100 divided by (20 minus 5)]*(MEDWO minus 5). A response of 1 in MEDWO score shows less medication worries all of the time and 5 as none of the time. The higher the score, the greater satisfaction to life and the less worry. The transformed dimension score for each domain was summarized and analyzed. LOCF was used as primary method of analysis. Measure type was considered as mean for adjusted mean and dispersion measure as 95% CI. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and at Weeks 24 and 48
Population: as for outcome 62
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Scores on a scale
  Week 24, n=292, 290: number analyzed (Participants) | 292 | 290
  Week 24, n=292, 290 | 4.2 [2.7 to 5.8] | -0.7 [-2.2 to 0.9]
  Week 48, n=292, 296: number analyzed (Participants) | 292 | 296
  Week 48, n=292, 296 | 4.0 [2.3 to 5.7] | -2.4 [-4.1 to -0.8]
Statistical Analysis 1: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p < 0.001, ANCOVA; Adjusted difference = 4.9, 95% CI 2-sided [2.8 to 7.1] — Treatment comparison at Week 24 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 2: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p < 0.001, ANCOVA; Adjusted difference = 6.4, 95% CI 2-sided [4.0 to 8.8] — Treatment comparison at Week 48 for the groups CAB LA+ RPV LA and current ART is presented

78. Secondary Outcome: Change From Baseline in DISWO Using HATQoL
Description: The HATQoL questionnaire was used to assess the health related QoL (HRQoL). It comprises of three dimensions: LISAT, medication worries (MEDWO) and disclosure worries (DISWO). The total imputed value score for DISWO is calculated on a 0-100 scale using the formula: DISWO 100=[100 divided by (20 minus 5)]*(DISWO minus 5). A response of 1 in DISWO score shows less medication worries all of the time and 5 as none of the time. The higher the score, the greater satisfaction to life and the less worry. The transformed dimension score for each domain was summarized and analyzed. LOCF was used as primary method of analysis. Measure type was considered as mean for adjusted mean and dispersion measure as 95% CI. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and at Weeks 24 and 48
Population: as for outcome 62
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Scores on a scale
  Week 24, n=291, 290: number analyzed (Participants) | 291 | 290
  Week 24, n=291, 290 | 8.3 [5.6 to 11.0] | 3.0 [0.3 to 5.8]
  Week 48, n=291, 296: number analyzed (Participants) | 291 | 296
  Week 48, n=291, 296 | 4.6 [1.7 to 7.6] | 2.6 [-0.3 to 5.6]
Statistical Analysis 1: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.008, ANCOVA; Adjusted difference = 5.3, 95% CI 2-sided [1.4 to 9.1] — Treatment comparison at Week 24 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 2: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.347, ANCOVA; Adjusted difference = 2.0, 95% CI 2-sided [-2.2 to 6.2]; Treatment comparison at Week 48 for the groups CAB LA+ RPV LA and current ART is presented

79. Secondary Outcome: Change From Baseline in Health Status Using 12-item Short Form Survey (SF-12)
Description: The SF-12 questionnaire consists of 7 questions which measures the degree of general health status and mental health distress. Each question is scored 0-5, except for question 2 scored 0-3. The HRQoL using SF-12 for the total score, physical component summary (PCS) and the mental component summary (MCS) were assessed for the two treatment groups. Missing Total or the component scores was imputed using LOCF. The PCS/MCS are calculated using computer software purchased from QualityMetric (http://www.qualitymetric.com). The higher the score, the better will be the health status. Measure type was considered as mean for adjusted mean and dispersion measure as 95% CI. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and at Weeks 24 and 48
Population: as for outcome 62
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Scores on a scale
  Total score, Week 24, n=291, 289: number analyzed (Participants) | 291 | 289
  Total score, Week 24, n=291, 289 | 0.0 [-0.3 to 0.4] | -0.2 [-0.5 to 0.1]
  Total score, Week 48, n=293, 296: number analyzed (Participants) | 293 | 296
  Total score, Week 48, n=293, 296 | -0.0 [-0.4 to 0.3] | 0.0 [-0.3 to 0.4]
  MCS, Week 24, n=289, 286: number analyzed (Participants) | 289 | 286
  MCS, Week 24, n=289, 286 | 0.288 [-0.579 to 1.155] | -0.388 [-1.259 to 0.484]
  MCS, Week 48, n=291, 293: number analyzed (Participants) | 291 | 293
  MCS, Week 48, n=291, 293 | 0.260 [-0.638 to 1.158] | -0.375 [-1.270 to 0.520]
  PCS, Week 24, n=286, 288: number analyzed (Participants) | 286 | 288
  PCS, Week 24, n=286, 288 | 0.650 [0.087 to 1.213] | -0.047 [-0.608 to 0.514]
  PCS, Week 48, n=288, 295: number analyzed (Participants) | 288 | 295
  PCS, Week 48, n=288, 295 | 0.758 [0.184 to 1.332] | 0.062 [-0.505 to 0.629]
Statistical Analysis 1: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.344, ANCOVA; Adjusted difference = 0.2, 95% CI 2-sided [-0.2 to 0.7] — Treatment comparison of SF-12 total scores at Week 24 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 2: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.785, ANCOVA; Adjusted difference = -0.1, 95% CI 2-sided [-0.6 to 0.4] — Treatment comparison of SF-12 total scores at Week 48 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 3: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.282, ANCOVA; Adjusted difference = 0.676, 95% CI 2-sided [-0.557 to 1.909] — Treatment comparison of SF-12 MCS at Week 24 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 4: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.327, ANCOVA; Adjusted difference = 0.635, 95% CI 2-sided [-0.637 to 1.907] — Treatment comparison of SF-12 MCS at Week 48 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 5: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.086, ANCOVA; Adjusted difference = 0.697, 95% CI 2-sided [-0.100 to 1.494] — Treatment comparison of SF-12 PCS at Week 24 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 6: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p = 0.092, ANCOVA; Adjusted difference = 0.696, 95% CI 2-sided [-0.113 to 1.505] — Treatment comparison of SF-12 PCS at Week 48 for the groups CAB LA+ RPV LA and current ART is presented

80. Secondary Outcome: Change From Baseline in Total Treatment Satisfaction Using HIV Treatment Satisfaction Questionnaire (HIVTSQs) at Weeks 4b, 24 and 44
Description: The HIVTSQ for total treatment satisfaction score is computed with 1-11 items. These 1-11 items are summed to produce a score with a possible range of -33 to 33. The item 12 in the scale will be calculated as an individual score.The higher the score, the greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment.A score of 0 represents no change. A maximum of 5 items can be missing, the missing scores will be imputed with the mean of the completed item scores. If 6 or more items are missing, then the overall treatment satisfaction scale score should not be computed and will remain missing.LOCF was used as primary method of analysis. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value. Data has been presented with respect to actual treatment received to the participants
Time Frame: Baseline and at Weeks 4b, 24 and 44
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Scores on a scale
  Week 4b, n=295, 0: number analyzed (Participants) | 295 | 0
  Week 4b, n=295, 0 | 3.99 (8.982) |
  Week 24, n=300, 288: number analyzed (Participants) | 300 | 288
  Week 24, n=300, 288 | 6.39 (10.328) | 1.08 (8.510)
  Week 44, n=300, 294: number analyzed (Participants) | 300 | 294
  Week 44, n=300, 294 | 6.02 (10.808) | 0.54 (9.877)

81. Secondary Outcome: Change in Treatment Satisfaction Over Time Using HIVTSQ Change (HIVTSQc) at Week 48 in Q4W Arm
Description: as for outcome 80
Time Frame: Week 48
Population: ITT-E population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA+RPV LA (Q4W)
Number analyzed (Participants) | 275
Scores on a scale | 29.05 (6.978)

82. Secondary Outcome: Change From Baseline in Treatment Acceptance at Weeks 8, 24 and 48 Using "General Acceptance" Dimension of the Chronic Treatment Acceptance (ACCEPT) Questionnaire
Description: The ACCEPT questionnaire is a generic medication acceptance measure assessing how participants weigh advantages and disadvantages of long-term medication.The questionnaire consists of 25 items that capture six dimensions.3 questions that focus on general acceptance of study medication will be analyzed.Items on the scale are rated as 1-5 scores:1:totally disagree,2:somewhat disagree,3:somewhat agree, 4:totally agree and 5:I don't know.Total score of the dimension is calculated as the mean of the recoded items of the dimension and then linearly transformed to be on a scale from 0 to 100:score:Total Score=(mean of the recoded items in the dimension minus1)divided by2*100.LOCF was used as primary method of analysis.Measure type was considered as mean for adjusted mean and dispersion measure as 95% CI.Baseline value is defined as the latest pre-treatment assessment with a non-missing value.Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value
Time Frame: Baseline and at Weeks 8, 24 and 48
Population: as for outcome 62
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Scores on a scale
  Week 8, n=302, 287: number analyzed (Participants) | 302 | 287
  Week 8, n=302, 287 | 8.9 [6.3 to 11.6] | 1.0 [-1.7 to 3.8]
  Week 24, 303, 295: number analyzed (Participants) | 303 | 295
  Week 24, 303, 295 | 12.3 [9.9 to 14.8] | 5.5 [3.0 to 8.0]
  Week 48, n=302, 298: number analyzed (Participants) | 302 | 298
  Week 48, n=302, 298 | 13.7 [11.2 to 16.3] | 3.0 [0.4 to 5.6]
Statistical Analysis 1: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p < 0.001, ANCOVA; Adjusted difference = 7.9, 95% CI 2-sided [4.1 to 11.7] — Treatment comparison at Week 8 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 2: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p < 0.001, ANCOVA; Adjusted difference = 6.9, 95% CI 2-sided [3.3 to 10.4] — Treatment comparison Week 24 for the groups CAB LA+ RPV LA and current ART is presented
Statistical Analysis 3: Comparison: CAB LA+RPV LA (Q4W) vs Current ART; Test type: Other; p < 0.001, ANCOVA; Adjusted difference = 10.7, 95% CI 2-sided [7.1 to 14.4] — Treatment comparison at Week 48 for the groups CAB LA+ RPV LA and current ART is presented

83. Secondary Outcome: Change From 4b in Tolerability of Injection at Week 5, 40 and 41 Using Numeric Rating Scale (NRS) Within CAB LA+RPV LA Arm
Description: The NRS questionnaire is used to assess the tolerability of injections in CAB LA+RPV LA arm only. The questionnaire consists of one single question and will assess maximum level of pain experienced with the most recent injections ranking from no pain (0) to extreme pain (10). Missing scores was imputed using LOCF.
Time Frame: Weeks 4b, 5, 40 and 41
Population: ITT-E population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA+RPV LA (Q4W)
Number analyzed (Participants) | 278
Scores on a scale
  Week 5 | 2.0 (2.94)
  Week 40 | 0.5 (2.79)
  Week 41 | 0.4 (2.83)

84. Secondary Outcome: Change From Baseline in Individual Item Scores of HIVTSQc at Weeks 4b, 24 and 44
Description: HIVTSQc is a 12 item questionnaire. The individual treatment change item scores on HIVTSQc scale are rated as +3 ('much more satisfied', 'much more convenient', 'much more flexible',etc.) to -3 ('much less satisfied', 'much less convenient', 'much less flexible', etc.). The higher the score, the greater the improvement in satisfaction with each aspect of treatment and the lower the score, the greater the deterioration in satisfaction with each aspect of treatment. LOCF was used as primary method of analysis. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and Weeks 4b, 24 and 44
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
Number analyzed (Participants) | 308 | 308
Scores on a scale
  Item 1; Week 4b; n=294, 0: number analyzed (Participants) | 294 | 0
  Item 1; Week 4b; n=294, 0 | 0.3 (1.42) |
  Item 1; Week 24; n=300, 287: number analyzed (Participants) | 300 | 287
  Item 1; Week 24; n=300, 287 | 0.4 (1.46) | -0.1 (1.04)
  Item 1; Week 44; n=300, 293: number analyzed (Participants) | 300 | 293
  Item 1; Week 44; n=300, 293 | 0.5 (1.42) | -0.1 (1.21)
  Item 2; Week 4b; n=295, 0: number analyzed (Participants) | 295 | 0
  Item 2; Week 4b; n=295, 0 | 0.0 (0.60) |
  Item 2; Week 24; n=300, 287: number analyzed (Participants) | 300 | 287
  Item 2; Week 24; n=300, 287 | 0.1 (0.70) | 0.0 (0.68)
  Item 2; Week 44; n=300, 293: number analyzed (Participants) | 300 | 293
  Item 2; Week 44; n=300, 293 | 0.1 (0.84) | -0.1 (0.82)
  Item 3; Week 4b; n=295, 0: number analyzed (Participants) | 295 | 0
  Item 3; Week 4b; n=295, 0 | 0.4 (1.35) |
  Item 3; Week 24; n=300, 288: number analyzed (Participants) | 300 | 288
  Item 3; Week 24; n=300, 288 | 0.3 (1.47) | 0.1 (1.12)
  Item 3; Week 44; n=300, 294: number analyzed (Participants) | 300 | 294
  Item 3; Week 44; n=300, 294 | 0.3 (1.45) | 0.0 (1.26)
  Item 4; Week 4b; n=295, 0: number analyzed (Participants) | 295 | 0
  Item 4; Week 4b; n=295, 0 | 0.3 (1.21) |
  Item 4; Week 24; n=300, 288: number analyzed (Participants) | 300 | 288
  Item 4; Week 24; n=300, 288 | 0.5 (1.29) | -0.0 (1.16)
  Item 4; Week 44; n=300, 294: number analyzed (Participants) | 300 | 294
  Item 4; Week 44; n=300, 294 | 0.4 (1.30) | -0.1 (1.22)
  Item 5; Week 4b; n=295, 0: number analyzed (Participants) | 295 | 0
  Item 5; Week 4b; n=295, 0 | 0.5 (1.24) |
  Item 5; Week 24; n=300, 288: number analyzed (Participants) | 300 | 288
  Item 5; Week 24; n=300, 288 | 0.8 (1.32) | 0.1 (1.31)
  Item 5; Week 44; n=300, 294: number analyzed (Participants) | 300 | 294
  Item 5; Week 44; n=300, 294 | 0.8 (1.42) | 0.0 (1.37)
  Item 6; Week 4b; n=294, 0: number analyzed (Participants) | 294 | 0
  Item 6; Week 4b; n=294, 0 | 0.5 (1.63) |
  Item 6; Week 24; n=299, 288: number analyzed (Participants) | 299 | 288
  Item 6; Week 24; n=299, 288 | 0.8 (1.77) | 0.2 (1.79)
  Item 6; Week 44; n=299, 293: number analyzed (Participants) | 299 | 293
  Item 6; Week 44; n=299, 293 | 0.9 (1.72) | 0.2 (1.78)
  Item 7; Week 4b; n=295, 0: number analyzed (Participants) | 295 | 0
  Item 7; Week 4b; n=295, 0 | 0.2 (0.90) |
  Item 7; Week 24; n=300, 288: number analyzed (Participants) | 300 | 288
  Item 7; Week 24; n=300, 288 | 0.2 (0.94) | 0.1 (1.00)
  Item 7; Week 44; n=300, 294: number analyzed (Participants) | 300 | 294
  Item 7; Week 44; n=300, 294 | 0.2 (0.99) | 0.2 (1.08)
  Item 8; Week 4b; n=294, 0: number analyzed (Participants) | 294 | 0
  Item 8; Week 4b; n=294, 0 | 0.3 (1.21) |
  Item 8; Week 24; n=299, 288: number analyzed (Participants) | 299 | 288
  Item 8; Week 24; n=299, 288 | 0.7 (1.27) | 0.1 (1.20)
  Item 8; Week 44; n=299, 294: number analyzed (Participants) | 299 | 294
  Item 8; Week 44; n=299, 294 | 0.6 (1.31) | 0.0 (1.27)
  Item 9; Week 4b; n=294, 0: number analyzed (Participants) | 294 | 0
  Item 9; Week 4b; n=294, 0 | 0.4 (1.22) |
  Item 9; Week 24; n=299, 288: number analyzed (Participants) | 299 | 288
  Item 9; Week 24; n=299, 288 | 0.6 (1.27) | 0.1 (1.20)
  Item 9; Week 44; n=299, 294: number analyzed (Participants) | 299 | 294
  Item 9; Week 44; n=299, 294 | 0.5 (1.32) | 0.0 (1.25)
  Item 10; Week 4b; n=293, 0: number analyzed (Participants) | 293 | 0
  Item 10; Week 4b; n=293, 0 | 0.8 (1.44) |
  Item 10; Week 24; n=298, 287: number analyzed (Participants) | 298 | 287
  Item 10; Week 24; n=298, 287 | 1.2 (1.56) | 0.3 (1.38)
  Item 10; Week 44; n=298, 293: number analyzed (Participants) | 298 | 293
  Item 10; Week 44; n=298, 293 | 1.1 (1.64) | 0.2 (1.60)
  Item 11; Week 4b; n=292, 0: number analyzed (Participants) | 292 | 0
  Item 11; Week 4b; n=292, 0 | 0.4 (1.23) |
  Item 11; Week 24; n=297, 287: number analyzed (Participants) | 297 | 287
  Item 11; Week 24; n=297, 287 | 0.7 (1.31) | 0.1 (1.28)
  Item 11; Week 44; n=297, 293: number analyzed (Participants) | 297 | 293
  Item 11; Week 44; n=297, 293 | 0.6 (1.45) | 0.1 (1.38)
  Item 12; Week 4b; n=293, 0: number analyzed (Participants) | 293 | 0
  Item 12; Week 4b; n=293, 0 | 0.3 (1.41) |
  Item 12; Week 24; n=298, 287: number analyzed (Participants) | 298 | 287
  Item 12; Week 24; n=298, 287 | 0.0 (1.52) | 0.1 (1.14)
  Item 12; Week 44; n=298, 293: number analyzed (Participants) | 298 | 293
  Item 12; Week 44; n=298, 293 | 0.0 (1.58) | 0.2 (1.17)

85. Other Pre Specified Outcome: Number of Participants With Different Demographic Parameters for Inter-subject Variability
Description: Blood samples were planned to be collected at indicated time points for PK analysis of CAB LA and RPV LA. Demographic parameters including, but not limited to, age, sex, race, body weight, body mass index, and relevant laboratory parameters were planned to be evaluated as potential predictors of inter subject variability for pharmacokinetic parameters.
Time Frame: Upto Week 48
Population: PK Population. This was an exploratory Outcome Measure. Data will not be analyzed and reported.
Arm/Group | CAB LA | RPV LA
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: AEs and SAEs were collected in Safety population.
Arm/Group | CAB LA+RPV LA (Q4W) | Current ART
All-Cause Mortality (participants affected / at risk) | 0/308 | 1/308
Serious Adverse Events (participants affected / at risk) | 13/308 | 14/308
Other Adverse Events (participants affected / at risk) | 263/308 | 117/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA+RPV LA (Q4W) (N=308) | Current ART (N=308)
Hepatitis A (Infections and infestations) | 1 (1) | 1 (1)
Acute hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA+RPV LA (Q4W) (N=308) | Current ART (N=308)
Injection site pain (General disorders) | 231 (1208) | 0 (0)
Injection site nodule (General disorders) | 37 (54) | 0 (0)
Injection site induration (General disorders) | 30 (54) | 0 (0)
Pyrexia (General disorders) | 21 (29) | 9 (9)
Fatigue (General disorders) | 22 (29) | 6 (9)
Injection site swelling (General disorders) | 23 (48) | 0 (0)
Nasopharyngitis (Infections and infestations) | 52 (87) | 42 (58)
Upper respiratory tract infection (Infections and infestations) | 32 (48) | 25 (30)
Influenza (Infections and infestations) | 17 (19) | 14 (15)
Respiratory tract infection viral (Infections and infestations) | 11 (12) | 17 (23)
Headache (Nervous system disorders) | 34 (48) | 17 (19)
Diarrhoea (Gastrointestinal disorders) | 22 (24) | 15 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (22) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT02951052/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT02951052/SAP_002.pdf